

Enterics for Global Health: *Shigella* surveillance study (EFGH) statistical analysis plan and case report forms





#### **Table of Contents**

| PDF Page<br>Number | Contents |
|---|---|
| 3 - 28 | The Enterics for Global Health (EFGH) <i>Shigella</i> Surveillance Statistical Analysis Plan |
| 29 - 55 | The Enterics for Global Health (EFGH) <i>Shigella</i> Surveillance Statistical Analysis Plan: Tables & Figures |
| 56 - 199 | The Enterics for Global Health (EFGH) <i>Shigella</i> Surveillance Study Case Report Forms |



## Enterics for Global Health (EFGH) Statistical Analysis Plan Version 4.0





#### Table of Contents SECTION 1. ADMINISTRATIVE INFORMATION......3 Protocol Version 3 Abbreviations .......4 SECTION 2. INTRODUCTION ......5 SECTION 3. STUDY METHODS ......5 Sample Size \_\_\_\_\_\_6 Framework......6 SECTION 5. STUDY POPULATIONS......7 Recruitment 8 Definitions 9 Analysis Methods 11 References 25



#### **SECTION 1. ADMINISTRATIVE INFORMATION**

Title: Statistical Analysis Plan (SAP) for the Enterics for Global Health (EFGH) study

**SAP Version:** 4.0 (18 December 2024)

**Protocol Version:** 5.0 (09 June 2023)

#### **SAP Revision History:**

| SAP version (date) | Justification for Revision | Timing of SAP in relation to interim analysis |
|---|---|---|
| 2.0 (17 June 2024) | Adding complete secondary aim sections and | N/A |
| | revised SAP per consortium review | |
| 3.0 (03 October 2024) | Updated SAP with details following review | N/A |
| | by the Design, Analyze and Communicate | |
| | group at the Bill & Melinda Gates Foundation | |
| 4.0 (18 December 2024) | 4.0 (18 December 2024) Updated SAP to reflect method of variance | |
| | estimation to be used in primary analysis | |

#### **SAP Working Group**

| Name | EFGH Role |
|---|---|
| Faisal Ahmmed | Co-Investigator, icddr,b |
| Hannah Atlas | Co-Investigator, University of Washington (UW) |
| John Clemens | Co-Principal Investigator-Bangladesh, International Vaccine Institute (IVI) |
| Erika Feutz | Data Manager & Analyst, UW |
| Sean Galagan | Senior Data Manager & Analyst, UW |
| Jahangir Hossain | Co-Principal Investigator-the Gambia, The Medical Research Council Unit - The Gambia (MRCG) |
| Muhammed Jawwad | Co-Investigator, The Aga Khan University (AKU) |
| Karen Kotloff | Co-Principal Investigator-Mali, Kenya, the Gambia, The University of Maryland, Baltimore (UMB) |
| Donnie Mategula | Co-Investigator, Malawi-Liverpool-Wellcome Trust (MLW) |
| Christine McGrath | Co-Investigator, UW |
| Billy Ogwel | Co-Investigator, Kenya Medical Research Institute (KEMRI) |
| Dr. Patricia Pavlinac | Co-Principal Investigator-Coordination, UW |
| James Platts-Mills | Co-Investigator, The University of Virginia (UVA) |
| Elizabeth Rogawski-McQuade | Co-Investigator, Emory University |
| Francesca Schiaffino | Co-Investigator, UVA |
| Mili Tapia | Co-Investigator, UMB |
| Tahir Yousufzai | Co-investigator, AKU |

#### **Also Contributed to SAP Content**

| Name | EFGH Role |
|---------------------|------------------------------------------------|
| Chloe Morozoff | Implementation Science Analyst, UW |
| Arianna Rubin Means | Co-Investigator, University of Washington (UW) |
| Olivia Schultes | Data Manager & Analyst, UW |



#### **Abbreviations**

ΔLAZ/HAZ Linear growth

AIC Akaike information criterion AKU The Aga Khan University CI 95% confidence interval

CLSI Clinical and Laboratory Standards Institute

CT Cycle threshold

DCS Diarrhea case surveillance EFGH Enterics for Global Health ETEC Enterotoxigenic *E. coli* 

GEMS Global Enteric Multicenter Study
GLM Generalized Linear Models
HAZ Height for age Z-score
HUS Healthcare Utilization Survey

ICD-11 International Classification of Diseases 11<sup>th</sup> Revision

IMCI Integrated Management of Childhood Illness

IR Incidence rate

IRB Institutional Review Board

IQR Interquartile range

IVI International Vaccine Institute

JMP WHO/UNICEF Joint Monitoring Programme for Water Supply, Sanitation and Hygiene

KEMRI Kenya Medical Research Institute

LAZ Length for age Z-score

LRTI Lower respiratory tract infection

LSD Less-severe diarrhea LTFU Lost to follow-up

MAD Medically-attended diarrhea

MAL-ED Malnutrition and Enteric Disease Study mBGS Modified buffered glycerol saline

MDR Multidrug-resistant

MLW Malawi-Liverpool-Wellcome Trust

MRCG The Medical Research Council Unit - The Gambia

MSD Moderate-to-severe diarrhea
MUAC Mid-upper arm circumference
MVS Modified Vesikari score
NPV Negative predictive value
PPV Positive predictive value

PR Prevalence ratio

ROC Receiver operating characteristics

RR Relative risk

SAP Statistical analysis plan SD Standard deviation SES Socioeconomic status TAC TaqMan Array Card

UMB The University of Maryland, Baltimore

USD United states dollars
UVA The University of Virginia
UW University of Washington
WAZ Weight for age Z-score
WHO World Health Organization
WLZ Weight for length Z-score
XDR Extensively drug-resistant



#### **SECTION 2. INTRODUCTION**

#### **Background and Rationale**

In low- and middle-income countries, nearly one third of children experience at least one episode of *Shigella*-attributable diarrhea during their first two years of life. In addition to being a leading cause of diarrhea, this enteric bacterium is also associated with linear growth faltering, a precursor to stunting. Stunting is a marker of vulnerability to childhood infection, decreased vaccine efficacy and lifelong morbidity. Currently, several promising *Shigella* vaccines are in development. Eventual Phase 2b/3 *Shigella* vaccine trials will require a consortium of potential vaccine trial sites in settings with a high incidence of *Shigella*-attributed medically-attended diarrhea (MAD), high participant retention, and the laboratory capacity to confirm *Shigella* infection. The Enterics for Global Health (EFGH) *Shigella* surveillance study will employ cross-sectional and longitudinal study designs to establish updated incidence rates and document consequences of *Shigella* diarrhea within seven country sites in Africa, Asia, and Latin America. Specifically, we aim to:

#### Aims

- 1. **Primary Aim**: Determine the incidence of *Shigella*-attributed MAD in children 6 to 35 months of age in each of the EFGH country sites.
- 2. **Secondary Aim 1:** Determine the incidence of *Shigella* MAD by serotype, severity definition, laboratory method (culture vs. qPCR), age, and by season.
- 3. **Secondary Aim 2:** Describe the prevalence of resistance to commonly used antibiotics in *Shigella* isolates in each EFGH country site.
- 4. **Secondary Aim 3:** Determine the risk of death, hospitalization, persistent diarrhea, experiencing a subsequent diarrhea episode, and linear growth faltering in the three months following an episode of *Shigella* MAD.
- 5. **Secondary Aim 4:** Compare various severity definitions in their ability to predict risk of death/hospitalization or linear growth faltering among cases of MAD and *Shigella*-attributable MAD, respectively.
- 6. **Secondary Aim 5:** Quantify the cost incurred by families and health care systems due to *Shigella* morbidity and mortality.
- 7. **Secondary Aim 6:** Identify optimal laboratory methods for *Shigella* culture by:
  - a. Comparing the isolation rate of *Shigella* between two transport media for rectal swabs (Cary-Blair and modified Buffered Glycerol Saline [mBGS]).
  - b. Comparing the isolation rate of *Shigella* between two fecal sample types (rectal swabs and whole stool) among the subset of children who produced whole stool in The Gambia and Bangladesh country sites.

#### SECTION 3. STUDY METHODS

#### **Study Design**

The EFGH study will employ cross-sectional and longitudinal study designs to establish incidence and consequences of *Shigella* diarrhea. Children aged 6-35 months of age presenting with diarrhea at selected study health facilities will be recruited over a 24-month period and followed for three months. Randomly selected households will be visited within each EFGH site catchment area over the 24-month recruitment period to estimate the population of children aged 6-35 months in the catchment area. A healthcare utilization survey (HUS) will be conducted among households in the catchment area with one or more children in the 6-35-month age range to determine the proportion of diarrhea cases that present to EFGH study health facilities. The number of cases divided by the estimated number of children 6-35 months of age residing in the catchment area and time of surveillance will estimate the crude incidence rate of *Shigella* diarrhea in 6-35 months of age. This incidence rate will be adjusted by the proportion of eligible children



enrolled and the proportion of eligible children with diarrhea who sought care at an EFGH recruiting facility.

#### Sample Size

The minimum number of confirmed *Shigella* cases (numerator) and minimum size of the source population within health facility catchment area (denominator) required to estimate *Shigella* incidences and 95% confidence intervals with specified precision (half-widths of 0.25 cases per 100 child-years) within children aged 6-35 months were estimated. To ensure appropriate precision in estimates of serotype and antibiotic susceptibility of *Shigella* isolates, we aim recruit at least 65 children with culture-confirmed *Shigella* diarrhea at each EFGH site. We assumed that 4.8% of diarrhea cases will be *Shigella* culture-positive in the EFGH study, requiring that we enroll 1400 children presenting to health facilities with diarrhea over the 24-month period (~58 per month). The size of the catchment area population (>97,000) was determined assuming an unadjusted *Shigella* incidence rate of 0.63 per 100 child-years (unadjusted for health care seeking behavior) and 95% confidence interval precision of 0.25 (half-width).

#### Framework

Not applicable.

#### **Interim Statistical Analysis and Stopping Guidance**

Interim "Data Readouts" presenting preliminary study results will be generated on a biannual basis and shared with study investigators and the BMGF. As this study is not a randomized trial and there is no intervention, there is no stopping guidance.

#### **Timing of Final Analysis**

The primary study publication will be prepared for the primary aim when every enrolled child has completed their three-month follow-up visit or is deemed lost to follow-up and all data for the primary aim has been cleaned (anticipated publication submission in May of 2025).

Figure A. Timeline of study activities

| | 2022 | | | 2023 | | | 2024 | | | 2025 | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Key Activity | Q1 | Q2 | Q3 | Q4 | Q1 | Q2 | Q3 | Q4 | Q1 | Q2 | Q3 | Q4 | Q1 | Q2 |
| Diarrhea case surveillance (24 | | | | | | | | | | | | | | |
| months recruitment + 3 months | | | | | | | | | | | | | | |
| final follow-up) | | | | | | | | | | | | | | |
| Population enumeration activities | | | | | | | | | | | | | | |
| Healthcare utilization survey | | | | | | | | | | | | | | |
| Data cleaning | | | | | | | | | | | | | | |
| Data analysis | | | | | | | | | | | | | | |
| Publication preparations | | | | | | | | | | | | | | |
| Dissemination of results | | | | | | | | | | | · | | | |

#### Longitudinal follow-up

The schedule of study procedures is outlined in Figure A. Regularly scheduled clinical visits include those at enrollment and at follow-up (week four and month three) and are defined as a 14-day period in which visits are considered completed (24-37 days post-enrollment for the week four visit and 84-97 days post-enrollment for the month three visit). Additionally, visits are allowed for up to 30 days past the visit window (38-67 days post-enrollment for the week 4 visit and 98-127 days post-enrollment for the month 3 visit) though may be excluded from analyses (**Table B**).

| Table B. Allowable windows for longitudinal follow-up | | |
|---|---|---|
| Visit Window Allowable visits | | |
| Week four follow-up visit | 24-37 days post-enrollment. | 38-67 days post-enrollment. |
| Month three follow-up visit 84-97 days post-enrollment. 98-127 days post-enrollment. | | |

Version: 4.0, 18 December 2024



#### **SECTION 4. STATISTICAL PRINCIPLES**

#### **Confidence Intervals and P-values**

#### Level of Statistical Significance

All statistical tests will be two-sided using a 5% significance level (alpha of 0.05).

#### Type I Errors

We will not adjust the alpha for multiple testing in the primary or secondary aims. For secondary aims that involve multiple hypothesis tests, we will frame the results as exploratory and acknowledge type-I error in the limitations sections.

#### Confidence Intervals to be Reported

Two-sided 95% confidence intervals will be used. The specific calculation of confidence intervals is described under each specific aim.

#### **Protocol Deviations**

#### <u>Definition of protocol deviations</u>

The following are pre-defined major protocol deviations with a direct bearing on the primary outcome:

• Errors in applying inclusion/exclusion criteria that are discovered after enrollment, including lack of informed consent.

The following are pre-defined minor protocol deviations:

- Missed sample collection (stool/rectal swab, blood spot) due to participant refusal or other barrier to sample collection (such as visit occurring over phone).
- Missed anthropometry assessment due to follow-up visit occurring over the phone

#### Description of which protocol deviations will be summarized

Protocol deviations will be classified as major and minor. The number (and percentage) of participants with major and minor protocol deviations will be summarized by study site in relevant analyses with details of the deviation provided. No statistical tests will be performed.

#### **Analysis Populations**

All children with non-missing outcome data (for each relevant aim) will be included in primary and secondary analyses.

Missing data for symptom variables will be assumed as absence of a given symptom in primary analyses.

#### SECTION 5. STUDY POPULATIONS

#### **Diarrhea Case Surveillance Screening**

The total number pre-screened, screened, and enrolled in Diarrhea Case Surveillance (DCS) will be reported along with summary of reasons for exclusion into the study.

#### **DCS** Eligibility

Children aged 6 to 35 months old presenting at an EFGH facility with diarrhea (three or more abnormally loose or watery stools per 24 hours) (Table C).

**Table C.** Description of study population and criteria for the inclusion and exclusion of DCS enrollment.



| Study Population | Children aged 6 to 35 months old presenting at an EFGH facility with diarrhea (three |
|---|---|
| J 1 | or more abnormally loose or watery stools in the previous 24 hours). |
| Inclusion Criteria | <ul> <li>Primary caregiver and child plan to remain at their current residence for at least the next four months</li> <li>Primary caregiver is able to provide informed consent (legal age or emancipated minor) and provides consent within a common language for which translations are available</li> <li>Child resides within the pre-defined study area</li> <li>Fewer than four hours have passed since the child presented to a health facility</li> <li>Diarrhea episode is: <ul> <li>Acute (onset within seven days of study enrollment) and</li> <li>Represents a new episode (onset after at least two diarrhea-free days)</li> </ul> </li> <li>Caregiver is willing to have child participate in follow-up visits at week four and month three</li> <li>Willingness to have samples collected from the child (rectal swabs at enrollment)</li> <li>Site enrollment cap has not been met</li> </ul> |
| | Child is not being referred to a non-EFGH facility at the time of screening |
| Exclusion Criteria | <ul> <li>Children younger than six months or 36 months or older</li> <li>Diarrhea does not meet the study definition (three or more abnormally loose or watery stools in the previous 24 hours)</li> <li>Primary caregiver unable to provide informed consent or refuses to provide consent</li> <li>Primary caregiver refuses verbal consent to screening procedures</li> <li>Child does not reside in the study catchment area</li> <li>four or more hours have passed since child presented to the study facility</li> <li>Diarrhea episode is not acute (&gt;7 days) or does not represent a new episode (&lt;2 diarrhea free days)</li> <li>Caregiver unwilling to have child participate in follow-up at four weeks and three months</li> <li>Caregiver unwilling to have samples collected at enrolment (rectal swabs)</li> <li>Site enrolment cap has been met</li> <li>Child is being referred to a non-study facility</li> </ul> |

#### **Population Enumeration and HUS Eligibility**

All households residing in the study catchment area and where an adult household member provides verbal consent will be eligible to participate in population enumeration activities. Children who are (1) 6-35 months of age, (2) had diarrhea (three or more unusually loose or watery stools during a 24-hour period) in the past 14 days, and (3) whose primary caretakers provides written or verbal informed consent (per site procedures and institutional review board [IRB] requirements) will complete the HUS.

#### Recruitment

Children will be passively recruited from study outpatient facilities for DCS enrollment. Prior to the screening process, potential participants will be pre-screened for eligibility by the study staff.

Per CONSORT guidelines, we will report the number of individuals who (**Figure 1**):

- 1. Underwent pre-screening
- 2. Underwent screening



- 3. Did not undergo screening (and reasons)
- 4. Met inclusion criteria
- 5. Did not meet inclusion criteria (and reasons)
- 6. Enrolled in the study
- 7. Not enrolled in study (and reasons)
- 8. Completed week four and month three follow-up visits

#### Withdrawal/Follow-Up

#### Withdrawal

Withdrawal of consent will be tabulated by country site using the following categories: withdrawal but allow prior collected data/ samples to be used and withdrawal and disallow already collected data/samples to be utilize.

#### Missed Visits/Loss to follow-up

Week four visits (defined as study visits 24 to 67 days after enrollment) and month three visits (defined as study visits 84 to 127 days after enrollment) that were missed will be tabulated in categories of completely missed, visit occurred but outside of window, visit occurred over phone by country site. Lost to follow-up (LTFU) will be defined as missing both the week four and month three visit.

#### **SECTION 6. ANALYSIS**

#### **Definitions**

- 1. **Diarrhea** defined as three or more abnormally loose or watery stools in a 24-hour period.
- 2. **Diarrhea episode** will be defined as the period of days in which the above definition is met followed by two diarrhea-free days.
- 3. **Culture-confirmed** *Shigella* **diarrhea case** will be defined as a case of acute diarrhea presenting to an EFGH facility in which *Shigella* was isolated from either of the cultured fecal sample collected by rectal swab and transported in mBGS or Cary-Blair media.
- 4. **qPCR-confirmed** *Shigella* **diarrhea case** will be defined as a case of acute diarrhea presenting to an EFGH facility in which *Shigella* DNA was identified in the fecal sample by qPCR (cycle threshold [CT] <31.1 for rectal swab or CT<29.8 for whole stool) by the TaqMan Array Card (TAC) assay.
- 5. **Shigella attributed diarrhea case** will be defined as a case of acute diarrhea presenting to an EFGH facility in which *Shigella* was confirmed by either culture or qPCR (as outlined in #3 and #4 above).
- 6. **Dysentery** will be defined for DCS as a caregiver report of blood in the stool during the index diarrhea episode or a clinician diagnosis during the enrollment procedures and for the HUS as caregiver report of blood in the stool.
- 7. **Watery diarrhea** will be defined for DCS as the lack of caregiver report of blood in the stool during screening, enrollment and during the diarrhea episode, and no dysentery diagnosis by the clinician among enrolled participants in the DCS, and for the HUS as the lack of caregiver report of blood in the stool for children whose caregiver reported diarrhea in the previous 14 days.
- 8. **Severity of diarrhea** will be defined according to multiple definitions (dysentery/watery diarrhea, hospitalized diarrhea, modified Vesikari score [MVS], moderate or severe diarrhea by MVS or dysentery, the Global Enteric Multicenter Study [GEMS] moderate-to-severe diarrhea [MSD] or less-severe diarrhea [LSD], GEMS-*Shigella*, Clark or the Malnutrition and Enteric Disease Study [MAL-ED] for incidence rate and consequence comparisons.



- 9. **Deaths** occurring within the three-month follow-up period will be assessed by caregiver report at each scheduled visit or during upcoming visit phone reminders. Date and cause of death will be obtained from caregiver history, hospital records or death certificate, when available. The death certificate will be considered the gold standard for date of death. If a child died in the three-month period, but this information was not known until up to five months (two months beyond scheduled three-month visit), this will be included as death. Deaths occurring outside of the three-month window will not be included. Causes of death will be determined by a panel of International Classification of Diseases 11<sup>th</sup> revision (ICD-11) trained clinicians using information from the child's death certificate (if available), caregiver interview (if available), and case notes from the child's care team.
- 10. **Hospitalization** will be assessed at the week four and month three visits by caregiver recall and hospital records (gold standard) when available. Date and time of admission, length of hospital stay, presenting signs/symptoms, and treatment received will be obtained. Hospitalizations that are a continuation of management from a previous hospitalization (such as referrals) will be excluded from the analysis. For the purpose of standardization across sites, hospitalization will be defined as an overnight stay (child was on the ward from at least 12am to 6am or self-discharged prior to that timeframe).
- 11. **Loss to follow-up (LTFU)** will be defined as not having attended both the week four and month three follow-up visits after two months of actively tracing the child.
- 12. **Linear growth** will be defined as the change in mean length/height-for-age Z-score (ΔLAZ/ΔHAZ) from enrollment to three months. The 2006 World Health Organization (WHO) reference population will be used to calculate HAZ from the average of two repeated length/height (cm) measures per child per time point.
- 13. **Duration of diarrhea/dysentery/vomiting/fever** will be determined as the number of days a child has the symptoms within an episode of diarrhea. Because an episode is defined by two diarrhea-free days, the duration of each symptom may differ from the duration of the diarrhea episode (for example if there is one diarrhea free day within an episode). Notably this is distinct from the duration of the episode.
- 14. **Duration of diarrhea episode** will be defined as the number of days between when the caregiver reported the child's diarrhea starting and the last day of diarrhea prior to the two consecutive diarrhea-free days concluding the episode.
- 15. **Prolonged diarrhea** will be defined as seven or more days of diarrhea within the index diarrhea episode beginning from diarrhea onset.
- 16. **Persistent diarrhea** will be defined as 14 or more days of diarrhea within the index diarrhea episode beginning from diarrhea onset.
- 17. **Chronic diarrhea** will be defined as 30 or more days of diarrhea within the index diarrhea episode beginning from diarrhea onset.
- 18. **Extended case fatality** will be calculated as the proportion of enrolled participants that experience a mortality event from any cause during the three months of EFGH follow-up.
- 19. **Stunting** will be defined as a length-for-age Z-score (LAZ, children <24 months of age) or height-forage Z-score (HAZ, children ≥24 months of age) <-2.
- 20. **A subsequent diarrhea/dysentery episode** will be defined as new diarrhea/dysentery episodes (>48 hours after a diarrhea-free period).
- 21. **Cost per episode treated** will be calculated using the direct and indirect costs of *Shigella*-associated MAD per outpatient and inpatient episode, from the household, health system, and societal perspectives.



22. Antibiotic resistance will be based on zone size (from disc diffusion) values for each tested antibiotic and categorized as susceptible, intermediate, or resistant according to the most recent Clinical and Laboratory Standards Institute (CLSI) interpretive standards at the time of data analysis. Resistant and intermediate categories will be collapsed into a non-susceptible category to create a dichotomous variable. Multidrug-resistant (MDR) will be defined as resistance to at least three of the following medications: Ampicillin, Azithromycin, Ceftriaxone, Ciprofloxacin, Nalidixic Acid, Pivemicellinam, and Trimethroprim-Sulfamethoxazole. Extensively drug-resistant (XDR) will be defined as resistance to Ampicillin, Azithromycin, Ciprofloxacin, Ceftriaxone and Trimethoprim-Sulfamethoxazole. Resistance to all WHO recommended treatments will be defined as resistance to Azithromycin, Ciprofloxacin and Ceftriaxone.

#### **Analysis Methods**

#### **Statistical Analysis**

- **1. Primary Aim.** *To determine the incidence of* Shigella-attributed diarrhea in children 6 to 35 months of age in each of the EFGH country sites.
  - a. <u>Statistical Analysis:</u> The adjusted incidence of *Shigella* will be calculated as the sum of total confirmed *Shigella* diarrhea cases divided by the child-years at risk of children 6-35 months of age in the defined catchment area, adjusting for healthcare-seeking behavior and children who were eligible but not enrolled (*w*<sub>n</sub>). Crude incidence rates as well as incidence rates adjusted for enrollment but not care-seeking will also be presented. Analyses will be conducted separately using both culture-confirmed *Shigella* and attributable *Shigella* by molecular methods (TAC). All incidence rates will first be calculated using the number of *Shigella* cases and defined population size at the facility level, adjusted for the facility-specific enrollment adjustment, summed to determine the total enrollment-adjusted incidence rate, and then adjusted for care-seeking to determine the final adjusted incidence (**Table 3**). Pooled incidence across all country sites will be computed by taking the population-weighted average incidence using the estimated population in the catchment area.

Child-years at risk to *Shigella* is determined by the defined population size and the facility-specific period of follow-up ( $days_j/365.25$ ; approximately two years). The first is the estimated number of children 6-35 months of age in the catchment area which will be determined by totaling the number of children in this age range enumerated during population enumeration activities and extrapolating this estimate to study clusters not visited and households that were not reached ( $w_d$ ).

Among children 6-35 months of age who had diarrhea in the past 14 days and whose caregiver consented the HUS, the healthcare seeking adjustment,  $w_{\rm HC}$  is defined as the proportion of children with a similar syndrome who sought care for diarrhea at an EFGH-facility. The healthcare seeking adjustment will be estimated for each enrolled case using the estimated coefficients from a 'propensity to seek care' weighting model fit to data from children reporting diarrhea in the previous two weeks in the HUS. The propensity score model will be a multivariate logistic regression model where the outcome is report of healthcare seeking at a primary healthcare facility and predictors will include variables hypothesized to have an association with healthcare seeking and that are captured in both diarrhea case surveillance in the HUS (EFGH country site, age, sex, days with fever, days with vomiting, maximum number of vomiting episodes in one day, maximum number of stools in one day, blood in stool, and wealth quintile).. The propensity to seek care model in the HUS will use any care-seeking at a primary healthcare facility and will then be



adjusted for the site-specific difference in overall care-seeking and care-seeking to EFGH facilities ( $w_{HC at EFGH}$ ).

In sensitivity analyses, we will restrict the weighting model to cases of diarrhea from the HUS within the past seven days instead of 14 days as seven-day recall is likely less biased than 14-day recall (although will inevitably be less precise because of fewer episodes included). Because children who have more severe diarrhea are more likely to seek care, we expect to upweight diarrhea cases enrolled with less severe diarrhea more heavily than diarrhea cases enrolled with more severe diarrhea.



Cases with Shigella who enrolled in EFGH

Cases with Shigella who sought care at EFGH who sought care at EFGH facility

Which at EFGH = 
$$1/\%$$
 sought care at EFGH facility

Which at EFGH =  $1/\%$  sought care at EFGH proposity score which sold who sought care at EFGH

Which at EFGH =  $1/\%$  sought care at EFGH proposity score which sold which

The enrollment adjustment will be episode and facility-specific based on DCS enrollment procedures. Specifically, it will be computed separately for dysentery and watery diarrhea (defined as caregiver report of blood in the stool during screening) and for each facility. The enrollment adjustment is defined as the percentage of children who were enrolled among the estimated number of children six to 35 months of age living in the catchment area who met the study definition of diarrhea and therefore would have been eligible for



study participation but screened out due to lack of consent, no longer being at the facility, or other administrative reasons (i.e. presented overnight or during a weekend when EFGH screening did not occur). This adjustment is split into two parts: prescreening ( $w_{\text{screen}}$ ) and screening  $(w_{\text{enroll}})$ . The screening adjustment determines the percentage enrolled of those who were theoretically eligible (6-35 months, living in catchment area, and met diarrhea definition) to account for children who were not enrolled due to caregiver refusal or withdrawal of consent, limited staff of clinic capacity, the respondent not planning to remain in the study area four months, the child being enrolled in another interventional study, more than four hours having passed since the child began screening procedures, the child being referred to a non-EFGH facility or the child not being enrolled due to the enrollment cap. The prescreening adjustment determines the percentage of children 6-35 months of age whose caregiver or clinical records indicated they presented with diarrhea, dysentery or gastroenteritis and who were not already enrolled in EFGH who were screened to account for children who did not get screened due to verbal refusal by the caregiver or the child not being present in the facility. Because it is unknowable whether or not these children would have been eligible had they undergone full screening, we will apply the observed eligibility proportion from screening to those pre-screened. The final enrollment adjustment is taken by multiplying the screening and prescreening adjustments. Summaries of the calculation of denominators and adjustments will be presented in supplementary tables.

<u>Confidence intervals</u> around the primary aim of adjusted incidence of *Shigella* (as well as secondary aims presenting stratified *Shigella* incidence by age, serogroup, serotype, disease severity and seasonality) will be generated using boot strapping.

#### b. Sensitivity analyses:

- i. We will restrict the care seeking adjustment to cases of diarrhea within the past seven days instead of 14 days as seven-day recall is likely less biased than 14-day recall (although will inevitably be less precise because of fewer episodes included).
- ii. As the enrollment adjustment does not consider, as potentially eligible, children who are currently enrolled in EFGH and in the three-month follow-up period, we will estimate the potential impact of this exclusion on the diarrhea incidence by estimating, through follow-up visit and unscheduled visit questionnaires, the proportion of enrolled cases who presented to EFGH facilities with diarrhea who would otherwise meet the EFGH eligibility criteria. We will estimate incidence rates that include these subsequent diarrhea episodes to estimate the upper bound of incidence rates (such as might be observed in a prospective cohort study).
- iii. Attributable *Shigella* by TAC will be defined as a rectal swab ipaH CT<31.1, however a sensitivity analysis using a cutoff of CT<30.0 will be conducted.

#### Statistical Analysis of Secondary Aims

- 1. **Secondary Aim #1:** Determine the incidence of *Shigella* by serotype, severity definition, laboratory method (culture vs. qPCR), age, and by season.
  - a. <u>Statistical Analysis:</u> Enrollment- and healthcare seeking-adjusted <u>Shigella</u> incidence following the protocol incidence calculation as measured by culture and qPCR will be stratified by the following factors:
    - i. Serogroup and Serotype (Table 1.1, Figure 1.1):
      - 1. Shigella species (S. boydii, S. dysenteriae, S. flexneri, S. sonnei or undetermined), S. flexneri serotype (1a, 1b, 1d, 2a, 2b, 3a, 3b, 4a, 4b, 5a,



- 5b, 6, 7a, X, Y, non-typable and other), *S. dysenterarie* serotype (1 or non-type 1) and combined bivalent and quadrivalent vaccine target indicators (defined as *Shigella* positive for *S. flexneri* 2a or *S. sonnei*, and *S. flexneri* 2a, 3a or 6 or *S. sonnei*, respectively).
- 2. The denominator for this sub-analysis will be the overall denominator for the primary endpoint.
- 3. Serotype distribution will be visualized graphically either as pie charts or as a map with country-level pie-charts (**Figure 1**, not shown).

#### ii. Age (Table 1.2):

- 1. Stratified by age at enrollment visit (6-8 months, 9-11 months, 12-17 months, 18-23 months or 24-35 months).
- 2. The denominator for this sub-analysis will be the estimated child-years at risk in the catchment area for each age stratification.
- iii. **Diarrhea severity definition:** *Shigella* incidence will be stratified by the following diarrhea severity definitions (**Table 1.2**):
  - 1. **Dysentery vs. watery diarrhea** will be defined according to whether or not dysentery was present during the diarrheal episode.
  - 2. **Hospitalized diarrhea** defined as the child being admitted to hospital (overnight stay) during the diarrheal episode.
  - 3. Modified Vesikari Score (MVS) defined as in PATH Vesikari Clinical Severity Scoring System Manual<sup>4</sup>: Duration of diarrhea: 1-4 days (1 point), 5 days (2 points)  $\geq$ 6 days (3 points); Max # of stool in 24 hour period: 1-3 (1 point), 4-5 (2 points), ≥6 (3 points); Duration of vomiting: 1 day (1 point), 2 days (2 points),  $\geq$ 3 days (3 points); max # of vomiting episodes in 24 hour period: 1 (1 point), 2-4 (2 points), >5 (3 points); Axillary temperature 36.6-37.9°C (1 point), 38.0-38.4°C (2 points), ≥38.5°C (3 points); dehydration defined using WHO dehydration categories of some and severe as per Integrated Management of Childhood Illness<sup>5</sup> (IMCI) guidelines, some dehydration (2 points), severe dehydration (3 points); treatment: rehydration (1 point), hospitalization (2 points). The scores will be summed and categorized as severe illness (11+ points), moderate illness (9-10 points), mild illness (0-8 points). If pre- or post-rehydration weights are not known to calculate % dehydration, WHO dehydration categories of some and severe as per IMCI guidelines will be used.
  - 4. **Moderate or severe diarrhea by MVS or dysentery** will be defined as a MVS of 9+ points or presence of visible blood in stool (Pavlinac, Vaccines, 2022).<sup>6</sup> Secondary analyses will use a more stringent cut-off of 11 points and a less stringent cut-off of seven points.
  - 5. GEMS MSD and LSD will be defined as in Kotloff, Lancet GH, 2019.<sup>7</sup> Moderate-to-severe diarrhea (MSD) defined as presenting to a health facility with diarrhea and severe or some dehydration (by WHO criteria), visible blood in stool, or inpatient admission. Less-severe-diarrhea (LSD) defined as presenting to a health facility without MSD.
  - 6. **GEMS-Shigella** will be defined as in Pavlinac, CID, 2021.<sup>8</sup> Duration of diarrhea 1-3 days (0 points), 4-5 days (2 points), ≥6 days (3 points); WHO-defined dehydration categories: severe (8 points), some (4 points), none (0 points); inpatient admission (5 points). The scores will be summed and categorized as mild (<6 points), moderate (6-8 points), and severe (9+ points).



- 7. **Clark score** will be defined as in Clark, JID, 1988.<sup>9</sup> Duration of diarrhea: 1-4 days (1 point), 5-7 days (2 points), >7 days (3 points); Max # of stool in 24 hour period: 2-4 (1 point), 5-7 (2 points), >7 (3 points); Duration of vomiting: 2 days (1 point), 3-5 days (2 points), >5 days (3 points); max # of vomiting episodes in 24 hour period: 1-3 (1 point), 4-6 (2 points), >6 (3 points); Duration of reported fever: 1-2 days (1 point), 3-4 days (2 points), ≥5 days (3 points); Rectal temperature 38-38.2°C (1 point), 38.3-38.7°C (2 points), ≥38.8°C (3 points); behavioral signs: Irritable/less playful (1 point), Lethargic/listless (2 points), Seizures (3 points). The scores will be summed and categorized as mild (2-8 points), moderate to severe (9+ points).
- 8. **MAL-ED score** will be defined as in Lee, J Pediatr Gastroenterol Nutr., 2016<sup>10-11</sup> Duration of diarrhea: 2-4 days (1 point), 5-7 days (2 points), ≥8 days (3 points); Max # of stool in 24 hour period: <5 loose stools/24 hours (1 point), 5-7 loose stools/24 hours (2 points), ≥8 stools/24 hours (3 points); Duration of vomiting: 1 day (1 point), 2 days (2 points), ≥3 days (3 points); duration of reported fever: 1+ days (1 point); Confirmed temperature: ≥37.5°C (confirmed by field worker) (2 points); Dehydration: Some (2 points), severe (3 points). The scores will be summed and categorized as non-severe (<6 points) or severe (6+ points)
- 9. The denominator for each subgroup of this sub-analysis will be the overall child-years at risk of *Shigella* in the catchment area (same as the primary analysis).

#### iv. Diarrhea season:

- 1. Seasonality will be presented graphically (**Figure 1.2** [not shown]) as monthly or quarterly incidence.
- 2. The denominator for this sub-analysis will be the estimated child-years at risk in the catchment area for each study month or quarter.
- b. The adjusted incidence rate and 95% confidence interval will be reported for each stratification both overall and by country.
- c. To describe the prevalence *Shigella* and other important enteric pathogens (see below) among participants enrolled in EFGH, the proportion of participant samples testing positive for each pathogen will be calculated among participants who had a stool sample tested by TAC:
  - i. Pathogens tested and attributable CT thresholds:
    - 1. *Shigella* (CT<31.1)
    - 2. Adenovirus 40/41 (CT<25.5)
    - 3. *Cryptosporidium* (CT<27.1)
    - 4. Norovirus GII (CT<26.6)
    - 5. Rotavirus (CT<34.2)
    - 6. Heat stabile toxin-producing *E. coli* (ST-ETEC, CT<27.9)
    - 7. Typical enteropathogenic *E. coli* (tEPEC, CT<20.7)
    - 8. *Campylobacter jejuni* (CT<20.7)
    - 9. Astrovirus (CT<26.7)
    - 10. Sapovirus (CT<24.4)
    - 11. Vibrio cholerae (CT<33.9)
    - 12. Salmonella (CT<33.3)
    - 13. *Aeromonas* (CT<23.6)
    - 14. Cyclospora cayetanensis (CT<33.9)
    - 15. Entamoeba histolytica (CT<32.6)
    - 16. *Cystoisospora belli* (CT<34.4)



- ii. Prevalences will be calculated for all participants with MAD and among the following subsets:
  - 1. Among participants presenting with moderate or severe diarrhea (by the Modified Vesikari Score 9+) and/or dysentery.
  - 2. Among participants who tested positive for *Shigella*-attributable MAD (among non-*Shigella* pathogens).
  - 3. Among participants who did not test positive for *Shigella*-attributable MAD (among non-*Shigella* pathogens).



- 2. **Secondary Aim** #2: Describe the prevalence of resistance to commonly used antibiotics in Shigella isolates in each EFGH country site.
  - a. <u>Statistical Analysis:</u> The proportion of *Shigella* culture positive stool samples that are resistant to the medications listed below will be calculated by EFGH region and EFGH study site (**Table 2.1**, **Figure 2.1** [not shown]):
    - Ampicillin
    - Azithromycin
    - Ceftriaxone
    - Ciprofloxacin
    - Nalidixic acid
    - Pivemicellinam
    - Trimethoprim-sulfamethoxazole

Resistance will be defined as "non-susceptibility", or resistant or intermediate zone size classifications according to the most recent CLSI guidelines at the time of analysis. Resistance will be computed for all of the above antibiotics for all sites, by region (South America [Peru], West Africa [The Gambia and Mali], East Africa [Kenya and Malawi], and Asia [Pakistan and Bangladesh]), and among *S. sonnei* positive samples and *S. flexneri* positive samples. Additionally, we will present the percentage of multi-drug resistant *Shigella* (MDR, resistant to three or more antibiotics), extensively drug resistant *Shigella* (XDR, resistant to all of the following: Azithromycin, Ciprofloxacin, Ceftriaxone, Trimethoprim-sulfamethoxazole, and Ampicillin), and resistance to all WHO recommended treatments (resistant to all of the following: Azithromycin, Ciprofloxacin, and Ceftriaxone).

b. <u>Confidence intervals</u> around non-susceptibility proportions will be determined assuming a binomial distribution.



3. **Secondary Aim #3:** Determine the risk of all-cause mortality, hospitalization, persistent diarrhea, experiencing a subsequent diarrhea episode, and change in linear growth in the three months following an episode of MAD.

#### a. Statistical Analysis:

Deaths will be described individually in terms of *Shigella* attribution and overall (**Table 3.1**). Extended all-cause case fatality including ICD-11 cause, age, enrollment site, time from enrollment to death, and *Shigella* attribution will be described (**Table 3.2**). A Fisher's exact test will be used to test whether the proportion of children who died differed between those with and without *Shigella* at enrollment. The cumulative incidence of all-cause mortality will be plotted using the Kaplan-Meier survival function, both overall and stratified by *Shigella*-attribution (**Figure 3.1** [not shown]). Participants will be censored at date of death, last known alive date, or latest follow-up date. Models will not be adjusted because of the anticipated small number of outcomes.

The risk of hospitalization, risk of experiencing subsequent diarrhea episodes, and prevalence of persistent diarrhea will be described by leading attributable cause of the index MAD episode. Shigella will either be split into Shigella with appropriate antibiotic treatment and Shigella without appropriate antibiotic treatment or treated as a mediator and addressed using a formal mediation analysis (Table 3.3). The relative risks comparing subsequent diarrhea episodes and hospitalizations among children stratified by the likely etiology of diarrhea at enrollment will be determined using a modified-Poisson model with robust standard errors using a dichotomized outcome (did the outcome occur during follow-up or not) and Wald chi-square tests of the two-way comparison. The proportion of children with persistent diarrhea will be compared overall and by the likely etiology of diarrhea at enrollment, using log-binomial regression (or modified-Poisson regression with robust standard errors if any model does not converge). All multivariate models will adjust for site, age, maternal education, wealth quintile, and breastfeeding. For all outcomes of interest, we will test for effect modification between attribution of any bacterial targets and appropriate antibiotic use, and if no evidence is observed (p>0.05) that target will be combined into a single category regardless of antibiotic treatment. In this primary analysis, hospitalizations occurring at any point between enrollment and follow-up will be included.

Hospitalizations that occur during the index diarrhea episode will be disaggregated from those occurring after the index diarrhea episode has resolved to separately estimate enteric pathogen associations with short- and longer-term severe illnesses (**Table 3.4**). A supplementary analysis will additionally include stratification of risk of subsequent diarrhea by whether or not the subsequent diarrhea episodes were medically-attended. Finally, a supplementary analysis will compare the risk of hospitalization, risk of subsequent diarrhea, and prevalence of persistent diarrhea among children with *Shigella*, by culture-positive *Shigella* vs. culture-negative/TAC-attributable *Shigella*. Multivariate supplementary tables described here will be adjusted for site, age, maternal education, wealth quintile, and breastfeeding.

The distribution of LAZ/HAZ at enrollment, week four, and month three will be presented as boxplots stratified by likely etiology at enrollment of the top five most prevalent attributable enteric pathogens by qPCR (**Figure 3.2** [not shown]). Supplemental tables will display these values stratified by site.



The mean and standard deviation of LAZ/HAZ from enrollment to week four follow-up and enrollment to month three follow-up will be presented among surviving children by likely etiology at enrollment of the top five most prevalent attributable enteric pathogens by qPCR, including *Shigella* stratified by receiving appropriate antibiotics and untreated. Other bacterial pathogens will be similarly stratified by antibiotic use if there is evidence of effect modification (p<0.05) (Table 3.5). Two sets of linear regression models, one modelling enrollment to week four and another from enrollment to month three, will be used to model the association between likely MAD etiology and linear growth (\Delta LAZ/HAZ) in the months following the diarrhea episode among surviving children. Models will include adjustment for site, age, sex, maternal education, wealth quintile, breastfeeding, days from enrollment to relevant follow-up visit and baseline LAZ/HAZ. Lowess curves will be generated to show mean  $\Delta LAZ/HAZ$  between the timepoints (enrollment, week four, and month three) by likely MAD etiology at enrollment (Figure 3.3 [not shown]). We will report prevalence of stunting (LAZ/HAZ<-2) at enrollment, week four follow up, and month three follow up by likely etiology of MAD at enrollment, including Shigella stratified by receiving appropriate antibiotics and untreated. Other bacterial pathogens will be similarly stratified by antibiotic use if there is evidence of effect modification (p<0.05). Prevalence ratios (PR) adjusted for site, age, sex, maternal education, wealth quintile, breastfeeding, and baseline LAZ/HAZ will be generated to describe the association between diarrhea etiology and stunting (Table 3.6). An alluvial plot will be generated to show the proportion of stunted and non-stunted at enrollment, week four follow up, and month three follow up and transition of stunting status between study visits (Figure 3.4 [not shown]). Supplementary tables will report both LAZ/HAZ and stunting analyses stratified by site, by Shigella species (S. flexneri, S. sonnei, S. boydii, dysenteriae), and by diagnostic method (culture positive vs. culture negative/TACattributable). For all analyses utilizing LAZ/HAZ data, individual LAZ/HAZ greater than 6.0 or less than -6.0 will be excluded as implausible values. 12 Also excluded will be any height decrease of greater than 1.5cm or height increase of greater than 6cm between enrollment and month three follow-up. 13



4. **Secondary Aim** #4: Compare various severity definitions in their ability to predict risk of death/hospitalization or linear growth faltering among cases of medically attended diarrhea and Shigella-attributable medically attended diarrhea, respectively.

Based on signs and symptoms collected from EFGH cases, we will construct diarrhea severity definitions as described above in Secondary Aim 1. Scores will be categorized as originally constructed (i.e. mild, moderate, and severe). We will describe the mean scores and frequencies/percentages of children falling in all severity definition categories both overall, and among children with *Shigella*-attributed diarrhea by site and overall (**Table 4.1**). In supplementary tables, we will report further stratification by age at enrollment and laboratory method (for *Shigella*-attributable MAD only).

As GEMS and MVS +/- dysentery are severity scores of particular interest for informing *Shigella* vaccine trial clinical endpoints, we will compare the components and symptoms that make up these scores with and without the combination of meeting the GEMS definition of MSD and moderate or severe diarrhea (9+ points) by the MVS +/- dysentery among children with *Shigella*-attributed diarrhea (**Table 4.2**). In supplementary tables, we will present this table further stratified by culture positivity.

To evaluate the scores' associations with poor outcomes, we will dichotomize scores into moderate or severe vs. mild diarrhea (for GEMS-Shigella, MVS, Clark and MVS +/- dysentery), severe vs. mild diarrhea (for MAL-ED) or MSD vs. less-severe-diarrhea (LSD) (for GEMS). We will calculate the diagnostic accuracy (sensitivity, specificity, positive predictive value [PPV], and negative predictive value [NPV]) of severe vs. non-severe diarrhea (by each severity score definition) in identifying children who die or were hospitalized during the initial episode (**Table 4.3**). Diagnostic accuracy will be reported overall and stratified by appropriate antibiotic treatment. As part of secondary analysis, we will look at all hospitalizations and deaths occurring throughout the three-month follow-up. We will report the performance of scores for all MAD as well as in the subset of children with Shigella-attributed diarrhea. Primary analyses will consider death or hospitalization as a combined outcome, and secondary analyses will report these outcomes separately. We will additionally explore varying cut-offs used for score-based severity definitions by conducting Receiver Operating Characteristics (ROC) analyses to identify cut-points that maximally distinguish those children who had experienced a death or hospitalization from those that did not (**Figure 4.1**).

We will also evaluate scores' association with linear growth. We will perform a linear regression of each dichotomized score on the change in length-for-age or height-for-age z-score (ΔLAZ/HAZ) from baseline to month three, adjusting for baseline LAZ/HAZ (**Table 4.4**). We will use generalized estimating equations to account for multiple enrollments of the same child. We will report model results among all MAD as well as children with *Shigella*-attributed diarrhea, and results will be further stratified by antibiotic use or with antibiotic use treated as a mediator. We will compare the magnitude of association (beta values) between scores.

Because other EFGH analysis (biomarker sub-study) will evaluate the combination of signs/symptoms and inflammatory biomarkers in their ability to distinguish *Shigella* from non-*Shigella*-attributed diarrhea, we will not address that question in this aim.



5. **Secondary Aim #5**: Quantify the cost incurred by families and health care systems due to Shigella morbidity and mortality.

For each child enrolled in the study, we will collect data on medical and non-medical resources used to treat the episode of diarrhea, using child medical records and standardized questionnaires administered to caregivers. Direct medical costs include medical resources used in the treatment of diarrhea. We will estimate the costs of drugs and diagnostics used in diarrhea management, by applying a standardized country-specific unit cost from National Price Lists to each treatment administered or prescribed in medical records. In situations where data is missing from National Price Lists, we will estimate unit costs using a mean value from local pharmacies and health facilities. We will also estimate service delivery costs: operational costs for medical visits, such as health workers' salaries or maintenance of facility equipment. To estimate these costs, we will apply standardized country-specific unit costs from WHO-CHOICE<sup>14</sup> to each visit based on the level of care (inpatient vs. outpatient) and number of days admitted (inpatient only). Standardized questionnaires include questions regarding whether medical resources were paid for by the caregiver or funded by the public health system. Direct non-medical costs include non-medical fees incurred by caregivers, such as costs to travel to the health facility. We will estimate non-medical fees through caregiver direct reports from standardized questionnaires. Indirect (non-medical) costs include caregiver time lost from work while caring for their sick child. To estimate indirect costs, we will apply a national average wage rate from the International Labor Organization (https://www.ilo.org) to caregiverreported time lost from work from standardized questionnaires.

We will estimate the <u>average cost per episode of Shigella-attributable MAD</u>, referred to henceforth as the "cost per episode", by averaging costs across *Shigella-*positive cases, including cases of culture-confirmed *Shigella* and/or *Shigella* confirmed by molecular methods (TAC). We will present the mean and standard deviation (SD) of costs per episode, from the household perspective (including out-of-pocket medical and non-medical fees incurred by caregivers), the health system perspective (medical resources funded by the public health system), and the societal perspective (both household and health system costs). We will stratify societal costs by client and visit characteristics, as described in **Table 5.1**. Costs will be presented in 2024 US dollars (USD) to allow for comparability across sites. We will inflate costs incurred in earlier years to 2024 values using GDP price deflators from the World Bank and convert local currencies to equivalent USD values using midyear currency values. Additional sub-analyses will be conducted to determine costs per episode of MAD associated with *Shigella* serotypes, other diarrheal pathogens, and other stratifications as relevant.

To identify the effects of visit characteristics on costs per episode of *Shigella* MAD, we will use multivariate Generalized Linear Models (GLMs). GLMs require explicit specification of the distribution of the dependent variable and the link function describing how independent variables are functionally related to the dependent variable. We will use the modified Park test<sup>14</sup>, common to health econometrics, to identify the GLM distribution and link function. Our final model will be determined from the modified Park test results but will be initially tested using a gamma distribution with log link<sup>15</sup>:

$$\ln (Y_i) = \beta_0 + \beta_1 Country_i + \beta_2 Severity_i + \beta_3 X_i$$

where the cost per episode (*Y*) for a given child, *i*, is a function of the country in which the child was treated (*Country*), the severity of diarrhea (*Severity*), and other client or visit characteristics (*X*). Other client or visit characteristics will be selected based on descriptive results from Table 5.1, with model variables being selected when variability across categories is evident. Models will be run separately per costing perspective. Coefficients, confidence intervals, and p-values will be presented for all independent variables (**Table 5.2**).

We will estimate the annual economic burden of Shigella MAD in each EFGH country site (c). The



estimated adjusted incidence of *Shigella* MAD (from the primary aim) and the estimated population sizes of children 6-35 months (converted to person-years) will be used to estimate the number of annual *Shigella* MAD episodes per country site. We will then apply the average cost per episode of *Shigella* MAD to the number of estimated episodes per year. The annual economic burden will be calculated separately per costing perspective (**Table 5.3**). We will produce estimates per site, standardized to 100,000 population size to allow for comparability across catchment areas.

$$\text{Annual } \textit{Shigella} \; \text{MAD } \text{costs}_c = \frac{\textit{Shigella} \; \text{MAD episodes}_c}{100 \; \text{person years}} \times \; \text{person years}_c \; \times \; \text{cost per episode}_c$$



- 6. **Secondary Aim #6**: To identify optimal laboratory methods for Shigella culture by:
  - a. comparing the isolation rate of Shigella between two transport media for rectal swabs (Cary-Blair and mBGS)

We will calculate the proportion of rectal swab samples from Cary-Blair and mBGS media from which *Shigella* was isolated overall and per site as well as stratified by serotype (**Table 6.1**). A two-sided 95% confidence interval around each proportion will be calculated assuming a Binomial distribution. Proportions will be compared using a McNemar's test of superiority to determine if one media is superior to the other in terms of *Shigella* isolation rates.

b. comparing the isolation rate of Shigella between two fecal sample types (rectal swabs and whole stool) among the subset of children who produced whole stool in the Gambia and Bangladesh country sites.

We will calculate the proportion of <u>rectal swab</u> samples from which *Shigella* was isolated and the proportion of <u>whole stool</u> samples from which *Shigella* was isolated, matched by media type (Cary-Blair or mBGS), overall and per site and stratified by *Shigella* species (**Table 6.2**). A two-sided 95% confidence interval for the absolute difference in proportions will be calculated using McNemar's test. When assessing non-inferiority, the lower bound of the 95% confidence interval will be compared to the non-inferiority margin of an absolute difference of 0.01.



#### Statistical Software

All analyses will be conducted using STATA or R and the software used reported in all analysis write-ups.

#### References

#### References to be Provided for Non-standard Statistical Methods

All methods being proposed are standard.

#### Data Management Plan

Procedures relating to data entry, management, and quality assurance and control are outlined in the EFGH Data Management Plan.

#### Statistical Master File

The Statistical Master File is maintained by the EFGH Central Data Management Team.

#### Referenced Literature

- 1. Rogawski McQuade ET, Shaheen F, Kabir F, et al. Epidemiology of *Shigella* infections and diarrhea in the first two years of life using culture-independent diagnostics in 8 low-resource settings. *PLoS Negl Trop Dis* 2020; **14**(8): e0008536.
- 2. Nasrin D, Blackwelder WC, Sommerfelt H, et al. Pathogens associated with linear growth faltering in children with diarrhea and impact of antibiotic treatment: The Global Enteric Multicenter Study. *J Infect Dis* 2021.
- 3. Anderson JD, Bagamian KH, Muhib F, et al. Burden of enterotoxigenic *Escherichia coli* and shigella non-fatal diarrhoeal infections in 79 low-income and lower middle-income countries: a modelling analysis. *Lancet Glob Health* 2019; **7**(3): e321-e30.
- 4. PATH. Vesikari Clinical Severity Scoring System Manual, 2011.
- 5. Integrated management of childhood illness: conclusions. WHO Division of Child Health and Development. *Bull World Health Organ* 1997; **75 Suppl 1**: 119-28.
- 6. Pavlinac PB, Rogawski McQuade ET, Platts-Mills JA, et al. Pivotal *Shigella* Vaccine Efficacy Trials-Study Design Considerations from a Shigella Vaccine Trial Design Working Group. *Vaccines (Basel)* 2022; **10**(4).
- 7. Kotloff KL, Nasrin D, Blackwelder WC, et al. The incidence, aetiology, and adverse clinical consequences of less severe diarrhoeal episodes among infants and children residing in low-income and middle-income countries: a 12-month case-control study as a follow-on to the Global Enteric Multicenter Study (GEMS). *Lancet Glob Health* 2019; 7(5): e568-e84.
- 8. Pavlinac PB, Platts-Mills JA, Tickell KD, et al. The Clinical Presentation of Culture-positive and Culture-negative, Quantitative Polymerase Chain Reaction (qPCR)-Attributable Shigellosis in the Global Enteric Multicenter Study and Derivation of a Shigella Severity Score: Implications for Pediatric Shigella Vaccine Trials. *Clin Infect Dis* 2021; **73**(3): e569-e79.
- 9. Clark HF, Borian FE, Bell LM, Modesto K, Gouvea V, Plotkin SA. Protective effect of WC3 vaccine against rotavirus diarrhea in infants during a predominantly serotype 1 rotavirus season. *J Infect Dis* 1988; **158**(3): 570-87.
- 10. Lee GO, Richard SA, Kang G, et al. A Comparison of Diarrheal Severity Scores in the MAL-ED Multisite Community-Based Cohort Study. *J Pediatr Gastroenterol Nutr* 2016; **63**(5): 466-73.



### Enterics for Global Health (EFGH) Statistical Analysis Plan – Tables and Figures Version 4.0





#### **Table of Contents**

| Primary AimPrimary Aim | 3 |
|---|---|
| Figure 1: Diarrhea case surveillance participant screening, enrollment and follow-up. | 3 |
| Table 1: Baseline participant characteristics | 4 |
| Table 2: Baseline characteristics of population enumeration | |
| Table 3: Shigella Incidence by country and method of ascertainment | |
| Secondary Aim 1 | |
| Table 1.1: Shigella incidence by species and serotype | 8 |
| Table 1.2: Shigella incidence by age and diarrhea severity | 9 |
| Table 1.3: Shigella incidence by severity | 10 |
| Table 1.4: Prevalence of enteric pathogens detected by molecular diagnostics. | 11 |
| Secondary Aim 2 | 12 |
| Table 2.1: Country and region antibiotic-non-susceptibility | 12 |
| Secondary Aim 3 | 13 |
| Table 3.1: All-cause case fatality | 13 |
| Table 3.2: Causes of death | 13 |
| Table 3.3: Hospitalization, subsequent diarrhea episodes, and persistent diarrhea | 14 |
| Table 3.4: Risk of hospitalization stratified by during index episode and after index episode | 15 |
| Table 3.5: Mean change in LAZ/HAZ | 16 |
| Table 3.6: Prevalence of stunting | 17 |
| Secondary Aim 4 | |
| Table 4.1: Moderate to Severe MAD by site | 18 |
| Table 4.2: Clinical characteristics of moderate-to-severe MAD | 19 |
| Table 4.3: Diagnostic accuracy of severity scores | 20 |
| Table 4.4: Severity scores and relationship to change in LAZ/HAZ | 21 |
| Figure 4.1: ROC curves for severity scores | 22 |
| Secondary Aim 5 | 23 |
| Table 5.1: Cost per episode of MAD | 23 |
| Table 5.2: Factors associated with cost | 24 |
| Table 5.3: Annual costs of Shigella-associated MAD | 25 |
| Secondary Aim 6 | 26 |
| Table 6.1: Culture Positivity by serotype | 26 |
| Table 6.2: Rectal swab and whole stool comparison | 2.7 |



## Primary Aim

Figure 1: Diarrhea case surveillance participant screening, enrollment and follow-up.



Figure 1. EFGH CONSORT diagram. <sup>a</sup> Reasons participants were not screened or did not meet eligibility do not sum to total as participants could have screened out for multiple reasons. b Among enrolled participants who attended the Week Four visit or missed the Week Four visit but not due to death, withdrawal or lost to follow-up (LTFU).




#### **Table 1: Baseline participant characteristics**

| emographics | Rangladach | | heal Case Su | | | | The Cambia | Total |
|---|---|---|---|---|---|---|---|---|
| | Bangladesh | Kenya | Malawi | Mali | Pakistan | Peru | The Gambia | Total |
| otal enrolled: N | | | | | | | | |
| emale sex: n (%) | | | | | | | | |
| ge (months): n (%) | | | | | | | | |
| - 8 | | | | | | | | |
| – 11 | | | | | | | | |
| 2 – 17 | | | | | | | | |
| 8 - 23 | | | | | | | | |
| 4 – 35 | | | | | | | | |
| ge in months: median (IQR) | | | | | | | | |
| lighest maternal education achieved: n (%) | | | | | | | | |
| ess than primary school | | | | | | | | |
| oranic school only | | | | | | | | |
| rimary school or greater<br>inknown or declined | | | | | | | | |
| ccompanying caregiver employment: n (%) | | | | | | | | |
| ot employed<br>mployed | | | | | | | | |
| nknown | | | | | | | | |
| Children <5 years in household: median (IQR) | | | | | | | | |
| ge at end of exclusive breastfeeding: median (IQR) | | | | | | | | |
| Vealth index: median (IQR) | | | | | | | | |
| Vater, Sanitation and Hygiene (WASH) characteristics | | | | | | | | |
| rinking water source <sup>a</sup> : n (%) | | | | | | | | |
| nproved source | | | | | | | | |
| nimproved source | | | | | | | | |
| irface water | | | | | | | | |
| nknown or other source | | | | | | | | |
| anitation access <sup>b</sup> : n (%) | | | | | | | | |
| nproved source | | | | | | | | |
| nimproved source | | | | | | | | |
| pen defecation | | | | | | | | |
| nknown or other source | | | | | | | | |
| rinking water treatment: n (%) <sup>c</sup> | | | | | | | | |
| oil | | | | | | | | |
| leach/chlorination | | | | | | | | |
| plar disinfection | | | | | | | | |
| et stand and settle | | | | | | | | |
| train through a cloth<br>ilter (ceramics/sand/composite/LifeStraw) | | | | | | | | |
| ther method | | | | | | | | |
| linical characteristics | | | | | | | | |
| ymptoms at enrollment <sup>c</sup> : n (%) | | | | | | | | |
| ysentery <sup>d</sup> | | | | | | | | |
| edema | | | | | | | | |
| igns of LRTI <sup>e</sup> | | | | | | | | |
| tiff neck | | | | | | | | |
| eneralized rash | | | | | | | | |
| onvulsions | | | | | | | | |
| ethargy or unconscious | | | | | | | | |
| almar pallor | | | | | | | | |
| ehydration <sup>f</sup> : n (%) | | | | | | | | |
| one | | | | | | | | |
| evere | | | | | | | | |
| ome evere nmunization status: n (%) <sup>c</sup> | | | | | | | | |
| evere nmunization status: n (%)° eceived age-appropriate vaccinations, per country guidelines | | | | | | | | |
| evere nmunization status: n (%) <sup>c</sup> eceived age-appropriate vaccinations, per country guidelines eceived rotavirus vaccine | | | | | | | | |
| evere mmunization status: n (%) <sup>c</sup> eccived age-appropriate vaccinations, per country guidelines eccived rotavirus vaccine are seeking prior to enrollment visit: n (%) <sup>c</sup> | | | | | | | | |
| nnunization status: n (%)° cceived age-appropriate vaccinations, per country guidelines eccived rotavirus vaccine are seeking prior to enrollment visit: n (%)° mmunity health worker | | | | | | | | |
| evere munization status: n (%) <sup>c</sup> seceived age-appropriate vaccinations, per country guidelines seceived rotavirus vaccine are seeking prior to enrollment visit: n (%) <sup>c</sup> ommunity health worker rug seller | | | | | | | | |
| evere munization status: n (%) <sup>c</sup> seceived age-appropriate vaccinations, per country guidelines seceived rotavirus vaccine are seeking prior to enrollment visit: n (%) <sup>c</sup> mmunity health worker rug seller salth outpost | | | | | | | | |
| evere mmunization status: n (%)° eceived age-appropriate vaccinations, per country guidelines eceived rotavirus vaccine are secking prior to enrollment visit: n (%)° mmunity health worker rug seller ealth outpost patient health facility | | | | | | | | |
| evere mmunization status: n (%) <sup>c</sup> ecevived age-appropriate vaccinations, per country guidelines eceived rotavirus vaccine are seeking prior to enrollment visit: n (%) <sup>c</sup> ommunity health worker rug seller ealth outpost patient health facility utpatient health facility | | | | | | | | |
| evere munization status: n (%) <sup>c</sup> seceived age-appropriate vaccinations, per country guidelines seceived rotavirus vaccine are seeking prior to enrollment visit: n (%) <sup>c</sup> summunity health worker rug seller ealth outpost patient health facility utpatient health facility surmacist | | | | | | | | |
| evere mnunization status: n (%) <sup>c</sup> eceived age-appropriate vaccinations, per country guidelines eceived rotavirus vaccine are seeking prior to enrollment visit: n (%) <sup>c</sup> ommunity health worker rug seller ealth outpost patient health facility utpatient health facility armacist eligious or traditional healer | | | | | | | | |
| evere mmunization status: n (%) <sup>c</sup> ceceived age-appropriate vaccinations, per country guidelines eceived rotavirus vaccine are seeking prior to enrollment visit: n (%) <sup>c</sup> ommunity health worker rug seller ealth outpost patient health facility utpatient health facility arrmacist eligious or traditional healer ther | | | | | | | | |
| evere mmunization status: n (%) <sup>c</sup> ceceived age-appropriate vaccinations, per country guidelines eceived rotavirus vaccine are secking prior to enrollment visit: n (%) <sup>c</sup> ommunity health worker rug seller ealth outpost patient health facility utpatient health facility narmacist eligious or traditional healer ther ospitalized: n (%) <sup>g</sup> | R) | | | | | | | |
| evere mnunization status: n (%) <sup>c</sup> eccived age-appropriate vaccinations, per country guidelines eccived rotavirus vaccine are seeking prior to enrollment visit: n (%) <sup>c</sup> ommunity health worker rug seller ealth outpost patient health facility utpatient health facility narmacist eligious or traditional healer ther ospitalized: n (%) <sup>g</sup> uration of diarrhea prior to care seeking (days): median (IQ) | R) | | | | | | | |
| evere mmunization status: n (%) <sup>c</sup> seceived age-appropriate vaccinations, per country guidelines seceived rotavirus vaccine are seeking prior to enrollment visit: n (%) <sup>c</sup> sommunity health worker trug seller sealth outpost patient health facility utpatient health facility utpatient health facility sarmacist sligious or traditional healer ther sospitalized: n (%) <sup>g</sup> uration of diarrhea prior to care seeking (days): median (IQ) foldified Vesikari score (MVS) <sup>n</sup> : median (IQR), n (%) ild (0-8 points) | R) | | | | | | | |
| evere mmunization status: n (%) <sup>c</sup> seceived age-appropriate vaccinations, per country guidelines seceived rotavirus vaccine are seeking prior to enrollment visit: n (%) <sup>c</sup> sommunity health worker trug seller sealth outpost patient health facility utpatient health facility utpatient health facility sarmacist sligious or traditional healer ther sospitalized: n (%) <sup>g</sup> uration of diarrhea prior to care seeking (days): median (IQ) foldified Vesikari score (MVS) <sup>n</sup> : median (IQR), n (%) ild (0-8 points) | R) | | | | | | | |
| evere mmunization status: n (%) <sup>c</sup> eceived age-appropriate vaccinations, per country guidelines eceived rotavirus vaccine are seeking prior to enrollment visit: n (%) <sup>c</sup> ommunity health worker rug seller ealth outpost patient health facility utpatient health facility turpatient health facil | R) | | | | | | | |
| evere mmunization status: n (%) <sup>c</sup> ceceived age-appropriate vaccinations, per country guidelines eceived rotavirus vaccine are seeking prior to enrollment visit: n (%) <sup>c</sup> ommunity health worker rug seller ealth outpost patient health facility utpatient health facility utpatient health facility armacist eligious or traditional healer ther ospitalized: n (%) <sup>c</sup> urration of diarrhea prior to care seeking (days): median (IQ oddfied Vesikari score (MVS) <sup>c</sup> : median (IQR), n (%) ild (0-8 points) odderate (9-10 points) evere (11+ points) | R) | | | | | | | |
| evere mmunization status: n (%) <sup>c</sup> ceceived age-appropriate vaccinations, per country guidelines eceived rotavirus vaccine are seeking prior to enrollment visit: n (%) <sup>c</sup> ommunity health worker rug seller ealth outpost patient health facility utpatient health facility utpatient health facility narmacist eligious or traditional healer ther ospitalized: n (%) <sup>g</sup> uration of diarrhea prior to care seeking (days): median (IQ lodified Vesikari score (MVS) <sup>h</sup> : median (IQR), n (%) ild (0-8 points) loderate (9-10 points) evere (11+ points) loderate or severe diarrhea by MVS or dysentery <sup>i</sup> : n (%) EMS <sup>i</sup> : median (IQR), n (%) | R) | | | | | | | |
| evere mmunization status: n (%) <sup>c</sup> ceceived age-appropriate vaccinations, per country guidelines eceived rotavirus vaccine are seeking prior to enrollment visit: n (%) <sup>c</sup> ommunity health worker rug seller ealth outpost patient health facility utpatient health facility utpatient health facility utpatient health facility arrmacist eligious or traditional healer ther ospitalized: n (%) <sup>c</sup> urration of diarrhea prior to care seeking (days): median (IQ lodified Vesikari score (MVS) <sup>c</sup> : median (IQR), n (%) lid (0-8 points) loderate (9-10 points) evere (11+ points) loderate or severe diarrhea by MVS or dysentery <sup>i</sup> : n (%) EMS!: median (IQR), n (%) loderate to severe diarrhea (MSD) | R) | | | | | | | |
| evere mmunization status: n (%) <sup>c</sup> ceceived age-appropriate vaccinations, per country guidelines eceived rotavirus vaccine are seeking prior to enrollment visit: n (%) <sup>c</sup> ommunity health worker rug seller ealth outpost patient health facility utpatient health facility utpatient health facility utpatient health facility arrmacist eligious or traditional healer ther ospitalized: n (%) <sup>c</sup> urration of diarrhea prior to care seeking (days): median (IQ lodified Vesikari score (MVS) <sup>c</sup> : median (IQR), n (%) lid (0-8 points) loderate (9-10 points) evere (11+ points) loderate or severe diarrhea by MVS or dysentery <sup>i</sup> : n (%) EMS!: median (IQR), n (%) loderate to severe diarrhea (MSD) | R) | | | | | | | |
| evere mmunization status: n (%) <sup>c</sup> ecevived age-appropriate vaccinations, per country guidelines eceived rotavirus vaccine are seeking prior to enrollment visit: n (%) <sup>c</sup> ommunity health worker rug seller ealth outpost patient health facility utpatient health facility utpatient health facility armacist eligious or traditional healer ther ospitalized: n (%) <sup>g</sup> uration of diarrhea prior to care seeking (days): median (IQ lodlifed Vesikari score (MVS) <sup>g</sup> : median (IQR), n (%) (idd (0-8 points) ioderate (9-10 points) evere (11+ points) loderate or severe diarrhea by MVS or dysentery <sup>i</sup> : n (%) EMS <sup>g</sup> : median (IQR), n (%) loderate to severe diarrhea (MSD) ess severe diarrhea (LSD) | R) | | | | | | | |
| evere mmunization status: n (%) <sup>c</sup> ecevived age-appropriate vaccinations, per country guidelines eceived rotavirus vaccine are seeking prior to enrollment visit: n (%) <sup>c</sup> ommunity health worker rug seller ealth outpost patient health facility utpatient nearther deligious or traditional healer ther ospitalized: n (%) <sup>g</sup> uration of diarrhea prior to care seeking (days): median (IQ dolffied Vesikari score (MVS) <sup>h</sup> : median (IQR), n (%) iddefate (9-10 points) evere (11+ points) toderate (9-10 points) toderate (9-10 points) toderate or severe diarrhea by MVS or dysentery <sup>i</sup> : n (%) EMS: median (IQR), n (%) toderate to severe diarrhea (MSD) sess severe diarrhea (LSD) EMS-Shigella score <sup>k</sup> : median (IQR), n (%) | R) | | | | | | | |
| evere | R) | | | | | | | |
| evere mmunization status: n (%) <sup>c</sup> ceceived age-appropriate vaccinations, per country guidelines eceived rotavirus vaccine are seeking prior to enrollment visit: n (%) <sup>c</sup> ommunity health worker rug seller galth outpost patient health facility utpatient dealth facility utpatient health facility utpatient | R) | | | | | | | |
| invere imunization status: n (%) <sup>c</sup> ceceived age-appropriate vaccinations, per country guidelines seceived rotavirus vaccine are seeking prior to enrollment visit: n (%) <sup>c</sup> mmunity health worker rug seller calth outpost patient health facility attraction traditional healer ther sopitalized: n (%) <sup>c</sup> uration of diarrhea prior to care seeking (days): median (IQ odified Vesikari score (MVS) <sup>c</sup> ; median (IQR), n (%) id (0-8 points) oderate (9-10 points) vere (11+ points) oderate or severe diarrhea by MVS or dysentery <sup>i</sup> : n (%) EMS <sup>1</sup> : median (IQR), n (%) oderate to severe diarrhea (MSD) sss severe diarrhea (LSD) EMS-Shigella score <sup>c</sup> ; median (IQR), n (%) id (<6 points) oderate (6-8 points) oderate (6-9 points) vere (9+ points) lark score; median (IQR), n (%) | R) | | | | | | | |
| were munization status: n (%) creatived age-appropriate vaccinations, per country guidelines believed rotavirus vaccine mre seeking prior to enrollment visit: n (%) munity health worker ug seller patient health facility tipatient health facility armacist eligious or traditional healer her popitalized: n (%) mation of diarrhea prior to care seeking (days): median (IQ odified Vesikari score (MVS) median (IQR), n (%) id (0-8 points) oderate (9-10 points) vere (11+ points) oderate or severe diarrhea by MVS or dysentery median (IQR), n (%) EMS median (IQR), n (%) | R) | | | | | | | |




None

| | Bangladesh | Kenya | Malawi | Mali | Pakistan | Peru | The Gambia | Total |
|---|---|---|---|---|---|---|---|---|
| Non-severe (<6 points) | - | | | | | | | |
| Severe (6+ points) | | | | | | | | |
| Anthropometry | | | | | | | | |
| LAZ/HAZ: median (IQR) | | | | | | | | |
| MUAC: median (IQR) | | | | | | | | |
| WAZ: median (IQR) | | | | | | | | |
| WLZ: median (IQR) | | | | | | | | |
| Stunted <sup>n</sup> : n (%) | | | | | | | | |
| Severe | | | | | | | | |
| Moderate | | | | | | | | |
| None | | | | | | | | |
| Wasted°: n (%) | | | | | | | | |
| Severe | | | | | | | | |
| Moderate | | | | | | | | |
| None | | | | | | | | |
| Underweight <sup>p</sup> : n (%) | | | | | | | | |
| Severe | | | | | | | | |
| Moderate | | | | | | | | |

HAZ: height for age Z-score, IQR: interquartile range, JMP: WHO/UNICEF Joint Monitoring Programme for Water Supply, Sanitation and Hygiene, LAZ: length for age Z-score, LRTI; lower respiratory tract infection, LSD: less-sever-diarrhea, MSD: moderate-to-severe diarrhea, MUAC: mid-upper arm circumference, MVS: modified Vesikari score, WAZ: weight for age Z-score, WHO: world health organization, WLZ: weight for length Z-score.

- a Drinking water source was classified according to the WHO/UNICEF Joint Monitoring Programme for Water Supply, Sanitation and Hygiene (JMP) as surface water (water from a river, dam, lake, pond, stream, canal or irrigation channel), unimproved (unprotected wells or springs), or improved (water piped into the dwelling, yard or plot, public taps or standpipes, tube wells or boreholes, protected dug wells or springs, rainwater collection, water from a tanker-truck, water from a cart with a small tank or drum, filtered or unfiltered water kiosks, bottled water, or sachet water
- b Sanitation access was classified according to the JMP as open defecation (no facility, bush or field), unimproved (flush toilets to elsewhere, pit latrines without slab floor, bucket toilets or hanging toilets/latrines), or improved (flush toilets to piped sewer systems, septic tanks or unknown location, ventilated improved pit latrines, pit latrines with slab floors, or composting toilets).
- <sup>c</sup> Columns do not sum to 100% as multiple options could be selected.
- <sup>d</sup> Blood in the stool as reported by caregiver during the diarrheal episode or by clinical diagnosis
- One or more of the following signs indicative of lower respiratory infection: cough, difficulty breathing, chest in-drawing, chest auscultation, central cyanosis, oxygen saturation <90%, or severe respiratory distress.
- f Based on WHO criteria. Severe dehydration = At least two of the following signs: lethargy, abnormally sunken eyes, drinks poorly, skin pinch >2 seconds. Some dehydration = At least two of the following signs: restless/irritable, abnormally sunken eyes, drinks eagerly, skin pinch 1-2 seconds.
- <sup>g</sup> Defined as an overnight stay (child was on the ward from at least 12am to 6am or self-discharged prior to that timeframe
- <sup>b</sup> Defined as in PATH Vesikari Clinical Severity Scoring System Manual: Duration of diarrhea: 1-4 days (1 point), 5 days (2 points) ≥6 days (3 points); Max # of stool in 24 hour period: 1-3 (1 point), 4-5 (2 points), ≥6 (3 points); Duration of vomiting: 1 day (1 point), 2 days (2 points), ≥3 days (3 points); max # of vomiting episodes in 24 hour period: 1 (1 point), 2-4 (2 points), ≥5 (3 points); Axillary temperature 36.6-37.9°C (1 point), 38.0-38.4°C (2 points), ≥38.5°C (3 points); dehydration 1-5% (2 points), ≥6% (3 points); treatment: rehydration (1 point), hospitalization (2 points), ≥6% (3 points); dehydration 1-5% (2 points), ≥6% (3 points); dehydration 1-5% (2 points), ≥6% (3 points); dehydration 1-5% (2 points), ≥6% (3 points); dehydration (1 point), bospitalization (2 points), ≥6% (3 points); dehydration 1-5% (2 points), ≥6% (3 points); dehydration 1-5% (2 points), ≥6% (3 points); dehydration (3 points); dehydration 1-5% (2 points), ≥6% (3 points); dehydration (3 points); dehydration 1-5% (2 points), ≥6% (3 points); dehydration (3 points); dehydration 1-5% (2 points), ≥6% (3 points); dehydration (3 points); dehydration (3 points); dehydration 1-5% (2 points), ≥6% (3 points); dehydration (3 points); dehydration 1-5% (2 points), ≥6% (3 points); dehydration (3 points); deh
- Defined as in Pavlinac, Vaccines, 2022 as a MVS of 9+ or presence of visible blood in stool. N=x could not be assessed due to missing data for diarrhea duration.
- Defined as in Kotloff, Lancet GH, 2019. Moderate-to-severe diarrhea (MSD) defined as presenting to a health facility with diarrhea and severe or some dehydration (by WHO criteria), visible blood in stool, or inpatient admission. Less-severe-diarrhea (LSD) defined as presenting to a health facility without MSD.
- <sup>k</sup> Defined as in Pavlinac, CID, 2021. Duration of diarrhea through day of presentation: 1-3 days (0 points), 4-5 days (2 points), ≥6 days (3 points); WHO-defined dehydration categories: severe (8 points), some (4 points), none (0 points); inpatient admission (5 points).<sup>7</sup>
- Defined as in Clark, JID, 1988. Duration of diarrhea: 1-4 days (1 point), 5-7 days (2 points) >7 days 3 points); Max # of stool in 24 hour period: 2-4 (1 point), 5-7 (2 points), >7 (3 points); Duration of vomiting: 2 days (1 point), 3-5 days (2 points), >5 days (3 points); max # of vomiting episodes in 24 hour period: 1-3 (1 point), 4-6 (2 points), >6 (3 points); Duration of reported fever: 1-2 days (1 point), 3-4 days (2 points), >5 days (3 points); Rectal temperature 38-38.2° (2 (1 point), 3-3.3-38.7° (2 points), >38.8° (3 points); behavioral signs: Irritable/less playful (1 point), Lethargic/listless (2 points), Seizures (3 points). N=x could not be assessed due to missing data for diarrhea duration.
- m Defined as in Lee, BMJ Open, 2014: Duration of diarrhea: 2-4 days (1 point), 5-7 days (2 points), ≥8 days (3 points); Max # of stool in 24 hour period: <5 loose stools/24 hours (1 point), 5-7 loose stools/24 hours (2 points), ≥8 stools/24 hours (3 points); Duration of vomiting: 1 day (1 point), 2 days (2 points), ≥3 days (3 points); duration of reported fever: 1+ days (1 point); Confirmed temperature: ≥37.5°C (confirmed by field worker) (2 points); Dehydration: Some (2 points), severe (3 points). N=x could not be assessed due to missing data for diarrhea duration.
- <sup>n</sup> Severe stunting: HAZ/LAZ < -3, Moderate stunting:  $-3 \le HAZ/LAZ < -2$ .
- ° Severe wasting: WLZ < -3 or MUAC < 11.5, Moderate wasting: -3 ≤ WLZ < -2 or 11.5 ≤ MUAC < 12.5.
- <sup>p</sup> Severely underweight: WAZ < -3, Moderately underweight:  $-3 \le WAZ < -2$ .



#### Table 2: Baseline characteristics of population enumeration

| Table 2. Demographic and Clinical Characteristics of the Popul | ation Enumeratio | n and Heal | thcare Utiliza | ation Surv | ey, by study si | te. | | |
|---|---|---|---|---|---|---|---|---|
| Indicator | Bangladesh | Kenya | Malawi | Mali | Pakistan | Peru | The Gambia | Overall |
| Population Enumeration | | | | | | | | |
| Total clusters demarcated: n | | | | | | | | |
| Study area: m <sup>2</sup> | | | | | | | | |
| Clusters enumerated: n (%) | | | | | | | | |
| Cluster enumerated | | | | | | | | |
| No households present in the cluster | | | | | | | | |
| Could not enumerated cluster due to safety or other reasons | | | | | | | | |
| Not enumerated | | | | | | | | |
| Total individuals enumerated: n | | | | | | | | |
| Children 6-35 months of age enumerated: n | | | | | | | | |
| Caregiver reported children 6-35 months of age had diarrhea | | | | | | | | |
| in the past two weeks: n (%) | | | | | | | | |
| Yes | | | | | | | | |
| No | | | | | | | | |
| Don't know | | | | | | | | |
| Caregiver of child 6-35 months of age with diarrhea consented | | | | | | | | |
| to HUS: n (%) | | | | | | | | |
| Yes, consented | | | | | | | | |
| No, refused | | | | | | | | |
| No, caregiver not available for consent no successful revisit | | | | | | | | |
| Care-seeking for diarrhea: n (%) <sup>a</sup> | | | | | | | | |
| Did not seek care<br>Sought care at an EFGH facility | | | | | | | | |
| Sought care at an EFGH facility Sought care at a different outpatient hospital or health center | | | | | | | | |
| Sought care at a different outpatient nospital or health center | | | | | | | | |
| Sought care at an inpatient nospital of health center Sought care at a health outpost | | | | | | | | |
| Sought care at a health outpost Sought care at a drug seller or pharmacist | | | | | | | | |
| Sought care at a traditional or religious healer | | | | | | | | |
| Other | | | | | | | | |
| Days between diarrhea onset and care seeking: median (IQR) | | | | | | | | |
| Demographic indicators of children in the HUS | | | | | | | | |
| Female sex: n (%) | | | | | | | | |
| Age (months): n (%) | | | | | | | | |
| 6 – 8 | | | | | | | | |
| 9 – 11 | | | | | | | | |
| 12 – 17 | | | | | | | | |
| 18 - 23 | | | | | | | | |
| 24 - 35 | | | | | | | | |
| Age in months: median (IQR) | | | | | | | | |
| Clinical characteristics | | | | | | | | |
| Symptoms during diarrheal illness: n (%) <sup>a</sup> | | | | | | | | |
| Blood in stool | | | | | | | | |
| Irritable | | | | | | | | |
| Very thirsty | | | | | | | | |
| Sunken eyes | | | | | | | | |
| Wrinkled skin | | | | | | | | |
| Drinks eagerly, thirsty | | | | | | | | |
| Unable to drink or drank poorly | | | | | | | | |
| Lethargic, unconscious, or hard to stay awake | | | | | | | | |

HUS: healthcare utilization survey, IQR: interquartile range.

a Column does not sum to total as surveyed participants may have sought care from multiple sources or reported multiple clinical symptoms.



Table 3: Shigella Incidence by country and method of ascertainment

| | Confirn | ned <i>Shigella</i> case | es: n | Shigella MAD incidence | | |
|---|---|---|---|---|---|---|
| EFGH Country | Watery<br>diarrhea | Dysentery | Total | Crude IR (CI) | Enrollment-<br>adjusted IR <sup>a</sup> (CI) | Adjusted IR <sup>b</sup><br>(CI) |
| Culture-confirmed Sh | | Dysentery | Total | Crude III (CI) | aujusteu IIV (CI) | (CI) |
| Bangladesh | 0 | | | | | |
| Kenya | | | | | | |
| Malawi | | | | | | |
| Mali | | | | | | |
| Pakistan | | | | | | |
| Peru | | | | | | |
| The Gambia | | | | | | |
| Total <sup>d</sup> | | | | | | |
| Shigella attributable b | y molecular di | agnostics <sup>e</sup> | | | | |
| Bangladesh | | | | | | |
| Kenya | | | | | | |
| Malawi | | | | | | |
| Mali | | | | | | |
| Pakistan | | | | | | |
| Peru | | | | | | |
| The Gambia | | | | | | |
| Totald | | | | | | |

CI: 95% confidence interval, CT: cycle threshold, IR: incidence rate, MAD: medically-attended diarrhea, mBGS: Modified buffered glycerol saline.

<sup>&</sup>lt;sup>a</sup> The number of confirmed *Shigella* watery diarrhea cases per 100 child-years adjusted for enrollment plus the number of confirmed *Shigella* dysentery cases per 100 child-years at risk adjusted for enrollment.

<sup>&</sup>lt;sup>b</sup> The number of confirmed *Shigella* watery diarrhea cases per 100 child-years, adjusted for care-seeking and enrollment plus the number of confirmed *Shigella* dysentery cases per 100 child-years at risk, adjusted for care-seeking and enrollment.

<sup>&</sup>lt;sup>c</sup> Includes isolates from rectal swabs transported in mBGS or Cary-Blair media.

<sup>&</sup>lt;sup>d</sup> Totals are the sum of country-level estimates weighted to the proportion of child-years contributing to the combined denominator.

<sup>&</sup>lt;sup>e</sup> Defined as an ipaH cycle threshold (CT) < 31.1.

Culture<sup>a</sup> TAC<sup>b</sup> Total

Culture<sup>a</sup> TAC<sup>b</sup> The Gambia



# Secondary Aim 1

Table 1.1: Shigella incidence by species and serotype

Enrollment- and Healthcare Seeking-Adjusted Shigella MAD Incidence Rate (CI) Culture<sup>a</sup> TAC<sup>b</sup> Culture<sup>a</sup> TAC<sup>b</sup> Culture<sup>a</sup> TAC<sup>b</sup> Culture<sup>a</sup> TAC<sup>c</sup> Culture<sup>a</sup> TAC<sup>c</sup> Culture<sup>a</sup> TAC<sup>c</sup> Pakistan Malawi Table 1.1. Adjusted Shigella incidence stratified by Shigella species and serotype. Kenya Bangladesh Alternate quadrivalent vaccine targetse Quadrivalent vaccine targets<sup>d</sup> Bivalent vaccine targets<sup>c</sup> Non-typable S. dysentariae 2a 2b 3a 3b 4a 4b 5a 5b S. flexneri S. boydii Other Serotype S. Aexneri and S. sonnei

CI: 95% confidence interval, CT: cycle threshold, MAD: medically-attended diarrhea, TAC: TaqMan array card.

Undetermined1


<sup>&</sup>lt;sup>a</sup> S. flexneri 7a is not assessed by culture.

<sup>&</sup>lt;sup>b</sup> Defined as an ipaH cycle threshold (CT) < 31.1. S. boydii and S. dysentariae are not assessed by TAC.

<sup>°</sup> S. flexneri 2a or S. sonnei.

<sup>&</sup>lt;sup>d</sup> S. flexneri 2a, 3a, or 6 or S. sonnei.

<sup>&#</sup>x27;S. flexneri 1b, 2a or 3a or S. sonnei.

Undetermined by culture means any serotypes/subserotypes not listed in the table. Undetermined by TAC means Shigella detected by PCR but molecular criteria to assign species/serotype to S. sonnei or S. flexneri was not met.



# Table 1.2: Shigella incidence by age and diarrhea severity

| Table 1.2. Adjusted Shigella incidence stratified by participant age | tified by partici | pant age and | diarrhea se | and diarrhea severity definition. | tion. | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 0 | | Enrollment: and Healthcare Seeking-Adjusted Shigella MAD Incidence Rate (CI) | and Hea | theare Seek | ino-Adiust | ed Shipella | AAD Incid | ence Rate (C | 1 | | | | İ |
| B | Bangladesh | Kenya | | Malawi | | Mali | 6 | Pakistan | | Peru | ì | The Gambia | ıbia | Total | |
| Strata Cult | Culture TAC <sup>a</sup> | Culture | $AC^a$ | Culture TAC <sup>a</sup> | | Culture TAC <sup>a</sup> | | Culture TAC <sup>a</sup> | | Culture | $TAC^a$ | Culture | g. | Culture T | $TAC^a$ |
| Age at enrollment (months) | | | | | | | | | | | | | | | |
| 8-9 | | | | | | | | | | | | | | | |
| 9 – 11 | | | | | | | | | | | | | | | |
| 12 - 17 | | | | | | | | | | | | | | | |
| 18 - 23 | | | | | | | | | | | | | | | |
| 24 - 35 | | | | | | | | | | | | | | | |
| Diarrhea severity classifications | | | | | | | | | | | | | | | |
| Dysentery | | | | | | | | | | | | | | | |
| Watery diarrhea | | | | | | | | | | | | | | | |
| Hospitalized | | | | | | | | | | | | | | | |
| Modified Vesikari score (MVS) <sup>b</sup> | | | | | | | | | | | | | | | |
| Mild illness (0-8 points) | | | | | | | | | | | | | | | |
| Moderate illness (9-10 points) | | | | | | | | | | | | | | | |
| Severe illness (11+ points) | | | | | | | | | | | | | | | |
| Moderate or severe diarrhea by | | | | | | | | | | | | | | | |
| MVS or dysentery <sup>c</sup> | | | | | | | | | | | | | | | |
| $\mathbf{GEMS}^{\mathrm{d}}$ | | | | | | | | | | | | | | | |
| Moderate-to-severe diarrhea (MSD) | | | | | | | | | | | | | | | |
| Less-severe-diarrhea (LSD) | | | | | | | | | | | | | | | |
| GEMS-Shigella score <sup>e</sup> | | | | | | | | | | | | | | | |
| Mild (<6 points) | | | | | | | | | | | | | | | |
| Moderate (6-8 points) | | | | | | | | | | | | | | | |
| Severe (9+ points) | | | | | | | | | | | | | | | |
| Clark scoref | | | | | | | | | | | | | | | |
| Mild (2-8 points) | | | | | | | | | | | | | | | |
| Moderate to severe (9+ points) | | | | | | | | | | | | | | | |
| MAL-ED score <sup>g</sup> | | | | | | | | | | | | | | | |
| Non-severe (<6 points) | | | | | | | | | | | | | | | |
| Severe (6+ points) | | | | | | | | | | | | | | | |
| CI: 95% confidence interval, CT: cycle threshold, LSD: less-severe-diarrhea, MAD: medically-attended diarrhea, MSD: moderate-to-severe diarrhea, MVS: modified Vesikari score, TAC: TaqMan array card, WHO: World Health | old, LSD: less-se | rere-diarrhea, | MAD: med | lically-attende | d diarrhe | a, MSD: mod | derate-to-se | vere diarrhea | , MVS: mo | dified Vesika | ıri score, T | AC: TaqMan | array card, | , WHO: World | Health |

<sup>1</sup> Defined as an ipaH cycle threshold (CT) < 31.1. S. boydii and S. dysentariae are not assessed by TAC. Organization.


b Defined as in PATH Vesikari Clinical Severity Scoring System Manual: Duration of diarrhea: 1-4 days (1 point), 5 days (2 points); ≥6 days (3 points); Max # of stool in 24 hour period: 1-3 (1 point), 4-5 (2 points), ≥6 days (2 points), ≥3 days (2 points); max # of vomitting episodes in 24 hour period: 1 (1 point), 2-4 (2 points), ≥6 (3 points); Axillary temperature 36.6-37.9°C (1 point), 38.0-38.4°C (2 points), ≥38.5°C (3 points); dehydration 1-5% (2 points); treatment: rehydration (1 point), hospitalization (2 points).

d Defined as in Kotloff, Lancet GH, 2019. Moderate-to-severe diarrhea (MSD) defined as presenting to a health facility with diarrhea and severe or some dehydration (by WHO criteria), visible blood in stool, or inpatient admission. Less-severe-diarrhea (LSD) defined as presenting to a health facility without MSD.

<sup>&</sup>lt;sup>†</sup>Defined as in Clark, IID, 1988. Duration of diarrhea: 1-4 days (1 point), 5-7 days (2 points) > 7 days (3 points); Max # of stool in 24 hour period: 2-4 (1 point), 5-7 (2 points); Duration of vomiting: 2 days (1 point), 3-4 days (2 points); Duration of reported fever: 1-2 days (1 point), 3-4 days (2 points); Pectal temperature (2 points); Pectal temperature (3 points); Duration of reported fever: 1-2 days (3 points); Pectal temperature (3 points); Pectal temperature (4 points); Pectal temperature (5 points); Pectal tem \* Defined as in Pavlinac, CID, 2021. Duration of diarrhea through day of presentation: 1-3 days (0 points), 4-5 days (2 points), 26 days (3 points); WHO-defined dehydration categories: severe (8 points), some (4 points), none (0 points); inpatient admission (5 points).

<sup>38-38.2°</sup>C (1 point), 38.3-38.7°C (2 points), 238.8°C (3 points), behavioral signs: Irritable/less playful (1 point), Lethargic/listless (2 points), Seizures (3 points).

\*\*Befined as in Lee, J Pediatr Gastroenterol Nutr., 2016. Duration of diarrhea: 2-4 days (1 points), 5-7 days (2 points); Max # of stool in 24 hour period: <5 loose stools/24 hours (1 point), 5-7 loose stools/24 hours.

<sup>(2</sup> points), 28 stools/24 hours (3 points); Duration of vomiting: 1 day (1 point), 2 days (2 points), 3 days (3 points); duration of reported fever: 1+ days (1 point); Confirmed temperature: 23.7.5°C (confirmed by field worker) (2 points); Dehydration: Some (2 points), severe (3 points).


### Table 1.3: Shigella incidence by severity

Table 1.3. Adjusted incidence of relevant vaccine Shigella serotypes and species by diarrhea severity.

| | | Enrollment- and Healthcare Seeking-Adjusted Shigella MAD Incidence Rate (CI) | althcare Seeking-Ad | justed <i>Shigella</i> MAD | Incidence Rate (CI) | | |
|---|---|---|---|---|---|---|---|
| Bangladesh | Kenya | Malawi | Mali | Pakistan | Peru | The Gambia | Total |
| Strata Culture TAC | Culture TAC <sup>a</sup> Cultur | Culture TAC <sup>a</sup> | Culture TACa | Culture TAC <sup>a</sup> | Culture TAC <sup>a</sup> | Culture TAC <sup>a</sup> | Culture TAC <sup>a</sup> |
| Bivalent vaccine targets (S. flexneri 2a & S. sonnei) | | | | | | | |
| GEMS moderate-to-severe diarrhea (MSD) <sup>b</sup> | | | | | | | |
| MVS moderate or severe diarrhea or dysentery <sup>c</sup> | | | | | | | |
| Quadrivalent vaccine targets (S. flexneri 2a, 3a & 6 & S. sonnei) | | | | | | | |
| GEMS MSD <sup>₺</sup> | | | | | | | |
| MVS moderate or severe diarrhea or dysentery° | | | | | | | |
| Quadrivalent vaccine targets (S. flexneri 1b, 2a & 3a & S. sonnei) | i) | | | | | | |
| GEMS MSD <sup>♭</sup> | | | | | | | |
| MVS moderate or severe diarrhea or dysentery° | | | | | | | |
| THE PERSON OF TH | TOTAL I THE THE THE TANK I TO THE TANK I TO | 1 256 | 1 11 11 77 | 1 400 | - : | 1. 131 2.1 2234 1 .1 | |

CI: 95% confidence interval, CT: cycle threshold, GEMS: Global Enteric Multicenter Study, MAD: medically-attended diarrhea, MSD: moderate-to-severe-diarrhea, MVS: modified Vesikari score, TAC: TaqMan array card, WHO: World Health Organization.


<sup>&</sup>lt;sup>a</sup> Defined as an ipaH cycle threshold (CT) < 31.1.

<sup>&</sup>lt;sup>b</sup> Defined as in Kotloff, Lancet GH, 2019. Moderate-to-severe diarrhea (MSD) defined as presenting to a health facility with diarrhea and severe or some dehydration (by WHO criteria), visible blood in stool, and/or inpatient admission.

<sup>&</sup>lt;sup>c</sup> Defined as in Pavlinac, Vaccines, 2022 as a MVS of 9+ or presence of visible blood in stool.



### Table 1.4: Prevalence of enteric pathogens detected by molecular diagnostics.

| | | Positive below the attributable cycle threshold (CT) cutoff: n/N (%) | |
|---|---|---|---|
| Enteric pathogen <sup>a</sup> | Bangladesh | Kenya Malawi Mali Pakistan Peru The Gambia | Total |
| All medically-attended diarrhea (MAD) | | | |
| Shigella (cycle threshold [CT]<31.1) | | | |
| Adenovirus 40/41 (CT<25.5) | | | |
| Cryptosporidium (CT<27.1) | | | |
| Norovirus GII (CT<26.6) | | | |
| Rotavirus (CT<34.2) | | | |
| ST-ETEC (CT<27.9) | | | |
| tEPEC (CT<20.7) | | | |
| Campylobacter jejuni (CT<20.7) | | | |
| Astrovirus (CT<26.7) | | | |
| Sapovirus (CT<24.4) | | | |
| V. cholerae (CT<33.9) | | | |
| Salmonella (CT<33.3) | | | |
| Aeromonas (CT<23.6) | | | |
| Cyclospora cayetanensis (CT<33.9) | | | |
| Entamoeba histolytica (CT<32.6) | | | |
| Cystoisospora belli (CT<34.4) | 177 0 10 | | |
| Moderate or severe MAD by the Modifie | u Vesikari Scor | re (9+) +/- aysentery | |
| Shigella (CT<31.1) | | | |
| Adenovirus 40/41 (CT<25.5) | | | |
| Cryptosporidium (CT<27.1) | | | |
| Norovirus GII (CT<26.6) | | | |
| Rotavirus (CT<34.2)<br>ST-ETEC (CT<27.9) | | | |
| tEPEC (CT<20.7) | | | |
| Campylobacter jejuni (CT<20.7) | | | |
| Astrovirus (CT<26.7) | | | |
| Sapovirus (CT<24.4) | | | |
| V. cholerae (CT<33.9) | | | |
| Salmonella (CT<33.3) | | | |
| Aeromonas (CT<23.6) | | | |
| Cvclospora cavetanensis (CT<33.9) | | | |
| Entamoeba histolytica (CT<32.6) | | | |
| Cystoisospora belli (CT<34.4) | | | |
| Shigella-attributable MAD (CT<31.1) | | | |
| Adenovirus 40/41 (CT<25.5) | | | |
| Cryptosporidium (CT<27.1) | | | |
| Norovirus GII (CT<26.6) | | | |
| Rotavirus (CT<34.2) | | | |
| ST-ETEC (CT<27.9) | | | |
| tEPEC (CT<20.7) | | | |
| Campylobacter jejuni (CT<20.7) | | | |
| Astrovirus (CT<26.7) | | | |
| Sapovirus (CT<24.4) | | | |
| V. cholerae (CT<33.9) | | | |
| Salmonella (CT<33.3) | | | |
| Aeromonas (CT<23.6) | | | |
| Cyclospora cayetanensis (CT<33.9) | | | |
| Entamoeba histolytica (CT<32.6) | | | |
| Cystoisospora belli (CT<34.4) | 1 110 | | |
| Non-Shigella-attributable MAD (CT≥31. | <u>1 or no amplific</u> | cation) | |
| Adenovirus 40/41 (CT<25.5) | | | |
| Cryptosporidium (CT<27.1) | | | |
| Norovirus GII (CT<26.6) | | | |
| Rotavirus (CT<34.2) | | | |
| ST-ETEC (CT<27.9) | | | |
| tEPEC (CT<20.7) | | | |
| Campylobacter jejuni (CT<20.7) | | | |
| Astrovirus (CT<26.7) | | | |
| Sapovirus (CT<24.4) | | | |
| V. cholerae (CT<33.9) | | | |
| Salmonella (CT<33.3) | | | |
| Aeromonas (CT<23.6) | | | |
| Cyclospora cayetanensis (CT<33.9) | | | |
| Entamoeba histolytica (CT<32.6) | | | |
| Cystoisospora belli (CT<34.4) | | li MAD; modically attended distribus ST ETEC; heat stabile toyin producing E coli | |

CT: cycle threshold, tEPEC: typical enteropathogenic E. coli, MAD: medically-attended diarrhea, ST-ETEC: heat stabile toxin-producing E. coli.

<sup>a</sup> The top three most prevalent pathogens by site are highlighted in green.

<sup>b</sup> Defined as in Pavlinac, Vaccines, 2022 as a MVS of 9+ or presence of visible blood in stool.



### Table 2.1: Country and region antibiotic-non-susceptibility Secondary Aim 2

Total Peru South Asia total Pakistan Bangladesh Antibiotic non-susceptibility: % (CI)
West Africa total The Gambia Mali East Africa total Table 2.1. Country- and region-specific antibiotic non-susceptibility to culture-confirmed Shigella isolates Malawi Kenya Resistance to all WHO recommended treatments<sup>a</sup> Extensive drug resistance (XDR) Trimethoprim-sulfamethoxazole Multidrug resistance (MDR)<sup>b</sup> All *Shigella* isolates S. sonnei
Ciprofloxacin
All Shigella isolates S. sonnei

Nalidixic acid
All Shigella isolates Ampicillin All Shigella isolates All *Shigella* isolates S. *flexneri* All *Shigella* isolates S. *flexneri* All Shigella isolates All Shigella isolates All Shigella isolates All Shigella isolates S. sonnei
Pivemicellinam Azithromycin S. sonnei Ceftriaxone S. flexneri S. flexneri Antibiotic S. flexneri S. flexneri S. flexneri S. flexneri S. flexneri S. flexneri S. sonnei


S. sonnei

1. S. sonnei

1. S. Sonnei

1. S. Sonnei

1. Sonnei

2. Sonnei

2. Sonnei

2. MDE: extensive drug resistance, WHO: World Health Organization.

3. WHO recommended treatments include Azithromycin, Ciprofloxacin, and Ceftriaxone.

4. WHO recommended treatments antibiotics.

5. Resistant to any three or more antibiotics.

6. Resistant to all of the following: azithromycin, ciprofloxacin, ceftiaxone, trimethoprim-sulfamethoxazole, and ampicillin.



### **Secondary Aim 3**

### Table 3.1: All-cause case fatality

**Table 3.1.** Extended all-cause case fatality among children enrolled in EEGH with and without Shigella

| Table 3.1. Laterided | an-cause case rata | iity aiiioii | g chinaren c | inoncu | III LI OII WI | ui aiia wii | mout snigetti | ı |
|---|---|---|---|---|---|---|---|---|
| attributed MAD. | | | | | | | | |
| | | | All-cau | se case f | fatality <sup>a</sup> : n/N | V (%) | | |
| | | | | | - | | The | |
| | Bangladesh | Kenya | Malawi | Mali | Pakistan | Peru | Gambia | Overall |
| Overall | | | | | | | | |
| $Shigella^b$ | | | | | | | | |
| No Shigella <sup>c</sup> | | | | | | | | |
| 2 5 1 72 2 5 11 11 | 1 1 1 1 1 70 4 | a | | 1 | | | | |

MAD: Medically-attended diarrhea, TAC: Taqman array card.

### Table 3.2: Causes of death

Table 3.2. ICD-11<sup>a</sup> causes of death<sup>b</sup> for all known mortality events occurring within the EFGH three-month follow-up period

| | Time since | Age at | Shigella | | Caus | es of Death | |
|---|---|---|---|---|---|---|---|
| | enrollment to | death | attribution at | Immediate | Distal | Most | Underlying |
| Site | death (days) | (months) | enrollment <sup>c</sup> | (1a) | (1b) | Distal (1c) | (2) |

ICD-11: International Classification of Diseases 11th Revision.

<sup>&</sup>lt;sup>a</sup> Death occurring within 3 months of EFGH follow-up.

<sup>&</sup>lt;sup>b</sup> By culture isolation or TAC ipaH <31.1.

<sup>&</sup>lt;sup>c</sup> By absence of culture isolation or ipaH ≥31.1.

<sup>&</sup>lt;sup>a</sup> International Classification of Diseases, Eleventh Revision (ICD-11), World Health Organization (WHO) 2019/2021 https://icd.who.int/browse11. Licensed under Creative Commons Attribution-NoDerivatives 3.0 IGO licence (CC BY-ND 3.0 IGO).

<sup>&</sup>lt;sup>b</sup> Causes of death are agreed upon by a panel of ICD-11 trained clinicians using information from the child's death certificate (if available), caregiver interview (if available), and case notes from the child's care team.

<sup>&</sup>lt;sup>c</sup> By culture isolation or TAC ipaH <31.1.



### Table 3.3: Hospitalization, subsequent diarrhea episodes, and persistent diarrhea

**Table 3.3.** Risk of hospitalization, subsequent diarrhea, and diarrhea persistence in the three months following medically attended diarrhea attributed to *Shigella* and other leading attributable causes of the index MAD.

| | | RR, PR | |
|---|---|---|---|
| | n/N (%) | Semi-Unadjusted <sup>a</sup> | Adjusted <sup>b</sup> |
| Persistent Diarrhea <sup>c</sup> | | | |
| Shigella, treated | | PR | aPR |
| No Shigella, treated | | Ref | Ref |
| Shigella, untreated | | PR | aPR |
| No Shigella, untreated | | Ref | Ref |
| Pathogen 1 <sup>d</sup> | | PR | aPR |
| No Pathogen 1 d | | Ref | Ref |
| Pathogen 2 <sup>d</sup> | | PR | aPR |
| No Pathogen 2 <sup>d</sup> | | Ref | Ref |
| Pathogen 3 <sup>d</sup> | | PR | aPR |
| No Pathogen 3 <sup>d</sup> | | Ref | Ref |
| Pathogen 4 <sup>d</sup> | | PR | aPR |
| No Pathogen 4 <sup>d</sup> | | Ref | Ref |
| Other attributable pathogen <sup>e</sup> | | PR | aPR |
| Other attributable pathogen not present <sup>e</sup> | | Ref | Ref |
| Hospitalization <sup>f</sup> | | | |
| Shigella, treated | | RR | aRR |
| No Shigella, treated | | Ref | Ref |
| Shigella, untreated | | RR | aRR |
| No Shigella, untreated | | Ref | Ref |
| Pathogen 1 <sup>d</sup> | | RR | aRR |
| No Pathogen 1 d | | Ref | Ref |
| Pathogen 2 <sup>d</sup> | | RR | aRR |
| No Pathogen 2 <sup>d</sup> | | Ref | Ref |
| Pathogen 3 <sup>d</sup> | | RR | aRR |
| No Pathogen 3 <sup>d</sup> | | Ref | Ref |
| Pathogen 4 <sup>d</sup> | | RR | aRR |
| No Pathogen 4 <sup>d</sup> | | Ref | Ref |
| Other attributable pathogen <sup>e</sup> | | RR | aRR |
| Other attributable pathogen not present <sup>e</sup> | | Ref | Ref |
| Subsequent Diarrhea Episodes <sup>g</sup> | | | |
| Shigella, treated | | RR | aRR |
| No Shigella, treated | | Ref | Ref |
| Shigella, untreated | | RR | aRR |
| No Shigella, untreated | | Ref | Ref |
| Pathogen 1 <sup>d</sup> | | RR | aRR |
| No Pathogen 1 d | | Ref | Ref |
| Pathogen 2 <sup>d</sup> | | RR | aRR |
| No Pathogen 2 <sup>d</sup> | | Ref | Ref |
| Pathogen 3 <sup>d</sup> | | RR | aRR |
| No Pathogen 3 <sup>d</sup> | | Ref | Ref |
| Pathogen 4 <sup>d</sup> | | RR | aRR |
| No Pathogen 4 <sup>d</sup> | | Ref | Ref |
| Other attributable pathogen <sup>e</sup> | | RR | aRR |
| Other attributable pathogen not present <sup>e</sup> | | Ref | Ref |

CI: 95% confidence interval, MAD: Medically-attended diarrhea, PR: prevalence ratio, RR: Relative risk.

<sup>&</sup>lt;sup>a</sup> Adjusted only for enrollment site

<sup>&</sup>lt;sup>b</sup> Adjusted for enrollment site, age, maternal education, breastfeeding history, and wealth quintile.

<sup>&</sup>lt;sup>c</sup> Persistence is defined by having 14 or more days of diarrhea during the index diarrhea episode.

<sup>&</sup>lt;sup>d</sup> Pathogens selected based on top five prevalent attributable pathogens by qPCR in the study population.

<sup>&</sup>lt;sup>e</sup>Includes [list qPCR available attributable pathogens excluding those listed in pathogens 1-4].

f Includes any hospitalizations in the month three follow-up period including during the child's index diarrhea episode prior to enrollment, at enrollment, within the child's index episode after enrollment, and after resolution of the index episode.

<sup>&</sup>lt;sup>g</sup> A subsequent diarrhea episode is defined as one or more days of three or more loose stools following two diarrhea-free days after the index diarrhea episode. Pathogen comparisons refer to the pathogen present at the child's index diarrhea episode and pathogen presence for the subsequent episode is unknown.



## Table 3.4: Risk of hospitalization stratified by during index episode and after index episode

**Table 3.4.** Risk of hospitalization during and following the resolution of a MAD episode stratified by leading attributable causes of the index MAD.

| | RR (CD | |
|---|---|---|
| (%) N/u | Semi-Unadjusted <sup>a</sup> | Adjusted <sup>b</sup> |
| Hospitalizations during the index diarrhea episode | | |
| Shigella, treated <sup>c</sup> | RR | aRR |
| No <i>Shigella</i> , treated <sup>c</sup> | Ref | Ref |
| Shigella, untreated <sup>c</sup> | RR | aRR |
| No <i>Shigella</i> , untreated <sup>c</sup> | Ref | Ref |
| Pathogen 1c | RR | aRR |
| No Pathogen 1 ° | Ref | Ref |
| Pathogen 2 <sup>c</sup> | RR | aRR |
| No Pathogen 2 ° | Ref | Ref |
| Pathogen 3 <sup>c</sup> | RR | aRR |
| No Pathogen 3 <sup>c</sup> | Ref | Ref |
| Pathogen 4 <sup>c</sup> | RR | aRR |
| No Pathogen 4 c | Ref | Ref |
| Other attributable pathogen <sup>d</sup> | RR | aRR |
| Other attributable pathogen not present <sup>d</sup> | Ref | Ref |
| Hospitalizations following resolution of index diarrhea episode | | |
| Shigella, treated <sup>c</sup> | RR | aRR |
| No <i>Shigella</i> , treated <sup>c</sup> | Ref | Ref |
| Shigella, untreated <sup>c</sup> | RR | aRR |
| No Shigella, untreated <sup>c</sup> | Ref | Ref |
| Pathogen 1 <sup>c</sup> | RR | aRR |
| No Pathogen 1 ° | Ref | Ref |
| Pathogen 2° | RR | aRR |
| No Pathogen 2 c | Ref | Ref |
| Pathogen 3 <sup>c</sup> | RR | aRR |
| No Pathogen 3 <sup>c</sup> | Ref | Ref |
| Pathogen 4° | RR | aRR |
| No Pathogen 4 c | Ref | Ref |
| Other attributable pathogen <sup>d</sup> | RR | aRR |
| Other attributable pathogen not present <sup>d</sup> | Ref | Ref |

CI: 95% confidence interval, ETEC: Enterotoxigenic E. coli, MAD: Medically-attended diarrhea, RR: Relative risk.


<sup>&</sup>lt;sup>a</sup> Adjusted only for enrollment site

<sup>&</sup>lt;sup>b</sup> Adjusted for enrollment site, age, maternal education, breastfeeding history, and wealth quintile. <sup>c</sup> Pathogens selected based on top five prevalent attributable pathogens by qPCR in the study population.

<sup>&</sup>lt;sup>d</sup> Includes [list qPCR available attributable pathogens excluding those listed in pathogens 1-4].



### Table 3.5: Mean change in LAZ/HAZ

**Table 3.5** Mean change in LAZ/HAZ and difference in LAZ/HAZ from enrollment to week four and enrollment to month three among participants by presence of leading etiologies of the index MAD.

| | | Mean ALAZ/HA | Mean ALAZ/HAZ from enrollment to: | enroll | enrollment to: |
|---|---|---|---|---|---|
| Species | n/N (%) | Week four (SD) | Month three (SD) | Week four (CI) <sup>a</sup> | Week four (CI) <sup>a</sup> Month three (CI) <sup>a</sup> |
| Shigella, treated <sup>c</sup> | | | | | |
| No Shigella, treated <sup>c</sup> | | | | Ref | Ref |
| Shigella, untreated <sup>c</sup> | | | | | |
| No Shigella, untreated <sup>c</sup> | | | | Ref | Ref |
| Pathogen 1 <sup>c</sup> | | | | | |
| No Pathogen 1 ° | | | | Ref | Ref |
| Pathogen 2° | | | | | |
| No Pathogen 2 ° | | | | Ref | Ref |
| Pathogen 3 <sup>c</sup> | | | | | |
| No Pathogen 3° | | | | Ref | Ref |
| Pathogen 4° | | | | | |
| No Pathogen 4 c | | | | Ref | Ref |
| Other attributable pathogen d | | | | | |
| Other attributable pathogen not present <sup>d</sup> | p. | | | Ref | Ref |
| CI: 95% confidence interval, HAZ: Height-for-age z-score, LAZ: Length-for-age z-score, MAD: Medically-attended diarrhea, SD: standard | leight-for-age z | -score, LAZ: Length- | -for-age z-score, MAD: 1 | Medically-attended di | arrhea, SD: standar |
| deviation | | | | | |

<sup>&</sup>lt;sup>a</sup> Adjusted for site, age, sex, maternal education, breastfeeding history, wealth quintile, baseline LAZ/HAZ, and days from enrollment to follow-


<sup>&</sup>lt;sup>b</sup> Pathogens selected based on top five prevalent attributable pathogens by qPCR in the study population. <sup>c</sup> Includes [list qPCR available pathogens excluding those listed in pathogens 1-4].



Table 3.6: Prevalence of stunting

Table 3.6. Prevalence of stunting at enrollment, week four follow-up, month three follow-up and association between diarrhea etiology and stunting among children by presence of leading etiologies of the index MAD.

| and stunting annoting children by presence of teaching chologies of the index party. | reading chologies c | TIME TIMES INTO | | | | |
|---|---|---|---|---|---|---|
| | Enrollment | Weel | Week four | Month three | three | i |
| | n/N (%) | n/N (%) | $aPR^a$ (CI) | (%) N/u | aPR <sup>a</sup> (CI) | |
| Shigella, treated <sup>c</sup> | | | | | | 1 |
| No Shigella, treated <sup>c</sup> | | | Ref | | Ref | |
| Shigella, untreated <sup>c</sup> | | | | | | I |
| No Shigella, untreated <sup>c</sup> | | | Ref | | Ref | |
| Pathogen 1 <sup>c</sup> | | | | | | I |
| No Pathogen 1 ° | | | Ref | | Ref | |
| Pathogen 2 <sup>c</sup> | | | | | | ı |
| No Pathogen 2 ° | | | Ref | | Ref | |
| Pathogen 3 <sup>c</sup> | | | | | | |
| No Pathogen 3 <sup>c</sup> | | | Ref | | Ref | |
| Pathogen 4 <sup>c</sup> | | | | | | |
| No Pathogen 4 ° | | | Ref | | Ref | |
| Other attributable pathogen <sup>d</sup> | | | | | | |
| Other attributable pathogen not present <sup>d</sup> | | | Ref | | Ref | |

CI: 95% confidence interval, MAD: medically-attended diarrhea.

<sup>a</sup> Adjusted for site, age, sex, maternal education, breastfeeding history, and wealth quintile. and enrollment LAZ/HAZ (baseline).

<sup>b</sup> Pathogens selected based on top five prevalent attributable pathogens by qPCR in the study population.

<sup>c</sup> Includes [list aPCR available pathogens excluding those listed in pathogens 1-4].




### **Secondary Aim 4**

### Table 4.1: Moderate to Severe MAD by site

| | | Proportion | n of MAD ca | ases meeti | ng severity de | efinitions | : n/N (%) | |
|---|---|---|---|---|---|---|---|---|
| Severity score | Bangladesh | Kenya | Malawi | Mali | Pakistan | Peru | The Gambia | Tota |
| All MAD | | | | | | | | |
| Modified Vesikari score (MVS)a, Median (IQR), n (%) | | | | | | | | |
| Mild illness (0-8 points) | | | | | | | | |
| Moderate illness (9-10 points) | | | | | | | | |
| Severe illness (11+ points) | | | | | | | | |
| Moderate or severe diarrhea by MVS or dysenteryb, n (%) | | | | | | | | |
| GEMS <sup>c</sup> , n (%) | | | | | | | | |
| Moderate-to-severe-diarrhea (MSD) | | | | | | | | |
| Less-severe-diarrhea (LSD) | | | | | | | | |
| GEMS-Shigella scored, Median (IQR), n (%) | | | | | | | | |
| Mild (<6 points) | | | | | | | | |
| Moderate (6-8 points) | | | | | | | | |
| Severe (9+ points) | | | | | | | | |
| Clark score <sup>e</sup> , Median (IQR), n (%) | | | | | | | | |
| Mild (2-8 points) | | | | | | | | |
| Moderate or severe (9+ points) | | | | | | | | |
| MAL-ED score <sup>f</sup> , Median (IQR), n (%) | | | | | | | | |
| Non-severe (<6 points) | | | | | | | | |
| Severe (6+ points) | | | | | | | | |
| Shigella-attributed MAD | | | | | | | | |
| MVS <sup>a</sup> , Median (IQR), n (%) | | | | | | | | |
| Mild illness (0-8 points) | | | | | | | | |
| Moderate illness (9-10 points) | | | | | | | | |
| Severe illness (11+ points) | | | | | | | | |
| Moderate or severe diarrhea by MVS or dysentery <sup>b</sup> , n (%) | | | | | | | | |
| GEMS <sup>c</sup> , n (%) | | | | | | | | |
| MSD | | | | | | | | |
| LSD | | | | | | | | |
| GEMS-Shigella score <sup>d</sup> , Median (IQR), n (%) | | | | | | | | |
| Mild (<6 points) | | | | | | | | |
| Moderate (6-8 points) | | | | | | | | |
| Severe (9+ points) | | | | | | | | |
| Clark score, Median (IQR), n (%) | | | | | | | | |
| Mild (2-8 points) | | | | | | | | |
| Moderate or severe (9+ points) | | | | | | | | |
| MAL-ED score <sup>f</sup> , Median (IQR), n (%) | | | | | | | | |
| Non-severe (<6 points) | | | | | | | | |
| Severe (6+ points) EMS: Global Enteric Multicenter Study, ISD: less severe diarri | | | | | | | | |

GEMS: Global Enteric Multicenter Study, LSD: less-severe-diarrhea, MAL-ED: Malnutrition and Enteric Disease Study, MSD: moderate-to-severe diarrhea, MVS: modified Vesikari score, WHO: World Health Organization.

<sup>a</sup> Defined as in PATH Vesikari Clinical Severity Scoring System Manual: Duration of diarrhea: 1-4 days (1 point), 5 days (2 points) ≥6 days (3 points); Max # of stool in 24 hour period: 1-3 (1 point), 4-5 (2 points), 26 (3 points); Duration of vomiting: 1 day (1 point), 2 days (2 points), 23 days (3 points); max # of vomiting episodes in 24 hour period: 1 (1 point), 2-4 (2 points), 25 (3 points); Axillary temperature 36.6-37.9°C (1 point), 38.0-38.4°C (2 points), 238.5°C (3 points); dehydration 1-5% (2 points), ≥6% (3 points); treatment: rehydration (1 point), hospitalization (2 points).

b Defined as in Pavlinac, Vaccines, 2022 as a MVS of 9+ or presence of visible blood in stool.

e Defined as in Kotloff, Lancet GH, 2019. Moderate-to-severe diarrhea (MSD) defined as presenting to a health facility with diarrhea and severe or some dehydration (by WHO criteria), visible blood in stool, or inpatient admission. Less-severe-diarrhea (LSD) defined as presenting to a health facility without MSD.

<sup>d</sup> Defined as in Pavlinac, CID, 2021. Duration of diarrhea through day of presentation: 1-3 days (0 points), 4-5 days (2 points), ≥6 days (3 points); WHO-defined

dehydration categories: severe (8 points), some (4 points), none (0 points); inpatient admission (5 points).

e Defined as in Clark, JID, 1988. Duration of diarrhea: 1-4 days (1 point), 5-7 days (2 points) > 7 days (3 points); Max # of stool in 24 hour period: 2-4 (1 point), 5-7 (2 points), >7 (3 points); Duration of vomiting: 2 days (1 point), 3-5 days (2 points), >5 days (3 points); max # of vomiting episodes in 24 hour period: 1-3 (1 point), 4-6 (2 points), >6 (3 points); Duration of reported fever: 1-2 days (1 point), 3-4 days (2 points), ≥5 days (3 points); Rectal temperature 38-38.2°C (1 point), 38.3-38.7°C (2 points), ≥38.8°C (3 points); behavioral signs: Irritable/less playful (1 point), Lethargic/listless (2 points), Seizures (3 points).

† Defined as in Lee, J Pediatr Gastroenterol Nutr., 2016: Duration of diarrhea: 2-4 days (1 point), 5-7 days (2 points), ≥8 days (3 points); Max # of stool in 24 hour

period: <5 loose stools/24 hours (1 point), 5-7 loose stools/24 hours (2 points), ≥8 stools/24 hours (3 points); Duration of vomiting: 1 day (1 point), 2 days (2 points),  $\geq$ 3 days (3 points); duration of reported fever: 1+ days (1 point); Confirmed temperature:  $\geq$ 37.5°C (confirmed by field worker) (2 points); Dehydration: Some (2 points), severe (3 points).




## Table 4.2: Clinical characteristics of moderate-to-severe Shigella-attributed MAD

Table 4.2. Clinical characteristics of children with Shigella-attributed diarrhea by GEMS and MVS and/or dysentery. Grey columns highlight discrepant clinical features between the two definitions (and what children would be missed if one definition were chosen and not the other).

| MVS moderate or severe diarrhea +/- dysentery <sup>a</sup> | _ | | • | |
|---|---|---|---|---|
| GEMS MSD <sup>b</sup> | + | 1 | + | |
| Symptom / severity score component | | | | |
| Shigella-attributed MAD (culture or TAC +), N | | | | |
| Hospitalized, n (%) | | | | |
| Dehydration, n (%) | | | | |
| None | | | | |
| Some | | | | |
| Severe | | | | |
| Dysentery, n (%) | | | | |
| Diarrhea duration (days)< Median (IQR) | | | | |
| Maximum number of stools in a 24-hour period, Median (IQR) | | | | |
| Fever, n (%) | | | | |
| Number of days with fever, Median (IQR) | | | | |
| Vomiting, n (%) | | | | |
| Number of days with vomiting, Median (IQR) | | | | |
| Maximum number of vomiting episodes in a 24-hour period, Median (IQR) | | | | |
| ALAZ/HAZ from enrollment to 3-month follow-up, Median (IQR) | | | | |
| CEMS. Clobal Estation Multisometry Birth for any and a room 1 AZ. I mough for any and MOD. and desired a room MOD. and the Mountains distributed to a room MOD. | to to correct discussion I CD: Loca | beilibear NAVA achande dienes | Monitori goon WIIIO. W. | ould Hoolth Ouganization |


GEMS: Global Enteric Multicenter Study, HAZ: Height-for-age z-score, LAZ: Length-for-age z-score, MSD: moderate-to-severe diarrhea, LSD: less-severe-diarrhea, MVS: modified Vesikari score, WHO: World Health Organization.

<sup>a</sup> Defined as in Pavlinac, Vaccines, 2022 as a MVS of 9+ or presence of visible blood in stool.

<sup>b</sup> Defined as in Kotloff, Lancet GH, 2019. Moderate-to-severe diarrhea (MSD) defined as presenting to a health facility with diarrhea and severe or some dehydration (by WHO criteria), visible blood in stool, or inpatient admission. Less-severe-diarrhea (LSD) defined as presenting to a health facility without MSD.



### Table 4.3: Diagnostic accuracy of severity scores

| Table 43. Diagnostic accuracy of dichotomized diarrhea severity scores of identifying hospitalization and/or mortality among all medically attended diarrhea (MAD) and Shigella-attributed MAD during index diarrhea episode. | severity scores of i | dentifying hos | pitalization | and/or mor | tality among a | Il medically a | ttended diarr | hea (MAD) a | nd Shigell | <i>a</i> -attributed | MAD during | index diarrhe | episode. | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Total $(N = )$ | | | | Any antibi | Any antibiotics prescribed $(N = 1)$ | pa | | | No antibio | No antibiotics prescribed $(N = 1)$ | _ | |
| Sensitivity | Sensitivity Specificity Accuracy | Accuracy | PPV | NPV | Sensitivity Specificity Accuracy | Specificity | Accuracy | PPV | Adn | ensitivity | Sensitivity Specificity Accuracy | Accuracy | PPV | NPV |
| | | | (12) | | | | | | | | | | | |
| MVS (moderate or severe) <sup>a</sup> | | | | | | | | | | | | | | |
| MVS (moderate or severe) and/or dysentery <sup>b</sup> | | | | | | | | | | | | | | |
| GEMS (MSD)° | | | | | | | | | | | | | | |
| GEMS-Shigella (moderate or severe) <sup>d</sup> | | | | | | | | | | | | | | |
| Clark score (moderate or severe) <sup>e</sup> | | | | | | | | | | | | | | |
| MAL-ED score (severe) <sup>f</sup> | | | | | | | | | | | | | | |
| Shigella-attributed MAD | | | | | | | | | | | | | | |
| MVS (moderate or severe) <sup>a</sup> | | | | | | | | | | | | | | |
| MVS (moderate or severe) and/or dysentery <sup>b</sup> | | | | | | | | | | | | | | |
| GEMS (MSD) <sup>c</sup> | | | | | | | | | | | | | | |
| GEMS-Shigella (moderate or severe) <sup>d</sup> | | | | | | | | | | | | | | |
| Clark score (moderate or severe) <sup>e</sup> | | | | | | | | | | | | | | |
| MAL-ED score (severe) <sup>f</sup> | | | | | | | | | | | | | | |
| CI: 95% confidence interval. GEMS: Global Enteric Multicenter Study. HAZ, Height-for-age z-score. LAZ: Length-for-age z-score. MAL-ED: Malnutrition and Enteric Disease Study. MSD: moderate-to-severe diarrhea. MVS: | ic Multicenter Stud | lv. HAZ: Heig | ht-for-age z- | score. LAZ: | Length-for-age | z-score. MA | ED: Malnut | rition and En | eric Diseas | e Study, MS | D: moderate-to | -severe diarrh | ea. MVS: | |

CI: 95% confidence interval, GEMS: Global Enteric Multicenter Study, HAZ: Height-for-age z-score, LAZ: Length-for-age z-score, MAL-ELY: Mannutrition and Enteric Disease Suudy, MSD. Incursace-to-severe dualities, 127 v. o. modified Vesikar score, WHO: World Health Organization.

\*Defined as in PATHY vesikaria System Manual as a MVS of 9+.

\*Defined as in Pavlinac, Vaccines, 2022 as a MAM Manual as a MVS of 9+.

\*Defined as in Retoff, Lancet GH, 2019. Moderate-to-severe diarrhea (MSD) defined as presenting to a health facility with diarrhea and severe or some dehydration (by WHO criteria), visible blood in stool, or inpatient admission.

\*Defined as in Pavlinac, CID, 2021 as a score of 9+.

\*Defined as in Clark, JID, 1988 as a score of 9+.

\*Defined as in Clark, JID, 1988 as a score of 6+.




# Table 4.4: Severity scores and relationship to change in LAZ/HAZ from enrollment to three-month follow-up

Table 4.4. Linear regression of dichotomized diarrhea severity scores and ALAZ/HAZ from enrollment to three-month follow-up among all medically attended diarrhea (MAD) and Shigella-attributed MAD. Generalized estimating equations used to account for multiple enrollments of the same child.

| | | Total | | Appropriate a | Appropriate antibiotics prescribed | ribed | No antibi | No antibiotics prescribed | |
|---|---|---|---|---|---|---|---|---|---|
| | | (N=) | | | (N=) | | | (N = ) | |
| Severity score <sup>a</sup> | β (CI) | p-value QIC | ÓIC | β (CI) | p-value QIC | QIC | β (CI) | p-value QIC | ÓIC |
| All MAD | | | | | | | | | |
| MVS (moderate or severe) <sup>b</sup> | | | | | | | | | |
| MVS (moderate or severe) and/or dysentery <sup>c</sup> | | | | | | | | | |
| GEMS (moderate-to-severe diarrhea [MSD]) <sup>d</sup> | | | | | | | | | |
| GEMS-Shigella (moderate or severe) <sup>e</sup> | | | | | | | | | |
| Clark score (moderate or severe) <sup>f</sup> | | | | | | | | | |
| MAL-ED score (severe) <sup>g</sup> | | | | | | | | | |
| Shigella-attributed MAD | | | | | | | | | |
| MVS (moderate or severe) <sup>b</sup> | | | | | | | | | |
| MVS (moderate or severe) and/or dysentery <sup>c</sup> | | | | | | | | | |
| GEMS (MSD) <sup>d</sup> | | | | | | | | | |
| GEMS-Shigella (moderate or severe) <sup>e</sup> | | | | | | | | | |
| Clark score (moderate or severe) <sup>f</sup> | | | | | | | | | |
| MAL-ED score (severe) <sup>§</sup> | | | | | | | | | |
| TO AN A THE LIP CONCLUDE A THE COLOR OF THE COLOR OF THE COLOR | | 134 44 178 1 70 | 1 1 1 1 | .4 | 1 100 | | 1. 1 3.6370 | 1. 11 2.1 121 | |

AIC: Akaike's information Criteria, CI: 95% confidence interval, GEMS: Global Enteric Multicenter Study, MAL-ED: Malnutrition and Enteric Disease Study, MSD: moderate-fo-severe diarrhea, MVS: modified Vesikari score, WHO: World Health Organization.

WHO: World Health Organization.

\*\*Befined as a played for baseline LAZ/HAZ.

\*\*Defined as in PATIVE vesikari its Scoring System Manual as a MVS of 9+.

\*\*Defined as in PATIVE Severity Scoring System Manual as a played in stool.

\*\*Defined as in Pativinac, Vaccines, 2022 as a MVS of 9+ or presence of visible blood in stool.

\*\*Defined as in Rotloff, Lancet GH, 2019. Moderate-to-severe diarrhea (MSD) defined as presenting to a health facility with diarrhea and severe or some dehydration (by WHO criteria), visible blood in stool, or inpatient admission.

<sup>e</sup> Defined as in Pavlinae, CID, 2021 as a score of 9+.

f Defined as in Clark, JID, 1988 as a score of 9+.

B Defined as in Lee, J Pediatr Gastroenterol Nutr., 2016 as a score of 6+.




### Figure 4.1: ROC curves for severity scores

Figure 4.1 (example output below). ROC curve for the four numeric severity scores (MVS, GEMS-Shigella, Clark score, MAL-ED score) on the outcome of hospitalization and/or mortality.



GEMS: Global Enteric Multicenter Study, MAL-ED: Malnutrition and Enteric Disease Study, MVS: modified Vesikari score, ROC; receiver operating characteristic, WHO: World Health Organization.

<sup>b</sup> Defined as in Kotloff, Lancet GH, 2019. Moderate-to-severe diarrhea (MSD) defined as presenting to a health facility with diarrhea and severe or some dehydration (by WHO criteria), visible blood in stool, or inpatient admission. Less-severe-diarrhea (LSD) defined as presenting to a health facility without MSD.

a Defined as in PATH Vesikari Clinical Severity Scoring System Manual: Duration of diarrhea: 1-4 days (1 point), 5 days (2 points) ≥6 days (3 points); Max # of stool in 24 hour period: 1-3 (1 point), 4-5 (2 points), ≥6 (3 points); Duration of vomiting: 1 day (1 point), 2 days (2 points), ≥3 days (3 points); max # of vomiting episodes in 24 hour period: 1 (1 point), 2-4 (2 points), ≥5 (3 points); Axillary temperature 36.6-37.9°C (1 point), 38.0-38.4°C (2 points), ≥38.5°C (3 points); dehydration 1-5% (2 points), ≥6% (3 points); treatment: rehydration (1 point), hospitalization (2 points).
b Defined as in Kotloff, Lancet GH, 2019. Moderate-to-severe diarrhea (MSD) defined as presenting to a health facility with diarrhea and severe or some dehydration

<sup>°</sup>Defined as in Clark, JID, 1988. Duration of diarrhea: 1-4 days (1 point), 5-7 days (2 points) >7 days (3 points); Max # of stool in 24 hour period: 2-4 (1 point), 5-7 (2 points), >7 (3 points); Duration of vomiting: 2 days (1 point), 3-5 days (2 points), >5 days (3 points); max # of vomiting episodes in 24 hour period: 1-3 (1 point), 4-6 (2 points), >6 (3 points); Duration of reported fever: 1-2 days (1 point), 3-4 days (2 points), ≥5 days (3 points); Rectal temperature 38-38.2°C (1 point), 38.3-38.7°C (2 points); ≥38.8°C (3 points); behavioral signs: Irritable/less playful (1 point), Lethargic/listless (2 points), Seizures (3 points).

d Defined as in Lee, J Pediatr Gastroenterol Nutr., 2016: Duration of diarrhea: 2-4 days (1 point), 5-7 days (2 points), ≥8 days (3 points); Max # of stool in 24 hour

d Defined as in Lee, J Pediatr Gastroenterol Nutr., 2016: Duration of diarrhea: 2-4 days (1 point), 5-7 days (2 points), ≥8 days (3 points); Max # of stool in 24 hour period: <5 loose stools/24 hours (1 point), 5-7 loose stools/24 hours (2 points), ≥8 stools/24 hours (3 points); Duration of vomiting: 1 day (1 point), 2 days (2 points), ≥3 days (3 points); duration of reported fever: 1+ days (1 point); Confirmed temperature: ≥37.5°C (confirmed by field worker) (2 points); Dehydration: Some (2 points), severe (3 points).



### **Secondary Aim 5** Table 5.1: Cost per episode of MAD

| Table 5.1. Cost per episode of medically attended A | <i>Shigella</i> diarrhea | a <sup>a</sup> | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | | | | D 2024: Mea | | | |
| | Bangladesh | Kenya | Malawi | Mali | Pakistan | Peru | The Gambia | Total |
| Costing perspective | | | | | | | | |
| Household <sup>b</sup> | | | | | | | | |
| Health system <sup>c</sup> | | | | | | | | |
| Societal <sup>d</sup> | | | | | | | | |
| Visit characteristics <sup>e</sup> | | | | | | | | |
| Visit type | | | | | | | | |
| Inpatient | | | | | | | | |
| Outpatient | | | | | | | | |
| Level of facility presented to | | | | | | | | |
| Primary | | | | | | | | |
| Secondary<br>Tertiary | | | | | | | | |
| Client demographics <sup>e</sup> | | | | | | | | |
| Sex | | | | | | | | |
| Female | | | | | | | | |
| Male | | | | | | | | |
| Age at enrollment (months) | | | | | | | | |
| 6—8 | | | | | | | | |
| 9—11 | | | | | | | | |
| 12—17 | | | | | | | | |
| 18—23 | | | | | | | | |
| 24—35 | | | | | | | | |
| Diarrhea severity <sup>e</sup> | | | | | | | | |
| Dysentery | | | | | | | | |
| Watery diarrhea | | | | | | | | |
| GEMS <sup>f</sup> | | | | | | | | |
| Less-severe diarrhea (LSD) | | | | | | | | |
| Moderate-to-severe diarrhea (MSD) | | | | | | | | |
| Severity by Modified Vesikari score (MVS) <sup>g</sup> | | | | | | | | |
| Mild (0-8 points) | | | | | | | | |
| Moderate (9-10 points) | | | | | | | | |
| Severe (11+ points) | | | | | | | | |
| MVS moderate or severe diarrhea and/or | | | | | | | | |
| dysentery <sup>h</sup> Anthropometry <sup>e</sup> | | | | | | | | |
| Stunted <sup>i</sup> | | | | | | | | |
| Severe | | | | | | | | |
| Moderate | | | | | | | | |
| None | | | | | | | | |
| Wastedi | | | | | | | | |
| Severe | | | | | | | | |
| Moderate | | | | | | | | |
| None | | | | | | | | |
| Underweight <sup>k</sup> | | | | | | | | |
| Severe | | | | | | | | |
| Moderate | | | | | | | | |
| None | | | | | | | | |
| LAZ: Length for age Z-score, LSD: less-severe diarrhea, M | ASD: Moderate-to | <ul> <li>severe diar</li> </ul> | rhea. MVS: M | Iodified Ve | sikari score. N | 1UAC: mi | d-upper arm circu | mference. |

SD: standard deviation, TAC: TaqMan Array Card, USD: US dollars, WAZ: Weight for age Z-score, WHO: World Health Organization, WLZ: Weight for length Z-

<sup>&</sup>lt;sup>a</sup> Children who tested positive for Shigella by culture and/or molecular (TAC) diagnostics.

<sup>&</sup>lt;sup>b</sup> Household perspective includes caregiver out-of-pocket costs and indirect costs (caregiver time lost from work).

<sup>&</sup>lt;sup>c</sup> Health system perspective includes costs of medical treatment funded by the public health system.

<sup>&</sup>lt;sup>d</sup> Societal costs include all costs presented in the household and health system perspectives.

<sup>&</sup>lt;sup>e</sup>Costs stratified per visit characteristic, client demographics, diarrhea severity, and anthropometry category are societal costs.

Defined as in Kotloff, Lancet GH, 2019. Moderate-to-severe-diarrhea (MSD) defined as presenting to a health facility with diarrhea and severe or some dehydration (by WHO criteria), visible blood in stool, or inpatient admission. Less-severe-diarrhea (LSD) defined as presenting to a health facility without MSD.

<sup>&</sup>lt;sup>g</sup> Defined as in PATH Vesikari Clinical Severity Scoring System Manual: duration of diarrhea: 1-4 days (1 point), 5 days (2 points) ≥6 days (3 points); max # of stool in 24 hour period: 1-3 (1 point), 4-5 (2 points),  $\geq$ 6 (3 points); duration of vomiting: 1 day (1 point), 2 days (2 points),  $\geq$ 3 days (3 points); max # of vomiting episodes in 24 hour period: 1 (1 point), 2-4 (2 points), ≥5 (3 points); axillary temperature 36.6-37.9°C (1 point), 38.0-38.4°C (2 points), ≥38.5°C (3 points); dehydration 1-5% (2 points), ≥6% (3 points); treatment: rehydration (1 point), hospitalization (2 points).

h Defined as in Pavlinac, Vaccines, 2022 as a MVS of 9+ or presence of visible blood in stool.

i Severe stunting: LAZ < -3, Moderate stunting:  $-3 \le LAZ < -2$ .

Severe wasting: WLZ < -3 or MUAC < 11.5, Moderate wasting:  $-3 \le$  WLZ < -2 or  $11.5 \le$  MUAC < 12.5.

<sup>&</sup>lt;sup>k</sup> Severely underweight: WAZ < -3, Moderately underweight:  $-3 \le WAZ < -2$ .



Table 5.2: Factors associated with cost

| Table 5.2. Factors associated with costs of medically-attended Shigella diarrhea. <sup>a</sup> | costs of medically | -attended Sh | igella diarrhea | l, a | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | House | Household perspective <sup>b</sup> | ive <sup>b</sup> | Health s | Health system perspective <sup>c</sup> | ective | Societa | Societal perspectived | eq |
| Parameter | Coefficient | $\overline{\mathbf{CI}}$ | p-value | Coeffi | CI | p-value | Coefficient | CI | p-value |
| Intercept | | | | | | | | | |
| Country | | | | | | | | | |
| Bangladesh | Reference - | | ı | Reference - | | 1 | Reference - | | |
| Kenya | | | | | | | | | |
| Malawi | | | | | | | | | |
| Mali | | | | | | | | | |
| Pakistan | | | | | | | | | |
| Peru | | | | | | | | | |
| The Gambia | | | | | | | | | |
| Diarrhea severity | | | | | | | | | |
| Mild | Reference - | | ı | Reference - | | 1 | Reference - | | 1 |
| Moderate | | | | | | | | | |
| Severe | | | | | | | | | |

CI: 95% confidence interval.

<sup>a</sup> Children who tested positive for *Shigella* by culture and/or molecular (TaqMan Array Card) diagnostics.

<sup>b</sup> Household perspective includes caregiver out-of-pocket costs and indirect costs (caregiver time lost from work).

<sup>c</sup> Health system perspective includes costs of medical treatment funded by the public health system.

<sup>d</sup> Societal costs include all costs presented in the household and health system perspectives.




### Table 5.3: Annual costs of Shigella-associated MAD

Table 5.3. Annual costs of medically-attended Shigella diarrhea<sup>a</sup> in country sites.

| | Peru The Gambia | |
|-----------------------------|-----------------|------------------------------|
| SD 2024 | Pakistan | |
| 000 population), USD 202 | Mali | |
| al costs per site (per 100, | Malawi | |
| Annual cos | Kenya | |
| | Bangladesh | |
| | Strata | Household costs <sup>b</sup> |

Health system costs<sup>c</sup>

Societal costs<sup>d</sup>

USD: US dollars.

<sup>a</sup> Children who tested positive for *Shigella* by culture and/or molecular (TaqMan Array Card ) diagnostics. <sup>b</sup> Household costs includes caregiver out-of-pocket costs and indirect costs (caregiver time lost from work). <sup>c</sup> Health system costs includes costs of medical treatment funded by the public health system. <sup>d</sup> Societal costs include all costs presented in the household and health system perspectives.




### **Secondary Aim 6 Table 6.1: Culture Positivity by serotype**

| Table 6.1. Shigella culture po | sitivity proportion by tr | ansport media type and EFGH s | | |
|---|---|---|---|---|
| | | Shigella culture po | ositivity <sup>a</sup> : % (CI) | |
| Country | N " | Cary Blair | mBGS | p-value <sup>b</sup> |
| All Shigella isolates | | | | |
| Bangladesh | | | | |
| Kenya | | | | |
| Malawi | | | | |
| Mali | | | | |
| Pakistan | | | | |
| Peru <sup>c</sup> | | | | |
| The Gambia | | | | |
| Overall | | | | |
| S. flexneri | | | | |
| Bangladesh | | | | |
| Kenya | | | | |
| Malawi | | | | |
| Mali | | | | |
| Pakistan | | | | |
| Peru <sup>c</sup> | | | | |
| The Gambia | | | | |
| Overall | | | | |
| S. sonnei | | | | |
| Bangladesh | | | | |
| Kenya | | | | |
| Malawi | | | | |
| Mali | | | | |
| Pakistan | | | | |
| Peru <sup>c</sup> | | | | |
| The Gambia | | | | |
| Overall | | | | |
| S. boydii | | | | |
| Bangladesh | | | | |
| Kenya | | | | |
| Malawi | | | | |
| Mali | | | | |
| Pakistan | | | | |
| Peru <sup>c</sup> | | | | |
| The Gambia | | | | |
| Overall | | | | |
| S. dysenteriae | | | | |
| Bangladesh | | | | |
| Kenya | | | | |
| Malawi | | | | |
| Mali | | | | |
| Pakistan | | | | |
| Peru <sup>c</sup> | | | | |
| The Gambia | | | | |
| Overall | | | | |

CI: 95% confidence interval, mBGS: modified buffered glycerol saline.

<sup>&</sup>lt;sup>a</sup> Culture *Shigella* culture positivity is defined as the percentage of enrolled participants with *Shigella* isolated from culture out of total participants with both rectal swabs cultured using both Cary-Blair and mBGS transport media.

<sup>&</sup>lt;sup>b</sup> McNemar's test of superiority.

<sup>&</sup>lt;sup>c</sup> Includes only participants enrolled after January 19, 2023 due to a laboratory error that made previous results incomparable across media types.



### Table 6.2: Rectal swab and whole stool comparison

Table 6.2. Shigella culture-positivity from rectal swab and whole stool samples, across sites involved in the whole stool/rectal swab comparison sub-study.

| | | | Shigella culture positivitya: (CI) | |
|---|---|---|---|---|
| Country | N | Rectal swab | Whole stool <sup>b</sup> | Difference |
| All Shigella isolates | | | | |
| Bangladesh | | | | |
| The Gambia | | | | |
| Overall | | | | |
| S. flexneri | | | | |
| Bangladesh | | | | |
| The Gambia | | | | |
| Overall | | | | |
| S. sonnei | | | | |
| Bangladesh | | | | |
| The Gambia | | | | |
| Overall | | | | |
| S. boydii | | | | |
| Bangladesh | | | | |
| The Gambia | | | | |
| Overall | | | | |
| S. dysenteriae | | | | |
| Bangladesh | | | | |
| The Gambia | | | | |
| Overall | | | | |
| CI: 95% confidence ir | nterval | | | |

CI: 95% confidence interval.

<sup>&</sup>lt;sup>a</sup> Shigella culture positivity is defined as the percentage of participants with Shigella isolated from culture out of total participants with both rectal swab and whole stool collected for the Shigella culture comparison.

<sup>&</sup>lt;sup>b</sup> Whole stool is collected among children who produce a sample while still at the enrollment facility.



Enterics for Global Health: Shigella Surveillance Study (EFGH)

### Diarrhea Case Surveillance Case Report Form Appendix



### Table of Contents

| CRF Number | CRF Name |
|------------|-----------------------------------------------------------|
| 01 | Pre-Screening |
| 02 | Screening |
| 03 | Pre-Enrollment |
| 04 | Enrollment |
| 04a | Medical Management |
| 04b | Wealth Index - Bangladesh |
| 04b | Wealth Index - The Gambia |
| 04b | Wealth Index - Kenya |
| 04b | Wealth Index - Malawi |
| 04b | Wealth Index - Mali |
| 04b | Wealth Index - Pakistan |
| 04b | Wealth Index - Peru |
| 04c | HIV Information (Mali, Malawi, Kenya Sites Only) |
| 04d | Daily record (For Participants with Overnight Stays Only) |
| 04e | Referral |
| 05 | Discharge |
| 06 | Diarrhea Diary |
| 07 | Follow-up |
| 08 | Unwell Child |
| 09 | Hospital Record Abstraction |
| 10a | Mortality |
| 10b | Mortality Interview |
| 11 | Study Close Out |
| 12 | Shigella Light Contact |
| 13 | Stool Sample Collection |
| 13b | Home Whole Stool Sample Collection |
| 14 | Blood Sample Collection |
| 18 | Diarrhea Case Surveillance Protocol Violation |
| 19 | Adverse Event |

**Purpose:** To assess screening eligibility.

**Instructions:** Please complete this pre-screening for all children appearing less than 5 years with diarrhea/dysentery/gastroenteritis who present to this health facility at any day/time should have this form completed. Plain text is for prompts for study staff, and *italics* are instructions for study staff.

| cor | completed. Plain text is for prompts for study staff, and italics are instructions for study staff. | | | | | | |
|---|---|---|---|---|---|---|---|
| A. | VISIT INFORMATION | | | | | | |
| | 1. | Screening ID | | | | _ - | ll |
| | | | | (Countr | (Country ID - Facility ID - Sequential Screening # - Staff ID) | | |
| | 2. | Date child presented to h | ealth facility: | | | 2 0 _ | (dd-mm-yyyy) |
| | | | | Unk | nown | | |
| | 3. | Approximate time child p | resented to | _ | | : min, 2 | 4:00 hr) |
| | | health facility: | | Unk | nown | 2 0 | 1/1/1 |
| | 4. | Pre-screening Date: | | 11_ | _ - - : | | |
| | 5. | Pre-screening Time: | | | | | 4:00 hr) |
| | 6. | Based on Q2/Q3 minus Q | | • | | | • |
| | | to the health facility? (if b | | | /60 minutes, indicat | | - |
| | | Unknown (if time of p | | - | | | ii iidais box) |
| | 7. | EFGH country site: | | | | ••• | |
| | / • | Bangladesh | | | | | |
| | | Pakistan | Peru | | The Gambia | Į. | |
| В. | PRE | E-SCREENING QUESTIONS | | | | | |
| | 8. | Did the child present to the recruitment facility during working hours? | | | | | |
| | | ☐ Yes (skip to Q10) | | | | | |
| | | ☐ No | | | | | |
| | 9. | Are the Pre-Screening que | estions being ansv | vered bas | ed on facility record | s or in r | eal-time? |
| | | Real-time | | | | | |
| | | Facility records (only o | applicable for child | dren prese | nting outside of wo | rking ho | urs) |
| | 10. | Please confirm diarrhea/o | lysentery/gastroe | nteritis is | one of the complair | nts of th | e child |
| | | Confirmed | | | | | |
| | | Not confirmed (ineligi | ble, skip to Sectioi | n C) | | | |
| | 11. | Age of the child according | to respondent or | record: | months (i | f outsid | e age range [6-35 |
| | | months], ineligible, skip to | Section C) | | | | |
| | | Missing (ineligible, ski | p to Section C) | | | | |
| | 12. | Is the child still present in | the facility? | | | | |
| | | Yes, the child is still pr | esent in the facilit | ty | | | |
| | | No, the child has alrea | dy left the facility | (ineligibl | e, proceed to Section | 1 C) | |
| | 13. | Is the child currently enro | lled in EFGH and i | nvolved i | n active follow up? | | |
| | | Yes (ineligible because | already enrolled, | , skip to S | ection C, complete U | nwell Cl | hild CRF [CRF 08]) |
| | | ☐ No | | | | | |
| C. | PRE | SCREENING ELIGIBILITY DE | TERMINATION | | | | |

Version: 6.0 (01-11-2022) 

| | 14. | Based on the responses above, is the child eligible t | o move on to the screening process? |
|---|---|---|---|
| | | Yes (complete Section D and continue to Screen | ing CRF [CRF 02]) |
| | | ☐ No (stop process after completing Section D) | |
| D. | D. FORM COMPLETION | | |
| | 15. | ID of person completing this form: | Date form completed: |
| | | | _ - - 2 0 _ (dd-mm-yyyy) |
| | 16. | ID of person reviewing this form: | Date form reviewed: |
| | | | _ - - 2 0 _ (dd-mm-yyyy) |
| | 17. | ID of person entering this form: | Date form entered: |
| | | | _ - - 2 0 _ (dd-mm-yyyy) |
| | 18. | ID of person conducting data verification: | Date of data verification: |


**Purpose:** *To determine study eligibility* 

**Instructions:** Please complete this screening for all children who are preliminarily eligible based on the Pre-Screening form. Plain text is for prompts for study staff, and *italics* are instructions for study staff.

| A. | VISI | T INFORMATION | | | | | |
|---|---|---|---|---|---|---|---|
| | 1. | Screening ID | | -<br>(Count | - - | | |
| | 2. | Screening Date: | | II_ | - | - 2 0 _ | (dd-mm-yyyy) |
| | 3. | Screening Time: | | II_ | : (hh : min, 24:00 hr) | | |
| | 4. | EFGH country site: | | 1 | | | |
| | | Bangladesh | Kenya | | Malawi | | Mali |
| | | Pakistan | Peru | | The Gambia | | |
| В. | RESI | SPONDENT INFORMATION & VERBAL SCREENING CONSENT | | | | | |
| | 5. | Is the child accompanied by a primary caregiver who is able to provide consent? | | | | | |
| | | Yes (conduct verbal screening consent) | | | | | |
| | | ☐ No (thank the respondent and stop screening process, skip to Section G) | | | | | |
| | 6. | What is the relationship of the respondent to the child being screened? | | | | | |
| | | ☐ Biological mother | gical mother | | | Adopt | ed mother |
| | | Adopted father Grandm | | other | other Grandfather | | father |
| | | Aunt Uncle | | | | Older | sister |
| | | Older brother | Other, s | pecify: _ | | | |
| | 7. | Did the respondent conse | nt to screening? | ) | | | |
| | | Yes (skip to Q8) | | | | | |
| | | Not applicable, screer | ing consent is n | ot requir | ed at this site (sk | rip to Q8) | |
| | | No, respondent did no | t provide conse | nt to scr | eening | | |
| | | 7a. If respondent did no | t provide conser | nt to scre | ening, why? | | |
| | | Not interested in skip to Section G) | n participating in | researc | h (thank the resp | ondent and | stop screening process, |
| | | | e (thank the resp | ondent ( | and stop screening | ng process, s | skip to Section G) |
| | | Caregiver too bu | sy (thank the re | sponden | t and stop screen | ing process | s, skip to Section G) |
| | | Child too sick (th | ank the respond | dent and | stop screening p | rocess, skip | to Section G) |
| | | Other (specify): | | | | | |
| | | (thank the responde | nt and stop scre | ening pr | ocess, skip to Sec | tion G) | |


| , | , | Y | | |
|---|---|---|---|---|
| | 8. | What is the [insert site-specific administrative unit] that this child lives in? ("lives" defined as having spent 7 or more days of the last 14 days there) | | |
| | | OR Other (specify): | | |
| | | Please refer to list of smallest administrative units and enter in corresponding code. If list does not | | |
| | | contain administrative unit, indicate "Other" and specify. | | |
| | 9. | Verification that the child lives in the catchment area (using site-specific verification process) | | |
| | | Verified child lives in catchment area | | |
| | | Verified child does not live in catchment area (ineligible) | | |
| | | Could not verify that child lives in catchment area (ineligible) | | |
| C. | BAS | IC INFORMATION ABOUT THE CHILD AND THE PRESENT ILLNESS EPISODE | | |
| | 10. | Child sex | | |
| | | Male | | |
| | | ☐ Female | | |
| | 11. | What is the child's date of birth? | | |
| | | 11a. Day: Unknown | | |
| | | 11b. Month: Unknown | | |
| | | 11c. Year: | | |
| | 12. | (if Day unknown | by study team calculation: mont<br>, assume 15 <sup>th</sup> of the month; if outside age ra | inge [6-35 months], ineligible) |
| | 12 | | le (all unknown; day + month unknown; year<br>according to respondent: month | |
| | 13. | Unknown (if | uknown & Q12 not calculable, ineligible) | |
| | 1.1 | | reported age to determine eligibility if mont | |
| | 14. | - | ually loose or watery stools has the child had | u III tile past 24 flours: |
| | | | 0, put "0" before digit; if < 3, ineligible) | |
| | 15. | | arrhea (defined as 3 or more abnormally loo | se/watery stool in a 24 hour period) start? |
| | | | _ - 2 0 (dd-mm-yyyy) | |
| | 16. | | how many days has the child had diarrhed<br>uring a 24 hour period)? Review memory aid | , - |
| | | days | (if <10, put "0" before digit; if >7 days, inelig | gible) |
| | 17. | Has there been a | any visible blood in the child's stool since the | e diarrhea started? |
| | | Yes | | |
| | | ☐ No (skip to Q | (20) | |
| | 18. | Within the last 2 | 4 hours, has there been visible blood in the | child's stools? |
| | | Yes | | |
| | | ☐ No (skip to Q | 220) | |
| | 19. | Including today, | how many days has the child had visible blo | od in their stools? |
| | | days | (if <10, put "0" before digit) | |


| | 20. | Does the respondent plan to remain in the study area with the child for the next 4 months? |
|---|---|---|
| | | ☐ Yes |
| | | ☐ No (ineligible) |
| | 21. | Is the child currently enrolled in an interventional study? |
| | | Yes (ineligible) |
| | | □ No |
| D. | STU | DY ELIGIBILITY DETERMINATION |
| | 22. | Diarrhea is one of the complaints of the child (see Pre-Screening CRF 01, Q10) |
| | | Yes (must be "Yes" to be eiligible) |
| | | □ No |
| | 23. | Accompanying respondent is able and willing to provide informed consent (see Q5) |
| | | Yes (must be "Yes" to be eiligible) |
| | | □ No |
| | 24. | Child is verified to live in catchment area (see Q9) |
| | | Yes (must be "Yes" to be eiligible) |
| | | □No |
| | 25. | The child is between 6-35 months of age (see Q12 or Q13) |
| | | Yes (must be "Yes" to be eiligible) |
| | | □No |
| | 26. | Child has had 3 or more unusually loose or watery stools in the past 24 hours (see Q14) |
| | | Yes (must be "Yes" to be eiligible) |
| | | □No |
| | 27. | Child has had 7 or fewer days of diarrhea (see Q16) |
| | | Yes (must be "Yes" to be eiligible) |
| | | □ No |
| | 28. | The respondent plans to remain in the study area with the child for the next 4 months (see Q20) |
| | | Yes (must be "Yes" to be eiligible) |
| | | □ No |
| | 29. | Child is <u>not</u> currently enrolled in an interventional study (see Q21) |
| | | Yes (must be "Yes" to be eiligible) |


| | | □ No | |
|---|---|---|---|
| E. | STU | DY ELIGIBILITY DETERMINATION | |
| | 30. | Is the child eligible for enrollment in the EFGH stud | y? (Responses to Q22-29 must all be "Yes") |
| | | Yes | |
| | | ☐ No (thank the respondent and stop screening process, skip to Section G) | |
| F. | отн | ER REASONS NOT ENROLLED (answered among tho | se who are eligible for enrollment) |
| | 31. | Has more than 4 hours passed since the child prese screening process (see Pre-Screening CRF 01, Q6) | ented to the health facility and the child started the |
| | | Yes (thank the respondent and stop screening process, complete Section G) | |
| | | □No | |
| | 32. | Has the enrollment cap already been met? | |
| | | Yes (thank the respondent and stop screening process, complete Section G) | |
| | | □ No | |
| | 33. | Is the child being referred to another facility? | |
| | | Yes, to an EFGH recruiting facility. | |
| | | ID EFGH recruiting facility that child is being referred: (If this child meets eligibility criteria, he/she can continue from the Pre-Enrollment CRF at the referall facility [the screening ID should remain the same]. Thank the respondent and stop the screening process, complete Section G). | |
| | | Yes, to a non-EFGH recruiting facility (thank the Section G) | respondent and stop screening process, complete |
| | | ☐ No (complete Section G and proceed to the info | rmed consent process) |
| G. | FOR | M COMPLETION | |
| | 34. | ID of person completing this form: | Date form completed: |
| | 35. | ID of person reviewing this form: | - - 2 0 (dd-mm-yyyy) Date form reviewed: _ - - 2 0 (dd-mm-yyyy) |
| | 36. | ID of person entering this form: | Date form entered: - - 2 0 (dd-mm-yyyy) |
| | 37. | ID of person conducting data verification: | Date of data verification: |


**Purpose:** To determine whether or not a potential participant was enrolled in the study (among those who were eligible and ready to be enrolled by the Screening Form)

**Instructions:** Please complete this form after a potential participant is deemed eligibile by Screening Form (CRF 02) and potential participant and caregiver have undergone the informed consent process. If a caregiver does not consent, that will be captured in this form. If a child screened eligible, then was referred to another EFGH recruiting facility, that child can be consented at the referred-to EFGH facility and pre-enrollment form completed using the screening ID assigned at the former facility. Plain text is for prompts for study staff, and *italics* are instructions for study staff.

| A. | PRE- | ENROLLMENT INFORMATION |
|---|---|---|
| | 1. | |
| | 2. | Was informed consent obtained from the caregiver? |
| | | Yes |
| | | □ No (skip to Q2b) |
| | | 2a. If yes, date consented: - - 2 0 (dd-mm-yyyy) (skip to Q3) |
| | | 2b. If no, why? |
| | | □ Not interested in participating in research (thank the respondent and stop screening process, skip to Section B) |
| | | ☐ Not enough time (thank the respondent and stop screening process, skip to Section B) |
| | | Caregiver too busy (thank the respondent and stop screening process, skip to Section B) |
| | | Child too sick (thank the respondent and stop screening process, skip to Section B) |
| | | Other (specify): |
| | 3. | (thank the respondent and stop screening process, skip to Section B) Was the child enrolled in the EFGH study? |
| | ٥. | |
| | | Yes (skip to Q5) |
| | | ∐ No |
| | 4. | Why was the child <u>not</u> enrolled in the EFGH study? |
| | | Caregiver withdrew consent (skip to Q6) |
| | | Child was eligible for enrollment but did not continue because of staff/clinic capacity (skip to Q6) |
| | | Child was eligible for enrollment but did not continue because of late timing of enrollment (skip to Q6) |
| | | ☐ Other (specify):(skip to Q6) |
| | 5. | Please assign the next available PID to the participant: |
| | 6. | Has the child been previously enrolled in EFGH? |
| | | Yes |
| | | ☐ No (skip to Section B) |


| | | 6a. | If yes, Previous PID: | _ |
|---|---|---|---|---|
| | | 6b | <i>If yes,</i> Date of enrollment: - - | - 2 0 <u> </u> ( <i>dd-mm-yyyy</i> ) |
| | | 6c. | . If yes, Facility the child recruited from (refer to facility list and enter facility code): | |
| | | | Unknown | |
| В. | FORI | M COMPLETION | | |
| | 7. | ID of | person completing this form: | Date form completed: |
| | | | _ - - 2 0 (dd-mm-yyyy) | |
| | 8. | ID of person reviewing this form: Date form reviewed: | | Date form reviewed: |
| | | - 2 0 (dd-mm-yyyy) | | |
| | 9. | ID of person entering this form: Date form entered: | | |
| | | - - 2 0 (dd-mm-yyyy) | | |
| | 10. | ID of | person conducting data verification: | Date of data verification: |
| | | 1 | 1 1 1 | _ - - 2 0 (dd-mm-yyyy) |

Please proceed to CRF 04 - Enrollment CRF


**Purpose:** To capture information about the enrolled participant at presentation or during the period leading up to presentation to the health facility (subsequent forms will ascertain information about what happens throughout the course of the facility visit). Instructions: Please complete this form after completing the Pre-Enrollment Form and participant been assigned a unique participant identification number (PID). Text in **bold** should be read to study participants, plain text is for prompts for study staff, and italics are instructions for study staff. PLEASE PLACE PARTICIPANT LABEL HERE (OPTIONAL): PARTICIPANT INFORMATION A. |\_\_\_|\_\_| 1. Participant ID \_\_|\_\_| - |\_\_\_| - | 2 | 0 |\_\_\_| (dd-mm-yyyy) 2. Date of Enrollment: \_\_|\_\_| : |\_\_\_| (hh : min, 24:00 hr) Time form is started: 3. 4. EFGH country site: ☐ Bangladesh ☐ Kenya ☐ Malawi □ Mali ☐ Pakistan ☐ Peru ☐ The Gambia DIARRHEA EPISODE INFORMATION (PRESENTATION) (Instructions to staff: Text in **bold** should be read verbatim, plain text is for prompts for study staff, and italics are instructions for study staff. Note: Diarrhea episode is defined as diarrhea (3 or more unusually loose or watery stools in a 24 hour period). Use memory aid to facilitate remembering days. 5. From the time this diarrhea episode started up until now, has there been any visible blood in the child's stool? □ Yes  $\square$  No (skip to Q6) ☐ Unknown (skip to Q6) If Yes, for how many days has there been blood in the child's stool 5a. \_| days (including today)? From the time this diarrhea episode started up until now, what is the maximum number of abnormally loose or 6. watery stools that the child produced in a single 24 hour period? | |loose stools From the time this diarrhea episode started up until now, has the child vomited? 7. □ Yes  $\square$  No (skip to Q8) If the child has had episodes of vomiting, how many 7a. | | days (if <10, put "0" before digit) days has the child vomited at least once?


| | Ĭ | Ţ : | | | <u> </u> | |
|---|---|---|---|---|---|---|
| | | 7b. | Thinking about the day when vomiting, how many times did period? | | 11 | times (if <10, put "0" before digit) |
| | 8. | From th | ne time this diarrhea episode s | tarted up until now, has the | e child felt h | not to the touch (fever)? |
| | | □ Yes | | | | |
| | | □ No (s | skip to Q9) | | | |
| | | 8a. | If child has had a fever during many days did the fever persi | • | 11 | days (if <10, put "0" before digit) |
| C. | MED | ICAL EXA | MINATION: ASSESSMENT OF D | DEHYDRATION AND THE CH | ILD'S GENEI | RAL CONDITION |
| | 9. | What is | the child's general condition? | | | |
| | | □ Well, | /Alert | ☐ Restless/Irritable | | ☐ Lethargic or Unconscious |
| | 10. | Assess t | the child's eyes and determine | if they are: | | de la constantina de |
| | • | □ Norn | nal (skip to Q11) | | ☐ Abnorn | nally sunken |
| | | lf child's eyes are determined to be abnormally sunken, please ask the caregiver: <b>Is the appearance</b> of your child's eyes abnormal? □ Yes (abnormal for child) □ No | | | | ne caregiver: Is the appearance of |
| | 11. | Describ | e the child's ability to drink or b | oreastfeed: | | |
| | | □ Norn | nal/Not Thirsty | ☐ Drinks eagerly/Thirsty | | ☐ Drinks poorly/Unable to drink |
| | 12. | Using a normal | | inch up the child's skin on tl | he abdomin | al wall and assess the skin's return to |
| | | □Imm | ediately | $\square$ 1 to <2 seconds (slowly) | | □ ≥2 seconds (very slowly) |
| | 13. | Dehydration assessment (to be completed based on data in Q9-Q12 above) | | | | |
| | | □ <u>Seve</u> | re dehydration | ☐ Some dehydration | | □ <u>No dehydration</u> |
| | | At least | two of the following signs | At least two of the following signs | | |
| | | (check o | all that apply): | (check all that apply): | | |
| | | ☐ Let | hargic or Unconscious | ☐ Restless/irritable | | |
| | | □Ab | normally sunken eyes based | ☐ Abnormally sunken e | yes based | |
| | | on cli | nician assessment and | on clinician assessment | and | |
| | | careg | iver confirmation | caregiver confirmation | | |
| | | ☐ Dri | nks poorly/unable to drink | ☐ Drinks eagerly/Thirsty | / | |
| | | ☐ Ski | n pinch goes back ≥2 seconds | ☐ Skin pinch goes back | 1 to <2 | |
| | | (very | slowly) | seconds (slowly) | | |
| | | Please assess the following physical signs: | | | | |


| 14. | Vital signs | | | |
|---|---|---|---|---|
| | 14a. Temperature (taken using the Exergen thermometer): . °C | | | |
| | 14b. | Heart rate: beats per minute | | |
| | 14c. | Respiratory rate: breaths per minute | | |
| 15. | Tears | | | □Normal □Decreased □Absent |
| 16. | Jaundi | ce/yellow eyes | | ☐ Yes ☐ No |
| 17. | Cough | | | ☐ Yes ☐ No |
| 18. | Difficu | Ity breathing | | ☐ Yes ☐ No |
| 19. | Chest i | n-drawing | | ☐ Yes ☐ No |
| 20. | Stridor | - | | ☐ Yes ☐ No |
| 21. | Stiff ne | eck | | ☐ Yes ☐ No |
| 22. | Genera | alized rash | | ☐ Yes ☐ No |
| 23. | Runny | nose | | ☐ Yes ☐ No |
| 24. | Convul | lsions | | ☐ Yes ☐ No |
| 25. | Lethar | gy or Unconscious | | ☐ Yes ☐ No |
| 26. | Chest a | auscultation signs suggestive of pneumonia | | ☐ Yes ☐ No |
| 27. | Centra | l cyanosis | | ☐ Yes ☐ No |
| 28. | Oxygen saturation <90% (pulse oximetry) | | ☐ Yes ☐ No ☐ Not available | |
| 29. | Severe respiratory distress | | ☐ Yes ☐ No | |
| 30. | Palmar pallor | | ☐ Yes ☐ No | |
| 31. | Ear pain | | ☐ Yes ☐ No | |
| 32. | Pus drainage from ear canal | | ☐ Yes ☐ No | |
| 33. | Tender | r swelling behind the ear | | ☐ Yes ☐ No |
| 34. | Signs o | of abscess | | ☐ Yes ☐ No |
| 35. | Signs o | of oedema | | ☐ Yes ☐ No |
| | 35a. | If yes: | | |
| | | $\square$ Oedema on both feet/ankles (mild) | | |
| | | ☐ Oedema on both feet/ankles, lower legs, hand | ls, c | or lower arms <i>(moderate)</i> |
| | ☐ Generalized oedema, including both feet, legs, hands, arms, and face (severe) | | | |
| 36. | Tick all diagnoses applicable (check all that apply) | | | |
| | ☐ Diarrhea ☐ Dysentery | | | Dysentery |
| | ☐ Gastroenteritis ☐ Anemia | | Anemia | |
| | ☐ Sickle cell ☐ HIV | | | |
| | Malaria Urinary Tract Infection | | | |
| | Suspected sepsis Tuberculosis | | | |
| | | per respiratory tract infection | | Fever of unknown origin/Febrile illness |
| | | ner lower respiratory tract infections | | Pneumonia |
| | ⊨ ∐∐ ACι | utely unwell, unknown cause | | Meningitis |


| | | | Asthma | Poisoning/ herba | al intoxication |
|---|---|---|---|---|---|
| | | | Moderate acute malnutrition/ moderate wasting | | Inutrition/ severe wasting |
| | | | None | Soft tissue/skin i | |
| | | | Other 1 (specify): | Other 2 (specify) | |
| | | | REMINDER: Record any therapies initiated in | the Medical Manager | ment CRF (CRF 04b) |
| D1. | CHIL | D PRE | SENTATION ANTHROPOMETRY (PRIOR TO ANY REH | YDRATION OR NO RE | HYDRATION REQUIRED) |
| | 37. | Will this child be rehydrated in the facility? | | | |
| | | ПΥ | es and pre-rehydration weight and MUAC able to be | collected (complete S | ections D1, D2 & D3) |
| | | ПΥ | es and pre-rehydration weight and MUAC are NOT at | ole to be collected <i>(co</i> | mplete Section D2 & D3) |
| | | | lo (complete Section D1 & D2, then skip to Q52) | | · |
| | 38. | a. | What is the child's mid upper arm circumference (M measurement) | | . (cm) |
| | | b. Arm from which MUAC is being measured (please ensure the <u>same</u> arm is used to collect 1 <sup>st</sup> , 2 <sup>nd</sup> , and 3 <sup>rd</sup> measurements) | | □ Right □Left | |
| | | C. | What is the child's MUAC? (2 <sup>nd</sup> measurement) | nt) _ . (cm) | |
| | | If measurement 2 differs from measurement 1, subtract the lower measurement from the higher measurement | | | |
| | | and, if the difference is 0.3cm or greater, obtain a third measurement | | | |
| | | d. What is the child's MUAC? (3 <sup>rd</sup> measurement, if applicable) (cm) | | | |
| | | ☐ Not applicable | | | |
| | | (3 <sup>rd</sup> measurement not indicated) | | | |
| | | Comments: | | | |
| | 39. | Hov | v is the child's weight being recorded? | | |
| | | | dult scale, child only (child is ≥24 months OR able to | stand on the scale alo | ne; skip to Q43a) |
| | | ПΑ | dult scale, child and caregiver together (child is <24 r | months OR unable to s | stand on the scale alone) |
| | 40. | а. | What is the weight of child and caregiver (1st measu | ırement) | . (kg) |
| | | b. | What is the weight of the caregiver alone (1st measu | urement) | . (kg) |
| | | c. | What is the <u>calculated</u> weight of the child(Q40a mir | nus Q40b) | . (kg) |
| | 41. | a. | What is the weight of child and caregiver (2 <sup>nd</sup> meason | urement) | (kg) |
| | | b. | What is the weight of the caregiver alone (2 <sup>nd</sup> meas | | . (kg) |
| | | c. | What is the <u>calculated</u> weight of the child <i>(Q41a mi</i> measurement) | | . (kg) |
| | | lj | f measurement 2 (Q41c) differs from measurement 1( | ** | • |
| | | measurement and if the difference is 0.2 kg or greater, obtain a third measurement; otherwise skip to Q44 | | | |


| | 42. | | What is the weight of child and caregiver (3 <sup>rd</sup> measurement) | _ _(kg) |
|---|---|---|---|---|
| | | | | ☐ Not applicable (3 <sup>rd</sup> measurement not indicated) |
| | | b. | What is the weight of the caregiver alone (3 <sup>rd</sup> measurement) | |
| | | D. | what is the weight of the caregiver alone (5.4 measurement) | |
| | | | | measurement not indicated) |
| | | c. | What is the calculated weight of the child (Q42a minus Q42b) (3 <sup>rd</sup> | |
| | | С. | measurement) | □ Not applicable |
| | | | medsarement, | (3 <sup>rd</sup> measurement not indicated) |
| | | Con | nments: | (5 measurement not maleuteu) |
| | | | If the child is ≥24 months AND able to stand on the s | cale alone: |
| | 43. | _ | | |
| | 43. | a. | What is the child's weight? (1st measurement) | . (kg) |
| | | b. | What is the child's weight? (2 <sup>nd</sup> measurement) | . (kg) |
| | | If measurement 2 differs from measurement 1, subtract the lower measurement from the higher measurement if the difference is 0.2 kg or greater, obtain a third measurement | | |
| | c. What is the child's weight? (3 <sup>rd</sup> measurement, if applicable) | | . (kg) | |
| | | | | ☐ Not applicable |
| | | · | | (3 <sup>rd</sup> measurement not indicated) |
| | | Comments: | | |
| D2. | CHILD | LENC | GTH/HEIGHT (All participants, irrespective of rehydration status) | |
| | 44. | Hov | v is the child's length (if <24 months) / height (if ≥24 months) being recorde | ed? |
| | | ☐ Recumbent length (if <24 months) | | |
| | | ☐ Standing height (if ≥24 months and able to stand) | | |
| | | a. | What is the length/height of the child? (1st measurement) | . (cm) |
| | | b. | What is the length/height of the child? (2 <sup>nd</sup> measurement) | . (cm) |
| | | | If measurement 2 differs from measurement 1, subtract the lower | measurement from the higher |
| | | | measurement and if the difference is 0.5 cm or greater, obto | nin a third measurement |
| | | | What is the length/height of the child? (3 <sup>rd</sup> measurement, if applicable) | . (cm) |
| | | c. | | ☐ Not applicable |
| | | | | (3 <sup>rd</sup> measurement not indicated) |


| | | Con | nments: | |
|---|---|---|---|---|
| D3. | | | ST-REHYDRATION ANTHROPOMETRY (complete ONLY if child was rehydrat skip to Section F) | ted [partially or fully] in the facility, |
| | 45. | | s rehydration therapy completed at the facility? | |
| | | □Y | es, child was fully rehydrated at the facility | |
| | | □١ | lo, child was not fully rehydrated and is being sent home with rehydration | therapy (ORS) |
| | 46. | a. | What is the child's MUAC? (1st measurement) | . (cm) |
| | | b. | Arm from which MUAC is being measured | □ Right □Left |
| | | С | What is the child's MUAC? (2 <sup>nd</sup> measurement) | (cm) |
| | | If | measurement 2 differs from measurement 1, subtract the lower measuren | nent from the higher measurement |
| | | | and, if the difference is 0.3 cm or greater, obtain a third | measurement. |
| | | d. | What is the child's MUAC? (3 <sup>rd</sup> measurement, if applicable) | . (cm) |
| | | | | ☐ Not applicable |
| | | (3 <sup>rd</sup> measurement not indicated) | | |
| | | Comments: | | |
| | 47. | Hov | v is the child's weight being recorded? | |
| | | $\square$ Adult scale, child only (child is $\ge$ 24 months AND able to stand on the scale alone; skip to Q51a) | | |
| | | □ A | dult scale, child and caregiver together (child is <24 months OR unable to s | stand on the scale alone) |
| | 48. | a. | What is the weight of child and caregiver (1st measurement) | . (kg) |
| | | b. | What is the weight of the caregiver alone (1st measurement) | . (kg) |
| | | c. | What is the <u>calculated</u> weight of the child (Q48a minus Q48b) | . (kg) |
| | 49. | a. | What is the weight of child and caregiver (2 <sup>nd</sup> measurement) | (kg) |
| | | b. | What is the weight of the caregiver alone (2 <sup>nd</sup> measurement) | . (kg) |
| | | c. | What is the <u>calculated</u> weight of the child_ $(Q49a \text{ minus } Q49b)$ (2 <sup>nd</sup> measurement) | . (kg) |
| | | IJ | measurement 2 (Q49c) differs from measurement 1(Q48c), subtract the lo | |
| | | | measurement and if the difference is 0.2 kg or greater, obtain | |
| | 50. | a. | What is the weight of child and caregiver (3 <sup>rd</sup> measurement) | _ (kg) |
| | | | | ☐ Not applicable |
| | | | | (3 <sup>rd</sup> measurement not indicated) |


| | · | · | | |
|---|---|---|---|---|
| | | b. | What is the weight of the caregiver alone (3 <sup>rd</sup> measure) | ment) . (kg) |
| | | | | ☐ Not applicable |
| | | | | (3 <sup>rd</sup> measurement not indicated) |
| | | c. | What is the calculated weight of the child (Q50a minus | Q50b) (3 <sup>rd</sup> . (kg) |
| | | | measurement) | ☐ Not applicable |
| | | | | (3 <sup>rd</sup> measurement not indicated) |
| | | Con | nments: | |
| | 51. | a. | What is the child's weight? (1st measurement) | . (kg) |
| | | b. | What is the child's weight? (2 <sup>nd</sup> measurement) | _ . (kg) |
| | | lf | measurement 2 (Q51b) differs from measurement 1 (Q52 | La), subtract the lower measurement from the higher |
| | | | measurement and if the difference is 0.2 kg ( | or greater, obtain a third measurement |
| | | c. | What is the child's weight? (3 <sup>rd</sup> measurement, if applica | able) (kg) |
| | | | | ☐ Not applicable |
| | | | | (3 <sup>rd</sup> measurement not indicated) |
| | | Comments: | | |
| F. | | | <b>ALTH HISTORY</b> (Instructions to staff: Text in <b>bold</b> should be italics are instructions for study staff) | e read verbatim, plain text is for prompts for study |
| | 52. | | nere a known or suspected cholera epidemic in the study | area at present? |
| | | □ Y | ′es | |
| | | | No. | |
| | | | Jnknown | |
| | F2 | | | |
| | 53. | | syour child ever been diagnosed with any of the following | |
| | | □F | Rheumatic heart disease | ☐ Leukemia |
| | | | iickle cell anemia | ☐ Tuberculosis |
| | | | HIV | ☐ Other 1 (specify): |
| | | | Other 2 (specify): | ☐ None |
| | | | Breastfeeding Histo | pry |
| | T | | your child ever breastfed? | |
| | 54. | Has | your omia over breastrea. | |
| | 54. | Has<br>□ Y | | |


| | | □ Unknown (skip to Q59) | | | |
|---|---|---|---|---|---|
| | 55. | Other than breastmilk, has your child <u>ever</u> consumed any of the following since their birth? | | | |
| | | Water (fluid) | ☐ Yes | □ No | ☐ Unknown |
| | | Formula (fluid) | ☐ Yes | □ No | ☐ Unknown |
| | | Processed milk (fluid) | ☐ Yes | □ No | ☐ Unknown |
| | | Cow/goat/camel/donkey milk (fluid) | ☐ Yes | □ No | ☐ Unknown |
| | | Sweetened water (fluid) | ☐ Yes | □ No | ☐ Unknown |
| | | Tea (fluid) | ☐ Yes | □ No | ☐ Unknown |
| | | Fruit juice (fluid) | ☐ Yes | □ No | ☐ Unknown |
| | | Porridge (semi-solid food) | ☐ Yes | □ No | ☐ Unknown |
| | | Rice (solid food) | ☐ Yes | □ No | ☐ Unknown |
| | | Other liquid not listed (specify): | ☐ Yes | □ No | □ Unknown |
| | | Other semi-solid foods not listed (specify): | □ Yes | □ No | □ Unknown |
| | | Other solid food not listed (specify): | ☐ Yes | □ No | ☐ Unknown |
| | 56. | Instructions to staff: If the caregiver answered "Yes" to any rows in Q55, skip to Q57. If the caregiver answered "No" to all questions in Q55: According to your answers, your child was exclusion breastfed immediately before (or up until) this diarrheal episode (that is, your child has only ever been go breast milk). If caregiver responds that this statement is incorrect, then correct questions in Q55 to show what child has received other than breastmilk). | | | |
| | | $\square$ Yes, caregiver confirmed that this child was exclus | ively breastfed up un | til this illness episo | de (skip to Q59) |
| | | ☐ No, the caregiver stated this child was not exclusive or more foods and/or fluids marked in Q55 | vely breastfed until th | is illness episode a | nd the child received 1 |
| | 57. | If answered "Yes" to one or more <u>fluids</u> defined in Q55 please ask the caregiver: Thinking about the time immediately before (or up until) this illness episode, how old was your child when they first had fluids other than breastmilk (such as water, tea, formula, or milk)? | | | |
| | | months (if <10, put "0" before digit) □ Ur | nknown | | |
| | 58. | If answered "Yes" to one or more <u>foods</u> defined in Q55 please ask the caregiver: Thinking about the time immediately before (or up until) this illness episode, how old was your child when they first had semi-solid or solid foods (such porridge, rice, or other foods)? | | | |
| | | months (if <10, put "0" before digit) □ Ur | nknown | | |
| | | Immunizatio | on History | | |
| | 59. | Is the child's immunization record available? | | | |
| | | □Yes | | | |
| 1 | 1 | I and the second | | | |

| | | □ No (skip to Q62) | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | Note: If caregiver has access to the child's immunization record but did not bring the immunization record to the | | | | | | |
| | | Enrollment Visit, please remind them to bring it to the Week 4 Follow Up Visit and information will be abstracted in | | | | | | |
| | | Follow Up CRF (CRF 07) | | | | | | |
| | 60. | Using the immunization record, indica | te ho | w many dose | es of the following va | ccines tl | ne child has recei | ved? |
| | | (enter 0 if none, 9 if unknown. If a vac | cine v | was given as | s part of a composite | vaccine | but not alone (e. | g. measles as |
| | | part of MMR or MR vaccine, mark "0" to the component (e.g. measles) and "1" to the composite (MMR) | | | | | | R) |
| | | Rotavirus vaccine | | lI | Bacille Calmette-G | iuerin (E | 3CG) | II |
| | | Polio vaccine (OPV or IPV) | | 11 | Rubella vaccine | | | II |
| | | Pentavalent vaccine (DPT+HiB+HBV) | | 11 | HiB vaccine (Hemo | philus i | influenzae) | II |
| | | S. pneumococcus vaccine (PCV) | | 11 | Hepatitis A vaccino | е | | II |
| | | Measles vaccine | | 11 | Hepatitis B vaccine | 2 | | II |
| | | MR vaccine (measles+rubella) | | 11 | Typhoid fever vac | cine | | II |
| | | MMR vaccine (measles+mumps+rubel | la) | 11 | Varicella vaccine | | | II |
| | | Yellow fever vaccine | | 11 | Meningococcal A | vaccine | | II |
| | | DPT vaccine (Diphteria+pertussis+teta | nus) | 11 | Malaria vaccine (R | TS,S) | | II |
| | 61. | How many doses of Vitamin A has the | child | received? | (enter 9 if un | known) | | |
| | | REMINDER TO MALI, MALAWI, AN | | | • | | Information CRF | (CRF 04c) |
| | | befo | re pro | ceeding with | h the enrollment ques | tions | | |
| | CARE | GIVER INFORMATION (Instructions to s | staff: ` | Text in <b>bold</b> . | should be read verbat | im, plai | n text <i>is for prom</i> | pts for study |
| G. | | and italics are instructions for study sto | | | | | | |
| | 62. | What is the age of the accompanying | caregi | ver? | | | | |
| | | years □ Unknown | | | | | | |
| | 63. | What does the accompanying caregive | er do 1 | for work on | a typical day? | | | |
| | | ☐ Not employed | □ H <sub>ℓ</sub> | ousewife | | ☐ Stud | dent | |
| | | ☐ Business (self-employed) | ☐ Bı | usiness (othe | er employer) | ☐ Pro | fessional (e.g. tea | acher. lawver) |
| | | ☐ Casual laborer | | armer | . , , | □Unk | | · |
| | | ☐ Other (specify):) | | | | | | |
| | 64. | What is the highest level of formal sch | nooling | g achieved h | by the child's mother? | | | |
| | 04. | □ None | | | rimary school | | ☐ Declined to a | ncwor |
| | | | | | | | | iiswei |
| | | ☐ Some secondary school | | | school or greater | | □ Unknown | |
| | | ☐ Koranic school only | Ш | Primary sch | ool only | | | |
| | 65. | What is the highest level of formal sch | oolin | g achieved b | y the child's father? | | | |
| | | □ None | | Less than pr | rimary school | | ☐ Declined to a | nswer |
| | | Some secondary school ☐ Secondary school or greater ☐ Unknown | | | | | | |

| | | ☐ Koranic school only | ☐ Primary school only | |
|---|---|---|---|---|
| | ADD | ITIONAL INFORMATION ON THE CHILD | 'S HOUSEHOLD ENVIRONMENT (Instru | ctions to staff: Text in <b>bold</b> should be |
| Н. | read | verbatim, plain text is for prompts for s | tudy staff, and italics are instructions fo | or study staff) |
| | | Household, Wo | ater, Sanitation, and Hygiene Informa | tion |
| | 66. | How many children under 5 years of a | ge are living in the child's household (i | ncluding this child)? |
| | | _ children under 5 years of age | (if <10, put "0" before digit) | |
| | 67. | What is the main source of drinking w | rater for the members of the household | d (check one) |
| | | ☐ Piped water into dwelling ☐ Piped into compound/yard/plot ☐ Piped to neighbor | | |
| | | ☐ Public tap/standpipe | ☐ Tube well or borehole | ☐ Protected well |
| | | ☐ Unprotected well | ☐ Water from spring (protected) | ☐ Water from spring (unprotected) |
| | | ☐ Rainwater | ☐ Tanker-truck | ☐ Cart with small tank/drum |
| | | ☐ Water kiosk (filtered) | Water kiosk (un filtered) | ☐ Bottled water |
| | | ☐ Sachet water | ☐ Surface water (river/dam/lake/ | ☐ Other (specify): |
| | | | pond/canal/irrigation channel) | |
| | 68. | Does the household do anything to make the water safer to drink? | | |
| | | ☐ Yes ☐ No (skip to Q70) ☐ Unknown (skip to Q70) | | |
| | 69. | If yes, what does the household usual | ly do to make the water safer to drink? | (Check all that apply) |
| | | ☐ Boil | ☐ Add bleach/chlorine | ☐ Solar disinfection |
| | | ☐ Let it stand and settle | ☐ Strain through a cloth | ☐ Filter (ceramic/sand/ |
| | | | | composite/LifeStraw) |
| | | ☐ Other, specify: | | |
| | 70. | | he household is (currently) using for <u>h</u> | <u>vgiene</u> (such as hand-washing, |
| | | showering, or brushing teeth) or cook | | |
| | | ☐ Piped water into dwelling | ☐ Piped into compound/yard/plot | ☐ Piped to neighbor |
| | | ☐ Public tap/standpipe | ☐ Tube well or borehole | ☐ Protected well |
| | | ☐ Unprotected well | ☐ Water from spring (protected) | ☐ Water from spring (unprotected) |
| | | ☐ Rainwater | ☐ Tanker-truck | ☐ Cart with small tank/drum |
| | | ☐ Water kiosk (filtered) | ☐ Water kiosk (unfiltered) | ☐ Bottled water |
| | | ☐ Sachet water | ☐ Surface water (river/dam/lake/ | ☐ Other (specify): |
| | | | pond/canal/irrigation channel) | |
| | 71. | Does the household do anything to m | ake the water safer for hygiene and co | oking? |
| | | ☐ Yes | □ No (skip to Q73) | ☐ Unknown (skip to Q73) |
| | 72. | | ly do to make the water safer for hygie | |
| | | ☐ Boil | ☐ Add bleach/chlorine | ☐ Solar disinfection |
| | | ☐ Let it stand and settle | ☐ Strain through a cloth | ☐ Filter (ceramic/sand/ |
| | | | | composite/LifeStraw) |
| | | ☐ Other (specify): | | |

| | 73. | What kind of toilet facility do members of the household usually use? (Check one) | | | | |
|---|---|---|---|---|---|---|
| | | ☐ Flushed or pour flush to piped | ☐ Flushed or pou | ır flush to septic | ☐ Flushed or po | our flush to |
| | | sewer system | tank | | somewhere els | е |
| | | ☐ Flushed or pour flush, don't know where | ☐ Ventilated imp | roved pit latrine | ☐ Pit latrine wi | th slab floor |
| | | ☐ Pit latrine without slab floor | ☐ Composting toilet | | ☐ Bucket toilet | |
| | | ☐ Hanging toilet/hanging latrine | ☐ Open defecation | on/bush/field | □ Other (specif | fy): |
| | 74. | Does the household share this toilet fa | acility with other h | ouseholds? | | |
| | | ☐ Yes | | | | |
| | | □ No (skip to Q76) | | | | |
| | 75. | How many households use this toilet f | acility? | (if <10, | put "0" before dig | git) □ Unknown |
| | 76. | Please ask the caregiver verbally: Whe | en do you usually v | vash your hands? (c | heck all that apply | ) |
| | | ☐ Before eating ☐ After handling domestic animals | | | | |
| | | ☐ Before cooking | | ☐ After cleaning a | aning a child who defecated | |
| | | ☐ Before you nurse or prepare baby's | food | ☐ After you defec | cate | |
| | | ☐ Never (skip to Q78) | | ☐ Other (specify): | | |
| | 77. | When you wash your hands, what do you usually use? | | | | |
| | | ☐ Water only | | ☐ Water and soap | ) | |
| | | ☐ Water and ashes | | ☐ Water and mud | or clay | |
| | | ☐ Other (specify): | | | | |
| | | REMINDER: Please comple<br>before pro | | Wealth CRF (CRF 04b<br>nrollment questions | -[site specific]) | |
| I. | | R CARESEEKING BEHAVIOR (Instruction | | <b>old</b> should be read v | <i>erbatim,</i> plain tex | t is for prompts for |
| | | staff, and italics are instructions for stu | | | | anima da dha alimia |
| | 78. | During this episode of diarrhea, did yo today? | ou seek any other | medical care for you | ar child before col | ning to the clinic |
| | | □ Yes | | | | |
| | | □ No (skip to Q87) | | | | |
| | 79. | If yes, where did you seek other medi | cal treatment and | how many times? (/ | Not including the d | current clinic visit. |
| | | Check all that were visited and report put "99") | number of times vi | sited. If <10, put "0" | as first digit. If tim | nes visited unknown |
| | | ☐ Traditional healer | _ times | ☐ Religious healer | | _ times |
| | | ☐ Drug seller | _ times | ☐ Pharmacist | | _ times |
| | | ☐ Community health worker | _ times | ☐ Health outpost | | _ times |

| | ☐ Health facility (outpatient ca | re) _ | _ times | □ He | alth facility (in | npatient care) | _ times |
|---|---|---|---|---|---|---|---|
| | ☐ Other (specify): | | | | | times | |
| 80. | Did your child receive any test | s prior to comir | ng to clinic | ? | | | |
| | □ Yes | | | | | | |
| | ☐ No (skip to Q83) | | | | | | |
| <br>81. | If yes, Please indicate from the | list below whi | ch tests yo | ur chil | d received wh | nen you sought | care prior to coming |
| | to the health facility today? | | | | | | |
| | ☐ Stool culture ☐ Microscopy | | | | | | |
| | ☐ Rotavirus antigen test | ☐ Cr | yptosporidiur | m/giardia antige | n test | | |
| | □Other (specify): | | | | | | |
| 82. | If yes, Did you pay for any of the tests your child received? | | | | | | |
| | ☐ Yes, purchased one or more | all were pr | ovided | for free | ☐ Don't know | | |
| 83. | Did your child receive any trea | tment(s) when | you sough | nt care | prior to comi | ng to clinic? | |
| | □ Yes | | | | | | |
| | □ No (skip to Q86) | | | | | | |
| 84. | If yes, Please indicate from the | list below which | ch treatme | ents yo | ur child recei | ved when you so | ought care prior to |
| | coming to the health facility to | day? (check all | that apply | ′) | | | |
| | ☐ Oral rehydration solution (O | RS) | □ Zinc | | | ☐ Anti-diarrhe | al |
| | ☐ RUSF or locally made supple | mentary food | ☐ ReSo | oMal | ſal □ Anti-malarial | | |
| | ☐ Albendazole | | □ Meb | endazo | ndazole | | |
| | ☐ Other 1 (specify): | | ☐ Othe | er 2 <i>(sp</i> | 2 (specify): | | |
| | ☐ Antibiotic(s) (specify below, | check all that a | oply) | | | | |
| | ☐ Amoxicillin | ☐ Azithromyo | cin | | Ampicillin | | gmentin/<br>noxiclav |
| | ☐ Ceftriaxone | ☐ Ciprofloxad | in (Cipro) | | Cefuroxime | □ Ce | fixime |
| | ☐ Clarithromycin | ☐ Clindamyci | n | | Chlorampheni | icol 🗆 Co | trimoxazole (Septrin) |
| | ☐ Doxycycline | ☐ Erythromy | cin | | Gentamicin | □ Pe | nicillin |
| | ☐ Pyrazinamide | ☐ Streptomy | cin | □1 | etracycline | □Ur | known |
| | ☐ Other 1 (specify): | ☐ Other 2 (sp | ecify): | | Other 3 (speci | fy): | |
| 85. | Did you purchase any of these | treatments? | | | | | |
| | ☐ Yes, purchased them | | | | No, they we | ere provided for | free |
| | ☐ No, received leftover medica | itions from som | eone else | | ☐ Do not recall | | |
| <br>86. | Once you made the decision to from someone? | seek care outs | side the ho | ouseho | ld for your ch | ild, did you nee | d to seek permission |
| 1 | | | | | | | |

| | | ПΥ | es | | | | |
|---|---|---|---|---|---|---|---|
| | | | lo (skip to Q87) | | | | |
| | | 86a. | If yes, from whom (check all that | t apply): | | | |
| | | | ☐ Head of household | | | ☐ Other house | ehold member |
| | | | ☐ Family member outside of the | household | | ☐ Community | leader |
| | | | ☐ Religious leader | | | ☐ Pharmacist | or drug seller |
| | | | ☐ Other (specify): | | | | |
| J. | INFORMATION ON COST OF VISIT AND TRANSPORTATION TO THE FACILITY (Instructions to staff: Text in bold should be | | | | | | |
| J. | read | verbo | atim, plain text is for prompts for s | tudy staff, and ita | alics ar | re instructions f | or study staff) |
| | 87. | Approximately how much time did it take you and this child to get to the health facility today? (if <10, put "0" | | | | | |
| | | before digit) | | | | | |
| | | days OR | | | | | |
| | | _ uays On _ llouis On _ llillilutes 🗆 Doll t know | | | | | |
| | 88. | What method of transportation did you and your child use to travel to the facility? (check all that apply) | | | | | |
| | | □V | Valked | ☐ Motorbike | | | ☐ Private or shared car |
| | | □ P | ersonal vehicle | ☐ Shared van/b | ous/tax | ti | ☐ Other (specify): |
| | 89. | Арр | roximately how much did you pa | y for your transp | ortatio | on to the clinic | for this visit? (If personal vehicle |
| | | repo | orted in Q88, include cost of gas; re | eport cost numeri | ically i | n local currency | ; if none, put "0") |
| | | | □Unknow | n | | | |
| к. | FOR | м со | MPLETION | | | | |
| | 90. | ID o | of person completing this form: | 1 1 1 | Date | form complete | d: |
| | | | <u> </u> | '' | | • | 2 0 _ <i>(dd-mm-yyyy)</i> |
| | 91. | ID o | f person reviewing this form: | _ | Date | form reviewed | : |
| | | | | | _ | - - | 2 0 <u> </u> <i>(dd-mm-yyyy)</i> |
| | 92. | ID o | of person entering this form: | | Date | form entered: | |
| | | | | | | - - | 2 0 <u> </u> (dd-mm-yyyy) |
| | 93. | ID o | f person conducting data verificat | ion: | Date | of data verifica | tion: |
| | | | | | | - - | 2 0 <i>(dd-mm-yyyy)</i> |

**Purpose:** To ascertain information on clinical management during the enrollment facility visit for all enrolled participants from the point of presentation through the point of being ready to leave the facility/discharge. Instructions: Please complete the following information for all enrolled participants. Text in **bold** should be read to study participants, plain text are prompts for study staff, and italics are instructions for study staff. This form will remain open throughout the entirety of the child's stay during their enrollment visit. PLEASE PLACE PARTICIPANT LABEL HERE (OPTIONAL): A. **PARTICIPANT INFORMATION** 1. Participant ID 2. Date of Enrollment: |:|\_\_\_| (hh: min, 24:00 hr) 3. Time form is started: 4. EFGH country site: ☐ Bangladesh ☐ Malawi ☐ Mali ☐ Kenya ☐ The Gambia □ Peru ☐ Pakistan В. **ADMISSION INFORMATION** Was the child admitted to an inpatient ward (i.e. for an overnight stay) during this visit? 5. ☐ Yes Date of admission: |\_\_\_| - |\_\_ | - | 2 | 0 |\_\_\_| (dd-mm-yyyy) ☐ Same as date of enrollment (Q2) Time admitted to inpatient ward: |\_\_\_| : |\_\_\_| (hh : min, 24:00 hr) □Unknown (skip to Section C) □ No Was the child primarily seen in: ☐ Outpatient ward ☐ Emergency room  $\square$  Other (specify): C. DIAGNOSTIC TESTS RECEIVED DURING FACILITY VISIT 7. Did the child receive any of the following stool tests during their facility visit? (check all that apply) ☐ Stool culture (SEPARATE from culture planned for EFGH) ☐ Microscopy ☐ Rotavirus antigen test ☐ Cryptosporidium/giardia antigen test ☐ Other (*specify*): □ None MEDICAL MANGEMENT DURING FACILITY VISIT AND PRESCRIBED FOR DISCHARGE PERIOD D. To the staff completing this form: Are you one of the treating clinicians?

| | <ul><li>☐ Yes, I am part of this child's clinical team</li><li>☐ No, I am abstracting this information from the child's medical record</li></ul> | | |
|---|---|---|---|
| <br>9. | | Was oral rehydration solution (ORS) or ReSoMal (half strength ORS) administered during the visit? | |
| <br>J. | □ Yes | | |
| | ☐ No, child received other rehydration therapy (skip to Q10) | | |
| | | , not necessary for this child (skip to Q10) | ~/ |
| | | , not available due to stock out (skip to Q10) | |
| | □ No | , specify) | (skip to Q10) |
| | 9a. | Type of oral rehydration initiated: | |
| | | ☐ Low osmolarity ORS solution | |
| | | (Glucose: 75mmol, Sodium: 75 mmol, Chloride: 6 | 55mmol, Potassium: 20mmol) |
| | | icddr,b ORS solution | g, Sodium citrate: 1.45 g, Anhydrous Glucose: 6.75 g) |
| | | □ ReSoMal/Half-strength ORS | g, Soutum citiate. 1.43 g, Annyurous Giucose. 6.73 g) |
| | | (Glucose: 125mmol, Sodium: 45 mmol, Chloride: | 70mmol, Potassium: 40mmol) |
| | | ☐ High osmolarity (original formulation) ORS | , |
| | (Glucose: 111mmol, Sodium:90 mmol, Chloride: 80mmol, Potassium: 20mmol) | | |
| | □ Other (specify type & composition): | | |
| | 9b. | How was it administered: ☐ Orally ☐ Nasogastr | rically |
| | 9c. Date ORS or ReSoMal initiated: - - 2 0 (dd-mm-yyyy) | | |
| <br> | | ☐ Same as date of enrollment (Q2) | |
| | 9d. | Time ORS or ReSoMal initiated: : | |
| | 9e. | Date ORS or ReSoMal completed: - - | |
| | 9f. | ☐ Same as date of enrollment (Q2) ☐ Continuir Time ORS or ReSoMal completed: : | |
| | <i>J</i> 1. | ☐ Continuing ☐ Unknown | |
| | 9g. | <u> </u> | (hrs) (Auto-generated from date/time of |
| | | initiation to date/time of completion. If $<10$ , put | 0 before the last digit ie 4 hours would be "04") |
| | 9h. | If answer to 9g is less than 4 hours: Why? | |
| | | $\square$ Caregiver did not want to remain in the facility | y |
| | | ☐ Other (specify): | |
| | 9i. | Total number of packets of ORS or ReSoMal offered to the child during visit: | □ Unknown |
| | Ωi | What volume of water was each packet mixed | ☐ Not applicable (ie packets not used) mL (note standard is 1,000 mL) |
| | 9j. | with: | ☐ Unknown |
| | 9k. | Total volume of ORS or ReSoMal offered to the | mL |
| | | child during the visit: | (autogenerated as # packets × volume water mixed |
| | 0, | W II | with packet) |
| | 91. | Was there any mixed ORS/ReSoMal remaining that the child did not drink? | ☐ Yes ☐ No (skip to Q9o) |

| <br>Ī | _ | \A/I | |
|---|---|---|---|
| | 9m. | What volume was left over that the child did not drink? | mL |
| | 9n. | Total volume of ORS or ReSoMal consumed by | |
| | | the child during the visit: | (autogenerated as volume offered – volume |
| | | | remaining or volume offered if none remained) |
| | 9o. | Was the ORS administered during the facility visit | provided by the health facility (free of charge) or did |
| | | the caregiver need to buy it either at the health f | acility or elsewhere? |
| | | $\square$ Provided free by facility or national health insu | rance |
| | | ☐ Provided by EFGH | |
| | | $\square$ Caregiver needed/needs to buy it either at the | health facility or elsewhere |
| | | ☐ Other (specify): | |
| | | □ Unknown | |
| <br>10. | Wher | the child was ready to leave or was discharged, w | as the child instructed to continue oral rehydration |
| | treatr | ment at home? | |
| | ☐ Yes | S | |
| | □ No | (skip to Q11) | |
| | | If yes, please provide counseling to the caregiver | on how to prepare and deliver the ORS |
| | 10a. | How many packets of at-home ORS were prescrib | ped? . packets |
| | | | (half packets can be indicated with ".5") |
| | | | ☐ Unknown |
| | | | ☐ Not applicable (i.e. packets not used) |
| | 10b. | Was the prescribed ORS/ReSoMal for the disch | narge period provided by the health facility (free of |
| | | charge), or does the caregiver need to buy the OF | RS/ReSoMal at the health facility or elsewhere? |
| | | $\square$ Provided free by facility or national health insu | rance |
| | | ☐ Provided by EFGH | |
| | | $\square$ Caregiver needed/needs to buy it either at the | health facility or elsewhere |
| | | ☐ Other (specify): | |
| | | □ Unknown | |
| 11. | Was I | V rehydration administered during the visit? | |
| | ☐ Yes | S | |
| | □ No | , contraindication (skip to Q12) | |
| | □ No | , child received other rehydration therapy (skip to | Q12) |
| | | , not necessary for this child (skip to Q12) | , |
| | | , not available due to stock out (skip to Q12) | |
| | | , specify: | (skip to Q12) |
| | | Type of IV (check all administered): | ( |
| | 11a. | ☐ Normal saline ☐ Dextrose ☐ Ringer's lactate so | lution □Cholera saline□ Other (specify): |
| | 11b. | Date IV rehydration initiated: - | - 2 0 (dd-mm-yyyy) |
| | | ☐ Same as date of enrollment (Q2) | |
| | 11c. | Time IV rehydration initiated: : | <i>(hh : min, 24:00 hr)</i> □ Unknown |
| | 11d. | Date IV rehydration completed: - | - 2 0 (dd-mm-yyyy) |
| | | ☐ Same as date of enrollment (O2) | |

| | 11e. Time IV rehydration completed: : (hh : min, 24:00 hr) □ Continuing □ Unknown | | |
|---|---|---|---|
| | 11f. | Duration of IV rehydration (hrs) (Auto-generated ) | from date/time of initiation to date/time |
| | 111. | of completion. If <10, put 0 before the last digit ie 4 hours wo | |
| | 11g. | Size of one IV bag: mL (if between 1-999, put "0999") | |
| | 118. | If multiple IVs were administered, report volume of the average of all IVs administered. | |
| | 11h. | Total number of IV bags received: . □ Unknown | · |
| | 11i. | Total volume administered during visit: n of each bag but can be edited by staff. If between 1-999, put | |
| | | ☐ Unknown | 0999 / |
| | 11j. | Was the IV(s) administered during the facility visit provided b | y the health facility (free of charge) or did |
| | 11). | the caregiver need to buy it either at the health facility or else | |
| | | IVs administered) | ewilete. (effect all that apply if mattiple |
| | | ☐ Provided free by facility or national health insurance | |
| | | ☐ Provided by EFGH | |
| | | ☐ Caregiver needed/needs to buy it either at the health facili | ty or elsewhere |
| | | ☐ Other (specify): | |
| | | □ Unknown | |
| 12. | Was z | inc supplementation administered during the visit? | ☐ Yes ☐ No (skip to Q13) |
| | 12a. | Date zinc initiated: - - 2 0 _ | (dd-mm-yyyy) |
| | | ☐ Same as date of enrollment (Q2) | |
| | 12b. | Date zinc completed: - - 2 0 | |
| | | $\square$ Same as date of enrollment (Q2) $\square$ Continuing $\square$ Unknow | |
| | 12c. | Amount of zinc administered per day during facility visit: (If child vomited after receiving zinc and another dose was ad | |
| | | dose) | ministered consider only the post volint |
| | 12d. | Was the zinc administered during the facility visit provided by | |
| | | the caregiver need to buy it either at the health facility or else | ewhere? |
| | | ☐ Provided free by facility or national health insurance ☐ Provided by EFGH | |
| | | • | tu or alsowhere |
| | | ☐ Caregiver needed/needs to buy it either at the health facili | |
| | | ☐ Other (specify): | |
| <br>12 | \ | | : |
| <br>13. | | the child was ready to leave or was discharged, was the child | instructed to take zinc at nome: |
| | ☐ Yes | | |
| | | , contraindicated (skip to Q14) | |
| | | , received other nutritional product (skip to Q14) | |
| | | not necessary for this child (skip to Q14) | |
| | | , not available due to stock out (skip to Q14) | (11 - 21) |
| | ⊔ No | other reason (specify): | (skip to Q14) |
| | 13a. | What was the prescribed daily dose of at-home zinc supplementation? | mg |
| | 401 | What was the prescribed duration of at-home zinc | |
| | 13b. | supplementation? | days □ Unknown |

| | 13c. Was the prescribed zinc for the discharge period provided by the health facility (free of charge) or does the caregiver need to buy the zinc either at the health facility or elsewhere? | | | | |
|---|---|---|---|---|---|
| | ☐ Provided free by facility or national health insurance | | | | |
| | ☐ Provided by EFGH | | | | |
| | ☐ Caregiver needed/needs to buy it either at the health facility or elsewhere | | | | |
| | | ☐ Other (specify): | • | • | |
| | | ☐ Unknown | | | |
| 14. | Were | supplementary or therapeu | itic foods administered | during the visit? | |
| | ☐ Yes | s (skip to Q16) | | | |
| | □ No | (skip to Q18) | | | |
| | ☐ Un | known | | | |
| 15. | If Unk | known, why? | | | |
| | | | andled by a separate u | nit & records are not availab | |
| | | her (specify): | ., | | (skip to Q18) |
| 16. | Kow | is below refer to supplement | tary or therapeutic food<br>visi | ds and micronutrients admin<br>it | istered during the facility |
| | Name (check box if administered) Date initiated Daily dose administered during Date completed | | | | |
| | (dd-mm-yyyy) facility visit (circle unit) (dd-mm-yyyy) | | | | |
| | □F75 (in-patient cases only) - - mL - | | | | |
| | □F100 (in-patient cases only) | | | | |
| | □RUS | F | - -<br> 2 0 | (mg/gram/sachet) | |
| | | | | ☐ Unknown | ☐ Continuing |
| | | | - - | (mg/gram/sachet) | - - |
| | □RUT | F | 2 0 | Unknown | ☐ Continuing |
| | | | 1 1 1 1 1 | | - - - - |
| | □RUS | F (locally made) | 2 0 | (mg/gram/sachet) | 2 0 _ |
| | | | | □ Unknown | ☐ Continuing |
| | □RUT | F (locally made) | _ - - - - | (mg/gram/sachet) | 2 0 |
| | | | 2 0 | ☐ Unknown | ☐ Continuing |
| | | | | (1 | _ - |
| | ⊔Mul | tiple micronutrients | 2 0 | (mg/gram/sachet) ☐ Unknown | 2 0 <br> Continuing |
| 17 | Were | the foods or micronutrients | administered during t | he facility visit provided by t | |
| 17. | | | | health facility or elsewhere? | |
| | multi | ole treatments administered | ) | | |
| | □ Pro | ovided free by facility or nati | onal health insurance | | |
| | ☐ Pro | ovided by EFGH | | | |
| | ☐ Cai | regiver needed/needs to bu | y it either at the health | facility or elsewhere | |
| | | ner (specify): | | • | |
| | | known | | | |
| 4.6 | | | e or was discharged w | as the child instructed to tal | ce supplementary or |
| 18. | When the child was ready to leave or was discharged, was the child instructed to take supplementary or therapeutic foods or micronutrients at home? | | | | |

| | ☐ Yes ☐ No (skip to Q21) | | | | | |
|---|---|---|---|---|---|---|
| 19. | Rows below refe | er to supplementar | y or therapeutic food | ds or micronutrie | nts prescribed for th | ne discharge period |
| | Name (check | ( box if prescribed) | - | ose prescribed<br>ge period <i>(circle u</i> | | Prescribed duration<br>(if <10, put "0" before digit) |
| | □RUSF | | (mg/gram/sach | <br>et) □ Unknown | da | ays 🗆 Unknown |
| | □RUTF | | (mg/gram/sach | <br>et) □ Unknown | da | ays 🗆 Unknown |
| | □RUSF (locally n | nade) | (mg/gram/sach | et) 🗆 Unknown | da | ays 🗆 Unknown |
| | □RUTF (locally n | nade) | (mg/gram/sach | <br>et) □ Unknown | da | ays 🗆 Unknown |
| | □Multiple micro | nutrients | (mg/gram/sach | <br>et) □ Unknown | da | ays 🗆 Unknown |
| 20. | Was/were the prescribed foods/micronutrients for the discharge period provided by the health facility (free of charge) or does the caregiver need to buy the foods either at the health facility or elsewhere? (check all that apply if multiple treatments prescribed) | | | | | |
| | <ul> <li>□ Provided free by facility or national health insurance</li> <li>□ Provided by EFGH</li> <li>□ Caregiver needed/needs to buy it either at the health facility or elsewhere</li> <li>□ Other (specify):</li> <li>□ Unknown</li> </ul> | | | | | |
| 21. | Were antibiotics administered during the visit? ☐ Yes ☐ No (skip to Q24) | | | | | |
| 22. | | Rows below r | refer to antibiotics ac | dministered <u>durin</u> | <u>q</u> the facility visit | |
| | Name<br>(check box if<br>administered) | Route of administration (check one | Date initiated<br>(dd-mm-yyyy) | mg | Frequency/day<br>(check one) | Date completed (dd-mm-yyyy) |
| | □Amoxicillin | □ IV □Oral □ IM □Other(specify): | _ - _ <br>- 2 0 _ | mg | □ 1x □2x<br>□3x □4x<br>Other: | - <br>- 2 0 <br> Continuing |
| | | Indication: □Diarrhe | a □Dysentery □Sepsis. | □Lower respiratory | infection | on |
| | □Azithromycin | □ IV □Oral □ IM | _ - <br>- 2 0 | mg | □ 1x □2x<br>□3x □4x<br>Other: | - <br>- 2 0 <br> Continuing |
| | | Indication: □Diarrhe | a □Dysentery □Sepsis. | □Lower respiratory | | on |
| | □Ampicillin | □ IV □Oral □ IM | _ - _ <br>- 2 0 _ | mg | □ 1x □2x<br>□3x □4x<br>Other: | - <br>- 2 0 <br> Continuing |
| | | Indication: □Diarrhe | a □Dysentery □Sepsis. | □Lower respiratory | | on |
| | □Augmentin/Co-<br>amoxiclav | □ IV □Oral □ IM | _ - _ <br>- 2 0 _ | mg<br>□ Unknown | ☐ 1x ☐2x<br>☐3x ☐4x<br>Other: | - <br>- 2 0 <br>Continuing |

| | Indication: $\square$ Diarrhea $\square$ Dysentery $\square$ Sepsis. | □Lower respiratory in | fection $\square M$ | lalnutrition |
|---|---|---|---|---|
| | Other (specify) | | | |
| □Cefixime | □ IV □Oral □ IM - - | mg | □ 1x □ | |
| | □Other( <i>specify</i> ): - 2 0 | □ Unknown | □3x □ | |
| | | □ Unknown | Other: | ☐ Continuing |
| | Indication: □Diarrhea □Dysentery □Sepsis. | □Lower respiratory in | fection $\square M$ | alnutrition |
| | □Other (specify) | | | |
| □Ceftriaxone | □ IV □Oral □ IM _ - | | □ 1x □ | 12x - |
| | □Other(specify): - 2 0 | mg | □3x □ | |
| | Liother (speedy). | ☐ Unknown | Other: | ☐ Continuing |
| | Indication: □Diarrhea □Dysentery □Sepsis. | | <del></del> | |
| | Other (specify) | Lower respiratory in | irection bivi | lamutition |
| Cinnefferencia | □ IV □Oral □ IM - | | | 12x - |
| • | | mg | □ 1x □ | |
| (Cipro) | $\square$ Other(specify): $\begin{vmatrix} - & 2 & & 0 & & & & & & & & & & & & & &$ | ☐ Unknown | □3x □ | |
| | | | Other: | Continuing |
| | Indication: $\square$ Diarrhea $\square$ Dysentery $\square$ Sepsis. | □Lower respiratory in | ifection $\square M$ | alnutrition |
| | Other (specify) | | | |
| □Cefuroxime | □ IV □Oral □ IM - - | mg | □ 1x □ | |
| | □Other( <i>specify</i> ): - 2 0 | | □3x □ | |
| | | ☐ Unknown | Other: | Continuing |
| | Indication: □Diarrhea □Dysentery □Sepsis. | □Lower respiratory in | fection $\square M$ | lalnutrition |
| | ☐Other (specify) | , , | | |
| □Clarithromycin | □ IV □Oral □ IM - - | | | 12x - |
| ciariciii oiriyeiri | □Other(specify): - 2 0 | mg | □3x □ | |
| | Liother (specify). | ☐ Unknown | Other: | ☐ Continuing |
| □Clindamycin | | | □ 1x □ | |
| — CililualityCili | | mg | | |
| | □Other( <i>specify</i> ): - 2 0 | ☐ Unknown | □3x □ | ☐ Continuing |
| | Indication: □Diarrhea □Dysentery □Sepsis. | <del>-</del> | Other: | |
| | | Lower respiratory in | irection Livi | lainutrition |
| | Other (specify) | | | 10 |
| □Chloramphenicol | □ IV □Oral □ IM _ - - | mg | □ 1x □ | |
| | □Other( <i>specify</i> ): - 2 0 | □ Unknown | □3x □ | |
| | | i | Other: | Continuing |
| | Indication: $\square$ Diarrhea $\square$ Dysentery $\square$ Sepsis. | □Lower respiratory in | ifection $\square M$ | alnutrition |
| | Other (specify) | | | |
| | □ IV □Oral □ IM - - | mg | □ 1x □ | |
| Septrin/trimethopri | □Other( <i>specify</i> ): - 2 0 | □ Unknown | □3x □ | |
| m-sulfamethoxazole | | LI OTIKITOWII | Other: | ☐ Continuing |
| | Indication: □Diarrhea □Dysentery □Sepsis. | □Lower respiratory in | fection DM | alnutrition |
| | | | il CCCIOII LIVI | |
| □Doxycycline | | | III CCCIOII LIVI | |
| | □Other (specify) | | | 2x |
| | □Other (specify)<br>□ IV □Oral □ IM - | mg | | |
| , , | □Other (specify) | mg | □ 1x □ | <sub>]4x</sub> - 2 0 |
| , , | □ Other (specify). □ IV □ Oral □ IM - - □ Other(specify): - 2 0 | mg | ☐ 1x ☐ ☐ 3x ☐ ☐ Other: | - 2 0 <br>☐ Continuing |
| , , | □Other (specify) □ IV □Oral □ IM □ □ - □ □Other(specify): - 2 0 □ □ Indication: □Diarrhea □Dysentery □Sepsis. | mg | ☐ 1x ☐ ☐ 3x ☐ ☐ Other: | - 2 0 <br>☐ Continuing |
| | □Other (specify) □ IV □Oral □ IM □ □ - □ □ □Other(specify): - 2 0 □ □ Indication: □Diarrhea □Dysentery □Sepsis. □Other (specify) | mg | ☐ 1x ☐ | - 2 0 Continuing |
| □Erythromycin | □Other (specify) □ IV □Oral □ IM _ - _ □Other(specify): - 2 0 _ Indication: □Diarrhea □Dysentery □Sepsis. □Other (specify) □ IV □Oral □ IM _ - _ | mg | ☐ 1x ☐ ☐ 3x ☐ ☐ Other: | - 2 0 Continuing |
| | □Other (specify) □ IV □Oral □ IM □ □ - □ □ □Other(specify): - 2 0 □ □ Indication: □Diarrhea □Dysentery □Sepsis. □Other (specify) | mg ☐ Unknown ☐Lower respiratory in mg ☐ Unknown | 1x | - 2 0 Continuing Ialnutrition 12x |
| | □Other (specify) □ IV □Oral □ IM _ - _ □Other(specify): - 2 0 _ Indication: □Diarrhea □Dysentery □Sepsis. □Other (specify) □ IV □Oral □ IM _ - _ | mg ☐ Unknown ☐Lower respiratory in mg ☐ Unknown | ☐ 1x ☐ ☐ 3x ☐ ☐ Other: | - 2 0 Continuing |
| | □Other (specify) □ IV □Oral □ IM _ - _ □Other(specify): - 2 0 _ Indication: □Diarrhea □Dysentery □Sepsis. □Other (specify) □ IV □Oral □ IM _ - _ | mg Unknown Lower respiratory ir mg Unknown | ☐ 1x ☐ | - 2 0 Continuing Ialnutrition I2x |
| | □ Other (specify) □ IV □ Oral □ IM _ - _ _ □ Other(specify): - 2 0 _ Indication: □ Diarrhea □ Dysentery □ Sepsis. □ Other (specify) □ IV □ Oral □ IM _ - _ _ □ Other(specify): - 2 0 _ | mg Unknown Lower respiratory ir mg Unknown | ☐ 1x ☐ | - 2 0 Continuing Ialnutrition I2x |
| | □Other (specify) □ IV □Oral □ IM □ | mg Unknown Lower respiratory in mg Unknown Lower respiratory in | ☐ 1x ☐ | - 2 0 Continuing |
| □Erythromycin | □ Other (specify) □ IV □ Oral □ IM □ □ □ □ □ □ Other(specify): □ 2 0 □ □ □ Indication: □ Diarrhea □ Dysentery □ Sepsis. □ Other (specify) □ IV □ Oral □ IM □ □ □ □ □ □ Other(specify): □ □ 2 0 □ □ □ Indication: □ Diarrhea □ Dysentery □ Sepsis. □ Other (specify) | mg Unknown Lower respiratory ir mg Unknown Lower respiratory ir | ☐ 1x ☐ | 2 0 |
| □Erythromycin | □Other (specify) □ IV □Oral □ IM □ | mg Unknown Lower respiratory in mg Unknown Lower respiratory in mg mg Unknown | 1x | 2 0 |
| □Erythromycin | □Other (specify) □ IV □Oral □ IM □ | mg Unknown Lower respiratory in mg Unknown Lower respiratory in mg mg Unknown | 1x | 2 0 |

| | | □Other (specify) | | | |
|---|---|---|---|---|---|
| | □Metronidazole<br>(Flagyl) | □ IV □Oral □ IM - - - | mg | ☐ 1x ☐2x<br>☐3x ☐4x<br>Other: | _ - <br>- 2 0 _ <br> Continuing |
| | | Indication: □Diarrhea □Dysentery □Sepsis. □Other (specify) | □Lower respiratory | infection | tion |
| | □Penicillin | □ IV □Oral □ IM - - □ Other(specify): | mg | ☐ 1x ☐2x<br>☐3x ☐4x<br>Other: | _ - <br>- 2 0 _ <br> Continuing |
| | | Indication: □Diarrhea □Dysentery □Sepsis. □Other (specify) | □Lower respiratory | infection | tion |
| | □Pyrazinamide | □ IV □Oral □ IM - - □ Other(specify): - 2 0 □ | mg | □ 1x □2x<br>□3x □4x<br>Other: | _ - <br>- 2 0 _ <br> Continuing |
| | | Indication: □Diarrhea □Dysentery □Sepsis. □Other (specify) | □Lower respiratory | infection Malnutri | tion |
| | □Streptomycin | □ IV □Oral □ IM - - - - - □Other(specify): - 2 0 | mg | □ 1x □2x<br>□3x □4x<br>Other: | - <br>- 2 0 <br> Continuing |
| | | Indication: □Diarrhea □Dysentery □Sepsis. □Other (specify) | ☐Lower respiratory | infection | tion |
| | □Tetracycline | □ IV □Oral □ IM - - - - <br>□Other(specify): - 2 0 | mg | □ 1x □2x<br>□3x □4x<br>Other: | _ - <br>- 2 0 _ <br>Continuing |
| | | Indication: □Diarrhea □Dysentery □Sepsis. □Lower respiratory infection □Malnutrition □Other (specify) □ | | | |
| | □Other1<br>(specify): | □ IV □Oral □ IM - - - | mg | □ 1x □2x<br>□3x □4x<br>Other: | - <br>- 2 0 <br>Continuing |
| | | Indication: □Diarrhea □Dysentery □Sepsis. □Other (specify) | ☐Lower respiratory | | tion |
| | □Other2<br>(specify): | □ IV □Oral □ IM - - - - - - □Other(specify): - 2 0 | mg | ☐ 1x ☐2x<br>☐3x ☐4x<br>Other: | _ - <br>- 2 0 _ <br> Continuing |
| | | Indication: □Diarrhea □Dysentery □Sepsis. □Other (specify) | □Lower respiratory | infection | tion |
| | □Other3<br>(specify): | □ IV □Oral □ IM □Other(specify): - 2 0 □ | mg | □ 1x □2x<br>□3x □4x<br>Other: | - <br>- 2 0 <br> Continuing |
| | | Indication: □Diarrhea □Dysentery □Sepsis. □Other (specify) | □Lower respiratory | infection | tion |
| 23. | | otics administered during the facility vi<br>eed to buy them either at the health fac | | | |
| | ☐ Provided by E☐ Caregiver nee | e by facility or national health insurance<br>EFGH<br>eded/needs to buy it either at the healt<br>y): | h facility or elsew | here | |
| 24. | | was ready to leave or was discharged, | was the child inst | ructed to take ant | ibiotics at home? |

| | ☐ Yes<br>☐ No (skip to Q27) | | | |
|---|---|---|---|---|
| 25. | Rows below refer to antibiotics <u>prescribed for</u> the discharge period | | | od |
| | Name (check box if prescribed) | mg | Frequency/day<br>(check one) | Prescribed duration<br>(if <10, put "0" before digit) |
| | □Amoxicillin | mg ☐ Unknown | ☐ 1x ☐2x ☐3x ☐4x<br>Other (specify): | days<br>□ Unknown |
| | | | sentery □Sepsis. □Lower respiratory infe | |
| | □Azithromycin | mg | ☐ 1x ☐2x ☐3x ☐4x<br>Other ( <i>specify</i> ): | days<br>□ Unknown |
| | | Indication: □Diarrhea □Dys □Other (specify) | sentery □Sepsis. □Lower respiratory infe | ction |
| | □Ampicillin | | ☐ 1x ☐2x ☐3x ☐4x<br>Other (specify): | |
| | | Indication: □Diarrhea □Dys □Other (specify) | sentery □Sepsis. □Lower respiratory infe | ction |
| | □Augmentin/Co-amoxiclav | | ☐ 1x ☐2x ☐3x ☐4x<br>Other ( <i>specify</i> ): | |
| | | Indication: □Diarrhea □Dys □Other (specify) | sentery □Sepsis. □Lower respiratory infe | |
| | □Cefixime | mg | ☐ 1x ☐2x ☐3x ☐4x<br>Other ( <i>specify</i> ): | days<br>□ Unknown |
| | | Indication: □Diarrhea □Dys □Other (specify) | sentery □Sepsis. □Lower respiratory infe | |
| | □Ceftriaxone | mg | ☐ 1x ☐2x ☐3x ☐4x<br>Other ( <i>specify</i> ): | days<br>□ Unknown |
| | | Indication: □Diarrhea □Dys □Other (specify) | sentery □Sepsis. □Lower respiratory infe | |
| | □Ciprofloxacin (Cipro) | mg | ☐ 1x ☐2x ☐3x ☐4x<br>Other (specify): | days<br>□ Unknown |
| | | Indication: □Diarrhea □Dys □Other (specify) | sentery □Sepsis. □Lower respiratory infe | ction Malnutrition |
| | □Cefuroxime | mg | ☐ 1x ☐2x ☐3x ☐4x<br>Other (specify): | days<br>□ Unknown |
| | | Indication: □Diarrhea □Dys □Other (specify) | sentery □Sepsis. □Lower respiratory infe | ction Malnutrition |
| | □Clarithromycin | mg | ☐ 1x ☐2x ☐3x ☐4x<br>Other (specify): | days □ Unknown |
| | | Indication: □Diarrhea □Dys □Other (specify) | sentery □Sepsis. □Lower respiratory infection | |
| | □Clindamycin | mg ☐ Unknown | ☐ 1x ☐2x ☐3x ☐4x<br>Other (specify): | days □ Unknown |
| | | Indication: □Diarrhea □Dys □Other (specify) | sentery □Sepsis. □Lower respiratory infe | |
| | □Chloramphenicol | mg ☐ Unknown | ☐ 1x ☐2x ☐3x ☐4x<br>Other (specify): | days<br>Unknown |
| | | Indication: □Diarrhea □Dys □Other (specify) | sentery □Sepsis. □Lower respiratory infe | ction |
| | ☐Cotrimoxazole/ Septrin/<br>trimethoprim-sulfamethoxazole | mg | ☐ 1x ☐2x ☐3x ☐4x<br>Other (specify): | days<br>□ Unknown |
| | | Indication: □Diarrhea □Dys | sentery □Sepsis. □Lower respiratory infe | ction Malnutrition |

| | | □Other (specify) | | |
|---|---|---|---|---|
| | □Doxycycline | mg ☐ Unknown | ☐ 1x ☐2x ☐3x ☐4x<br>Other (specify): | days |
| | | | entery Sepsis. Lower respiratory infec | |
| | | □Other (specify) | | |
| | □Erythromycin | mg | ☐ 1x ☐2x ☐3x ☐4x<br>Other (specify): | days<br>□ Unknown |
| | | Indication: □Diarrhea □Dyso □Other (specify) | entery □Sepsis. □Lower respiratory infe | ction Malnutrition |
| | □Gentamicin | mg | ☐ 1x ☐2x ☐3x ☐4x<br>Other ( <i>specify</i> ): | days |
| | | Indication: □Diarrhea □Dyse □Other (specify) | entery □Sepsis. □Lower respiratory infe | ction |
| | □Metronidazole (Flagyl) | mg ☐ Unknown | ☐ 1x ☐2x ☐3x ☐4x<br>Other (specify): | days<br>□ Unknown |
| | | Indication: □Diarrhea □Dyso□Other (specify) | entery □Sepsis. □Lower respiratory infe | ction |
| | | mg | □ 1x □2x □3x □4x | days |
| | □Penicillin | ☐ Unknown | Other (specify): | ☐ Unknown |
| | | Indication: □Diarrhea □Dyso □Other (specify) | entery □Sepsis. □Lower respiratory infe | ction |
| | □Pyrazinamide | mg | ☐ 1x ☐2x ☐3x ☐4x<br>Other (specify): | days<br>□ Unknown |
| | | Indication: □Diarrhea □Dyso □Other (specify) | entery □Sepsis. □Lower respiratory infe | ction Malnutrition |
| | □Streptomycin | mg | ☐ 1x ☐2x ☐3x ☐4x<br>Other ( <i>specify</i> ): | days<br>□ Unknown |
| | | Indication: □Diarrhea □Dyso □Other (specify) | entery □Sepsis. □Lower respiratory infe | |
| | □Tetracycline | mg | ☐ 1x ☐2x ☐3x ☐4x<br>Other (specify): | days<br>□ Unknown |
| | | Indication: □Diarrhea □Dyso □Other (specify) | entery □Sepsis. □Lower respiratory infe | ction Malnutrition |
| | □Other1 (specify): | mg ☐ Unknown | ☐ 1x ☐2x ☐3x ☐4x<br>Other <i>(specify):</i> | days<br>□ Unknown |
| | | Indication: □Diarrhea □Dyse □Other (specify) | entery □Sepsis. □Lower respiratory infe | ction |
| | □Other2 (specify): | mg<br>□ Unknown | ☐ 1x ☐2x ☐3x ☐4x<br>Other ( <i>specify</i> ): | days<br>□ Unknown |
| | | Indication: □Diarrhea □Dyso □Other (specify) | entery □Sepsis. □Lower respiratory infe | ction |
| | □Other3 (specify): | mg ☐ Unknown | ☐ 1x ☐2x ☐3x ☐4x<br>Other <i>(specify):</i> | days<br>□ Unknown |
| | | Indication: □Diarrhea □Dyso □Other (specify) | entery □Sepsis. □Lower respiratory infe | ction |
| 26. | Was/were the prescribed | antibiotics for the dischar | ge period provided by the health f | acility (free of charge) |
| 20. | or does the caregiver nee | • | her at the health facility or elsewh | ere? (check all that |
| | • | y or national health insura | nce | |
| | ☐ Provided by EFGH | | | |
| | ☐ Caregiver needed/nee | ds to buy it either at the he | ealth facility or elsewhere | |
| | ☐ Other (specify): | | | |

| | □ Unknown | | | | | |
|---|---|---|---|---|---|---|
| 27. | Was an anti-helm | inth initiated during the | visit? | □ Ye | s<br>o (skip to Q30) | |
| 28. | | Rows below refer to a | nti-helminth ( | admini | stered during the faci | ility visit |
| | Name<br>(check box if<br>administered) | Date initiated (dd-mm-yyyy) | mg | | Frequency | Date completed (dd-mm-yyyy) |
| | ☐ Albendazole | _ - - - | <br>□ Unknov | mg<br>wn | ☐ Hourly ☐ Daily ☐ Other(specify): | - - |
| | □ Mebendazole | | <br>□ Unknov | mg<br>wn | ☐ Hourly ☐Daily ☐Other(specify): | _ - - - - - |
| | ☐ Other (specify): | _ - - - - | Unknov | mg<br>wn | ☐ Hourly ☐Daily ☐Other( <i>specify</i> ): | _ - - - - - |
| 29. | Were the anti-helminths administered during the facility visit provided by the health facility (free of charge) or did the caregiver need to buy it either at the health facility or elsewhere? (check all that apply if multiple anti-helminths administered) | | | | | |
| | <ul> <li>□ Provided free by facility or national health insurance</li> <li>□ Provided by EFGH</li> <li>□ Caregiver needed/needs to buy it either at the health facility or elsewhere</li> <li>□ Other (specify):</li> <li>□ Unknown</li> </ul> | | | | | |
| 30. | When the child was ready to leave or was discharged, was the child instructed to take anti-helminths at home | | | ake anti-helminths at home? | | |
| | ☐ Yes ☐ No (skip to Q33) | | | | | |
| 31. | Rows below refer to anti-helminths prescribed for the discharge period | | | e period | | |
| | Name (check bo | ox if prescribed) | Dose prescribed for the discharge period | | · · | Prescribed duration<br><10, put "0" before digit) |
| | ☐ Albendazole | - | mg 🗆 Unknown _ | | known | _ days □ Unknown |
| | ☐ Mebendazole | | mg 🗆 Unknown | | known | _ days □ Unknown |
| | ☐ Other(specify): | | m | g 🗆 Un | known | _ days □ Unknown |
| 32. | charge) or does th | escribed anti-helminths for<br>ne caregiver need to buy<br>ultiple anti-helminths pre | the anti-heln | | • | health facility (free of acility or elsewhere? <i>(check</i> |
| | ☐ Provided by EF | y facility or national hea<br>GH<br>ed/needs to buy it eithe | | | ty or elsewhere | |

| | , | · | | | | |
|---|---|---|---|---|---|---|
| | | □ Other (specify): | | | | |
| | | □ Unknown | | | | |
| | 33. | Were any other treatments given during the facility visit and/or prescribed (excluding analgesics)? | | | | |
| | | ☐ Yes | | | | |
| | | □ No (skip to Q36) | | | | diada anno anniad Na |
| | 34. | Rows below refer to treatments administ<br>need to record analgesics (paracetamol), | | | | aiscnarge perioa. No |
| | | Treatment | Administered | | | d at discharge |
| | | (check box if administered or prescribed) | Aummsteret | i dui ilig visit | FTESCTIDE: | at discridige |
| | | <u>Antimalarial</u> | | | | |
| | | □Artemether lumefantrine | ☐ Yes | □ No | ☐ Yes | □ No |
| | | □Paludrine | ☐ Yes | □ No | ☐ Yes | □ No |
| | | □Artesunate | ☐ Yes | □ No | ☐ Yes | □ No |
| | | □Quinine | ☐ Yes | □ No | ☐ Yes | □No |
| | | □Proguanil | ☐ Yes | □ No | ☐ Yes | □No |
| | | Other treatments (excluding analgesics, inc | luding blood trans | fusion, probiotics) | <u> </u> | |
| | | □Other 1 (specify): | □ Yes | □ No | ☐ Yes | □ No |
| | | ☐ Other 2 (specify): | □Yes | □No | □ Yes | □ No |
| | | ☐ Other 3 (specify): | □Yes | □No | □ Yes | □ No |
| | 35. | Were any of the treatments prescribed for the discharge period provided by the health facility (free of charge) or did the caregiver need to buy it either at the health facility or elsewhere? (check all that apply if multiple treatments prescribed) | | | | |
| | | ☐ Provided free by facility or national health insurance | | | | |
| | | ☐ Provided by EFGH | | | | |
| | | $\square$ Caregiver needed/needs to buy it eit | her at the health | facility or elsew | here | |
| | | ☐ Other (specify): | | | | |
| | | □ Unknown | | | | |
| E. | FOR | M COMPLETION | | | | |
| | 36. | ID of person completing this form: | _11 | Date form comp | oleted:<br> - 2 0 _ | _ (dd-mm-yyyy) |
| | 37. | ID of person reviewing this form: | ll | Date form revie | wed:<br> - 2 0 _ | _ (dd-mm-yyyy) |
| | 38. | ID of person entering this form: | II | Date form enter | red:<br> - 2 0 | (dd-mm-yyyy) |
| | 39. | ID of person conducting data verification | on: | Date of data ver | rification:<br> - 2 0 | (dd-mm-yyyy) |

### Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name/Country Site CRF 04b— Wealth Index Form (Bangladesh)

Purpose: To collect household wealth information at the Bangladesh site. Instructions: Please complete this form for all households that are included in the Healthcare Utilization Survey at the Bangladesh EFGH site. Text in **bold** should be read to study participants, plain text is for prompts for study staff, and italics are instructions for study staff. Participant ID: |\_\_\_|\_\_|\_\_|\_\_| PLEASE PLACE PARTICIPANT LABEL HERE (OPTIONAL): **WEALTH INDEX** ☐ Yes ☐ No Does your household have a television? 1. 2. Does your household have a refrigerator? Yes No Does your household have an almirah/wardrobe? Yes No 3. Does your household have an electric fan? Yes No 4. 5. What is the main material of the floor? (select one) Cement ☐ Earth/sand Other material What is the main material of the exterior walls? (select one) Cement Other material What is the main material of the roof? (select one) Cement Other material **ADDITIONAL QUESTIONS** Yes No Does your household have an oven? 8. 9. Does your household have a motor bike? Yes No Yes No 10. Does your household have a car? Yes No 11. Does your household have an AC? Yes No 12. Does your household have a sewing machine? Yes No Does your household have a bi-cycle? 13. 14. Does your household have a dining table? Yes No Yes No 15. Does your household have a sofa? Does your household have a radio? Yes No 16.

# Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name/Country Site CRF 04b— Wealth Index Form (Bangladesh)

| | 17. | Household ownership? | |
|---|---|---|---|
| | | Own | Rented |
| | | Occupied | |
| | 18. | Source of drinking water | |
| | | Own tap Own tube well Own well Own hand pump Communal tap Communal tube well Others | <ul> <li>Communal hand pump</li> <li>Bottled water</li> <li>Water vendor</li> <li>Stored in reservoir</li> <li>Pond/canal/river</li> <li>Shared tap/tube well/well in HH</li> </ul> |
| | 19. | Shared latrine | Yes No |
| | 20. | Latrine type | |
| | | Sanitary latrine with flush | Sanitary latrine without flush |
| | | Non-sanitary/no water seal latrine | ☐ No latrine/use open space |
| C. | FORN | / COMPLETION | |
| | 21. | ID of person completing this form: | Date form completed: - - 2 0 (dd-mm-yyyy) |
| | 22. | ID of person reviewing this form: | Date form reviewed: - - 2 0 (dd-mm-yyyy) |
| | 23. | ID of person entering this form: | Date form entered:<br> - - 2 0 (dd-mm-yyyy) |
| | 24. | ID of person conducting data verification: | Date of data verification:<br> - - 2 0 <i>(dd-mm-yyyy)</i> |

# Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name/Country Site CRF 04b— Wealth Index Form (The Gambia)

**Purpose:** To collect household wealth information at The Gambia site.

| Gambia<br>are inst | | at are included in the Healthcare Utilization Survey at The ipants, plain text is for prompts for study staff, and <i>italics</i> Participant ID: |
|---|---|---|
| A. W | EALTH INDEX | |
| | DETERMINE IF THE RESPONDENT LIVES IN AN URB | AN OR RURAL AREA |
| | Urban | Rural |
| 1. | Does your household have a sofa? | Yes No |
| 2. | Does your household have a wardrobe? | Yes No |
| 3. | Does your household have a television? | Yes No |
| 4. | Does your household have a refrigerator? | Yes No |
| 5. | Does your household have a DVD / VCD player? | Yes No |
| 6. | Does your household have a satellite dish? | Yes No |
| 7. | Does any member of your household own: a bicycle? | Yes No |
| 8. | What is the main source of drinking water for me | embers of your household? (select one) |
| | Public tap / Standpipe | Other water source |
| | Piped to yard | |
| 9. | What kind of toilet facility do members of your h | ousehold usually use? |
| | Flush to septic tank | Other toilet type |
| | Pit latrine w/o slab/ Open Pit | |
| 10 | . What is the main material of the floor in your ho | usehold? (select one) |
| | Ceramic tile | Other floor material |
| 11 | . What is the main material of the exterior walls of | f your household? (select one) |
| | Ceramic tile | Other wall material |

# Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name/Country Site CRF 04b— Wealth Index Form (The Gambia)

| | 12. | How many of the following animals does your household own: Cattle? | None | 1 or more | |
|---|---|---|---|---|---|
| | 13. | Milk cows or bulls? | None | 1 or more | |
| | 14. | Horses, donkeys, or mules? | None | 1 or more. | 5 or more |
| | 15. | Goats? | None | 1 or more | |
| | 16. | Sheep? | None | 1 or more | |
| В. | ADD | ITIONAL QUESTIONS | | | |
| | 17. | Does your household have a functioning television? | Yes No | | |
| | 18. | Does your household have a functioning radio? | Yes No | | |
| | 19. | Does your household have a functioning refrigerator/fridge? | Yes No | | |
| | 20. | Does any member of your household own: a functioning motorcycle/scooter? | Yes No | | |
| | 21. | Does your household have functioning animal-<br>drawn cart? | Yes No | | |
| | 22. | What is the main material of the roof in your househo | old? (select one) | | |
| | | ☐ Thatch/Palm leaf | ☐ Metal/Tin/ | Cement | |
| | | Other roof material | | | |
| | 23. | Does your household own any chicken, Guinea fowl, ducks, turkeys or geese? | Yes No | | |
| C. | FORI | M COMPLETION | | | |
| | 24. | ID of person completing this form: | Date form com | | (dd-mm-yyyy) |
| | 25. | ID of person reviewing this form: | Date form revie | ewed: | (dd-mm-yyyy) |
| | 26. | ID of person entering this form: | Date form ente | red: | (dd |
| | 27. | ID of person conducting data verification: | Date of data ve | | |

#### Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name/Country Site CRF 04b— Wealth Index Form (Kenya)

CRF 04b— Wealth Index Form (Kenya) Purpose: To collect household wealth information for participants enrolled at the Kenya site. Instructions: Please complete this form for all participants enrolled at the Kenya EFGH site. Text in bold should be read to study participants, plain text is for prompts for study staff, and italics are instructions for study staff. PLEASE PLACE PARTICIPANT LABEL HERE (OPTIONAL): Participant ID: | | | | | | **WEALTH INDEX** A. Yes No (skip Q14) 1. Does your household have electricity? 2. Does your household have a television? Yes No (skip Q15) Yes No 3. Does your household have a sofa? 4. Does your household have a cupboard? Yes No 5. Yes No (skip Q16) Does your household have a DVD player? Yes No (skip Q17) 6. Does your household have a radio? Yes No 7. Does your household have a table? 8. Does your household have a clock? Yes No (skip Q18) 9. What is the main material of the floor of your dwelling? (select one) Cement Other Earth/sand What is the main material of the external walls of your dwelling? (select one) 10. Dung/mud/soil Other What is the main material of the roof of your dwelling? (select one) 11. ☐ Thatch/grass/makuti Other 12. What type of fuel does your household mainly use for cooking? (select one) Wood Other LPG/Natural gas What kind of toilet facility do members of your household usually use? (select one) 13. Other No facility/bush/field В. **ADDITIONAL QUESTIONS** Yes No 14. Does your household have a functioning electricity?

15. Does your household have a functioning television? ☐ Yes ☐ No Yes No Does your household have a functioning DVD player? 16. Does your household have a functioning radio? ☐ Yes ☐ No 17. Yes No 18. Does your household have a functioning clock? FORM COMPLETION Date form completed: 19. ID of person completing this form: | | | |\_\_|\_| - |\_\_| - | 2 | 0 |\_\_| (dd-mm-yyyy)


# Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name/Country Site CRF 04b— Wealth Index Form (Kenya)

| 20 | ID of person reviewing this form: | Date form reviewed: |
|---|---|---|
| 20. | <u> </u> | _ - - 2 0 _ (dd-mm-yyyy) |
| 21 | ID of person entering this form: | Date form entered: |
| <b>ZI</b> . | | _ - - 2 0 (dd-mm-yyyy) |
| 22 | ID of person conducting data verification: | Date of data verification: |
| ZZ. | | _ - - 2 0 (dd-mm-yyyy) |

# Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name/Country Site CRF 04b — Wealth Index Form (Malawi)

Purpose: To collect household wealth information at the Malawi site.

| <b>Instructions:</b> Please complete this form for all households that are included in the Healthcare Utilization Survey at the Malawi EFGH site. Text in <b>bold</b> should be read to study participants, plain text is for prompts for study staff, and <i>italics</i> are instructions for study staff. | | | |
|---|---|---|---|
| PL | EASE | PLACE PARTICIPANT LABEL HERE (OPTIONAL): | Participant ID: |
| A. | WEA | ALTH INDEX | |
| | 1. | Does your household have electricity? | Yes No |
| | 2. | Does your household have a radio? | Yes No |
| | 3. | Does your household have a television? | ☐ Yes ☐ No |
| | 4. | Does your household have a bed with a mattress? | ☐ Yes ☐ No |
| | 5. | Does your household have a sofaset? | ☐ Yes ☐ No |
| | 6. | Does any member of this household own: a mobile phone? | Yes No |
| | 7. | Does any member of this household have a bank a | ccount? Yes No |
| | 8. | What is the main material of the floor in your hous | sehold? (select one) |
| | | Earth/sand | Cement |
| | | Other floor material | |
| | 9. | What is the main material of the roof in your house | ehold? (select one) |
| | | ☐ Thatch/palm leaf | Metal |
| | | Other roof material | |
| | 10. | What type of fuel does your household mainly use | for cooking? (select one) |
| | | Wood | Other type of fuel |
| В. | FOR | M COMPLETION | |
| | 11. | ID of person completing this form: | Date form completed: _ - - 2 0 _ (dd-mm-yyyy) |
| | 12. | ID of person reviewing this form: | Date form reviewed: - - 2 0 (dd-mm-yyyy) |
| | 13. | ID of person entering this form: | Date form entered: |
| | 14. | ID of person conducting data verification: | _ - - 2 0 <i>(dd-mm-yyyy)</i> Date of data verification: _ - _ _ - 2 0 _ _ <i>(dd-mm-yyyy)</i> |

# Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name/Country Site CRF 04b — Wealth Index Form (Mali)

Purpose: To collect household wealth information at the Mali site.

| Mali<br>instr | <b>Instructions:</b> Please complete this form for all households that are included in the Healthcare Utilization Survey at the Mali EFGH site. Text in <b>bold</b> should be read to study participants, plain text is for prompts for study staff, and <i>italics</i> are instructions for study staff. | | |
|---|---|---|---|
| , | | PLACE PARTICIPANT LABEL HERE (OPTIONAL): | Participant ID: |
| A. | WEA | ALTH INDEX | |
| | 1. | In your house, do you have electricity? | Yes No |
| | 2. | In your house, do you have a television? | Yes No |
| | 3. | In your house, do you have a bed? | Yes No |
| | 4. | In your house, do you have a fan? | Yes No |
| | 5. | In your house, do you have a cupboard | Yes No |
| | 6. | In your house, do you have a CD/DVD player? | Yes No |
| | 7. | In your house, do you have a refrigerator? | Yes No |
| | 8. | In your house, do you have a chair? | Yes No |
| | 9. | In your house, do you have a motorcycle or scooter? | Yes No |
| | 10. | In your house, do you have soap, washing powder, or ash/sand/dirt for washing your hands? | Yes No |
| | 11. | Does any member of this household have a bank acco | unt? Yes No Don't know |
| | 12. | Where is your principal source of drinking water locat | ed? (select one) |
| | | Outside of the plot | Within the plot |
| | 13. | What is the distance to the principal source of drinkin | g water? (select one) |
| | | Less than 30 minutes round trip | More than 30 minutes round trip |
| | 14. | Main material of exterior walls of the house? (select of | ne) |
| | | Brick | Other |
| | 15. | Main material of roof of house? (select one) | |
| | | Cement | Mud with wood |
| | | Other | |

# Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name/Country Site CRF 04b — Wealth Index Form (Mali) ial of floor of house? (select one)

| | 16. | Main material of floor of house? (select one) | |
|---|---|---|---|
| | | Earth/sand floor | Ceramic tile floor |
| | | Other | |
| | 17. | In your house, what is the main fuel used for cooking | ? (select one) |
| | | ☐ Charcoal ☐ Wood | Other |
| | 18. | Does your household own any pigs? | Yes No |
| | 19. | Does your household own any camels or dromedaries | s? Yes No |
| | 20. | Does your household own any Guinea fowl, ducks, tu geese? | rkeys or Yes No |
| В. | FOR | M COMPLETION | |
| | 21. | ID of person completing this form: | Date form completed: |
| | 22. | ID of person reviewing this form: | Date form reviewed: |
| | | ID of person entering this form: | _ - - 2 0 (dd-mm-yyyy) Date form entered: |
| | 23. | 10 of person entering this form. | |
| | <ul><li>23.</li><li>24.</li></ul> | ID of person conducting data verification: | - - 2 0 (dd-mm-yyyy) Date of data verification: |

### Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name/Country Site CRF 04b— Wealth Index Form (Pakistan)

Purpose: To collect household wealth information at the Pakistan site. Instructions: Please complete this form for all households that are included in the Healthcare Utilization Survey at the Pakistan EFGH site. Text in **bold** should be read to study participants, plain text is for prompts for study staff, and italics are instructions for study staff. Participant ID: |\_\_\_|\_\_|\_\_| PLEASE PLACE PARTICIPANT LABEL HERE (OPTIONAL): **WEALTH INDEX** A. Yes No 1. Does your household have a refrigerator? Does your household have a washing machine? Yes No 2. 3. Does your household have a sofa? Yes No Yes No Does your household have a chair? 4. 5. Does your household have an Almirah/cabinet? ☐ Yes ☐ No ☐ Yes ☐ No Does your household have a computer? 6. 7. Does your household have an internet connection? Yes No Yes No 8. Does your household have a bed? Does any member of this household have a bank 9. Yes No account? What type of fuel does your household mainly use for cooking? (select one) 10. Other Wood What is the main material of the roof in your household? (select one) Other Cement/RCC 12. What is the main material of the walls in your household? (select one) Cement Other В. FORM COMPLETION Date form completed: ID of person completing this form: |\_\_\_|\_\_| 13. |\_\_|\_| - |\_\_| - | 2 | 0 |\_\_|\_| (dd-mm-yyyy) Date form reviewed: ID of person reviewing this form: |\_\_\_|\_\_| 14. |\_\_|\_| - |\_\_| - | 2 | 0 |\_\_|\_| (dd-mm-yyyy) ID of person entering this form: |\_\_\_|\_\_| Date form entered: 15. |\_\_|\_| - |\_\_| - | 2 | 0 |\_\_|\_| (dd-mm-yyyy) Date of data verification: 16. ID of person conducting data verification: |\_\_\_|\_\_| |\_\_|\_| - |\_\_| - | 2 | 0 |\_\_| (dd-mm-yyyy)

Purpose: To collect household wealth information at the Peru site. Instructions: Please complete this form for all households that are included in the Healthcare Utilization Survey at the Peru EFGH site. Text in **bold** should be read to study participants, plain text is for prompts for study staff, and italics are instructions for study staff. PLEASE PLACE PARTICIPANT LABEL HERE (OPTIONAL): Participant ID: |\_\_\_|\_\_|\_\_|\_\_| **WEALTH INDEX** A. Yes No 1. Does your household have a computer? Does your household have a bookshelf? Yes No 2. Yes No Does your household have windows with curtains or blinds? 3. Yes No Does your household have a sofa? 4. What type of toilet does your household use? (select one) 5. Indoor connected to public sewer Other What type of material is the roof made of in your household? (select one) Reinforced concrete Other 7. What type of material are the walls made of in your household? (select one) Other Brick or cement block В. FORM COMPLETION Date form completed: 8. ID of person completing this form: |\_\_\_|\_\_| |\_\_|\_| - |\_\_| - | 2 | 0 |\_\_| (dd-mm-yyyy) Date form reviewed: ID of person reviewing this form: | | | 9. |\_\_|\_| - |\_\_| - | 2 | 0 |\_\_|\_| (dd-mm-yyyy) Date form entered: ID of person entering this form: |\_\_\_|\_\_| 10. |\_\_|\_| - |\_\_| - | 2 | 0 |\_\_| (dd-mm-yyyy) ID of person conducting data verification: Date of data verification: 11. |\_\_|\_| - |\_\_| - | 2 | 0 |\_\_|\_| (dd-mm-yyyy) |\_\_\_|\_\_|

**Purpose:** To ascertain information on HIV information for enrolled participants and biological mother (if present). Instructions: Please complete this form for all enrolled participants at the Malawi, Mali, and Kenya sites ONLY. If the participant underwent HIV testing at the enrollment visit, this form should be initiated at the enrollment visit but completed once results are available (including viral load and/or CD4 results), assuming results are not available at the time of enrollment. Plain text is for prompts for study staff, and italics are instructions for study staff. PLEASE PLACE PARTICIPANT LABEL HERE (OPTIONAL): A. PARTICIPANT INFORMATION 1. Participant ID \_\_|\_\_|\_\_| 2 Date of Enrollment: |\_\_\_|\_\_| - |\_\_\_| - | 2 | 0 |\_\_\_| (dd-mm-yyyy) |\_\_\_|\_| - |\_\_\_| - | 2 | 0 |\_\_\_| (dd-mm-yyyy) 3. Date of Form Completion: **Note**: Date corresponds to when the entire form is completed (not intiated). If results are pending, this question will not be answered until results are available and this form is complete. EFGH country site: 4. ☐ Kenya ☐ Malawi ☐ Mali В. HIV INFORMATION, BIOLOGICAL MOTHER Is the accompanying caregiver the child's biological mother? 5. ☐ Yes | No (skip to Q13) What is the source of information for the mother's most recent HIV status? 6. A rapid test done at the clinic during the enrollment visit (complete remaining questions when results are available) A PCR test done at the clinic during the enrollment visit (complete remaining questions when results are available) Previous laboratory report Previous hospital record Maternal health passport, MCH booklet, or other similar document | Mother self-report Not applicable (results not known and testing not being performed) What is the enrolled child's biological mother's HIV status? Reminder to offer HIV testing in accordance 7. with guidelines and record result here. Negative or non-reactive (skip to Q19, end of form) Positive or reactive Unknown (skip to Q13) Declined to state (skip to Q13)

| | 8. | Is the | e a viral load result available for the mother? |
|---|---|---|---|
| | | Ye | S |
| | | ☐ No | o (skip to Q9) |
| | | 8a. | If yes, number of copies at most recent test: copies/mL. Undetectable |
| | | | <i>If yes,</i> date of most recent viral load test: - - 2 0 (dd-mm- |
| | | 8b. | yyyy) |
| | | | Unknown |
| | 9. | <u></u> | re a CD4 count or percentage available for the mother? |
| | | ∐ Ye | |
| | | | o (skip to Q10) |
| | | 9a. | <i>If yes,</i> CD4: _percent <u>OR</u> count |
| | | 9b. | <i>If yes,</i> date of CD4 test: - - 2 0 (dd-mm-yyyy) ☐ Unknown |
| | 10. | Is the | mother currently receiving highly active anti-retroviral therapy (HAART)? |
| | | Ye | S |
| | | ☐ No | o (skip to Q12) |
| | | = | nknown (skip to Q12) |
| | | | eclined to state (skip to Q12) |
| | | 11. | If yes, date initated: - - 2 0 (dd-mm-yyyy) Unknown |
| | 12. | <u></u> | mother currently receiving infection prophylaxis with cotrimoxazole (Septrin)? |
| | | Ye | |
| | | | o (skip to Q13) |
| | | 12a. | If yes, date initated: _ - _ - 2 0 (dd-mm-yyyy) Unknown |
| C. | HIV I<br>unkn | | MATION, CHILD (To be completed if the child if the biological mother is HIV-infected or HIV status |
| | 13. | What | is the source of information on the child's most recent HIV status? |
| | | | rapid test done at the clinic during the enrollment visit (complete remaining questions when |
| | | | s are available) |
| | | | PCR test done at the clinic during the enrollment visit (complete remaining questions when results |
| | | | vailable) |
| | | | evious laboratory report |
| | | Previous hospital record | |
| | | Child health passport, MCH booklet, or other similar document | |
| | | | rbal report from the caregiver ot applicable (results not known and testing not being performed) |
| | 14. | | is the child's HIV status? Reminder to offer HIV testing in accordance with guidelines and record |
| | | result | |
| | | ☐ Ne | egative or non-reactive (skip to Q17) |
| | | □ Ро | sitive or reactive |
| | | Ur | ıknown (skip to 17) |

| | 15. | Is there a viral load result available for this child? | | |
|---|---|---|---|---|
| | | ☐ Yes ☐ No (skip to Q16) | | |
| | | 15a. If yes, number of copies at most recent test: copies/mL Undetectable | | |
| | | 15b. <i>If yes</i> , date of most recent viral load test: - - 2 0 (dd-mm- | | |
| | | yyyy) | | |
| | | | Same as date of enrollment (Q2) Un | |
| | 16. | 16. Is there a CD4 count or percentage available for this child? Yes | | |
| | ☐ No (skip to Q17) | | | |
| | | 16a. | If yes, most recent CD4 result: pe | rcent <u>OR</u> count |
| 16b. If yes, date of most recent CD4 test: - - 2 0 _ Unknown | | | | |
| | 17. | Is the | child currently receiving any of the following: | |
| | | ПН | ighly active anti-retroviral therapy (HAART) or | anti-retroviral therapy (ART) for treatment (known |
| | HIV-infected children) | | | |
| | | Anti-retroviral (ARV) prophylaxis for prevention of HIV | | |
| ☐ None (skip to Q18) | | | | |
| | Unknown (skip to Q18) | | | |
| | | 17a. If yes, date initated: - 2 0 (dd-mm-yyyy) Unknown | | |
| | 18. | 18. Is the child currently receiving infection prophylaxis with cotrimoxazole (Septrin)? | | |
| | Yes | | | |
| | | □ N | o (skip to Section C) | |
| | | U | nknown (skip to Section C) | |
| | | 18a. If yes, date initated: - - 2 0 (dd-mm-yyyy) | | |
| | | Unknown | | |
| D. | FOR | RM COMPLETION | | |
| | 19. | ID of | person completing this form: | Date form completed: |
| | | l | l <u>l_</u> l | _ - - 2 0 _ (dd-mm-yyyy) |
| | 20. | ID of | person reviewing this form: | Date form reviewed: |
| | | | | _ - - 2 0 (dd-mm-yyyy) |
| | 21. | ID of person entering this form: | | Date form entered: |
| | | | | _ _ - _ - 2 0 (dd-mm-yyyy) |
| | 22. | ID of | person conducting data verification: | Date of data verification: |

#### Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name/Country Site CRF 04d— Daily Record (For Participants with Overnight Stays Only)

| <b>Purpose:</b> To document daily clinical events among participants with overnight stays. | | | | |
|---|---|---|---|---|
| to b<br>the<br>from<br>pro | pe com<br>partici<br>n the p<br>mpts f | ns: To be completed at the beginning of each day pleted on the same day of enrollment, but is to be ipant is hospitalized during the weekend/holidays participant's medical record when available. Text or study staff, and italics are instructions for stud | completed each day thereafter that the<br>(outside of working hours), the informa<br>in <b>bold</b> should be read to study particip | ne child is in the hospital. If ation can be abstracted |
| A. | PART | TICIPANT INFORMATION | | |
| | 1. | Participant ID | | |
| | 2. | Date of Enrollment | _ - - 2 0 _ | (dd-mm-yyyy) |
| | 3. | EFGH country site: | | |
| | | ☐ Bangladesh | ☐ Kenya | |
| | | □ Malawi | □ Mali | |
| | | ☐ Pakistan | □ Peru | |
| | | ☐ The Gambia | | |
| В. | CLIN | ICAL EVALUATION INFORMATION | | |
| | 4. | Date seen: - - 2 0 | _ (dd-mm-yyyy) | |
| | 5. | Time seen: : (hh : min, 24:00 hr) | | |
| | 6. | ID of Study Staff performing clinical evaluation: | | |
| | 61.151 | □ Non-EFGH study staff performed clinical evaluation (information being abstracted from medical record) | | |
| C. | | NICAL SIGNS (PHYSICAL EXAM) | | |
| | 7. | What is the source of the information? | | |
| | | ☐ Physical exam being performed in real time ☐ Medical record | | |
| | 8. | Temperature: . °C □ Missing | | |
| | 9. | Heart Rate: beats per minute. ☐ Missing | | |
| | 10. Respiratory Rate: breaths per minute | | | |
| | 11. What is the child's general condition? | | | |
| | | ☐ Well/Alert ☐ Restless/Irritab | e Unconscious | ☐ Missing |
| | 12. | Assess the child's eyes and determine if they are: | | |

#### Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name/Country Site CRF 04d— Daily Record (For Participants with Overnight Stays Only)

| | | , | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | ☐ Normal (skip to Q13) | | | ☐ Abnormally sunken | | ☐ Missii | ☐ Missing (skip to Q13) |
| | | 11a. If child's eyes are determined to be abnormally sunken, please ask the caregiver: Is the appearance of your child's eyes abnormal? | | | | | er: Is the appearance of | |
| | | | $\square$ Yes (abnormal for child) | | | | | |
| | | | □ No | | | | | |
| | 13. | Describe the child's ability to drink or breastfeed: | | | | | | |
| | | ☐ Normal/Not Thirsty | | ☐ Drink | ☐ Drinks eagerly/Thirsty ☐ Drindrink | | ly/Unable to | ☐ Missing |
| | 14. | Using a thumb and forefinger, gently pinch up the child's skin on the abdominal wall and assess the skin's retu<br>to normal: | | | | | | nd assess the skin's return |
| | | ☐ Immediately | | ☐ 1 to <2 seconds (slowly) | | □ ≥2 seconds (very slowly) | | ☐ Missing |
| | 15. | Dehyd | ration assessment (to | be compl | leted based on data | in Q10-Q14 abo | ive) | |
| | | ☐ Severe dehydration At least two of the following signs (check all that apply): | | At least t | □ Some dehydration □ No At least two of the following signs (check all that apply): | | <u>iion</u> | ☐ Could not be determined based on information available |
| | | ☐ Leth | argic or Unconscious | ☐ Restle | ess/irritable | | | |
| | | ☐ Sunken eyes | | ☐ Sunke | Sunken eyes | | | |
| | | ☐ Drinks poorly/unable to | | ☐ Drink | s eagerly/Thirsty | y/Thirsty | | |
| | | drink | | ☐ Skin p | inch goes back 1 to | | | |
| | | ☐ Skin | pinch goes back ≥2 | <2 secon | nds (slowly) | | | |
| | | second | ls (very slowly) | | | | | |
| D. | CLIN | CLINICAL EVENTS IN THE LAST 24 HOURS (MEDICAL RECORDS AND/OR CAREGIVER INTERVIEW) | | | | | | |
| | 16. | What is the source of the information? | | | | ☐ Medical record ☐ Caregiver report | | |
| <b>.</b> | 17. | Numbe | er of unusually loose | stools passed in last | 24 hours | (/ | if <10, put "0" before digit) | |
| | 17. | | ·<br> | | ·<br> | | ☐ Missing | 5 10 100 100 |
| | 18. | | Of the unusually loose or watery stools passed in the last | | | 24 hours, | f <10, put "0" before digit) | |
| | | now m | how many had visible blood in them? | | | ☐ Missing | | if <10 nut "0" hafara digit |
| | 19. | Number of vomiting episodes in last 24 hours | | | (if <10, put "0" before digit) ☐ Missing | | | |
| | REN | MINDER: Record any therapies initiated/completed in the Medical Management Form [CRF 04a] on a daily basis | | | | | | |
| E. | FORI | FORM COMPLETION | | | | | | |
| | 20. | ID of p | ID of person completing this form: | | | | Date form completed: _ - 2 0 _ (dd-mm-yyyy) | |
| | 21. | ID of person reviewing this form: | | | | Date form re | Date form reviewed: _ - - 2 0 (dd-mm-yyyy) | |
| | 22. | ID of person entering this form: | | | | Date form entered: _ - 2 0 _ (dd-mm-yyyy) | | |
| | 23. | ID of p | ID of person conducting data verification: | | | Date of data | | ) |

Purpose: To be completed after a child is enrolled in EFGH but is referred to another facility prior to their completion of the Discharge Form during their enrollment visit. Instructions: Please complete this form for any children who are enrolled in EFGH (assigned a Participant ID) and who are referred to another facility prior to completion of the "Discharge Form". Note: For children who are referred, two Medical Management Forms may be completed. Plain text is for prompts for study staff, and italics are instructions for study staff. PLEASE PLACE PARTICIPANT LABEL HERE (OPTIONAL): **Referral Information** A. Participant ID 1. |\_\_|\_| - |\_\_| - | 2 | 0 |\_\_| (dd-mm-yyyy) Date of Referral 2. |\_\_\_| : |\_\_\_| (hh : min, 24 hr) 3. Time of Referral Unknown 4. Is the child being referred to an EFGH recruiting site or a non-EFGH recruiting site? No, not an EFGH recruiting site Yes, to an EFGH recruiting site What facility is the child being referred to? 5. ☐ Name of EFGH recruiting site x ☐ Name of EFGH recruiting site x ☐ Name of EFGH recruiting site x ☐ Name of EFGH recruiting site x Other (specify):\_\_ Reason for referral (check all that apply) 6. ☐ Requires specific treatments or services that are not ☐ Requested by caregiver available ☐ Requires overnight stay ☐ Cost  $\square$  Other (specify): Diagnosis(es) when referred (check all that apply): 7. ☐ HIV Anemia Urinary Tract Infection Sickle cell Tuberculosis Malaria Fever of unknown origin Suspected sepsis Dysentery Acutely unwell, unknown cause Other Gastroenteritis Diarrhea Meningitis/ encephalitis Upper respiratory tract infection Poisoning/ herbal intoxication Pneumonia Other lower respiratory tract infections (other than Malnutrition pneumonia) COVID-19 Asthma

| | | ☐ Unknown ☐ Other (specify): | | | |
|---|---|---|---|---|---|
| В. | | TO THE FACILITY, COSTING INFORMATION, AND TRANSPORTATION HOME FROM THE FACILITY (Text in bold ld be read verbatim, plain text is for prompts for study staff, and italics are instructions for study staff) | | | |
| | 8. | Is the caregiver able and willing to continue wit | Is the caregiver able and willing to continue with the remaining interview questions? | | |
| | | □ Yes | | | |
| | | □ No (skip to Section C) | | | |
| | 9. | Did you miss any income-generating activities because of this child's health facility visit? | | | |
| | | □ Yes | | | |
| | | □ No (skip to Q12) | | | |
| | 10. | Approximately how much time have you misse | ed from income ger | nerating activi | ties? |
| | | hours <u>OR</u> days | | | |
| | 11. | What type of income generating activities? | | | |
| | | ☐ Salaried work | rk | | |
| | | ☐ Non-wage earnings (e.g. trading, personal bu | ☐ Other (spe | ner (specify): | |
| | 12. | Did anyone else visit the child during the child's stay at the health facility? | | | |
| | | □Yes | | | |
| | | □No (skip to Q13) | | | |
| | 10 | 12a. Approximately how many <u>adults</u> visited your child during his/her stay? | | | |
| | 13. How much did your child's stay at the health facility cost you in total? This includes medical costs, to and household costs such as food and hotels. | | | | |
| | | Total amount paid and/or owed (in local currency): | | | |
| | 14. | How much of those costs were spent on the following fees and materials? This includes money you've alread spent or still owe. (check "Yes" for all costs and report amount paid or owed numerically in local currency. Lead row blank if the caregiver did not pay for the fee/material or does not recall. If respondent does not know except, please ask for an estimate. Check "Unknown" if respondent cannot estimate amount. | | | |
| | | Clinical registration fee | | | |
| | | Lab tests or diagnostics | Amount: | | |
| | | Medical supplies purchased in the facility | Amount: | | |
| | | (e.g., needles, gloves) □ Unknown Medical supplies purchased outside of facility □ Yes, needed to pay for this Amount: | | | |
| | | Medical supplies purchased outside of facility (e.g., needles, gloves) □ Yes, needled to pay for this Amount: | | | |
| | | Doctor/nurse/health worker fees | | | |
| | | □ Unknown | | | |
| | | Medications administered during visit (e.g. ☐ Yes, needed to pay for this antibiotics, multivitamins) ☐ Unknown | | | |
| | | antibiotics, multivitamins) | | | |

| | | Medications to bring home ( multivitamins) | ☐ Yes, needed to pay for this | | | Amount: | | |
|---|---|---|---|---|---|---|---|--|
| | | Food for yourself or other fa | ☐ Yes, needed to pay for this | | | Amount: | | |
| | | Lodging for yourself or other | ☐ Yes, needed to pay for this | | | Amount: | | |
| | | Childcare | ☐ Yes, needed to pay for this | | | Amount: | | |
| | | Other (specify): | | ☐ Yes, needed to pay for this | | or this | Amount: | |
| | 15. | If your child becomes ill after facility? | er discharge, will it | be easy or o | hallenging fo | or you to | <b>4</b> | |
| | | Easy (skip to Q17) | | | Cha | llenging | | |
| | 16. | Why will it be challenging to | seek care again a | t a health fa | cility? (check | all that | apply) | |
| | | ☐ Money | Religion | | Transport | | | |
| | | Work | Distance | | ☐ Caring for other children | | | |
| | | Family members | Quality of car | e | Other (specify): | | | |
| | 17. | What method of transporta (check all that apply) | our child plai | n to use to tr | avel hon | ne from the facility today? | | |
| | | ☐ Walk | ☐ Motorbike | | ☐ Private or shared car | | | |
| | | ☐ Personal vehicle | ☐ Shared van/bu | s/taxi | ☐ Other (specify): | | | |
| C. | SCHE | EDULED FOLLOW UP VISIT DATES (to be completed by study staff and remind caregiver of scheduled visits) | | | | | | |
| | 18. | Next scheduled Week 4 visit | l_ | _ - - 2 0 (dd-mm-yyyy) | | | | |
| | 19. | Next scheduled Month 3 visi | l_ | _ _ - | - 2 | 0 _ <i>(dd-mm-yyyy)</i> | | |
| | PI | lease copy the scheduled follow up visit information into the Participant Information Card and give to caregiver. | | | | | | |
| D. | FORM | M COMPLETION | | | | | | |
| | 20. | ID of person completing this form: | | | Date form completed: _ - - 2 0 (dd-mm-yyyy) | | | |
| | 21. | ID of person reviewing this f | _ Da | Date form reviewed: - - 2 0 (dd-mm-yyyy) | | | | |
| | 22. | ID of person entering this fo | Da | Date form entered: _ - - 2 0 (dd-mm-yyyy) | | | | |
| | 23. | ID of person conducting data | Da | Date of data verification: | | | | |
| | | | | _ _ - . | - 2 | 0 _ <i>(dd-mm-yyyy)</i> | | |
| | - | : To be o | | ght care at | the study clinic (inpatient or outpatient) is ready | | | | |
|---|---|---|---|---|---|--|--|--|--|
| out<br>(cor<br>who<br>mis<br>inst | patie<br>mplet<br>ateve<br>sing.<br>ructio | nt this in<br>the Referi<br>r questi<br>Text in<br>ons for s | means when the child is ready to leave the<br>ral CRF (CRF 04e instead). If a participant is di<br>ions possible with the medical records/faci | facility). D<br>ischarged d<br>ility logs av | who is being discharged from the facility (for not complete this form if a child was referred during non-working hours, please aim to complete vailable; otherwise, indicate if information was ext are prompts for study staff, and italics are | | | | |
| A. | STA | ATUS AT | DISCHARGE | | | | | | |
| | 1. | Partic | ipant ID | 11_ | | | | | |
| | 2. What was the outcome of the child when leaving the | | | | e facility/health center? | | | | |
| | ☐ Improved or healthy (skip to Q3) | | | No better/same as when presenting to Q3) | | | | | |
| | | ☐ Worse (skip to Q3) | | | Died in facility | | | | |
| | | Ur | nknown <i>(skip to Q3)</i> | | Other (specify):(skip to Q3) | | | | |
| | | ШМ | issing (only applicable for participants disch | arged durin | g non-working hours) | | | | |
| | | 2a. | If the child died, what was the date of dea | (dd-<br>(skip<br>CRF | - - 2 0 <br>mm-yyyy)<br>to Section E and complete CRF10a - Mortality<br>and CRF 11 - Study Close Out CRF)<br>Jnknown/Missing | | | | |
| | 3. | Date | of Discharge | | - _ - 2 0 _ <i>(dd-mm-yyyy)</i><br>Unknown/Missing | | | | |
| | 4. | Time | of Discharge | I | _ : (hh: min, 24 hr)<br>Unknown/Missing | | | | |
| | 5. | Has th | <b>.</b> | f, or is the o | caregiver taking the child home against medical | | | | |
| | | ☐ Di | scharged by clinician (skip to Section B) | | Self-discharge | | | | |
| | | Ur | nknown/Missing | | | | | | |
| | 6. | Is the | caregiver present? | | | | | | |
| | | □ Yes | 5 | | | | | | |
| | | □No | (skip to Section B) | | | | | | |

| | 7. | Ask caregiver: What are the important factors in you was recommended by your child's provider? (Read | | |
|---|---|---|---|---|
| | | Child recovered | Caregiv | er needed to return to work |
| | | Cost of medical care too expensive | Caregiv<br>responsibil | er needed to return to domestic<br>ities |
| | | ☐ Transportation availability | Poor qu | ality care at health facility |
| | | Child not getting better | Other ( | specify): |
| В. | FINA | AL DIAGNOSIS(ES) AT DISCHARGE | | |
| | 8. | Final diagnosis(es) at discharge (check all that apply) | r): | |
| | | Anemia | | ☐ HIV |
| | | Sickle cell | Urinary | Tract Infection |
| | | Malaria | Tuberc | ulosis |
| | | Suspected sepsis | Fever of | f unknown origin |
| | | Dysentery | Acutely | , unwell, unknown cause |
| | | ☐ Diarrhea | Gastroenteritis | |
| | | Upper respiratory tract infection | gitis/ encephalitis | |
| | | Pneumonia | neumonia Poisoning/ herbal intoxication | |
| | | Other lower respiratory tract infections (other than pneumonia) | Malnut | rition |
| | | Asthma | COVID-19 | |
| | | Unknown/Missing | Other (specify): | |
| | | lf caregiver not present, as i | ndicated in Q | 6, skip to Section D. |
| C. | bold | T TO THE FACILITY, COSTING INFORMATION, AND TR<br>I should be read verbatim, plain text is for prompts for | study staff, ( | and italics are instructions for study staff) |
| | | e: If participant was referred from another EFGH facili<br>s incurred during the facility visit where the child was i | | |
| | 9. | Did you miss any income-generating activities bed | , | • • |
| | | □ Yes | | |
| | | □ No (skip to Q12) | | |
| | 10. | 10. Approximately how much time have you missed from income generating activities? | | |
| | | hours <u>OR</u> days | | |
| | 11. | What type of income generating activities? | | |
| | | ☐ Salaried work | | ☐ Hourly work |
| | | ☐ Non-wage earnings (e.g. trading, personal busing | ess, etc.) | ☐ Other (specify): |

| 12. | Did anyone else visit the ch | nild during the chi | ld's stay at t | the health f | facility? | |
|---|---|---|---|---|---|---|
| | □Yes | | | | | |
| | □No (skip to Q13) | | | | | |
| | 12a. Approximately how many <u>adults</u> visited your child during his/her stay? | | | | | |
| 13. | | | | | | ides medical costs, transport, |
| 15. | and household costs such as | - | active cost y | ou iii totui: | Till3 lilela | ides inculcal costs, transport, |
| | Total amount paid and/or o | wed (in local curr | ency): | | | ☐ None (skip to Q15) |
| 14. | | s" for all costs and l<br>ay for the fee/mate | report amoun<br>erial or does n | t paid or ow<br>ot recall. If i | ed numeri<br>responden | includes money you've already cally in local currency. Leave row t does not know exact cost, |
| | Clinical registration fee | | ☐ Yes, nee | ded to pay | for this | Amount: |
| | | | | | | □ Unknown |
| | Lab tests or diagnostics | | ☐ Yes, nee | eded to pay | for this | Amount: |
| | Medical supplies purchased | in the facility | ☐ Yes, needed to pay for this | | | ☐ Unknown Amount: |
| | (e.g., needles, gloves) | Till the facility | Tes, fleeded to pay for this | | | ☐ Unknown |
| | Medical supplies purchased | outside of | ☐ Yes, nee | eded to nav | for this | Amount: |
| | facility (e.g., needles, gloves | | | caca to pay | 101 11113 | ☐ Unknown |
| | Doctor/nurse/health worke | | ☐ Yes, nee | eded to pay | for this | Amount: |
| | | | | . , | | □ Unknown |
| | Medications administered of | during visit (e.g. | ☐ Yes, nee | eded to pay | for this | Amount: |
| | antibiotics, micronutrients) | | | | | □ Unknown |
| | Medications to bring home | (e.g. antibiotics, | ☐ Yes, nee | eded to pay | for this | Amount: |
| | micronutrients ) | | | | | □ Unknown |
| | Food for yourself or other fa | amily members | ☐ Yes, needed to pay for this | | | Amount: |
| | | | | | | Unknown |
| | Lodging for yourself or othe<br>members | er family | ☐ Yes, needed to pay for this | | | Amount: |
| | members | | ☐ Yes, needed to pay for this | | | Amount: |
| | Childcare | | □ 1es, 11et | eded to pay | 101 11115 | ☐ Unknown |
| | | | ☐ Yes, nee | eded to pay | for this | Amount: |
| | Transportation | | | p , | | □ Unknown |
| | Other (specify): | | ☐ Yes, nee | eded to pay | for this | Amount: |
| | | | | | | ☐ Unknown |
| 15. | If your child becomes ill afte facility? | r discharge, will it | be easy or c | hallenging f | or you to | seek care again at a health |
| | Easy (skip to Q17) | | | | Cha | allenging |
| 16. | Why will it be challenging t | o seek care again | at a health | facility? (cl | heck all th | nat apply) |
| | Money | Religion | | ☐ Transp | ort | |
| | Work | Distance | | Caring | Caring for other children | |
| | ☐ Family members ☐ Quality of care | | | Other: | | |

| | 17. What method of transportation do you and your child plan to use to travel home from the facility tod (check all that apply) | | | | |
|---|---|---|---|---|---|
| | | ☐ Walk ☐ Motorbike | | ☐ Private or shared car | |
| | | ☐ Personal vehicle | ☐ Shared van/bus/tax | i | ☐ Other (specify): |
| D. | SCHEDULED FOLLOW UP VISIT DATES (to be completed by study staff and remind caregiver of scheduled visits) | | | | |
| | 18. | Next scheduled Week 4 visit date: | | | _ - - 2 0 (dd-mm-yyyy) |
| | 19. | Next scheduled Month 3 vi | isit date: | | - _ - 2 0 (dd-mm-yyyy) |
| | Ple | Please copy the scheduled follow up visit information into the Participant Information Card and give to caregiver to take home (if caregiver is present). | | | |
| E. | FORM | M COMPLETION | | | |
| | 20. | ID of person completing th | is form: | Date form completed: | |
| | | | | | - - 2 0 (dd-mm-yyyy) |
| | 21. | ID -f this | .f | Date | form reviewed: |
| | | ID of person reviewing this | form: | | - _ - 2 0 (dd-mm-yyyy) |
| | 22. | ID of person entering this f | antonia a thio forman I I I I | | form entered: |
| | | ib of person entering this i | OIIII. | _ _ | - _ - 2 0 (dd-mm-yyyy) |
| | 23. | ID of person conducting da | nta verification: | Date | of data verification: |
| | | | | | - _ - 2 0 (dd-mm-yyyy) |

**Purpose:** The diarrhea diary will be given to the caregivers of children enrolled in the EFGH study on the day of enrollment. Day 0 is filled out by both caregiver and study staff together on the day of enrollment for practice. The first entry into the diary (Day 1) will be completed on by the caregiver after the entry for Day 0. The diary will capture information about the diarrhea episode in the previous 24 hours leading up to presentation to the facility, during their enrollment visit, and after the child leaves the facility to document the full severity of the diarrhea episode. The caregiver or her designee (such as a school aged child also living in the house) will complete the form daily, for a 14-day period beginning on the date of enrollment. The diary will be collected from the caregiver during the first follow-up visit, at the end of the 14 day period if the enrollment hospitalization lasts 14 days or greater, or picked up during a home visit. While study staff may counsel and remind caregivers on how to complete the diary, study staff should not fill in blank information as the diary is intended to reflect caregiver report only.

| PLEASE PLACE PARTICIPANT LABEL HERE (OPTIONAL): | OR write in Participant ID: |
|---|---|

**Instructions:** Please explain the following to the caregiver and work with the caregiver to fill out the first column "Day 0 - Previous 24 hours prior to Enrollment Visit" to reflect the child's signs and symptoms in the previous 24 hours leading up to presentation. The caregiver ALONE (not study staff) will then complete Days 1-14.

- Day: Period from the sunrise of a day to sunrise of the next day.
  - Please do not count any symptoms twice.
  - For Day 0, you should count the symptoms in previous 24 hours prior to the enrollment visit
  - For Day 1, you should count the symptoms since enrollment up until the sunrise of the next day. Please note that this may not be a full 24 hours period.
  - For Day 2 and onwards, please count the symptoms from sunrise of that day to sunrise of the next day.
  - Please note the dates using the format day (01-31)— month (01-12) year (2022 or 2023) (For example June 1, 2022 would be written as: 01-06-2022)
- Temperature: Refers to temperature collected either orally (thermometer inserted into the mouth), under the armpit, or forehead. Please note temperature taken on the forehead is DIFFERENT than if a child feels "hot to the touch."
  - If your child is still in the hospital and their temperature is being taken, that temperature reading can be reported.
  - If the study gave you a thermometer, please use it in the armpit of the child.
  - If the temperature is taken multiple times during the day, the highest should be recorded in the diary.
  - If you notice that your child is hot to touch on the forehead, please indicate that next to the appropriate box. Please answer this question even if you are also taking a thermometer reading.
- If your child has any of the signs shown in the figure, mark "X" in the box right to the figure for that day.
  - If your child is "normal" meaning s/he doesn't have any of the signs, make an "X" in the row corresponding to the smiling face( )
  - For "Medications", the smiley face ( ) indicates the child did <u>not</u> receive any ORS, Zinc supplements, or any antibiotics (ie absence of any medications)
  - For some symptoms (number of loose or watery stools and vomiting), please pay attention to the number of loose stools and vomiting and mark the box next to the highest number of loose stools or vomiting on that day.
- If you forget for a few days, try to start again on the correct day.
- Keep this form in a safe place and bring it to the health facility at the follow-up visit.

Version: 7.0 (09-06-2023) 

Enterics for Global Health – *Shigella* Surveillance Study (EFGH) CRF 06— Diarrhea Diary

| | | | | | | | | | | | | | | | 1 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| <b>(</b> 3 | DAY 14 - - 2 0 2 _ | - | | | | | | | | - | | | | | |
| <b>(</b> 3 | | - | | | | | | | | | | | | | Pag |
| <b>(</b> 3 | _ 2 0 2 - _ - _ 21 YAQ | | | | | | | | | | | | | | |
| <b>(</b> 3 | _ S 0 S - _ - - - 11 YAQ | | | | | | | | | | | | | | |
| <b>(</b> 3 | _ | | | | | | | | | | | | | | |
| <b>(</b> 3 | _ | | | | | | | | | | | | | | |
| <b>(</b> 3 | _ 2 0 2 - _ - 8 YAQ | | | | | | | | | | | | | | |
| <b>(</b> 3 | _ 2 0 2 - _ - _ 7 YAQ | | | | | | | | | | | | | | |
| <b>(</b> 3 | - - - - - - - 9 AAQ | | | | | | | | | | | | | | |
| <b>(</b> 3 | _ | | | | | | | | | | | | | | |
| <b>(</b> 3 | - | | | | | | | | | | | | | | |
| <b>(</b> 3 | - | - | | | | | | | | | | | | | |
| <b>(</b> 3 | - - - - - z vAa | | | | | | | | | | | | | | |
| <b>(</b> 3 | NAV 1 | | | | | | | | | | | | | | |
| <b>*</b> | Day 0 - Previous 24 hours<br>prior to enrollment Visit | | | | | | | | | | | | | | |
| | | _ | | 4 | * | * | * | * | + | | <b>3</b> | | 4 | + | |
| | | y Stool | | | * | 4 | 4 | 77 | 7 | | ing gri | | 7 | 4 | |
| | | Water | No loose or watery stool | | | | 4 | 4 | * | | No vomitting | | 4 | 4 | |
| | | ose or | ose or w | | | | | * | 7 | | ž | | 4 | 1 | |
| | | ally Lo | No loc | | | | | | * | | | | | | (200 |
| | | Number of Abnormally Loose or Watery Stool | | 07- | | | | | | - | | | | | 01-06-2 |
| | | er of A | | | 1 | 7 | | | | ng | | 1 | | | Varsion: 7 0 (01-06-2023) |
| | | Numb | | | | | | | | Vomiting | | | | | 1/orcio |
| | | | | | | | | | | | l | | | | |

Version: 7.0 (01-06-2023)


| <b>(</b> 3 | _ | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | _ | | | | | | | | |
| | _ | | | | | | | | |
| <b>(</b> 3 | _ S 0 S - _ _ - - 11 YAQ | | | | | | | | |
| <b>(</b> 3 | _ 2 0 2 - _ - - - 01 YAQ | | | | | | | | |
| <b>(</b> 3 | 2 0 2 - - - - e YAQ | | | | | | | | |
| <b>\$</b> | 2 0 2 - - _ - 8 YAQ | | | | | | | | |
| <b>(</b> 3 | _ 5 0 5 - _ - - - 7 YAQ | | | | | | | | |
| <b>(</b> 3 | _ | | | | | | | | |
| <b>©</b> | _ | | | | | | | | |
| <b>©</b> | 2 0 2 - - _ - 4 YAQ | | | | | | | | |
| <b>©</b> | 5 0 2 - - _ - £ YAQ | | | | | | | | |
| <b>©</b> | _ 2 0 2 - _ - _ | | | | | | | | |
| <b>\$</b> | * 2 0 2 - _ - _ YAQ<br>*May not be full 24—hour period | | | | | | | | |
| <b>*</b> | Day 0 - Previous 24 hours<br>prior to enrollment Visit | | | | | | | | |
| | | Blood in stool | | No oral rehydration solution (ORS) | Oral rehydration soluation (ORS) | No antibiotics | Antibiotics | No zinc | Zinc |
| | | Δ | | No oral reh | Oral rehydration | | | | |
| | | • | Medications | | | •€ | | • | |

| • | | io capture information about the enrolled particip<br>If multiple people are with the child, ask to speak | ant at follow-up visits. Ideally this form is completed by the primary with the primary caregiver. |
|---|---|---|---|
| | | | ripants at the Week 4 follow up visit and Month 3 follow up visit. Text rompts for study staff, and italics are instructions for study staff. |
| PLEA | SE PLA | ACE PARTICIPANT LABEL HERE (OPTIONAL): | |
| A. | PAR1 | TICIPANT INFORMATION | |
| | 1. | Participant ID: | |
| | 2. | Date of enrollment visit: (for reference) | - - 2 0 (dd-mm-yyyy) |
| | 3. | Date of follow up visit: | - - 2 0 (dd-mm-yyyy) |
| | 4. | Time form is started: | : (hh : min, 24:00 hr) |
| | 5. | EFGH country site: | |
| | | Bangladesh Kenya | Malawi Mali |
| | | Pakistan Peru | The Gambia |
| B. | FOLL | OW-UP VISIT INFORMATION | |
| | 6. | Follow up visit: | Week 4 Month 3 |
| | 7. | What is the relationship of the respondent to the | ne enrolled child? |
| | | ☐ Biological mother | Biological father |
| | | Grandmother | Grandfather |
| | | ☐ Aunt | Uncle |
| | | ☐ Older sister | Older brother |
| | | Other (specify): | |
| | 8. | Is the respondent the primary caregiver? | |
| | | Yes | |
| | | □ No | |
| | 9. | Where is this visit being conducted? | |
| | | ☐ Health facility | |
| | | Home | |
| | | Over the phone (only if home or health facil | ity not possible, skip to Section E) |
| | 10. | Is the child available for physical exam by the m | nedical team? (ask only for home/clinic visits) |
| | | Yes (skip to Section C) | |
| | | □ No | |
| | 11. | If no, why not? | |
| | | Child has moved (skip to Section E) | Child has passed away (stop form, skip to Section L: Form completion), complete CRF 10a - Mortality CRF and CRF 11 Study Close Out CRF) |

| | | | regiver refused to let study skip to Section E) | y staff see | Other (s | pecify): | |
|---|---|---|---|---|---|---|---|
| C. | ASSE | SSMEN | T OF THE CHILD'S GENERA | L CONDITION | | | |
| | Ask t | his Sect | ion only if the child is avail | able for physico | al exam by the | medical to | еат |
| | 12. | What | is the child's general condi | tion? | | | |
| | | ☐ Well/Alert ☐ Restless/Irritable ☐ Lethargic or Unconscious | | | | | |
| | 13. | Does the child appear unwell? | | | | | |
| | | ☐ Yes | (please complete CRF 08 - | Unwell Child Fo | orm) | | |
| | | □No | | | | | |
| D. | CHIL | D ANTH | ROPOMETRY (complete th | is section only | if the child is a | available fo | or a physical exam by study team) |
| | | | What is the child's mid up | oper arm circur | nference | | |
| | 14. | a. | (MUAC)? (1st measureme | ent) | | . (cm) | |
| | | | Arm from which MUAC is | being measure | ed | | |
| | | b. | (please ensure the <u>same</u> ( | arm is used to a | collect 1st, | ☐ Right ☐ Left | |
| | | | 2 <sup>nd</sup> , and 3 <sup>rd</sup> measurement | ts) | | | |
| | | c. | What is the child's mid up | I I | . (cm) | | |
| | | (MUAC)? (2 <sup>nd</sup> measurement) | | | | | |
| | | If m | If measurement 2 differs from measurement 1, subtract the lower measurement from the higher measurement | | | | |
| | | and, if the difference is 0.3cm or greater, obtain a third measurement. | | | | | |
| | | d. | | ild's mid upper arm circumference | | | _ . (cm) |
| | | ű. | (MUAC)? (3 <sup>rd</sup> measureme | ent, if applicable | e) | ☐ Not ap | oplicable (3 <sup>rd</sup> measurement not indicated) |
| | | Comm | nents: | | | | |
| | 15. | How i | s the child's weight being r | ecorded? | | | |
| | | ☐ Adı | ult scale, child only <i>(child is</i> | ≥24 months A | ND able to sta | ind on the : | scale alone; skip to Q19) |
| | | ☐ Adı | ult scale, child and caregive | r together <i>(chi</i> | ld is <24 mon | ths OR una | ble to stand on the scale alone) |
| | 16. | a. | What is the weight of ch | ild and caregive | er (1 <sup>st</sup> | 1 1 | 1 1 1 (1/2) |
| | | | measurement) | | | ll | _ . (kg) |
| | | b. | What is the weight of the | caregiver alon | e (1 <sup>st</sup> | 1 1 | _ . (kg) |
| | | | measurement) | | | I I | |
| | | c. | What is the <u>calculated</u> we | eight of the chil | ld <i>(Q16a</i> | 1 1 | . (kg) |
| | | | minus Q16b) | | | 11 | _[:][(\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\ |
| | 17. | a. | What is the weight of chi | ld and caregive | r (2 <sup>nd</sup> | 1 1 | _ . (kg) |
| | | | measurement) | | | '' | |
| | | b. | What is the weight of the | caregiver alon | e (2 <sup>na</sup> | | _ . (kg) |
| | | | measurement) | | LI (047 | '' | |
| | | C. | What is the <u>calculated</u> we<br>minus Q17b) (2 <sup>nd</sup> measur | • | ia (Q1/a | II | _ . (kg) |
| | | If m | <u> </u> | · | ement 1 (016 | c) subtrac | t the lower measurement from the higher |
| | | ''' | | - | | - | obtain a third measurement |

| | 18. | a. | What is the weight of child and caregiver (3 <sup>rd</sup> | . (kg) |
|---|---|---|---|---|
| | | | measurement) | ☐ Not applicable |
| | | | | (3 <sup>rd</sup> measurement not indicated) |
| | | b. | What is the weight of the caregiver alone (3 <sup>rd</sup> | . (kg) |
| | | | measurement) | ☐ Not applicable |
| | | | | (3 <sup>rd</sup> measurement not indicated) |
| | | c. | What is the calculated weight of the child (Q18a | . (kg) |
| | | | minus Q18b) (3 <sup>rd</sup> measurement) | ☐ Not applicable |
| | | | | (3 <sup>rd</sup> measurement not indicated) |
| | | Comr | ments: | |
| | 19. | a. | What is the child's weight? (1st measurement) | . (kg) |
| | | b. | What is the child's weight? (2 <sup>nd</sup> measurement) | . (kg) |
| | | If measurement 2 differs from measurement 1, subtract the lower measurement from the higher measurement | | |
| | | | and if the difference is 0.2 kg or grea | |
| | | c. | What is the child's weight? (3 <sup>rd</sup> measurement, if | . (kg) |
| | | | applicable) | ☐ Not applicable |
| | | | | (3 <sup>rd</sup> measurement not indicated) |
| | | Comr | ments: | |
| | 20. | How | is the child's length (if <24 months) / height (if ≥24 mo | nths) being recorded? |
| | | ☐ Re | cumbent length (if <24 months) | |
| | | □ Sta | anding height (if ≥24 months) | |
| | 24 | | What is the length/height of the child? (1st | 1 1 1/ |
| | 21. | a. | measurement) | _ (cm) |
| | | b. | What is the length/height of the child? (2 <sup>nd</sup> | 1 1 1/200 |
| | | D. | measurement) | . (cm) |
| | | If n | neasurement 2 differs from measurement 1, subtract ti | · |
| | | | and if the difference is 0.5cm or grea | |
| | | C. | What is the length/height of the child? (3 <sup>rd</sup> | . (cm) |
| | | | measurement, if applicable) | ☐ Not applicable |
| | | | | (3 <sup>rd</sup> measurement not indicated) |
| | | Comr | ments: | |
| E. | | | DYSENTERY RECOVERY AFTER LEAVING THE HEALTH | |
| | 1 | _ | | rolled in the EFGH study (upon returning home from the |
| | heal | th facili | ity visit) and relate to the child's recovery from the illne | ess they were enrolled with. |
| | 1 | | | |

| | · — | These questions are ONLY to be asked at the Week 4 follow-up visit (or the Month 3 follow-up visit if the Week 4 visit was missed). Caregiver should answer the below questions based on memory rather than the diarrhea diary card. | | |
|---|---|---|---|---|
| | 22. | 7 | gi <i>ver snould answer the below questions based c</i><br>e diarrhea diary card returned? | in memory rather than the diarrned diary cara. |
| | 22. | Yes | e diarrilea diary card returned: | |
| | | ☐ No | | |
| | | | andiaskie (fallanna visit talian alamakumbana | 1 |
| | | ☐ Not applicable (follow up visit taking place by phone) | | |
| | 23. | _ | ir child continue to have diarrhea (defined as 3 after leaving the health facility? | or more unusually loose or watery stools in a 24 hour |
| | | | arter reaving the health facility: | |
| | | Yes | (Alice to Continue E) | |
| | | | (skip to Section F) | |
| | | ļ | 't know (skip to Section F)) | |
| | 24. | | lid the diarrhea end? Refer to calendar to | |
| | | | ine date if # of days since leaving the facility | - |
| | | | nent) was known but not exact date. The end | (dd-mm-yyyy) |
| | | date is the last day of diarrhea before a diarrhea-free | | |
| | | period ( | of two days or more. | |
| | 25. | On the | worst day of diarrhea since leaving the health | |
| | | facility, | how many loose stools did the child have in | loose stools (if <10, put "0" before digit) |
| | | one day (24 hours)? | | |
| | 26. | Did the | child have blood in his/her stool during the dia | rrhea that continued after leaving the health facility? |
| | | Yes | | |
| | | ☐ No ( | skip to Q28) | |
| | | ☐ Don | 't know (skip to Q28) | |
| | 27. | How m | any days did the child have blood in stool? | days (if <10, put "0" before digit) |
| | 28. | Did the | child vomit any time during the episode of dia | rhea that continued after leaving the health facility? |
| | | Yes | | |
| | | ☐ No ( | skip to Q29) | |
| | | ☐ Don | 't know (skip to Q29) | |
| | | 28a. | How many days did the child vomit? | days (if <10, put "0" before digit) |
| | | | Thinking about the day when the child had | |
| | | 28b. | the most vomiting, how many times did s/he | (if <10, put "0" before digit) |
| | | | vomit in the day (24 hours)? | |
| | 29. | Did the | child have a fever (or feel hot to the touch) dur | ing the diarrhea that continued after leaving the health |
| | | facility? | • | |
| | | Yes | | |
| | | ☐ No ( | 'skip to Section F) | |
| | | ☐ Don | 't know (skip to Section F) | |
| | | 29a. | If yes, what was the highest temperature? | . °C |
| | | 29b. | How many days did s/he have the fever? | days |
| F. | MED | ICATION | S AFTER LEAVING THE FACILITY | |
| | This. | section (C | 230-Q33) is intended to capture what medication | s were used for the child's recovery from the diarrhea illness |
| | that | that led them to be enrolled in the EFGH study. These questions are only to be asked at the Week 4 follow-up visit (or the | | |

Month 3 follow-up visit if the Week 4 visit was missed). Prescribed treatments to be ascertained from the Medical Management CRF and ideally, pre-filled in the first column below prior to conducting the interview (to prime the interviewee on what medications were prescribed). Medications used and days used are to be answered by the caregiver. Note there may be some medications used that were not prescribed and those should be captured as well.

Name of the medications originally prescribed for the child during the discharge period (including those not)

Name of the medications originally prescribed for the child for the discharge period (including those not)

Name of the medications originally prescribed for the child during the discharge period (including those not)

Name of the medications originally prescribed for the child during the discharge period (including those not)

Name of the medications taken by your child, did your child, did your child, did your child receive some or all of the

| 30. | Name of the medications originally prescribed for the child for the discharge period (filled from Medical Management Form) | Name of medications actually taken by the child during the discharge period (including those not prescribed. Completed based on Caregiver report) | Among these medications taken by your child, did your child receive some or all of the medications for free? | Among these<br>medications <u>taken</u> by<br>your child, did you<br>purchase some or all of<br>the medications (at the<br>facility or elsewhere)? | Among these medications taken by the child, how many days did your child eat or drink the medication? |
|---|---|---|---|---|---|
| | □ ORS | □ ORS | ☐ Yes ☐ No ☐ Don't know | ☐ Yes<br>☐ No<br>☐ Don't know | days |
| | □ Zinc | □ Zinc | ☐ Yes<br>☐ No<br>☐ Don't know | ☐ Yes ☐ No ☐ Don't know | days |
| | □ RUSF | □ RUSF | ☐ Yes<br>☐ No<br>☐ Don't know | ☐ Yes<br>☐ No<br>☐ Don't know | days |
| | □ RUTF | □ RUTF | ☐ Yes<br>☐ No<br>☐ Don't know | ☐ Yes ☐ No ☐ Don't know | _days |
| | ☐ RUSF (locally made) | ☐ RUSF (locally made) | ☐ Yes<br>☐ No<br>☐ Don't know | ☐ Yes ☐ No ☐ Don't know | _days |
| | ☐ RUTF (locally made) | ☐ RUTF (locally made) | ☐ Yes<br>☐ No<br>☐ Don't know | ☐ Yes ☐ No ☐ Don't know | days |
| | | | <u>Antibiotics</u> | | |
| | ☐ Amoxicillin | ☐ Amoxicillin | ☐ Yes<br>☐ No<br>☐ Don't know | ☐ Yes<br>☐ No<br>☐ Don't know | days |
| | ☐ Azithromycin | ☐ Azithromycin | ☐ Yes ☐ No ☐ Don't know | ☐ Yes ☐ No ☐ Don't know | days □ Don't know |
| | ☐ Ampicillin | ☐ Ampicillin | ☐ Yes ☐ No ☐ Don't know | ☐ Yes ☐ No ☐ Don't know | days<br>□ Don't know |
| | ☐ Augmentin/Co-<br>amoxiclav | ☐ Augmentin/Co-<br>amoxiclav | ☐ Yes ☐ No ☐ Don't know | ☐ Yes ☐ No ☐ Don't know | _days □ Don't know |
| | ☐ Ceftriaxone | ☐ Ceftriaxone | ☐ Yes ☐ No ☐ Don't know | ☐ Yes ☐ No ☐ Don't know | _days<br>□ Don't know |

| ☐ Ciprofloxacin (Cipro) | ☐ Ciprofloxacin (Cipro) | ☐ Yes ☐ No ☐ Don't know | ☐ Yes ☐ No ☐ Don't know | _days □ Don't know |
|---|---|---|---|---|
| ☐ Cefixime | ☐ Cefixime | ☐ Yes ☐ No ☐ Don't know | ☐ Yes ☐ No ☐ Don't know | _days |
| ☐ Cefuroxime | ☐ Cefuroxime | ☐ Yes<br>☐ No<br>☐ Don't know | ☐ Yes ☐ No ☐ Don't know | days |
| ☐ Clarithromycin | ☐ Clarithromycin | ☐ Yes ☐ No ☐ Don't know | ☐ Yes ☐ No ☐ Don't know | days |
| ☐ Clindamycin | ☐ Clindamycin | ☐ Yes ☐ No ☐ Don't know | ☐ Yes ☐ No ☐ Don't know | _days |
| ☐ Chloramphenicol | ☐ Chloramphenicol | ☐ Yes ☐ No ☐ Don't know | ☐ Yes ☐ No ☐ Don't know | _days |
| ☐ Cotrimoxazole/<br>Septrin | ☐ Cotrimoxazole/<br>Septrin | ☐ Yes<br>☐ No<br>☐ Don't know | ☐ Yes ☐ No ☐ Don't know | days |
| ☐ Doxycycline | ☐ Doxycycline | ☐ Yes ☐ No ☐ Don't know | ☐ Yes ☐ No ☐ Don't know | _days |
| ☐ Erythromycin | ☐ Erythromycin | ☐ Yes ☐ No ☐ Don't know | ☐ Yes ☐ No ☐ Don't know | days |
| ☐ Gentamicin | ☐ Gentamicin | ☐ Yes ☐ No ☐ Don't know | ☐ Yes ☐ No ☐ Don't know | _days |
| ☐ Penicillin | ☐ Penicillin | ☐ Yes<br>☐ Don't know | ☐ Yes<br>☐ Don't know | days<br>□ Don't know |
| □ Pyrazinamide | ☐ Pyrazinamide | ☐ Yes ☐ No ☐ Don't know | ☐ Yes ☐ No ☐ Don't know | _days |
| ☐ Streptomycin | ☐ Streptomycin | ☐ Yes ☐ No ☐ Don't know | ☐ Yes ☐ No ☐ Don't know | days |
| ☐ Tetracycline | ☐ Tetracycline | ☐ Yes ☐ No ☐ Don't know | ☐ Yes ☐ No ☐ Don't know | days |
| ☐ Other1 (specify): | ☐ Other1 (specify): | ☐ Yes ☐ No ☐ Don't know | ☐ Yes ☐ No ☐ Don't know | _days |

| ☐ Other2 (specify): | ☐ Other2 (specify): | □ Yes | □Yes | days |
|---|---|---|---|---|
| | | □ No | □ No | ☐ Don't know |
| | | ☐ Don't know | ☐ Don't know | |
| ☐ Other3 (specify): | ☐ Other3 (specify): | ☐ Yes | ☐ Yes | days |
| | | □ No | □ No | ☐ Don't know |
| | | ☐ Don't know | ☐ Don't know | |
| | | <u>Antiprotozoals</u> | <u>i</u> | |
| | | □ Yes | □ Yes | l l ldove |
| ☐ Albendazole | ☐ Albendazole | □ No | □No | _days |
| | | ☐ Don't know | ☐ Don't know | □ Don't know |
| | | □ Yes | □Yes | |
| ☐ Mebendazole | ☐ Mebendazole | □ No | □No | days |
| | | ☐ Don't know | ☐ Don't know | ☐ Don't know |
| | | □ Yes | □ Yes | |
| ☐ Metronidazole | ☐ Metronidazole (Flagyl) | □ No | □No | days |
| (Flagyl) | (8)./ | ☐ Don't know | ☐ Don't know | ☐ Don't know |
| | | □ Yes | □ Yes | |
| ☐ Other (specify): | ☐ Other (specify): | □ No | □ No | days |
| | | ☐ Don't know | ☐ Don't know | ☐ Don't know |
| | | Boil ( know | Don't know | |
| | | <u>Antimalarial</u> | | |
| ☐ Artemether | ☐ Artemether | ☐ Yes | ☐ Yes | days |
| lumefantrine | lumefantrine | □ No | □ No | □ Don't know |
| Tamerantine | rameranemie | ☐ Don't know | ☐ Don't know | |
| | | ☐ Yes | ☐ Yes | <br> days |
| ☐ Paludrine | ☐ Paludrine | □ No | □ No | ☐ Don't know |
| | | ☐ Don't know | ☐ Don't know | L Boil ( kilow |
| | | □ Yes | ☐ Yes | days |
| ☐ Artesunate | ☐ Artesunate | □ No | □No | ☐ Don't know |
| | | ☐ Don't know | ☐ Don't know | □ Don't know |
| | | □ Yes | □ Yes | 1 1 12 |
| ☐ Quinine | ☐ Quinine | □ No | □ No | _days |
| | | ☐ Don't know | ☐ Don't know | ☐ Don't know |
| | | □ Yes | ☐ Yes | |
| ☐ Proguanil | ☐ Proguanil | □ No | □No | days |
| | | ☐ Don't know | ☐ Don't know | ☐ Don't know |
| | | 1 | | |
| | Other | treatments (excludin | g analgesics) | |
| ☐ Other1 (specify): | ☐ Other1 (specify): | □ Yes | ☐ Yes | _days |
| _ other (specify). | in other i (specify). | □ No | □ No | □ Don't know |
| | | ☐ Don't know | ☐ Don't know | |
| ☐ Other2 (specify): | ☐ Other2 (specify): | ☐ Yes | ☐ Yes | days |
| □ Other 2 (specify): | □ Otherz (specijy): | □ No | □ No | ☐ Don't know |
| | | ☐ Don't know | ☐ Don't know | LI DOIL CKIIOW |

| | | ☐ Other3 (specify): | ☐ Other3 (specify): | ☐ Yes<br>☐ No | | □ Yes<br>□ No | days |
|---|---|---|---|---|---|---|---|
| | | | | ☐ Don' | t know | ☐ Don't know | ☐ Don't know |
| | 31. | | ur child's stay at the heal | | • • | • | u in total? This includes |
| | | | nd/or owed (in local curre | | | | e (skip to Q33) |
| | 32. | spent or still owe. (c<br>row blank if the care | <b>costs were spent on the f</b><br>heck "Yes" for all costs an<br>giver <u>did not</u> pay for the f<br>n estimate in local curren | nd report<br>fee/mate | t amount pai<br>erial or does i | d or owed numerically<br>not recall. If responde | in local currency. Leave<br>ent does not know exact |
| | | Clinical registration fee | | | ☐ Yes, needed | I to pay for this | Amount: |
| | | Lab tests or diagnostics | | | ☐ Yes, needed | I to pay for this | Amount: |
| | | Medical supplies <u>purcha</u> gloves) | sed in the facility (e.g., needle | es, | ☐ Yes, needed | I to pay for this | Amount: |
| | | Medical supplies purcha needles, gloves) | sed <u>outside of facility</u> (e.g., | | ☐ Yes, needed | I to pay for this | Amount: |
| | | Doctor/nurse/health wo | rker fees | | ☐ Yes, needed | I to pay for this | Amount: |
| | | Medications administere multivitamins) | ed during visit (e.g. antibiotics | 5, | ☐ Yes, needed to pay for this | | Amount: |
| | | Medications to bring ho | me (e.g. antibiotics, multivitar | mins) | ☐ Yes, needed to pay for this Amo | | Amount: |
| | | Food for yourself or other | er family members | | ☐ Yes, needed to pay for this | | Amount: |
| | | Lodging for yourself or o | ther family members | | ☐ Yes, needed to pay for this | | Amount: |
| | | Childcare | | | ☐ Yes, needed to pay for this | | Amount: |
| | | Transportation | | | ☐ Yes, needed | I to pay for this | Amount: |
| | | ., ,,,, | | | | I to pay for this | Amount: |
| | 33. | _ | alth facility, about how m | | - | | _ |
| | | care for the child wh | ile they were ill with the | diarrhe | a episode th | ey were enrolled wit | h? |
| | | hours | <u>OR</u> days | | <u>OR</u> | □ None | |
| G. | NEW | ILLNESS SINCE LAST S | CHEDULED VISIT (EITHER | RENROL | LMENT OR V | VEEK 4) | |
| | | = | • | | | • | ther Enrollment or Week 4) |
| | _ | <u>excludes</u> the diarrheal illness for which the child was enrolled in the EFGH study . If an Unwell Child CRF was completed | | | | | |
| | for th | the participant, please reference the information from that CRF to complete this section. | | | | | |
| | | | New diarrhea/dyse | | | | |
| | 34. | | | | | | develop a new episode of |
| | | diarrhea, that is at diarrhea episode that started after at least 2 diarrhea free days? <u>Note</u> : Diarrhea episode is defined as diarrhea (3 or more unusually loose or watery stools in a 24 hour period). Use memory aid to facilitate | | | | | |
| | | remembering days. | 3 or more unusually loos | se or wa | tery stools in | a 24 nour perioa). U | se memory aid to facilitate |
| | | Yes No (skip to Q51) | | | | | |

| [ | | Doubling (Alin to 051) |
|---|---|---|
| | | ☐ Don't know (skip to Q51) |
| | 35. | How many new episodes of diarrhea did your child have since their last scheduled visit. Note: A new episode is |
| | <i></i> | defined by diarrhea beginning after at least 2 diarrhea-free calendar days. |
| | | (range 1-10) |
| | | child had more than 1 new episodes of diarrhea during the relevant follow-up period (between Enrollment and Week 4 or between |
| | | 4 and Month 3) ask the following questions about the <u>first</u> of those episodes. If the Week 4 visit was missed then the relevant follow-up |
| | | d is defined as between Enrollment and Month 3. When did the diarrhea start? Refer to calendar to |
| | 36. | |
| | 27 | determine date if # of days ago known (dd-mm-yyyy) |
| | 37. | When did the diarrhea end? Refer to calendar to - - 2 0 |
| | | determine date if # of days ago known (dd-mm-yyyy) |
| | | ☐ Ongoing |
| | 38. | Did the child have blood in stool during his/her diarrheal illness? (Use the memory aid to show pictures of each of |
| | | these symptoms) |
| | | Yes |
| | | <u></u> No |
| | | Don't know |
| | 39. | Did the child vomit at any time during the episode of diarrhea? |
| | | Yes |
| | | □ No |
| | | ☐ Don't know |
| | 40. | At any point during the diarrheal episode, did the child have any fever? (Fever meaning the child was hot to |
| | 40. | touch) |
| | | Yes |
| | | □ No |
| | | ☐ Don't know |
| | 41. | Did you seek care for the child's diarrhea outside your home? |
| | | Yes (skip to Q42) |
| | | □ No |
| | | 41a. If No to Q41, why not? (check all that apply then skip to Q51) |
| | | Child did not seem to need care |
| | | ☐ Clinic too far from home ☐ Cost for travel too high |
| | | Unable to find transport Other child at home could not be left alone |
| | | ☐ Flood or bad weather ☐ Other (on a rife) |
| | | Dolitical unrest |
| | 42. | When did you first seek care for the child's illness? Refer |
| | | to visual calendar aid carried by staff member to - - 2 0 |
| | | determine date relative to the date the episode started (as (dd-mm-yyyy) |
| | | recorded in Q36). |
| | 43. | If you sought care for the child for this diarrheal illness where did you go (check all that apply)? |
| | | ☐ Traditional healer ☐ Religious healer |

| , | | y | · |
|---|---|---|---|
| | | ☐ Drug seller | Pharmacist |
| | | Community health worker | Health outpost |
| | | Health facility (outpatient care) | Health facility (inpatient care) |
| | | Other (specify): | |
| | | If sought care at a health facility (either outpatient | or inpatient), continue to Q44. Otherwise, skip to Q51. |
| | 44. | What was the name of the hospital or health center th | at you visited? |
| | | EFGH recruiting facility, specify facility ID: | Other (specify): |
| | | <u> </u> | ☐ Don't remember |
| | 45. | When did you first visit the hospital or health | - - 2 0 |
| | | center? | (dd-mm-yyyy) |
| | | Refer to visual calendar aid carried by staff member to | Same as Q42 |
| | | determine date relative to the date the episode | |
| | | started. | |
| | 46. | Did the clinical team advise the child be hospitalized for | or treatment of diarrheal illness? |
| | | Yes | |
| | | No (skip to Q51) | |
| | 47. | | or treatment of diarrheal illness? (This question is intended |
| | | to differentiate between a child recommended to be add | mittea and actually damittea to the nospital) |
| | | Yes No (skip to Q51) | |
| | 40 | Date of admission: | |
| | 48. | - - 2 0 (dd-mm-yyy) | ,) |
| | | Same as date in Q45 | <i>''</i> |
| | | Don't remember | |
| | | | days |
| | 49. | How many days was the child admitted for? | Don't remember |
| | 50. | Was a Hospital Record Abstraction CRF (CRF 09) was co | <u> </u> |
| | | Yes | |
| | | ☐ No (complete a Hospital Record Abstraction CRF (CR | F 09)) |
| | | No, child was admitted to a non-EFGH facility (see Q | 44) |
| | | New other (non-diarrheal) illnesse | s since last scheduled study visit |
| | 51. | Since this child's last scheduled visit (either Enrollment | or Week 4), did your child become ill with any illness |
| | | besides diarrhea? | |
| | | Yes | |
| | | No (skip to Section H) | |
| | | Don't know (skip to Section H) | |
| | 52. | If yes, what was the illness your child had? | |
| | | Cough, respiratory distress | |
| | | Febrile illness | |
| | | Other (specify): | |
| | 53. | Did you seek any medical advice or treatment for this | illness? |

| , | r | · | | |
|---|---|---|---|---|
| | | Yes | | |
| | | ☐ No (skip to Section H) | | |
| | | Don't know (skip to Section H) | | |
| | 54. | If yes, from whom did you seek advice about care for | you | r child or where did you seek other medical treatment |
| | | (not including the current clinic visit) (check all that we | re co | onsulted) |
| | | ☐ Traditional healer | | Religious healer |
| | | Drug seller | | Pharmacist |
| | | Community health worker | | Health outpost |
| | | Health facility (outpatient care) | | Health facility (inpatient care) |
| | | Other (specify): | | |
| | | If sought care at a health facility (inpatient or ou | tpa | tient), continue to Q55. Otherwise, go to Section H |
| | | Immuniz | atic | n History. |
| | 55. | What was the name of the hospital or health center the | nat | you visited? |
| | | EFGH recruiting facility, specify facility ID: | | Other (specify): |
| | | LFGITTect ditting facility, specify facility 10. | _1 | ☐ Don't remember |
| | 56. | When did you first visit the hospital or health center? | | _ - - - 2 0 |
| | | Refer to visual calendar aid carried by staff member to | | (dd-mm-yyyy) |
| | | determine date relative to the date the episode started | | Don't remember |
| | 57. | Did the clinical team advise the child be hospitalized? | | |
| | 37. | Yes | | |
| | | No (skip to Q61) | | |
| | 58. | Was the child admitted (i.e, at least an overnight stay) | for | treatment of the illness? (This question is intended to |
| | | differentiate between a child recommended to be admi | | |
| | | Yes | | |
| | | □ No (skip to Q63) | | |
| | | Don't know (skip to Q63) | | |
| | 59. | Date of admission: | | |
| | | - - 2 0 (dd-mm-yyy | 'y) | |
| | | Same as date in Q56 | | |
| | | ☐ Don't remember | | |
| | 60. | How many days was the child admitted for? | | days OR 🗌 Don't remember |
| | | What was the diagnosis/diagnoses that your child rec | eive | ed at the health facility or hospital? (check all that |
| | 61. | apply) | | |
| | | ☐ Diarrhea | | Dysentery |
| | | Gastroenteritis | | HIV |
| | | ☐ Anemia | | Urinary Tract Infection |
| | | ☐ Sickle cell | | Tuberculosis |
| | | ☐ Malaria | | Fever of unknown origin/Febrile illness |
| | | Suspected sepsis | | ] Pneumonia |
| | | Upper respiratory tract infection | | Meningitis |
| | | Other lower respiratory tract infections | ÌГ | Poisoning/ herbal intoxication |

| ĺ | T | | | | |
|---|---|---|---|---|---|
| | | Acutely unwell, unknown cause | | Severe acute malnutrition/ severe wasting | |
| | | Asthma | | Moderate acute malnutrition/ moderate w | asting |
| | | Other 1 (specify): | | Other 2 (specify): | |
| | | ☐ None | | Don't know | |
| | 62. | Was a Hospital Record Abstraction CRF (CRF 0 | 9) complet | ed for this hospitalization? | |
| | | Yes | | | |
| | | No (complete a Hospital Record Abstractio | | | |
| | | No, child was admitted to a non-EFGH faci | | | |
| н. | | UNIZATION HISTORY (complete at Week 4 FU v | isit ONLY if | fimmunization record was not available at Enro | llment |
| | Visit) | | 11 | | |
| | 63. | Was the child's immunization record not avail | able at Enr | ollment and is available for abstraction now? | |
| | | Yes | | | |
| | | No (skip to Section I) | | | |
| | | Not applicable (skip to Section I) | | | |
| | 64. | • | • | s of the following vaccines the child has receive | |
| | | | - | art of a composite vaccine but not alone (e.g. m | |
| | | | omponent | (e.g. measles) and "1" to the composite (MMR) | <u> </u> |
| | | Rotavirus vaccine | | Bacille Calmette-Guerin (BCG) | 11 |
| | | Polio vaccine (OPV or IPV) | | Rubella vaccine | |
| | | Pentavalent vaccine (DPT+HiB+HBV) | | HiB vaccine (Hemophilus influenzae) | II |
| | | S. pneumococcus vaccine (PCV) | | Hepatitis A vaccine | |
| | | Measles vaccine | | Hepatitis B vaccine | |
| | | MR vaccine (measles+rubella) | | Typhoid fever vaccine | |
| | | MMR vaccine (measles+mumps+rubella) | | Varicella vaccine | |
| | | Yellow fever vaccine | | Meningococcal A vaccine | |
| | | DPT vaccine (Diphteria+pertussis+tetanus) | | Malaria vaccine (RTS,S) | |
| | 65. | How many doses of Vitamin A has the child re | | (enter 9 if unknown) | |
| I. | : | UNIZATION WILLINGNESS – WEEK 4 ONLY (con | - | <del>-</del> | |
| | 66. | When offered a new vaccine for your child, do | you typica | ally accept? | |
| | | Yes, always (skip to Q68) | | | |
| | | Sometimes | | | |
| | | Never | | | |
| | 67. | What deters you from accepting new vaccines | for your cl | niid? (select one) | |
| | | Vaccines are too expensive | | | |
| | | Vaccines are not available | | | |
| | | Do not think vaccines are safe | | | |
| | | Do not know about vaccines | | | |
| | | Other (specify): | | | - :12 |
| | 68. | | watery dia | ary and bloody diarrhea, would you agree to use | ) IT? |
| | | Yes (skip to visit-specific staff checks) | | | |

| 1 | | 1 | | | | |
|---|---|---|---|---|---|---|
| | | 68a. | ļ <u></u> | | ring reasons would deter yo | ou? (select one) |
| | | | ☐ Vaccines are too expensive | | | |
| | | | ☐ Vaccines are not available | | | |
| | | | ☐ D( | o not think vaccines | are safe | |
| | | | D | o not know about v | accines | |
| | | | | ther (specify): | | |
| J. | STUE | DY STAF | F CHEC | KS – WEEK 4 ONLY | | |
| | 69. | Please | e verify | the following proce | dures were completed as p | part of the follow-up visit: |
| | | Comp | oleted | Not completed | | |
| | | | | | Follow up CRF (CRF 07) co | mpleted |
| | | | | | Child length/height, weight Follow up CRF (CRF 07) | nt, and MUAC were collected and recorded in Section D of |
| | | | | | Dried blood Spot (DBS) collected, labelled as appropriate, and stored = Applicable only to sites participating in immune response sub-study and in whom the caregiver agreed to have blood sample taken. If not participating select "Not applicable to this visit") | |
| | | | | | Diarrhea diary returned | |
| | | | | | Diarrhea duration diary is information is clarified | reviewed with the caregiver and any missing or illegible |
| | | | | | Participant is reminded of | next scheduled follow up visit |
| | | | | | Appropriate reimburseme | nts issued |
| K. | STUE | OY STAF | F CHEC | KS – MONTH 3 ON | LY | |
| | 70. | Please | e verify | the following proce | dures were completed as p | part of the follow-up visit: |
| | | | | | Follow up CRF (CRF 07) co | mpleted |
| | | | | | Child length/height, weight Follow up CRF (CRF 07) | nt, and MUAC were collected and recorded in Section D of |
| | | | | | Appropriate reimburseme | nts issued |
| | | | | | Study Close Out CRF (CRF | 10) completed |
| L. | FORI | и сом | PLETIO | N | | |
| | 71. | ID of p | person | completing this for | m: | Date form completed: - - 2 0 (dd-mm-yyyy) |
| | 71. | ID of p | oerson | reviewing this form | : | Date form reviewed: _ - - 2 0 (dd-mm-yyyy) |
| | 72. | ID of p | person | entering this form: | ll | Date form entered:<br> - - 2 0 (dd-mm-yyyy) |
| | 73. | ID of person conducting data verification: | | rification: | Date of data verification: - - 2 0 (dd-mm-yyyy) | |

Purpose: To be completed when a study participant was deemed to be unwell during Shigella culture positive light contact; returned for a scheduled follow up visit and was determined to be unwell based on EFGH clinical team assessment; or the study participant sought care at the study clinic at a time other than the scheduled follow-up visits. Form to only be completed if child is physically present based on information ascertained, in real-time, during presentation. Instructions: Please complete this form for all enrolled participants who seek care at an EFGH recruiting facility outside of their scheduled follow-up visits, who are deemed unwell during their scheduled follow-up visit, or who have been asked to return to the facility for assessment after receiving a Shigella culture positive result. Please also complete an AE form if the illness is definitely, probably, or possibly related to study participation. Text in **bold** should be read to study participants, plain text is for prompts for study staff, and italics are instructions for study staff. PLEASE PLACE PARTICIPANT LABEL HERE (OPTIONAL): A. **PARTICIPANT INFORMATION** Participant ID: 2. Date the child presented to the facility: \_| - | 2 | 0 |\_\_\_| (dd-mm-yyyy) 3. Time form is started: (hh: min, 24:00 hr) 4. EFGH country site: ☐ Bangladesh ☐ Kenya ☐ Malawi ☐ Mali ☐ Pakistan ☐ Peru ☐ The Gambia What are the circumstances that lead to this unwell assessment? ☐ Child was identified to be unwell during a scheduled study follow up visit ☐ Child returned for care because he/she was experiencing symptoms or was ill ☐ Child was deemed unwell during *Shigella* culture positive light contact  $\square$  Other (specify): 6. I'm sorry to hear your child isn't feeling well. What are the primary health concerns of your child today? (check all that apply) ☐ Convulsing ☐ Fever/hotness of body ☐ Excessive crying ☐ Night sweats ☐ Ear problem ☐ Cough ☐ Eye problem  $\square$  *If yes,* Cough up blood? ☐ Not drinking and/or not eating ☐ Difficulty breathing/ wheeze ☐ Malaise ☐ Diarrhea ☐ Restless/irritable  $\square$  *If yes,* Blood in stool? ☐ Rash/itching ☐ Vomiting ☐ Swelling of the lips ☐ Trauma ☐ Other (*specify*): 7. When did this illness begin? |-|2|0| | (dd-mm-yyyy)

| | | - | tiple concerns reported in | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | on the date the first ill | | | | | | | | |
| | | Refer to calendar to determine date if # of | | | | | | | | | |
| | | days since illness began is known but not exact date | | | | | | | | | |
| В. | M | | EXAMINATION | | | | | | | | |
| υ. | 8. | | is the child's general cond | lition? | | | | | | | |
| | 0. | | ell/Alert | Restless/Irrit | tablo | | ТΠ | Lotha | argic or Unconsciou | | |
| | 9. | | s the child's eyes and dete | ······································ | | | | Letile | argic or officorisciou | | |
| | J. | | rmal (skip to Q10) | □ Abnormally | | | | Not r | ecorded (skip to Q | <br>10) | |
| | | 9a. | If child's eyes are determ | <del>-</del> | | iken i | | | | | on |
| | | Ju. | please ask the caregiver | | • | | | | - | rradeced in perso | 011, |
| | | | ☐ Yes (abnormal for chil | | <del>-</del> | | | • | | | |
| | | | □No | , | | | | | | | |
| | 10. | Descr | ibe the child's ability to dr | ink or breastfee | d: | | | | | | |
| | | □ No | rmal/Not Thirsty | ☐ Drinks eager | ly/Thirsty | / | | Drink | s poorly/ Unable to | o drink | |
| | 11. | Using | a thumb and forefinger, g | ently pinch up tl | he child's | skin | on th | ne ab | dominal wall and a | ssess the skin's | |
| | 11. | returr | n to normal: | | | | | | | | |
| | | | mediately | ☐ 1 to <2 second | nds (slow | ly) | | ≥2 se | conds(very slowly) | | |
| | | | ss the following physical si | | | | | | | | |
| | 12. | | erature (using Exergen Th | ermometer) | | <u> </u> | <u> </u> | <u> . </u> | _ °C | | |
| | 13. | Heart | | | | <u> </u> | <u> </u> | <u> </u> | beats per minute | | |
| | 14. | <del>-</del> | ratory rate | | | breaths per minute | | | | | |
| | 15. | Cough | | | | ☐ Yes ☐ No | | | | | |
| | 16. | | ulty breathing | | | ☐ Yes ☐ No | | | | | |
| | 17. | | in-drawing | | | ☐ Yes ☐ No | | | | | |
| | 18. | Strido | | | | ☐ Yes ☐ No | | | | | |
| | 19. | Stiff n | | | | ☐ Yes ☐ No | | | | | |
| | 20. | | ralized rash | | | ☐ Yes ☐ No | | | | | |
| | 21. | Runny | | | | □ Ye | | | | | |
| | 22. | Convu | | | | □ Ye | | | | | |
| | 23. | | rgy or Unconscious | | | □ Ye | | | | | |
| | 24. | Chest auscultation signs suggestive of pneumonia | | | | □ Ye | | | | | |
| | 25. | ļ | | | | □ Ye | | | | | |
| | 26. | ,,, | | | | ☐ Yes ☐ No ☐ Not available | | | | | |
| | 27. | | e respiratory distress | | | □ Ye | | | | | |
| | 28. | | r pallor | | | □ Ye | | | | | |
| | 29. | Ear pa | | | | □ Ye | | | | | |
| | 30. | | rainage from ear canal | | | □ Ye | | | | | |
| | 31. | | er swelling behind the ear | | | □ Ye | | | | | |
| | 32. | <u>.</u> | of abscess | | | □Y€ | | | | | |
| | 33. | Signs | Signs of oedema | | | □ Ye | es 🗆 | No | | | |

| | | 33a. | If yes: | | | | |
|---|---|---|---|---|---|---|---|
| | | | ☐ Oedema on both feet/ar | nkles <i>(mild)</i> | | | |
| | | | ☐ Oedema on both feet/ar | nkles, lower legs, h | ands, or | lower arms (moderate) | |
| | | | ☐ Generalized oedema, inc | cluding both feet, I | egs, hand | ds, arms, and face (severe | ?) |
| | 34. | Tick a | ll diagnoses applicable (as de | etermined by facili | lity standard of care, check all that apply) | | |
| | | ☐ Dia | arrhea (watery) | | ☐ Diarr | hea (dysentery) | |
| | | □An | emia | | □HIV | | |
| | | ☐ Sic | kle cell | | ☐ Urina | ary Tract Infection | |
| | | □Ма | alaria | | □ Tube | erculosis | |
| | | ☐ Sus | spected sepsis | | ☐ Feve | r of unknown origin/Febr | ile illness |
| | | □Up | per respiratory tract infectio | n | ☐ Pneu | ımonia | |
| | | ☐ Otl | her lower respiratory tract in | fections | ☐ Men | ingitis | |
| | | ☐ Acı | utely unwell, unknown cause | } | ☐ Poiso | oning/ herbal intoxication | |
| | | ☐ Ast | :hma | | ☐ Seve | re acute malnutrition/ se | vere wasting |
| | | | oderate acute malnutrition/ r | moderate | Soft | tissue/skin infection | |
| | | wasti | ng<br>her 1 <i>(specify)</i> : | | □ Otho | ar 2 (specify) | |
| | | Oti | iei 1 (specijy) | | | □ Other 2 (specify):<br>□ None | |
| | 35. | What | was the outcome of the illne | ess visit? | L NOITE | <b>-</b> | |
| | 33. | | ild was hospitalized (Complet | | | | |
| | | 1 | action Form [CRF 09]) | | ☐ Child was seen as an outpatient and returned home | | |
| | | .4 | her (specify): | | | | |
| | Skip | o to Sec | , , , | | as due to child returning after a Shigella culture positive | | |
| | | | | | | inwell or not yet recovere | |
| C. | | | ENT FOLLOWING LIGHT CON<br>whose Unwell Visit is becau | | | | • • • |
| | 36. | | new Shigella treatment presc | | | | ive contact, |
| | | ☐ Yes | i | | | | |
| | | | (skip to Section D: Form Con | npletion) | | | |
| | 27 | Name | · | Dose prescril | oed | Prescribed Duration | Drocorintian filled |
| | 37. | (check | box if prescribed) | (circle unit | ) | Prescribed Duration | Prescription filled |
| | | | (I) (C) | (ml | /mg) | days | □ Yes |
| | | ☐ Cip | rofloxacin (Cipro) | ☐ Unknow | n | ☐ Unknown | ☐ No<br>☐ Unknown |
| | | | | | | | Yes |
| | | ☐ Azit | thromycin | | /mg) | days | □ No |
| | | | ···· · | ☐ Unknow | n | ☐ Unknown | □ Unknown |
| | | | | /ml | /mg) | days | □ Yes |
| | | ☐ Cot | rimoxazole (Septrin) | (\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\ | | □ Unknown | □ No |
| | | | | LI OTINIOW | | L OTIKITOWIT | □ Unknown |
| | | | | (ml | /mg) | days | □ Yes |
| | | ⊔ Cef | triaxone | □ Unknow | | ☐ Unknown | □ No |
| | | | | | | □ Unknown | |

| | | □ Cefixime | (ml, | /mg)<br>n | days<br>□ Unknown | ☐ Yes<br>☐ No<br>☐ Unknown |
|---|---|---|---|---|---|---|
| | | ☐ Other 1 (specify): | (ml, | /mg)<br>n | days<br>Unknown | ☐ Yes<br>☐ No<br>☐ Unknown |
| | | ☐ Other 2 (specify): | (ml, | /mg)<br>n | days<br>Unknown | ☐ Yes<br>☐ No<br>☐ Unknown |
| | 38. | Were there any other recommend | led changes in the | child's cl | inical management? | |
| | | Yes | | | | |
| | | No (skip to Section D: Form Co | mpletion) | | | |
| | 39. | Please describe those changes in t | he child's clinical r | managem | ent (check all that apply) | |
| | | Change in recommended fluids | S | | | |
| | | Zinc prescribed | | | | |
| | | ☐ Nutritional therapy | | | | |
| | | Other (specify): | | | | |
| D. | FORI | M COMPLETION | | | | |
| | 40. | ID of person completing this form: | : | Date for | rm completed:<br> - - 2 0 _ | _ (dd-mm-yyyy) |
| | 41. | ID of person reviewing this form: | | Date for | rm reviewed:<br> - - 2 0 _ | _ (dd-mm-yyyy) |
| | 42. | ID of person entering this form: _ | | Date for | rm entered:<br> - - 2 0 _ | _ (dd-mm-yyyy) |
| | 43. | ID of person conducting data verif | ication: | Date of | data verification:<br> - - 2 0 _ | _ (dd-mm-yyyy) |

#### Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name/Country Site CRF 09— Hospital Record Abstraction Form

**Purpose:** To abstract important information from the child's medical record every time the child is hospitalized at an EFGH recruitment facility. If a child is only seen as an outpatient, do not complete this form.

**Instructions:** Please abstract the following information from the child's medical record as soon as staff learn of a hospitalization. Please use a separate form for every hospital admission other than a hospital admission that occurred as part of the child's enrollment visit. Please also complete an AE form if the illness is definitely, probably, or possibly related to study participation.

| PLE. | PLEASE PLACE PARTICIPANT LABEL HERE (OPTIONAL): | | | |
|---|---|---|---|---|
| A. | PAR | TICIPANT INFORMATION | | |
| | 1. | Participant ID | | l <u> </u> |
| | 2. | Date of Enrollment: | - - 2 | 0 (dd-mm-yyyy) |
| | 3. | Date of Form Completion: | - - 2 | 0 (dd-mm-yyyy) |
| | 4. | EFGH country site: | | |
| | | ☐ Bangladesh | ☐ Kenya | ☐ Malawi ☐ Mali |
| | | ☐ Pakistan | ☐ Peru | ☐ The Gambia |
| В. | ADN | IISSION INFORMATION | | |
| | 5. | Was the child admitted to | either an inpatient ward or | short-stay ward? |
| | | ☐ Inpatient ward | | |
| | | Complete the follow | ing for inpatient ward admis | |
| | | Date admitted to in | patient ward: | _ - - 2 0 (dd-mm-yyyy) |
| | | Time admitted to in | patient ward: | : (hh : min, 24:00 hr) ☐ Unknown |
| | | ☐ Short-stay ward (e.g. er | nergency room) | |
| | | Complete the follow | ing for short-stay ward adm | issions only. |
| | | Date admitted to sh | ort-stay ward: | - - 2 0 (dd-<br>mm-yyyy) |
| | | Time admitted to sh | ort-stay ward: | : (hh : min, 24:00 hr) □ Unknown |
| | 6. | What was the EFGH healt | n facility ID for the facility tha | at the child was admitted to? (refer to EFGH facility list) |
| | | <u> </u> | | |
| C. | DISC | HARGE INFORMATION | | |
| | 7. | What was the outcome of | the admission? | |
| | | Child was discharged | _ - 2 0 <u> </u> ( <i>dd-mm-yyyy)</i> □ Unknown<br> ( <i>hh : min, 24:00 hr</i> ) □ Unknown | |
| | | Child was referred | Time: : : Date: _ - | - 2 0 <i>(dd-mm-yyyy)</i> |
| | | Child died | Time: : | _ (hh : min, 24:00 hr) □ Unknown |
| | | | Date: - | _ - 2 0 <u> </u> ( <i>dd-mm-yyyy)</i> □ Unknown |

# Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name/Country Site CRF 09— Hospital Record Abstraction Form

| | | | Time: : | <i>(hh : min, 24:00 hr)</i> □ Unknown |
|---|---|---|---|---|
| | | | Date: - | - 2 0 <i>(dd-mm-yyyy)</i> □ Unknown |
| | | Child absconded | Time: : | |
| | 8. | Final Diagnosis(es) (check | all that apply) | |
| | | Diarrhea | | ☐ Dysentery |
| | | Gastroenteritis | | Anemia |
| | | Sickle cell | | HIV |
| | | ☐ Malaria | | ☐ Urinary Tract Infection |
| | | Suspected sepsis | | Tuberculosis |
| | | Upper respiratory trac | t infection | Fever of unknown origin/Febrile illness |
| | | Other lower respirator | y tract infections | Pneumonia |
| | | Acutely unwell, unkno | wn cause | Meningitis |
| | | Asthma | | Poisoning/ herbal intoxication |
| | | Moderate acute maln | utrition/ moderate wasting | Severe acute malnutrition/ severe wasting |
| | | ☐ None | | Soft tissue/skin infection |
| | | Other 1 (specify): | | U Other 2 |
| | | | | (specify): |
| D. | FOR | M COMPLETION | | |
| | 9. | ID of person completing t | nis form: | Date form completed: |
| | 10 | 1D ( ' | | _ _ - _ - 2 0 _ (dd-mm-yyyy) |
| | 10. | ID of person reviewing thi | s form: | Date form reviewed: |
| | 11. | ID of person entering this | form: | _ - - 2 0 (dd-mm-yyyy) Date form entered: |
| | 11. | ib of person entering this | 101111. 111 | _ - _ - 2 0 _ (dd-mm-yyyy) |
| | 12. | ID of person conducting d | ata verification: | Date of data verification: |
| | | | | _ - - 2 0 (dd-mm-yyyy) |

**Purpose:** To be completed when the staff learn a participant has passed away.

**Instructions:** Please complete this form for all participants who pass away. Note this form does <u>not</u> require a full caregiver interview. Please also complete an AE CRF if the mortality is definitely, probably, or possibly related to study participation. Please ensure a Study Close Out CRF is completed as soon as the staff are made aware of the death. Text in **bold** should be read to study participants, plain text is for prompts for study staff, and *italics* are instructions for study staff.

| 101 | Tot study start. | | | | | | |
|---|---|---|---|---|---|---|---|
| A. | PAR | TICIPANT INFORMATION | | | | | |
| | 1. | Participant ID: | | | | | |
| | 2. | Date of form completion: | | ll_ | - - 2 0 | (dd-mm-yyyy) | |
| | 3. | EFGH | country site: | | | | |
| | | □ Ва | ngladesh | ☐ Kenya | | ☐ Malawi | ☐ Mali |
| | | ☐ Pal | kistan | ☐ Peru | | ☐ The Gambia | |
| В. | INFC | RMAT | ION ABOUT THE DEA | TH | | | |
| | 4. | How | did the study staff lea | arn of the child's | death? | | |
| | | ☐ Ca | regiver attended reg | ularly scheduled | study visit | and informed study staf | f |
| | | ☐ Ca | regiver alerted study | staff of the deat | th outside o | of regularly scheduled co | ntacts |
| | | ☐ Stu | ıdy staff learned abo | ut the death froi | m commun | ity members outside of l | nealth facility |
| | | □ Не | alth facility staff info | rmed study staff | of the dea | th | |
| | | □ Ch | ild died while under I | FGH clinical tea | m's care | | |
| | | ☐ Other (specify): | | | | | |
| | 5. | Where did the death occur? | | | | | |
| | | ☐ Health facility | | | | | |
| | | □ Home | | | | | |
| | | ☐ On the way to the health facility | | | | | |
| | | □ Ot | □ Other (specify): | | | | |
| | 6. | Is a de | eath certificate or de | ath notification | form availa | ble? | |
| | | □Yes | 5 | | | | |
| | | □ No | (skip to Q10) | | | | |
| | | 6a. | If yes, is the caregiv | er willing to sha | re it or do | you have access to it? | |
| | | | □ Yes | | | | |
| | | □ No (skip to Q10) | | | | | |
| | 7. | Date of death listed on death certificate or death notification form: | | | | | |
| | | - - 2 0 (dd-mm-yyyy) □ Missing | | | | | |
| | 8. | Pleas | | | | n certificate or death not | ification form |
| | | Imme | diate (1a): | | | | |
| | | | mediate (1b): | | | | |
| | | Underlying (1c): | | | | | |

| | 9. | Please note other significant conditions contributing to the death, but not related to the disease or condition causing it (2) (then skip to Q15) | | |
|---|---|---|---|---|
| | | ☐ Missing | | |
| | 10. | If death certificate was <u>not</u> available, approximately | wh | nen did the death occur (based on caregiver report |
| | | or community knowledge)? | | , |
| | | - - 2 0 (dd-mr | т-у | <i>yyyy)</i> □ Unknown |
| | 11. | | | |
| | | ☐ Yes (Complete Section C. Treating Clinician Intervie | ew, | ) |
| | | □ No (skip to Section D) | | |
| C. | TDEA | TING CLINICIAN INTERVIEW | | |
| C. | | | | |
| | the c | The following section is intended to capture the open interview with the physician/clinician who was managing the child prior to their passing. Please listen closely to the physician's description of the events and enter them not the section below and then identify whether or not key terms were mentioned by the clinician. Check all terms mentioned by the physician in Q13. | | |
| | 12a. | Staff ID of person conducting clinician Interview: | _1. | |
| | 12b. | Please ask the physician: Can you please tell me in your own words about the events that led to the death? Record detailed notes of response in English, Spanish, or French; use additional paper as needed. If needed, probe for additional details on when respondent recognized symptoms, changed management plans, what diagnostic tests were performed etc. | | |
| | 13. Select any of the following words that were mentioned in the physician's narrative (check all that a | | | |
| | 13. | | ea | <u></u> |
| | | ☐ Abdominal pain ☐ Bleeding or hemorrhage | 늗늗 | Abdominal swelling<br>Cancer |
| | | Cough | ┝ | COVID-19/COVID |
| | | Dehydration | ┢ | Dengue fever |
| | | Diarrhea | Ī | Fever |
| | | Heart problems | Ē | Jaundice (yellow skin or eyes) |
| | | HIV/AIDS | | Malaria |
| | | Pneumonia | | Poisoning |
| | | Rash | | Seizure |

| | · | | · — |
|---|---|---|---|
| | | Shortness of breath/ difficulty breathing | Trauma/accident/injury |
| | | Typhoid | Sepsis |
| | | None of the above were mentioned | ☐Don't know |
| | | Other key words (specify 1-2): | |
| | 14. | Cause of death based on physician description | |
| | | Immediate (1a): | Not applicable |
| | | Intermediate (1b): | |
| | | Underlying (1c): | Not applicable |
| D. | CAR | EGIVER INTERVIEW | |
| | 15. | Is the caregiver willing to participate in a brief interv | iew? |
| | | ☐ Yes (when appropriate, proceed with Interview addition to the remaining question on this form) | and complete Mortality Interview CRF [CRF 10b] in |
| | | ☐ No (Complete Study Close Out CRF [CRF 11] in add | lition to Section E) |
| E. | FOR | M COMPLETION | |
| | 16. | ID of person completing this form: | Date form completed: - - _2 0 (dd-mm-yyyy) |
| | 17. | ID of person reviewing this form: | Date form reviewed: - - 2 0 (dd-mm-yyyy) |
| | 18. | ID of person entering this form: | Date form entered: - - - (dd-mm-yyyy) |
| | 19. | ID of person conducting data verification: | Date of data verification: |

#### Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name/Country Site CRF 10b— Mortality Interview CRF

**Purpose:** To be completed when a study participant passes away at a time that is acceptable to the caregiver

**Instructions:** Please complete this form for all enrolled participants who pass away at an appropriate time (based on site team's discretion) and who agree to be interviewed. Text in **bold** should be read to study participants, plain text is for prompts for study staff, and *italics* are instructions for study staff.

| A. | A. PARTICIPANT INFORMATION | | | | | |
|---|---|---|---|---|---|---|
| | 1. | Participant ID: | | | | |
| | 2. | Date of form completion: | | ll | - - 2 0 (dd-mm-yyyy) | |
| | 3. | Time form is started: | | ll | : (hh : min, 24 | 1:00 hr) |
| | 4. | EFGH country site: | | | | , |
| | | ☐ Bangladesh | ☐ Kenya | | ☐ Malawi | ☐ Mali |
| | | ☐ Pakistan | □ Peru | | ☐ The Gambia | |
| В. | INFO | RMATION ABOUT THE DEA | ГН | | | |
| | 5. | Did the caregiver give con | sent to the verb | al autopsy i | nterview? | |
| | | ☐ Yes | | | | |
| | | ☐ No (stop interview proc | ess, skip to Secti | ion E, Form | Complete) | |
| | 6. | How is the interview being | g conducted? | | | |
| | | ☐ In person at home | | | | |
| | | ☐ In person at an EFGH fa | cility | | | |
| | | ☐ By phone | | | | |
| | 7. | What was the timing of the death in relation to scheduled study follow up visits? | | | 5? | |
| | | ☐Between Enrollment and scheduled Week 4 follow up visits (i.e., Week 4 follow up visit did <u>not</u> occur) | | | | |
| | | ☐Between scheduled Week 4 follow up visit and scheduled Month 3 follow up visit (i.e., Month 3 follow | | | | |
| | | up visit did <u>not</u> occur) (Skij | | | | 1 10 1 11 |
| C. | | RHEA/DYSENTERY RECOVER<br>Been Enrollment and scheduk | | | ALIH FACILITY ( <u>complete d</u> | only if death occurred |
| | the he | 210 through Q16 relate to the period after the child was enrolled in the EFGH study (upon returning home from the health facility visit) and relate to the child's recovery from the illness they were enrolled with. If the caregiver as returned the Diarrhea Diary, that can be used in conjunction with the caregiver's recall to answer the | | | | |
| | Please state to the caregiver: We are so sorry to hear about your loss. Would you be willing to answer a few questions relating to the illness that led to your child's death? The interview will take approximately 10-15 minutes. If there are any questions you would prefer not to answer, you do not have to do so, and may stop the interview at any time. Note to staff: If at any point in the interview the caregiver wishes to stop, please ensure Section E is completed. | | | | | |
| | 8. | Are you [the caregiver] w | illing to proceed | with the ir | nterview? | |
| | | Yes | | | | |
| | | No (skip to Section E) | | | | |
| | 9. | Is the diarrhea diary card | available? | | | |
| | | ☐ Yes No | | | | |

### Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name/Country Site CRF 10b— Mortality Interview CRF

| | 10. | Did your child continue to have diarrhea (defined as 3 or more unusually loose or watery stools in a 24 hour period) after leaving the health facility? | |
|---|---|---|---|
| | | Yes | |
| | | No (skip to Section D) | |
| | | Don't remember (skip to Section D) | |
| | | Missing (skip to Section D) | |
| | 11. | <b>When did the diarrhea end?</b> Refer to calendar to determine date if # of days since leaving the facilit (enrollment) was known but not exact date. Also refer to the daily diary if returned. | y |
| | | - - 2 0 ( <i>dd-mm-yyyy</i> ) | |
| | 12. | On the worst day of diarrhea since leaving the health facility, how many loose stools did the child have | е |
| | | in one day (24 hours)? | |
| | | _ loose stools | |
| | 13. | Did the child have blood in his/her stool during the diarrhea that continued after leaving the health | h |
| | | facility? Yes | |
| | | ☐ No (skip to Q15) | |
| | | Don't remember (skip to Q15) | |
| | 14. | How many days since leaving the health facility did the child have blood in stool? | |
| | | days (if <10, put "0" before digit) | |
| | 15. | Did the child vomit any time during the episode of diarrhea that continued after leaving the health | |
| | | facility? | |
| | | Yes | |
| | | No (skip to Q16) | |
| | | Don't remember (skip to Q16) | |
| | | a. How many days did the child vomit? days (if <10, put "0" before digit) | |
| | | Thinking about the day when the child had the times in the day | |
| | | b. most vomiting, now many times did s/ne vomit (if < 10, nut "0" before digit) | |
| | 1.0 | in the day? | |
| | 16. | Did the child have a fever (or feel hot to the touch) during the diarrhea that continued after leaving the health facility? | e |
| | | ☐ Yes | |
| | | No (skip to Section D) | |
| | | Don't remember (skip to Section D) | |
| | | 16 a. If yes, what was the highest temperature? . . °C | ı |
| | | 16 b. How many days did s/he have the fever? days (if <10, put "0" before digit) | |
| D. | INTER | /IEW | |
| | The fo | lowing section is intended to capture the open interview with the caregiver about events and conditions | |
| | 1 | nding the participant's death. Please listen closely to the caregiver's description of the events and enter | |
| | | nto the section below and then identify whether or not key terms were mentioned by the caregiver. Chec | k |
| | † | ns mentioned by the caregiver in Q18. | |
| | 17a. | ID of person conducting Interview: _ | |
| | 17b. | Please ask the caregiver: Can you please tell me in your own words about the events that led to the death? | |

### Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name/Country Site CRF 10b— Mortality Interview CRF

| | | Record detailed notes of response in English, Spanish, or French; use additional paper as needed. If needed, probe for additional details on when respondent recognized symptoms, care sought, barriers to care, issues with transport, abnormalities, etc. | |
|---|---|---|---|
| | 18. | Select any of the following words that were mention | ned in the caregiver's narrative (check all that |
| | | apply): | |
| | | Abdominal pain | Abdominal swelling |
| | | Bleeding or hemorrhage | Cancer |
| | | Cough | COVID-19/COVID |
| | | Dehydration | Dengue fever |
| | | Diarrhea | Fever |
| | | Heart problems | Jaundice (yellow skin or eyes) |
| | | HIV/AIDS | Malaria |
| | | Pneumonia | Poisoning |
| | | Rash | Seizure |
| | | Sepsis | Shortness of breath/ difficulty breathing |
| | | Trauma/accident/injury None of the above were mentioned | ☐Typhoid ☐Don't know |
| | Other key words (specify 1-2): Cause of death based on interview (only applicable if interviewer is medically trained and ha | | if interviewer is modically trained and has |
| | 19. | completed WHO ICD training). | if interviewer is medically trained and has |
| | | Immediate (1a): | |
| | | Intermediate (1b): | |
| | | Underlying (1c): | |
| | | Not applicable | |
| | Than | | t time. We are very sorry to hear about the loss of your |
| | i | , | our child was sick. Please let me know if you have any |
| | | | th me with any further questions. END OF INTERVIEW. |
| E. | FORN | /I COMPLETION | |
| | | | Date form completed: |
| | 20. | ID of person completing this form: | _ - - 2 0 (dd-mm-yyyy) |
| | | | Date form reviewed: |
| | 21. | ID of person reviewing this form: | _ - - 2 0 (dd-mm-yyyy) |
| | | | Date form entered: |
| | 22. | ID of person entering this form: | _ - - 2 0 (dd-mm-yyyy) |
| | | ID of person conducting data verification: | Date of data verification: |
| | 23. | | |

| Pur | Purpose: To be completed when an enrolled participant is ready to be closed out of the study. | | | | | |
|---|---|---|---|---|---|---|
| | <b>Instructions:</b> Please complete this form for all enrolled participants at the time of study close out. Text in <b>bold</b> should be read to study participants, plain text is for prompts for study staff, and <i>italics</i> are instructions for study staff. | | | | | |
| PLE | PLEASE PLACE PARTICIPANT LABEL HERE (OPTIONAL): | | | | | |
| A. | PAR1 | TICIPANT INFORMATION | - | | | |
| | 1. | Participant ID: | | | | |
| | 2. | Date of form completion: | | | - - 2 0 | _ (dd-mm-yyyy) |
| | 3. | EFGH country site: | | | | |
| | | ☐ Bangladesh | ☐ Kenya | | ☐ Malawi | ☐ Mali |
| | | ☐ Pakistan | □ Peru | | ☐ The Gambia | |
| В. | STUE | DY CLOSE OUT | | | | |
| | 4. | Check all the scheduled follo | w up visits that h | ave occurre | d (check all that have occur | rred): |
| | | □ Week 4 | | | | |
| | | ☐ Month 3 | | | | |
| | 5. | What is the reason for study | close out? | | | |
| | | ☐ Participant completed Month 3 follow up visit | | | | |
| | | □ Voluntary withdrawal by caregiver (specify reason): | | | | |
| | | ☐ Planning to move out of study area ☐ Unhappy with study staff/procedures | | | | |
| | | ☐ Influence from another family member ☐ Unwilling to disclose/preferred not to state | | | | |
| | | ☐ Other (specify): | | | | |
| | | ☐ Eligibility revoked | | | | |
| | | ☐ Participant missed Month visit | 3 follow up visit | AND untrac | eable within 1 month of sch | neduled Month 3 follow up |
| | | If lost to follow up, dat | e of last known v | | f participant:<br>nm-yyyy) | |
| | | ☐ Participant died (please co | · | | | |
| | | ☐ Other reason (specify): | | <u> </u> | | |
| C. | FORI | RM COMPLETION | | | | |
| | 6. | ID of person completing thi | s form: | 1 1 | Date form completed: | |
| | 7. | | | _ ' ' | _ - - 2 <br>Date form reviewed: | 0 (dd-mm-yyyy) |
| | | ID of person reviewing this | torm: | 11 | _ - - 2 <br>Date form entered: | 0 (dd-mm-yyyy) |
| | 8. | ID of person entering this fo | orm: | l | _ - - 2 | 0 <i>(dd-mm-yyyy)</i> |
| | 9. | ID of person conducting dat | ta verification: | | Date of data verification: _ - 2 | |

#### Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name/Country Site CRF 12 - Shigella Light Contact Form

Purpose: To track light contact with enrolled participants with a positive Shigella culture result and capture information about their health status, whether or not they were contacted by the study staff and invited to return to the facility, and outcome of light contact. **Instructions:** Complete this form for any participants with a positive *Shigella* culture result. PLEASE PLACE PARTICIPANT LABEL HERE (OPTIONAL): A. **VISIT INFORMATION** 1. Participant ID \_\_\_|\_\_| - | 2 | 0 |\_\_\_| (dd-mm-yyyy) Enrollment Date: 2. Date of Form Completion: |-|2|0|\_\_\_|\_ (dd-mm-yyyy) 3. EFGH country site: 4. Bangladesh Kenya Malawi Mali Pakistan Peru The Gambia PARTICIPANT CONTACT INFORMATION В. Did you successfully make contact with the participant's caregiver? Yes No (skip to Q6) If yes, what was the date of contact |\_\_\_|\_| - |\_\_\_| - | 2 | 0 |\_\_\_| (dd-mm-yyyy) 5b. If yes, what method of contact was used? In-person at home In-person in the facility By phone Other (specify): If yes, At the time of light contact, how was the child doing? 5c. Child has improved since enrollment in the study (skip to Q7) Child is doing the same as when the child was enrolled in the study\* (skip to Q7) Child is doing worse\* (skip to Q7) Learned that child died (skip to Section D: Form Completion, complete CRF 11 - Study Close Out CRF and CRF 10a – Mortality CRF. Proceed with Mortality Interview if appropriate.) \*If the child is doing the same and/or worse, invite child and caregiver back to the health facility for further assessment. If they return to the facility, please complete CRF 08 - Unwell Child CRF. How many attempts were made to contact the caregiver? 6. \_| attempts

### Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name/Country Site CRF 12 - Shigella Light Contact Form

| С | OUT | TCOME OF LIGHT CONTACT | |
|---|---|---|---|
| | 7. | What was the outcome of the light contact? | |
| | | ☐ No further action by study staff, caregiver reported child's condition had improved | |
| | | Caregiver agreed to bring participant to EFGH facility for Unwell Child Visit (Complete CRF 08) | |
| | | Caregiver refused to bring participant to EFGH fa | ncility for Unwell Child Visit |
| | | Staff were not able to successfully contact the caregiver | |
| D. | FOR | FORM COMPLETION | |
| | 8. | ID of person completing this form: | Date form completed: |
| | | | _ - - 2 0 _ (dd-mm-yyyy) |
| | 9. | ID of person reviewing this form: | Date form reviewed: |
| | | | _ - - 2 0 _ (dd-mm-yyyy) |
| | 10. | ID of person entering this form: | Date form entered: |
| | | | _ - - 2 0 _ (dd-mm-yyyy) |
| | 11. | ID of person conducting data verification: | Date of data verification: |
| | | | _ - - 2 0 (dd-mm-yyyy) |
#### Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name/Country Site CRF 13 - Stool Sample Collection Form

**Purpose:** To capture information about fecal sample collection at the recruiting sites (separate Specimen Accession RCRF to be completed by central laboratory).

**Instructions:** Complete this form for all enrolled participants at Enrollment Visit.

| PL | EASE I | PLACE | PARTICIPANT LA | ABEL HERE (OPTIONAL): | PLEASE PLACE SPECIMEN ID LABEL HERE (OPTIONAL): |
|---|---|---|---|---|---|
| A. | VISIT | ΓINFO | RMATION | | |
| | 1. | Parti | cipant ID | | . |
| | 2. | Enro | llment Date: | _ - - 2 | 0 (dd-mm-yyyy) |
| | 3. | EFGH | l country site: | | |
| | | В | angladesh | | ☐ Kenya |
| | | □ N | ⁄lalawi | | ☐ Mali |
| | | □Р | akistan | | ☐ Peru |
| | | Т | he Gambia | | |
| В. | RECT | TAL SW | AB COLLECTION | N INFORMATION | |
| | 4. | How | many rectal swa | bs were collected? | |
| | | □ 0 | rectal swabs | | |
| | | 1 | rectal swab (dry | for TAC) | |
| | | 2 | rectal swabs (dr | y for TAC, mBGS) | |
| | | <u></u> 3 | rectal swabs (dr | y for TAC, mBGS, Cary-Blair, sk | ip to Q5) |
| | | 4a. | If <3 swabs we | re collected, why? | |
| | | | | Skip to Section C if | f 0 rectal swabs were collected |
| | 5. | Date | of swab collection | ·· | 2 0 (dd-mm-yyyy) |
| | 6. | Time | of swab collection | | same as date of enrollment (Q2) |
| | 7. | | | swabs collected have visible blo | |
| | ,. | <u> </u> | es | | |
| | | $+ \equiv -$ | lo | | |
| | 8. | Recta | al swab 1 (Dry sw | vab for freezing) | k if rectal swab 1 is missing (skip to Section C) |
| | | 8a. | | swab collected from? | |
| | | | Directly fro | m the child's rectum | |
| | | | ☐ Whole stoo | ol sample ( <i>only acceptable if dir</i> | rect swab is unable to be collected) |
| | | 8b. | Specimen ID: _ | | ☐ Not applicable |
| | 9. | Recta | al swab 2 (mBGS | transport media) | k if rectal swab 2 is missing (skip to Section C) |


#### Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name/Country Site CRF 13 - Stool Sample Collection Form

| | | 9a. | Where was the swab collected from? | |
|---|---|---|---|---|
| | | | ☐ Directly from the child's rectum | |
| | | | ☐ Whole stool sample ( <i>only acceptable if direct</i> | swab is unable to be collected) |
| | | 9b. | Time of placement in media: : | (hh : min, 24:00hr) |
| | | 9c. | Specimen ID: | ☐ Not applicable |
| | 10. | Recta | al swab 3 (Cary-Blair transport media) 🔲 Check | if rectal swab 3 is missing (skip to Section C) |
| | | 10a. | Where was the swab collected from? | |
| | | | ☐ Directly from the child's rectum | |
| | | | Whole stool sample (only acceptable if direct | swab is unable to be collected) |
| | | 10b. | Time of placement in media: : | (hh : min, 24:00 hr) |
| | | 10c. | Specimen ID: | Not applicable |
| C. | WHO | DLE STO | OOL COLLECTION INFORMATION | |
| | 11. | Was | whole stool collected prior to the child leaving the | health facility? |
| | | ☐ Y | es | |
| | | □ N | o (skip to Section D; For The Gambia, Peru, Malaw | i, Pakistan and Bangladesh sites – instruct caregivers about |
| | | home | e whole stool collection) | |
| | | 11a. | | |
| | | | ☐ Yes | |
| | | | No | |
| | | 11b. | Date of whole stool collection: - Date of collection is same as date of enrollment | |
| | | 11c. | Time of whole stool collection: : | |
| | | 11d. | Specimen ID: | ☐ Not applicable |
| | | + | angladesh and the Gambia sites complete Q11e; a | |
| | | 11e. | Time of placement in Cary-Blair media: | · |
| D. | SANA | DIETE | ANSPORT INFORMATION | 1 - 1 1 1 1 |
| <i>D</i> . | | | | 1 12101 1 1/dd mm man |
| | 12. | | specimens placed in cool box: - ate of placement in cool box is same as date of enro | |
| | 13. | <del> </del> | specimens placed in cool box: : | (hh : min, 24:00hr) |
| | 1/1 | Date | of departure from clinical site: - | - 2 0 <i>(dd-mm-yyyy)</i> |
| | 14. | | ate of departure is same as date of enrollment (Q2) | |
| | 15. | Time of departure from clinical site to lab: : (hh : min, 24:00 hr) | | |
| E. | FORI | M CON | IPLETION | |
| | 16. | ID of | person completing this form: | Date form completed: - - 2 0 (dd-mm-yyyy) |
| | 17. | ID of | person reviewing this form: | Date form reviewed: |
| | 18. | | | _ - - 2 0 (dd-mm-yyyy) Date form entered: |
| | | | person entering this form: | _ - - 2 0 _ (dd-mm-yyyy) |
| | 19. | ID of | person conducting data verification: | Date of data verification: |
| 1 | 1 | | | |


#### Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name/Country Site CRF 13b – Home Whole Stool Sample Collection Form

**Purpose:** To capture information about home whole stool sample collection within 24 hours of the enrollment visit at the recruiting sites (separate Specimen Accession CRF to be completed by central laboratory). Only applicable to Bangladesh, The Gambia, Pakistan, Malawi, and Peru sites.

**Instructions:** Complete this form for enrolled participants that have a stool sample collected within 24 hours of the enrollment visit (i.e. at a home visit).

| PL<br>[ | EASE F | PLACE | PARTICIPANT LABEL HERE (OPTIONAL): PLEASE PLACE SPECIMEN ID LABEL HERE (OPTIONAL): |
|---|---|---|---|
| A. | VISIT | INFO | RMATION |
| | 1. | Parti | cipant ID |
| | 2. | Enro | |
| | 3. | EFGH | d country site: |
| | | □в | angladesh |
| | | □ P | eru |
| В. | WHC | DLE ST | OOL COLLECTION INFORMATION |
| | 4. | Was | whole stool collected within 24 hours after discharge from the enrollment visit to the health facility? |
| | | □ Y | es (skip to 4b) |
| | | | lo |
| | | 4a. | If No, why not? (select one then skip to Section D) |
| | | | Child did not produce whole stool within 24 hours of leaving health facility (no home whole stool collection) |
| | | | Study resources not available for home visit to collect sample (e.g. after hours, no staff available) |
| | | | Study staff cannot contact the caregiver or no one was home during home visit |
| | | | Other (specify): |
| | | 4b. | Was there any blood visible in the whole stool? |
| | | | Yes |
| | | | □No |
| | | 4c. | Date caregiver reported whole stool passing: - - 2 0 (dd-mm-yyyy) |
| | | 4d. | Time caregiver reported whole stool passing: : (hh : min, 24:00 hr; approximate to the nearest hour if the caregiver does not know) |
| | | 4e. | Method of whole stool collection: |
| | | | Staff retrieved whole stool sample from child's home |
| | | | Caregiver brought whole stool sample to clinical site or recruitment facility |
| | | 4f. | Date of whole stool collection (either date returned by caregiver or date retrieved at home by staff): - - 2 0 (dd-mm-yyyy) |
| | | 4g. | Time of whole stool collection (either time returned by caregiver or time retrieved at home by staff): : (hh: min, 24:00 hr) |

Version: 1.0 (13-03-2023) 

#### Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name/Country Site CRF 13b – Home Whole Stool Sample Collection Form

| | | 4h. | Specimen ID: | ☐ Not applicable |
|---|---|---|---|---|
| | 5. | Whe | n was the whole stool sample placed in a cool box? | ) |
| | | IJ۷ | ☐Whole stool sample was placed in cool box upon pickup at home | |
| | | ١ | Whole stool sample was placed in cool box upon rec | ceipt at clinical site or recruitment facility |
| | | ١ | Whole stool sample was placed in cool box at centra | al laboratory |
| | | | Other (specify): | |
| C. | SAM | IPLE TRANSPORT INFORMATION | | |
| | 6. | Date of departure from clinical site to central laboratory: - - 2 0 (dd-mm-yyyy) Not applicable, whole stool sample transported directly from home to central laboratory | | |
| | 7. | Time of departure from clinical site to lab: : (hh: min, 24:00 hr) Not applicable, whole stool sample transported directly from home to central laboratory | | |
| D. | FOR | м сог | MPLETION | |
| | 8. | ID of | f person completing this form: | Date form completed: _ _ - _ - 2 0 _ _ (dd-mm-yyyy) |
| | 9. | ID of | person reviewing this form: | Date form reviewed: - - 2 0 (dd-mm-yyyy) |
| | 10. | ID of | person entering this form: | Date form entered: - - 2 0 (dd-mm-yyyy) |
| | 11. | ID of | f person conducting data verification: | Date of data verification: - - 2 0 (dd-mm-yyyy) |


#### Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name (Country Site) CRF 14 - Blood Sample Collection Form

**Purpose:** To capture information about blood sample collection at the recruiting sites (separate Specimen Accession form to be completed by central laboratory).

**Instructions:** Complete this form for all enrolled participants at Enrollment Visit and Week 4 visit (if blood collection is part of site protocol) PLEASE PLACE PARTICIPANT LABEL HERE (OPTIONAL): PLEASE PLACE SPECIMEN ID LABEL HERE (OPTIONAL): A. VISIT INFORMATION \_\_|\_\_|\_\_ 1. Participant ID Specimen ID: \_ Not applicable Specimen ID 2. \_\_|\_\_| - |\_\_\_| - | 2 | 0 |\_\_\_| (dd-mm-yyyy) Visit Date: Enrollment Week 4 Follow Up Visit 4. EFGH country site: 5. Bangladesh ☐ Kenya Malawi Mali Pakistan Peru The Gambia **BLOOD COLLECTION & TRANSPORT INFORMATION** Was a finger/heel prick of blood collected from the participant? Yes (skip to Q7) ☐ No 6a. If no, why? Caregiver refused (skip to Q12) \_\_\_\_ Other (specify): \_\_\_\_\_\_ (skip to Q12) How many dried blood spots were completely filled? 5 (skip to Q8) 4 3 □ 2

#### Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name (Country Site) CRF 14 - Blood Sample Collection Form

| | 8. | Date of blood collection: - - 2 0 (dd-mm-yyyy) Date of collection is same as visit date (Q2) | |
|---|---|---|---|
| | 9. | Time of blood collection: : (/ | hh : min, 24:00 hr) |
| | 10. | Date of departure from clinical site: $ _ _ _ - _ _ - 2 0 _ _ (dd-mm-yyyy)$ Date of departure is same as visit date (Q2) | |
| | 11. | Time of departure from clinical site to lab: _ | _ : (hh : min, 24:00 hr) |
| C. | FOR | M COMPLETION | |
| | 12. | ID of person completing this form: | Date form completed: |
| | 13. | ID of person reviewing this form: | Date form reviewed: - _ - 2 0 (dd-mm-yyyy) |
| | 14. | ID of person entering this form: | Date form entered: _ _ - _ _ - 2 0 _ _ (dd-mm-yyyy) |
| | 15. | ID of person conducting data verification: | Date of data verification: - - 2 0 (dd-mm-yyyy) |

#### Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name (Country Site) CRF 18— Diarrhea Case Surveillance Protocol Violation CRF

**Purpose:** To capture information about protocol violations that occurred from the start of study (for participants, the start of the study refers to the date participant ID (PID) was assigned) until the end of the study duration.

**Instructions:** Please complete this form for all protocol violations. If multiple PIDs are affected by the violation, please submit one form per PID. Please note that only protocol violations (not deviations) are reported here. As a reminder, a protocol violation is defined as a consistent variation in practice from study protocol/SOPs that may affect participant safety, participant willingness to participate in the study, and/or integrity of the research or study data. Protocol violation is a subset of protocol deviation. Please also complete a Note to File if the violation affected more than one participant at the same time. Please consult the Protocol Deviation/ Violation SOP for additional details.

| A. | PAR | TICIPANT AND SITE INFORMATION | ICIPANT AND SITE INFORMATION |
|---|---|---|---|
| | 1. | Screening ID: | - |
| | | | (Country ID - Facility ID - Sequential Screening # - Staff ID) |
| | 2. | Participant ID: | |
| | | | ☐ Not Applicable |
| | 3. | Date of screening: | - - 2 0 (dd-mm-yyyy) |
| | 4. | Date violation occurred: | - - 2 0 (dd-mm-yyyy) |
| | 5. | Date study staff was made aware of violation | - - 2 0 (dd-mm-yyyy) |
| | 6. | EFGH country site: | |
| | | ☐ Bangladesh ☐ Kenya | ☐ Malawi ☐ Mali |
| | | ☐ Pakistan ☐ Peru | ☐ The Gambia |
| В. | PRO | TOCOL VIOLATION REPORTING | |
| | 7. | Is the site PI aware of the violation? | |
| | | Yes | |
| | | □ No | |
| | 8. | Was this event reported to the site-specific IRB | ? |
| | | Yes | |
| | | ☐ No (skip to Q10) | |
| | 9. | If yes, date reported to local IRB: | _ - - - - - - - |
| | 10. | Was this event entered in the Protocol Deviation | on/ Violations Log? |
| | | Yes | |
| | | ☐ No | |
| | 11. | Was the participant informed of the Protocol V | iolation? |
| | | Yes | |
| | | ∐ No | |
| | | Not applicable | |
| C. | | CRIPTION OF PROTOCOL VIOLATION | |
| | 12. | Nature of violation (check all that apply) | |
| | | Consent not obtained or documented | Consent obtained using outdated consent form |

#### Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name (Country Site) CRF 18— Diarrhea Case Surveillance Protocol Violation CRF

| | | Failure to provide a copy of signed consent | Enrolment of subjects that do not meet the |
|---|---|---|---|
| | | form to the participant caregiver | inclusion/exclusion criteria |
| | | Undertaking of a study procedure not | Breach in confidentiality that may pose an immediate |
| | | approved by IRB | threat to the participant or caregiver |
| | | Loss of laptop or study equipment that | Failure to report a severe adverse event (SAE) to ethical |
| | | contains identifiable information about | review committees. |
| | | participant | |
| | | Other (please specify): | |
| | 13. | Brief summary of event (Description of event, locati | on it occurred if relevant): |
| | 10. | Brief Sammary of event (Bescription of eventy location | on to occurred in relevantly. |
| | 1.1 | What store have been taken to address this group? | |
| | 14. | What steps have been taken to address this event? | |
| | 15. | What steps have been taken to prevent further occ | urrences? |
| D. | EODI | M COMPLETION | |
| D. | | | Data farms as mulated. |
| | 16. | ID of person completing this form: | Date form completed: |
| | 4- | | _ _ - _ - 2 0 _ (dd-mm-yyyy) |
| | 17. | ID of person reviewing this form: | Date form reviewed: |
| | | | _ - _ - 2 0 _ (dd-mm-yyyy) |
| | 18. | ID of person entering this form: | Date form entered: |
| | | | _ - - 2 0 (dd-mm-yyyy) |
| | 19. | ID of person conducting data verification: | Date of data verification: |
| | | | _ - - 2 0 (dd-mm-yyyy) |

#### Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name (Country Site) CRF 18— Diarrhea Case Surveillance Protocol Violation CRF

#### Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name (Country Site) CRF 19— Adverse Event CRF

**Purpose:** To capture information about all adverse events (AE) definitely, probably, and possibly related to study participation occurring during the study participation period.

**Instructions:** Complete this form for all adverse events definitely, probably, and possibly related to study participation occurring during the study participation period. If an event was NOT related to study participation this form does not need to be completed or entered in REDCap. Consult the Adverse Event SOP for other details including AE guidance and reporting procedures.

| | , | | | | |
|---|---|---|---|---|---|
| A. | PART | FICIPANT AND SITE INFORMATION | | | |
| | 1 | Screening ID: | | - - _ | - |
| | 1. | Screening ib. | | (Country ID - Facility ID - S | Sequential Screening # - Staff ID) |
| | 2. | Participant ID: (if applicable) | I | | |
| | ۷. | rarticipant ib. (ij upplicubic) | | Not applicable (not enr | olled) |
| | 3. | Date of enrollment visit: (if applic | ahle) | - - | 2 0 (dd-mm-yyyy) |
| | ٥. | Date of efficient visit. (ij applic | | Not applicable (not enr | olled) |
| | 4. | Date of onset of AE | 1 | _ - - | 2 0 (dd-mm-yyyy) |
| | 5. | Time of onset of AE | I | : (hh | n : min, 24:00 hr) |
| | | Data of manufaction of AF | 1 | - - | 2 0 (dd-mm-yyyy) |
| | 6. | Date of resolution of AE | | Not resolved | |
| | _ | T' | | : (hh | ı : min, 24:00 hr) |
| | 7. | Time of resolution of AE | | Not resolved | |
| В. | AE D | ESCRIPTION AND REPORTING | | | |
| | 8. | Please describe the adverse even | t | | |
| | | Description of the adverse event | here | | |
| | 9. | AE Severity | | | |
| | Э. | | | (2) | |
| | | Mild (Grade 1) | Moderate ( | | Severe (Grade 3) |
| | | Life threatening (Grade 4) | Fatal (Grad | de 5) | |
| | 10. | Relationship of AE to study procedures | | | |

#### Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name (Country Site) CRF 19— Adverse Event CRF

| | | ☐ Definitely related | |
|---|---|---|---|
| | | Probably related | |
| | | ☐ Possibly related | |
| | 11. | Outcomes Attributed to the Event | |
| | | Resolved without sequelae | Resolved with sequelae |
| | | Recovering/Resolving | ☐ Not Recovered/Not Resolved |
| | | Resulted in death | Unknown |
| | 12. | Is this a Serious AE? | |
| | | Yes | |
| | | □No | |
| | 13. | Was this event reported to the site-specific IRB? | |
| | | Yes | |
| | | ☐ No (skip to Q15) | |
| | 14. | If yes, date reported | - - 2 0 (dd-mm-<br>yyyy) |
| | 15. | If Serious AE (Q12), was the SAE communicated to EFG | GH coordination team within 24 hours of event awareness? |
| | | Yes | |
| | | □ No | |
| | | Not applicable, AE not serious | |
| | 16. | Are there any additional notes about the AE? | |
| | | Comments and notes here | |
| C. | FOR | M COMPLETION | |
| | | ID of person completing this form: | Date form completed: - - 2 0 (dd-mm-yyyy) |
| | | ID of person reviewing this form: | Date form reviewed: - - 2 0 (dd-mm-yyyy) |
| | | ID of person entering this form: | Date form entered: - - 2 0 (dd-mm-yyyy) |
| | | ID of person conducting data verification: | Date of data verification: |



Enterics for Global Health: Shigella Surveillance Study (EFGH)

#### Population Enumeration & Healthcare Utilization Survey Case Report Form Appendix



#### Table of Contents

| CRF Number | CRF Name |
|------------|-----------------------------------------------------|
| 01 | Population Enumeration |
| 02a | Healthcare Utilization Survey |
| 02b | Wealth Index – Bangladesh |
| 02b | Wealth Index – The Gambia |
| 02b | Wealth Index – Kenya |
| 02b | Wealth Index – Malawi |
| 02b | Wealth Index – Mali |
| 02b | Wealth Index – Pakistan |
| 02b | Wealth Index – Peru |
| 03 | Revisit Household for Healthcare Utilization Survey |
| 04 | Cluster Completion |
| 20 | Population Enumeration & HUS Protocol Violation |

#### Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name/Country Site CRF 01— Population Enumeration

**Purpose:** Population Enumeration

**Instructions:** Complete this form for each household/domestic structure in identified cluster that appears inhabited after the person able to give consent (head of household/primary caregiver/adult household member) has been asked to provide verbal consent – OR – if after three attempts, the head of household/primary caregiver/adult household member (herein referred to as "adult household member") has not been home or available to ask for verbal consent. Text in **bold** should be read to study participants, plain text is for prompts for study staff, and italics are instructions for study staff.

| | ISIT INFORMATION | | |
|---|---|---|---|
| 1. | Date: _ - - 2 0 (dd- | -mm-yyyy) | |
| 2. | EFGH country site: | | |
| | □ Bangladesh | □ Kenya | |
| | □ Malawi □ | □ Mali | |
| | □ Pakistan □ | □ Peru | |
| | ☐ The Gambia | | |
| 3. | Cluster number: | | |
| | 3a. Sub-cluster number (applicable to Kenya and The Gambia only) | (1-4) | |
| | Household identifier (assigned if head of household/primary caregiver/adult | _ - 2 0 | <br> |
| 4. | household member have been asked for verbal consent - OR - if after three attempts, head of household/primary caregiver/adult household member have not been home or asked to consent): | (dd-mm-yyyy) | (Fieldworker (Sequential number) |
| 5. | Did the study team approach the household? | | |
| | ☐ Yes, met the adult household member (conduct verbal consent) | | |
| | ☐ Yes, adult household member is contactable by phone | | |
| | ☐ Yes, but adult household member was not home after | · — | |
| | ☐ Yes, but no one was ever home at each of the three attempts OR it appears or has been confirmed that no on | | |
| 6. | in the home during the ~ 2 week enumeration period Did the adult household member give verbal consent? | (ena of form) | |
| υ. | ☐ Yes | | |
| | ☐ No (skip to form completion) | | |
| | ☐ NA, adult household member/primary caregiver not ab | ole to provide consent (skip to form | n completion) |
| 7. | What is the name of the (insert site-specific adm | ministrative unit) that this house is | within? |
| | ☐ Other, specify: | | |
| 8. | How many people (including yourself, adults and children | currently live in the household? | |
| 9. | Does a child under 5 years of age (<60 months) currently | live in the household? | |
| <br> | □Yes | | |
| | □ No (skip to form completion) | | |

Page: 2 of 3

Enterics for Global Health – *Shigella* Surveillance Study (EFGH) Implementing Institution Name/Country Site Form 01— Population Enumeration

| | If 0, stop here. Questions below will be asked per each child under 5 years of age. The data system will automatically populate the number of rows below based on this answer. | Did this child experience diarrhea in the last two weeks (14 days) – that is 3 or more unusually loose or watery stools during a 24 hour period in the last 14 days? (only ask if the child is <60 months – automated question) | □ Yes<br>□ No (form complete)<br>□ Don't Know (form complete) | ☐ Yes<br>☐ No ( <i>form complete</i> ) |
|---|---|---|---|---|
| | l be asked per each c<br>iber of rows below bo | Age (auto<br>generated in real<br>time and<br>confirmed with<br>the caregiver) | months | months |
| | If 0, stop here. Questions below will be asked per each child under 5 years of will automatically populate the number of rows below based on this answer. | Date of birth/age | _ - - - <br> - - | - - - |
| MATION | | Child<br>Initials | | |
| CHILD INFORMATION | 0 months) | Child sex | ☐ Female | ☐ Female<br>☐ Male |
| | ars of age (<6<br>? | Is this person the primary caregiver of the child? | □ Yes | □ Yes |
| | How many children under 5 years of age (<60 months) currently live in the household? | What is the relationship of the person answering these questions to (name)? | <ul> <li>□ Biological mother</li> <li>□ Adopted mother</li> <li>□ Adopted father</li> <li>□ Grandmother</li> <li>□ Grandfather</li> <li>□ Uncle</li> <li>□ Older sister</li> <li>□ Older brother</li> <li>□ Other, specify:</li> </ul> | ☐ Biological mother<br>☐ Biological father |
| æi | How n<br>10. curren | Child 11. num | 7-1 | × |

# Enterics for Global Health – *Shigella* Surveillance Study (EFGH) Implementing Institution Name/Country Site Form 01— Population Enumeration

| □ Don't Know (form complete) | to form completion. | usehold that previously refused consent and then changed to include the original household identifier. |
|---|---|---|
| (dd-mm-yyyy) Day Missing Month Missing Year Missing | If one or more children are between 6 to <36 months of age and had diarrhea in the last 14 days, continue. If not, skip to form completion. Comments | If there is anything unique about this visit, please record a description in the comments section. If this was a household that previously refused consent and then changed their mind and requested to participate (provided consent), it is required to indicate that information here and to include the original household identifier. |
| ☐ Adopted mother ☐ Adopted father ☐ Grandmother ☐ Grandfather ☐ Aunt ☐ Uncle ☐ Older sister ☐ Older brother ☐ Other, specify: | If one or more children are between 6 to <36 months or Comments | If there is anything unique about this visit, plea. |

Page: 3 of 3 Version: 6.0 (01-11-2022)

Instructions: Complete the following questions for each child in the household between 6-35 months of age after consent is received. The questions should be answered by a household member who spends the most time with the child and is best able to recall symptoms related to the most recent diarrheal episode (likely the primary caregiver). Diarrhea is defined as 3 or more loose stools in a 24 hour period. A diarrheal episode is diarrhea that began after at least 2 days without diarrhea. Use the memory aid and ask the caregiver to answer the following questions thinking about the most recent episode of diarrhea. Text in bold should be read to study participants, plain text is for prompts for study staff, and italics are instructions for study staff.

A. VISIT INFORMATION

1. Date: |\_\_\_\_| - |\_\_\_| - |2 | 0 |\_\_\_| (dd-mm-yyyy)

| for | for study staff, and <i>italics</i> are instructions for study staff. | |
|---|---|---|
| A. | VISIT | NFORMATION |
| | 1. | Date: _ - - 2 0 (dd-mm-yyyy) |
| | 2. | FGH country site: |
| | | □ Bangladesh □ Kenya |
| | | Malawi Mali |
| | | Pakistan Peru |
| | | The Gambia |
| | 3. | Cluster number: |
| | | Sa. Sub-cluster number (applicable to Kenya and The Gambia only) (1-4) |
| | 4. | Household identifier - - |
| | т. | assigned for the lousehold enumeration): (dd-mm-yyyy) (Fieldworker ID) (Sequential number) |
| В. | DIAR | ARRHEA SIGNS AND SYMPTOMS (ODK will auto-generate this section for each eligible child) |
| | 5. | Child Initials & Age : ODK to autopopulate the list of children with initials and age who had diarrhea reported in section B of Form 01 — Child Initials Age (months) |
| | 6. | Who is answering the HUS questions on behalf of this child? Primary Caregiver of the Child Other Household Member |
| | 7. | What is the relationship of the respondent to the child? |
| | | Biological mother Biological father Adopted mother |
| | | Grandmother Grandfather Aunt |
| | | Uncle Older sister Older brother |
| | | Other, specify: |
| | 8. | Did the adult household member and/or primary caregiver give informed consent for participation in the nealthcare utilization survey? |
| | | ☐ Yes, verbal consent was obtained for the healthcare utilization survey |
| | | ☐ Yes, written informed consent was obtained for the healthcare utilization survey |
| | | ☐ No, declined consent (end of form) |
| | | ☐ No, primary caregiver is not available. Will revisit household to complete healthcare utilization survey (end of form. Complete HUS Revisit Form upon revisiting household) |

| position and the con- | | | | | |
|---|---|---|---|---|---|
| | 9. | Wher | n did the diarrhea start? Refer to calendar to | _ - _ | |
| | J. | deter | mine date if # of days ago known but not exact date | (dd-mm-yyyy) | |
| | | Wher | n did the diarrhea end? Refer to calendar to | _ - - | |
| | 10. | determine date if # of days ago known but not exact date | | (dd-mm-yyyy) | |
| | | | | Ongoing (days) | |
| | 11. | Durat | ion of diarrhea by date calculation (auto-generated) | (Add suggested range 1 to 14 in ODK) | |
| | | On the worst day of diarrhea during this episode, how many | | | |
| | 12. | loose stools did the child have in one day (24 hours)? | | | |
| | 13. | Did th | ne child have any of the following symptoms during h | is/her diarrheal illness? (Use the memory aid | |
| | | Ļ | ow pictures of each of these symptoms) | | |
| | | | in stool: | Yes No Don't Know | |
| | | | ple/less play: | Yes No Don't Know | |
| | | | en eyes: | Yes No Don't Know | |
| | | | kled skin: | Yes No Don't Know | |
| | | | s eagerly, thirsty: | Yes No Don't Know Yes No Don't Know | |
| | | | le to drink or drank poorly: rgic, unconscious, or hard to stay awake: | Yes No Don't Know Yes No Don't Know | |
| | | | - | | |
| | 14. | | ne child vomit at any time during the episode of diarr | nea : | |
| | | ∐ Y∈ | | | |
| | | | o (skip to Q15) | | |
| | | Do | on't know (skip to Q15) | | |
| | | 14a. | How many days did the child vomit? | (days) | |
| | | i-a. | now many days and the clind volint. | (Add suggested range 1 to 14 in ODK) | |
| | | 14b. | Thinking about the day when the child had the mos | t | |
| | | _ | vomiting, how many times did s/he vomit in the day | <u>_</u> | |
| | 15. | | y any point during the diarrheal episode, did the child | I have any fever? (Fever meaning the child | |
| | | was n | ot to touch) | | |
| | | | o (skip to Q16) | | |
| | | | on't know (skip to Q16) | | |
| | | | | °C | |
| | | 15a. | If yes, what was the highest temperature? | Temperature not collected | |
| | | 15b. | How many days did s/he have the fever? | days | |
| | 16. | Did y | ou seek care for the child's diarrhea outside your hom | ne? | |
| | | П Үе | es (skip to Q17) | | |
| | | ☐ No | | | |
| | | 16a. | If No to Q16, why not? | | - |
| | | | (If did not seek care for child's diarrhea outs | ide the home, form complete.) | |
| | | | - | | |
| | 17. | If you | sought treatment or care for the child for this illness | where did you go? (check all that apply) | |

| | <u>Facility</u> | | | Date first visited | | |
|---|---|---|---|---|---|---|
| | ☐ EFGH Facility X | | 11 | _ - - 2 0 _ (dd-mm-yyyy) | | |
| | ☐ EFGH Facility X | | ll_ | _ - - 2 0 _ (dd-mm-yyyy) | | |
| | Other health facility (outpat | tient care) | ll_ | - | - 2 0 _ | _ (dd-mm-yyyy) |
| | Other health facility (inpatie | ent care) | ll_ | - | - 2 0 _ | _ (dd-mm-yyyy) |
| | Other (specify, check all that | t apply) | | | | |
| | Traditional healer | | | | ligious healer<br> | |
| | ☐ Drug seller☐ Community Health w | vorker | | = | armacist<br>alth outpost | |
| | Other (specify): | | | | aitii outpost | |
| | What day of the child's diarrhea | a did the care | giver visit a l | nospital | or | |
| 18. | health center? (auto-generated | in ODK;If too | day, "00" will | be | | _ |
| 19. | displayed) Did the clinical team at any car | e provider a | dvise the chi | d he ho | snitalized during | his illness? |
| 19. | Yes | c provider de | avise the cili | u be ne | ospitulized during | |
| | ☐ No (skip to Q21) | | | | | |
| 20. | Was the child admitted to the | hospital (i.e. | at least an o | least an overnight stay) during this illness? | | |
| | Yes | | | | | |
| | ∐ No | | | | | |
| 21. | Did the child receive any of the | e following to | treat the di | arrhea? | check all that ap | oly) |
| | Intravenous fluids | | Yes | | ☐ No | ☐ Don't know |
| | A drinkable fluid made from | n a special | Yes | | ☐ No | ☐ Don't know |
| | packet called ORALITE or ORS Homemade fluid (such as t | hin watery | | | | |
| | porridge made from maize, r | - | | | <b>┌</b> ┐ | |
| | soup, sugar, salt water solution | n or yogurt- | ∐ Yes | Yes | | ☐ Don't know |
| | based drink) | | | | | □ Dow't know |
| | Antibiotic | | ☐ Yes (spe | Yes (specify) No Don't know | | □ Don t know |
| | If antibiotic was received | d, specify type | e received (ch | eck all | that apply): | |
| | ☐ Amoxicillin | ☐ Azithrom | ycin | ☐ Arte | sunate | ☐ Ampicillin |
| | ☐ Augmentin/ Co-<br>amoxiclav | □ Ceftriaxo | ne | ☐ Cipro | ofloxacin (Cipro) | ☐ Cefuroxime |
| | ☐ Clarithromycin | ☐ Clindamy | cin | □ Chlo | ramphenicol | ☐ Cotrimoxazole<br>(Septrin) |
| | ☐ Doxycycline | ☐ Erythrom | ycin | □ Gen | tamicin | ☐ Penicillin |
| | ☐ Pyrazinamide | □ Streptom | ycin | □ Tetr | acycline | □ Unknown |
| | ☐ Other (specify): | | | | | |

| ¥ | Antisecretory or antiemetics | Yes | ☐ No | Don't know |
|---|------------------------------|-------|------|--------------|
| | Zinc | ☐ Yes | ☐ No | Don't know |
| | Traditional medicine | ☐ Yes | ☐ No | Don't know |
| | None of the above | Yes | ☐ No | ☐ Don't know |

## Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name/Country Site CRF 02b— Wealth Index Form (Bangladesh)

**Purpose:** To collect household wealth information at the Bangladesh site.

**Instructions:** Please complete this form for all households that are included in the Healthcare Utilization Survey at the Bangladesh EFGH site. Text in **bold** should be read to study participants, plain text is for prompts for study staff, and *italics* are instructions for study staff.

| A. | WEALTH INDEX | | |
|---|---|---|---|
| | 1. | Does your household have a television? | Yes No |
| | 2. | Does your household have a refrigerator? | Yes No |
| | 3. | Does your household have an almirah/wardrobe? | ☐ Yes ☐ No |
| | 4. | Does your household have an electric fan? | ☐ Yes ☐ No |
| | 5. | What is the main material of the floor? (select one) | |
| | | Cement | ☐ Earth/sand |
| | | Other material | |
| | 6. | What is the main material of the exterior walls? (select one) | |
| | | Cement | Other material |
| | 7. | What is the main material of the roof? (select one) | |
| | | Cement | Other material |
| В. | ADDI | DDITIONAL QUESTIONS | |
| | 8. | Does your household have an oven? | Yes No |
| | 9. | Does your household have a motor bike? | ☐ Yes ☐ No |
| | 10. | Does your household have a car? | ☐ Yes ☐ No |
| | 11. | Does your household have an AC? | ☐ Yes ☐ No |
| | 12. | Does your household have a sewing machine? | ☐ Yes ☐ No |
| | 13. | Does your household have a bi-cycle? | ☐ Yes ☐ No |
| | 14. | Does your household have a dining table? | ☐ Yes ☐ No |
| | 15. | Does your household have a sofa? | ☐ Yes ☐ No |
| | 16. | Does your household have a radio? | ☐ Yes ☐ No |
| | 17. | Household ownership? | |
| | | Own | Rented |
| | | Occupied | |
| | 18. | Source of drinking water | |
| | | Own tap Own tube well | ☐ Communal hand pump ☐ Bottled water |

## Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name/Country Site CRF 02b— Wealth Index Form (Bangladesh)

| | | Own well Own hand pump Communal tap Communal tube well Others | <ul> <li>□ Water vendor</li> <li>□ Stored in reservoir</li> <li>□ Pond/canal/river</li> <li>□ Shared tap/tube well/well in HH</li> </ul> |
|---|---|---|---|
| | 19. | Shared latrine | Yes No |
| | 20. | Latrine type | |
| | | Sanitary latrine with flush | Sanitary latrine without flush |
| | | Non-sanitary/no water seal latrine | No latrine/use open space |
| C. | FORM | A COMPLETION | |
| | | /I COMPLETION | |
| | 21. | ID of person completing this form: | Date form completed: |
| | 21.<br>22. | | - - 2 0 (dd-mm-yyyy) Date form reviewed: |
| | | ID of person completing this form: | _ - - 2 0 _ (dd-mm-yyyy) |

## Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name/Country Site CRF 02b— Wealth Index Form (The Gambia)

**Purpose:** To collect household wealth information at The Gambia site.

**Instructions:** Please complete this form for all households that are included in the Healthcare Utilization Survey at The Gambia EFGH site. Text in **bold** should be read to study participants, plain text is for prompts for study staff, and *italics* are instructions for study staff.

| A. | WEA | ZEALTH INDEX | | |
|---|---|---|---|---|
| | | DETERMINE IF THE RESPONDENT LIVES IN AN URBAN | OR RURAL AREA | |
| | | Urban | Rural | |
| | 1. | Does your household have a sofa? | ☐ Yes ☐ N | 0 |
| | 2. | Does your household have a wardrobe? | Yes N | 0 |
| | 3. | Does your household have a television? | Yes N | 0 |
| | 4. | Does your household have a refrigerator? | Yes N | 0 |
| | 5. | Does your household have a DVD / VCD player? | Yes N | 0 |
| | 6. | Does your household have a satellite dish? | Yes N | 0 |
| | 7. | Does any member of your household own: a bicycle? | Yes N | 0 |
| | 8. | What is the main source of drinking water for memb | ers of your hous | sehold? (select one) |
| | | Public tap / Standpipe | Other wa | ter source |
| | | Piped to yard | | |
| | 9. | What kind of toilet facility do members of your hous | ehold usually us | se? |
| | | Flush to septic tank | Other toil | et type |
| | | Pit latrine w/o slab/ Open Pit | | |
| | 10. | What is the main material of the floor in your house | hold? (select one | e) |
| | | Ceramic tile | Other floo | or material |
| | 11. | What is the main material of the exterior walls of yo | ur household? ( | select one) |
| | | Ceramic tile | Other wa | ll material |
| | 12. | How many of the following animals does your household own: Cattle? | None | 1 or more |
| | 13. | Milk cows or bulls? | None | 1 or more |
| | 14. | Horses, donkeys, or mules? | None | 1 or more. 5 or more |
| | 15. | Goats? | None | 1 or more |

# Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name/Country Site CRF 02b— Wealth Index Form (The Gambia)

| | 16. | Sheep? | None 1 or more |
|---|---|---|---|
| В. | ADD | ITIONAL QUESTIONS | |
| | 17. | Does your household have a functioning television? | Yes No |
| | 18. | Does your household have a functioning radio? | Yes No |
| | 19. | Does your household have a functioning refrigerator/fridge? | Yes No |
| | 20. | Does any member of your household own: a functioning motorcycle/scooter? | Yes No |
| | 21. | Does your household have functioning animal-<br>drawn cart? | Yes No |
| | 22. | What is the main material of the roof in your househo | old? (select one) |
| | | ☐ Thatch/Palm leaf | Metal/Tin/Cement |
| | | Other roof material | |
| | 23. | Does your household own any chicken, Guinea fowl, ducks, turkeys or geese? | Yes No |
| C. | FORI | M COMPLETION | |
| | 24. | ID of person completing this form: | Date form completed: - - 2 0 (dd-mm-yyyy) |
| | 25. | ID of person reviewing this form: | Date form reviewed: _ - - 2 0 (dd-mm-yyyy) |
| | 26. | ID of person entering this form: | Date form entered: |
| | 27. | ID of person conducting data verification: | Date of data verification: - - 2 0 (dd-mm-yyyy) |

#### Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name/Country Site CRF 02b— Wealth Index Form (Kenya)

Purpose: To collect household wealth information for participants enrolled at the Kenya site.

**Instructions:** Please complete this form for all participants enrolled at the Kenya EFGH site. Text in **bold** should be read to study participants, plain text is for prompts for study staff, and *italics* are instructions for study staff.

| A. | WEA | /EALTH INDEX | |
|---|---|---|---|
| | 1. | Does your household have electricity? | Yes No (skip Q14) |
| | 2. | Does your household have a television? | Yes No (skip Q15) |
| | 3. | Does your household have a sofa? | Yes No |
| | 4. | Does your household have a cupboard? | Yes No |
| | 5. | Does your household have a DVD player? | Yes No (skip Q16) |
| | 6. | Does your household have a radio? | Yes No (skip Q17) |
| | 7. | Does your household have a table? | ☐ Yes ☐ No |
| | 8. | Does your household have a clock? | Yes No (skip Q18) |
| | 9. | What is the main material of the floor of your dwelling? | (select one) |
| | | Cement | Other |
| | | ☐ Earth/sand | |
| | 10. | What is the main material of the external walls of your o | dwelling? (select one) |
| | | ☐ Dung/mud/soil | Other |
| | 11. | What is the main material of the roof of your dwelling? | (select one) |
| | | ☐ Thatch/grass/makuti | Other |
| | 12. | What type of fuel does your household mainly use for co | poking? (select one) |
| | | Wood | Other |
| | | LPG/Natural gas | |
| | 13. | What kind of toilet facility do members of your househo | ld usually use? (select one) |
| | | ☐ No facility/bush/field | Other |
| B. | ADDI | TIONAL QUESTIONS | |
| | 14. | Does your household have a functioning electricity? | Yes No |
| | 15. | Does your household have a functioning television? | Yes No |
| | 16. | Does your household have a functioning DVD player? | Yes No |
| | 17. | Does your household have a functioning radio? | Yes No |
| | 18. | Does your household have a functioning clock? | Yes No |
| C. | FOR | M COMPLETION | |
| | 19. | ID of person completing this form: | Date form completed: - - 2 0 (dd-mm-yyyy) |
| | 20. | ID of person reviewing this form: | Date form reviewed: - - 2 0 (dd-mm-yyyy) |
| | 21. | ID of person entering this form: | Date form entered: - - 2 0 (dd-mm-yyyy) |
| | 22. | ID of person conducting data verification: | Date of data verification: |

#### Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name/Country Site CRF 02b — Wealth Index Form (Malawi)

Purpose: To collect household wealth information at the Malawi site.

**Instructions:** Please complete this form for all households that are included in the Healthcare Utilization Survey at the Malawi EFGH site. Text in **bold** should be read to study participants, plain text is for prompts for study staff, and *italics* are instructions for study staff.

| A. | WEA | LTH INDEX | |
|---|---|---|---|
| | 1. | Does your household have electricity? | Yes No |
| | 2. | Does your household have a radio? | Yes No |
| | 3. | Does your household have a television? | ☐ Yes ☐ No |
| | 4. | Does your household have a bed with a mattress? | ☐ Yes ☐ No |
| | 5. | Does your household have a sofaset? | ☐ Yes ☐ No |
| | 6. | Does any member of this household own: a mobile phor | ne? |
| | 7. | Does any member of this household have a bank accoun | nt? Yes No |
| | 8. | What is the main material of the floor in your household | 1? (select one) |
| | | Earth/sand | Cement |
| | | Other floor material | |
| | 9. | What is the main material of the roof in your household | ? (select one) |
| | | ☐ Thatch/palm leaf | Metal |
| | | Other roof material | |
| | 10. | What type of fuel does your household mainly use for co | ooking? (select one) |
| | | Wood | Other type of fuel |
| В. | FORM | M COMPLETION | |
| | 11. | ID of person completing this form: | Date form completed:<br> - _ - 2 0 (dd-mm-yyyy) |
| | 12. | ID of person reviewing this form: | Date form reviewed: |
| | 13. | ID of person entering this form: | _ - - 2 0 <i>(dd-mm-yyyy)</i><br>Date form entered: |
| | | ID of person conducting data verification: | _ - - 2 0 <i>(dd-mm-yyyy)</i> Date of data verification: |
| | 14. | | - - 2 0 (dd-mm-vvvv) |

#### Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name/Country Site CRF 02b — Wealth Index Form (Mali)

Purpose: To collect household wealth information at the Mali site.

**Instructions:** Please complete this form for all households that are included in the Healthcare Utilization Survey at the Mali EFGH site. Text in **bold** should be read to study participants, plain text is for prompts for study staff, and *italics* are instructions for study staff.

| A. | WEA | EALTH INDEX | |
|---|---|---|---|
| | 1. | In your house, do you have electricity? | Yes No |
| | 2. | In your house, do you have a television? | Yes No |
| | 3. | In your house, do you have a bed? | Yes No |
| | 4. | In your house, do you have a fan? | Yes No |
| | 5. | In your house, do you have a cupboard | Yes No |
| | 6. | In your house, do you have a CD/DVD player? | Yes No |
| | 7. | In your house, do you have a refrigerator? | Yes No |
| | 8. | In your house, do you have a chair? | Yes No |
| | 9. | In your house, do you have a motorcycle or scooter? | Yes No |
| | 10. | In your house, do you have soap, washing powder, or ash/sand/dirt for washing your hands? | Yes No |
| | 11. | Does any member of this household have a bank acco | unt? Yes No Don't know |
| | 12. | Where is your principal source of drinking water locat | ed? (select one) |
| | | Outside of the plot | ☐ Within the plot |
| | 13. | What is the distance to the principal source of drinkin | g water? |
| | | Less than 30 minutes round trip | More than 30 minutes round trip |
| | 14. | Main material of exterior walls of the house? (select of | ne) |
| | | Brick | Other |
| | 15. | Main material of roof of house? (select one) | |
| | | Cement | Mud with wood |
| | | Other | |
| | 16. | Main material of floor of house? (select one) | |
| | | Earth/sand floor | Ceramic tile floor |
| | | Other | |
| | 17. | In your house, what is the main fuel used for cooking? | (select one) |

#### Enterics for Global Health – Shigella Surveillance Study (EFGH) **Implementing Institution Name/Country Site**

#### CRF 02b — Wealth Index Form (Mali)

| | | ☐ Charcoal ☐ Wood | | Other |
|---|---|---|---|---|
| | 18. | Does your household own any pigs? | | Yes No |
| | 19. | Does your household own any came | els or dromedaries | ? Yes No |
| | 20. | Does your household own any Guin geese? | keys or Yes No | |
| В. | FORI | M COMPLETION | | |
| В. | <b>FORI</b> 21. | M COMPLETION ID of person completing this form: | | Date form completed: |
| В. | | | | |
| В. | 21. | ID of person completing this form: | _ | _ - - 2 0 <i>(dd-mm-yyyy)</i> Date form reviewed: |

#### Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name/Country Site CRF 02b— Wealth Index Form (Pakistan)

**Purpose:** To collect household wealth information at the Pakistan site.

**Instructions:** Please complete this form for all households that are included in the Healthcare Utilization Survey at the Pakistan EFGH site. Text in **bold** should be read to study participants, plain text is for prompts for study staff, and *italics* are instructions for study staff.

| A. | WEAI | LTH INDEX | |
|---|---|---|---|
| | 1. | Does your household have a refrigerator? | Yes No |
| | 2. | Does your household have a washing machine? | Yes No |
| | 3. | Does your household have a sofa? | Yes No |
| | 4. | Does your household have a chair? | Yes No |
| | 5. | Does your household have an Almirah/cabinet? | Yes No |
| | 6. | Does your household have a computer? | Yes No |
| | 7. | Does your household have an internet connection? | ☐ Yes ☐ No |
| | 8. | Does your household have a bed? | Yes No |
| | 9. | Does any member of this household have a bank account? | ☐ Yes ☐ No |
| | 10. | 0. What type of fuel does your household mainly use for cooking? (select one) | |
| | | Wood | Other |
| | 11. | What is the main material of the roof in your household? (select one) | |
| | | Cement/RCC | Other |
| | 12. | What is the main material of the walls in your household? (select one) | |
| | | Cement | Other |
| В. | FORM | RM COMPLETION | |
| | 13. | ID of person completing this form: | Date form completed: _ - - 2 0 _ (dd-mm-yyyy) |
| | 14. | ID of person reviewing this form: | Date form reviewed: |
| | 15. | ID of person entering this form: | - - 2 0 _ (dd-mm-yyyy) Date form entered: _ - - 2 0 _ (dd-mm-yyyy) |
| | 16. | ID of person conducting data verification: | Date of data verification: |

#### Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name/Country Site CRF 02b— Wealth Index Form (Peru)

**Purpose:** To collect household wealth information at the Peru site.

**Instructions:** Please complete this form for all households that are included in the Healthcare Utilization Survey at the Peru EFGH site. Text in **bold** should be read to study participants, plain text is for prompts for study staff, and *italics* are instructions for study staff.

| A. V | VEALT | ALTH INDEX | |
|---|---|---|---|
| | 1. | Does your household have a computer? | Yes No |
| | 2. | Does your household have a bookshelf? | Yes No |
| | 3. | Does your household have windows with curtains or b | olinds? Yes No |
| | 4. | Does your household have a sofa? | Yes No |
| | 5. | What type of toilet does your household use? (select of | one) |
| | | ☐ Indoor connected to public sewer | Other |
| | 6. | What type of material is the roof made of in your hou | sehold? (select one) |
| | | Reinforced concrete | Other |
| | 7. | What type of material are the walls made of in your h | ousehold? (select one) |
| | | Brick or cement block | Other |
| В. | FORM | M COMPLETION | |
| | 8. | ID of person completing this form: | Date form completed: _ - - 2 0 (dd-mm-yyyy) |
| | 9. | ID of person reviewing this form: | Date form reviewed: |
| | 10. | ID of person entering this form: | _ - - 2 0 (dd-mm-yyyy) Date form entered: |
| | 11. | ID of person conducting data verification: | - - 2 0 (dd-mm-yyyy) Date of data verification: _ - - 2 0 (dd-mm-yyyy) |

**Purpose:** Revisit the households that were placed on revisit list for Healthcare Utilization survey to assess eligibility of the child for Healthcare Utilization survey, obtain informed consent from the child's caregiver and conduct Healthcare Utilization survey.

**Instructions:** Complete the following questions for each child in the household that you are attempting to revisit. The questions should be answered by a household member who spends the most time with the child and is best able to recall symptoms related to the **most recent diarrheal episode (likely the primary caregiver)**. Diarrhea is defined as 3 or more loose stools in a 24 hour period. A diarrheal episode is diarrhea that began after at least 2 days without diarrhea. Use the memory aid and ask the caregiver to answer the following questions thinking about the most recent episode of diarrhea. Text in **bold** should be read to study participants, plain text is for prompts for study staff, and *italics* are instructions for study staff.

| A. | VISI | T INFORMATION | | | | |
|---|---|---|---|---|---|---|
| | 1. | Date: | _ - | - 2 0 | (dd-mm-yyyy) | |
| | 2. | EFGH country site: | | | | |
| | | ☐ Bangladesh | | ☐ Kenya | | |
| | | Malawi Malawi | | Mali | | |
| | | Pakistan | | Peru | | |
| | | ☐ The Gambia | | | | |
| | 3. | Cluster number: | | | | |
| | | 3a. Sub-cluster number (a The Gambia only) | pplicable to Kenya and | pplicable to Kenya and (1-4) | | |
| В. | REVI | /ISIT INFORMATION | | | | |
| | | Household identifier (same identifier as that | - <br> 2 0 | _ - | 111 | _ |
| | 4. | assigned for the household enumeration) (select from filtered dropdown list by cluster in the data system): | (dd-mm-yyyy) | | (Fieldworker ID) | (Sequential<br>number) |
| | | In the data system, select the to conduct the Healthcare | | o to Section D. If t | the Household ID is not i | |

| | CHILD INFORMATION | | | | | | |
|---|---|---|---|---|---|---|---|
| | How many children under 5 years of age (<60 months) currently live in the household? | years of age (<60 m | nonths) | | If O, stop here. Questions below will be asked per each child under 5 years of age. The data system will automatically populate the number of rows below based on this answer. | per each child<br>he number of n | under 5 years of age.<br>ows below based on |
| Child | What is the relationship of the person answering these questions to (name)? | Is this person<br>the primary<br>caregiver of the<br>child? | Child sex | Child<br>Initials | Date of birth/age | Age (auto<br>generated in<br>real time<br>and<br>confirmed<br>with the<br>caregiver) | Did this child experience diarrhea in the last two weeks (14 days) – that is 3 or more unusually loose or watery stools during a 24 hour period in the last 14 days? (only ask if the child is <60 months – automated question) |
| - | Biological mother Biological father Adopted mother Grandmother Grandfather Uncle Older sister Older brother Other, specify: | □ Yes | ☐ Female<br>☐ Male | | _ _ - _ - - - _ - _ | months | <ul><li> Yes</li><li> Complete)</li><li> Don't Know</li><li> (form complete)</li></ul> |

Page: 2 of 6


Enterics for Global Health – *Shigella* Surveillance Study (EFGH) Implementing Institution Name/Country Site CRF 03 – Revisit Household for Healthcare Utilization Survey

| <ul><li> Yes</li><li> Complete)</li><li> Don't Know</li><li> (form complete)</li></ul> | n E Form Completion. |
|---|---|
| months | skip to Section |
| _ _ - _ _ _ | If one or more children are between 6 to <36 months of age and had diarrhea in the last 14 days, continue to Section D. If not, skip to Section E Form Completion. |
| ale<br>- | and had diarrhe |
| Female Male | nths of age c |
| □ Yes | een 6 to <36 mor |
| Biological mother Biological father Adopted mother Grandmother Grandfather Uncle Older sister Older brother Other, specify: | If one or more children are betw |
| × | |

Page: 3 of 6


| D. | DIAR | RRHEA SIGNS AND SYMPTOMS (ODK will auto-generate this section for each eligible child) | | | | |
|---|---|---|---|---|---|---|
| | 7. | Did the adult household member and/or primary caregiver give informed consent for participation in the healthcare utilization survey? | | | | |
| | • | ☐ Yes, verbal consent was obtained for the healthcare utilization survey | | | | |
| | | ☐ Yes, written informed consent was obtained for the healthcare utilization survey | | | | |
| | | □ No, declined consent (end of form) | | | | |
| | | Child Initials & Age : | , , | | | |
| | _ | ODK to autopopulate the list of | children with initials and | | 1 1 1 | |
| | 8. | age who had diarrhea reported | in section C or in the | | Child Initials | Age (months) |
| | | previously completed Populatio | n Enumeration Form | | | |
| | 9. | Who is answering the HUS ques | tions on hehalf of this child | Pri | mary Caregiver of t | the Child |
| | Э. | Other Household Member | | | | |
| | 10. | What is the relationship of the respondent to the child? | | | | |
| | | ☐ Biological mother ☐ Biological father ☐ Adopted mother | | | | |
| | 1<br>1 | Grandmother | Grandfather | | Aunt | |
| | | Uncle | Older sister | | Older brother | r |
| | ************************************** | Other, specify: | | | | |
| | • | | | | | |
| | 11. | When did the diarrhea start? Refer to calendar to - - determine date if # of days ago known but not exact date (dd-mm-yyyy) | | | | |
| | | When did the diarrhea end? Refer to calendar to | | | | |
| | 12. | determine date if # of days ago known but not exact date (dd-mm-yyyy) | | | | |
| | | ☐ Ongoing | | | | |
| | 13. | Duration of diarrhea by date ca | lculation (auto-generated) | (Add sug | (days<br>ggested range 1 to | |
| | | On the worst day of diarrhea d | uring this episode, how ma | ny | | 1 1 - |
| | 14. | loose stools did the child have | in one day (24 hours)? | | | loose stools |
| | 15. | Did the child have any of the fo | ollowing symptoms during h | nis/her dia | arrheal illness? (Us | e the memory aid |
| | | to show pictures of each of thes | se symptoms) | | | |
| | | Blood in stool: | | ∐ Yes [ | No | |
| | | Irritable/less play: | | ∐ Yes [ | No Don't Kn | |
| | | Sunken eyes: Wrinkled skin: | | ∐ Yes [ | No Don't Kn | |
| | | | | Yes [ | No Don't Kn | |
| | | Drinks eagerly, thirsty: Unable to drink or drank poorly | , | Yes [ | No | |
| | | Lethargic, unconscious, or hard | | Yes | No Don't Kn | |
| | | | - | <u> </u> | | ~ · · |
| | 16. | Did the child vomit at any time | auring the episode of diarr | nea? | | |
| | | ☐ Yes | | | | |
| | | No (skip to Q18) | | | | |
| | | Don't know (skip to Q18) | | | | |

| | | 16a. How many days did the child vomit? | | | (days) (Add suggested range 1 to 14 in ODK) |
|---|---|---|---|---|---|
| | | 16b. | Thinking about the day when the child h vomiting, how many times did s/he vom | | |
| | 17. | At any any point during the diarrheal episode, did the child have any fever? (Fever meaning the child was hot to touch) | | | |
| | | ☐ Yes ☐ No (skip to Q18) | | | |
| | | Don't know (skip to Q18) | | | |
| | | 18a. | If yes, what was the highest temperature | e? | °C<br>Temperature not collected |
| | | 18b. | How many days did s/he have the fever | ? | days |
| | 18. | Did y | ou seek care for the child's diarrhea outsion | de your hom | e? |
| | | ☐ Yes (skip to Q19) ☐ No | | | |
| | | 18a. If No to Q18, why not? | | | |
| | | (If did not seek care for child's diarrhea outside the home, form complete.) | | | |
| | 19. | If you sought treatment or care for the child for this illness where did you go? (check all that apply) | | | |
| | | | <u>Facility</u> | | <u>Date first visited</u> |
| | | □ EFGH Facility X _ _ - _ - 2 0 _ _ (dd-mm-yyyy) | | | |
| | | ☐ EFGH Facility X _ _ - _ _ - 2 0 _ _ (dd-mm-yyyy) ☐ Other health facility (outpatient care) _ _ - _ _ - 2 0 _ _ (dd-mm-yyyy) | | | |
| | | ☐ Other health facility (inpatient care) _ - - 2 0 (dd-mm-yyyy) ☐ Other (specify, check all that apply) | | | |
| | | | Traditional healer | | Religious healer |
| | | | ☐ Drug seller ☐ Community Health worker | | Pharmacist<br>Health outpost |
| | | | Other (specify): | <b>L</b> | , meanin outpost |
| | | | day of the child's diarrhea did the caregive | | oital or |
| | 21. | health<br>displa | n center? (auto-generated in ODK;If today,<br>yed) | "00" will be | |
| | 22. | Did th | ne clinical team at any care provider adviso | e the child b | e hospitalized during this illness? |
| | | ☐ Ye | | | |
| | | | o (skip to Q24) | | |
| • | 23. | | he child admitted to the hospital (i.e. at le | east an overr | night stay) during this illness? |
| | | ☐ Ye | | | |
| | 24. | Did th | ne child receive any of the following to tre | at the diarrh | nea? (check all that apply) |

| | | Intravenous fluids | | Yes | | □No | | ☐ Don't know | |
|---|---|---|---|---|---|---|---|---|---|
| | | | nkable fluid made from<br>t called ORALITE or ORS | a special | Yes | | ☐ No | | ☐ Don't know |
| | | porrid | emade fluid (such as th<br>lge made from maize, ri<br>sugar, salt water solution<br>l drink) | ce, wheat, | Yes | | ☐ No | | ☐ Don't know |
| | | Antibi | iotic | | Yes (sp | ecify) | ☐ No | | ☐ Don't know |
| | | | If antibiotic was received | , specify type | e received (c | heck all | that apply): | | |
| | | | ☐ Amoxicillin | ☐ Azithrom | ycin | ☐ Arte | sunate | | Ampicillin |
| | | | ☐ Augmentin/ Co-<br>amoxiclav | ☐ Ceftriaxo | ne | ☐ Cipr | ofloxacin (Cipro) | | Cefuroxime |
| | | ☐ Clarithromycin ☐ | | ☐ Clindamy | rcin 🗆 Ch | | Chloramphenicol | | □ Cotrimoxazole<br>(Septrin) |
| | | ☐ Doxycycline | | ☐ Erythrom | nycin 🗆 Ge | | ntamicin $\Box$ | | Penicillin |
| | | ☐ Pyrazinamide ☐ S | | ☐ Streptom | ıycin 🗆 Tet | | racycline $\Box$ | | Unknown |
| | | ☐ Other (specify): | | | | | | | |
| | | Antise | ecretory or antiemetics | | Yes | | ☐ No | | ☐ Don't know |
| | | Zinc | | | Yes | | ☐ No | | ☐ Don't know |
| | | Tradit | cional medicine | | Yes | | ☐ No | | ☐ Don't know |
| | | None | of the above | | Yes | | ☐ No | | ☐ Don't know |
| E. | FORM | и сомі | PLETION | | | | | | |
| | 25. | ID of p | person completing this form | ı: | Date form complet | | m completed:<br>- _ - 2 0 | | |
| | 26. | ID of p | person reviewing this form: | _ | _1 | Date form reviewed: | | _ (dd-mm-yyyy) | |
| | 27. | ID of p | person entering this form: | | | | m entered:<br>- _ - 2 0 | ) | _ (dd-mm-yyyy) |
| | 28. | ID of p | person conducting data veri<br> | fication: | | | data verification:<br>- - 2 0 | | |
## Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name/Country Site CRF 04 — Cluster Completion Form

| Inst | Purpose: Document completion of all households in a cluster. Instructions: Complete this form after all households in an identified cluster have been approached/visited and no further attempts will be made. | | | |
|---|---|---|---|---|
| A. | . VISIT INFORMATION | | | |
| | 1. | Date: | ll | - _ - 2 0 (dd-mm-yyyy) |
| | 2. | EFGH country site: | | |
| | | □ Bangladesh | | □ Kenya |
| | | □ Malawi | | □ Mali |
| | | ☐ Pakistan | □ Peru | |
| | | ☐ The Gambia | | |
| | 3. | Cluster number: | 11_ | <u> </u> |
| | | 3a. Sub-cluster number (applicable to Kenya and The Gambia only) | (1-4) | |
| | 4. | Did the study team approach all households at least three times (if needed) and complete the PE and HUS CRF for each household in the cluster number noted above? | | |
| | | Yes No; there are no household structures in satellite image and expected population size is zero No; it was not possible to visit all households due to extreme weather or safety concerns Other (specify): | | |
| | 5. | How many unique households were visite | ed within th | is cluster? |

Version: 6.0 (01-11-2022) Page: 1 of 1

## Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name (Country Site) Population Enumeration & HUS Protocol Violation Form

**Purpose:** To capture information about Population Enumeration (PE) & Healthcare Utilization Survey (HUS)-related protocol violations that occurred from the start of study until the end of the study duration.

**Form Instructions:** Please complete this form for all PE & HUS protocol violations. If multiple IDs are affected by the violation, please list the affected IDs in the relevant section. Please note that only protocol violations (not deviations) are reported here. As a reminder, a <u>protocol violation</u> is defined as a consistent variation in practice from study protocol/SOPs that may affect participant safety, participant willingness to participate in the study, and/or integrity of the research or study data. <u>Protocol violation</u> is a subset of protocol deviation.

**Reporting Instructions:** To Report a PE & HUS Protocol Violation, please email the completed form to <a href="mailto:efgh@uw.edu">efgh@uw.edu</a> with the email subject "Site Name – PE & HUS Protocol Violation Report."

| | , | | · | | |
|---|---|---|---|---|---|
| A. | SITE | INFORMATION | | | |
| | 1. | EFGH country site: | | | |
| | | ☐ Bangladesh | Kenya | Malawi | Mali Mali |
| | | Pakistan | Peru | ☐ The Gambia | |
| | 2. | Date violation occurred: | | _ - - 2 0 _ | (dd-mm-yyyy) |
| | 3. | Date study staff was made a | ware of violation | _ - - 2 0 _ | (dd-mm-yyyy) |
| | 4. | Date reported by email to Efteam (efgh@uw.edu) | GH Coordination | _ - - 2 0 _ | (dd-mm-yyyy) |
| В. | PRO | TOCOL VIOLATION REPORTING | G | | |
| | 5. | Is the site PI aware of the vio | lation? | | |
| | | Yes | | | |
| | | ☐ No | | | |
| | 6. | Was this event reported to the site-specific IRB? | | | |
| | | Yes | | | |
| | | □ No (skip to Q8) | | | |
| | 7. | If yes, date reported to local IRB: _ - 2 0 (dd-mm-yyyy) | | | |
| | 8. | Was this event entered in the Protocol Deviation/ Violations Log? | | | |
| | | Yes | | | |
| | | □No | | | |
| | 9. | Was the participant informe | d of the Protocol V | iolation? | |
| | | Yes | | | |
| | | ☐ No | | | |
| | | ☐ Not applicable | | | |
| C. | DESC | CRIPTION OF PROTOCOL VIOLATION | | | |
| | 10. | Nature of violation (check al | l that apply) | | |
| | | Consent not obtained or | documented | Consent obtained using outda | ted consent form |
| | | Failure to provide a copy | of signed consent | Administration of Healthcare | Utilization Survey to |
| | | form to the participant cares | | household who did not meet the | inclusion/exclusion criteria |
| | | Undertaking of a study p | rocedure not | Breach in confidentiality | |

Version: 1.0 (01-11-2022) 

# Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name (Country Site) Population Enumeration & HUS Protocol Violation Form

| | | Loss of tablet or study equipment that contains identifiable information about Other (please specify): |
|---|---|---|
| | 11. | participant Who is affected by the violation? (select one) |
| | | Individual |
| | | Enter Affected Household ID: |
| | | _ - - 2 0 - _ - - (skip to Q13) |
| | | ☐ Site-wide |
| | | List affected Household IDs: |
| | 12. | Brief summary of event (Description of event, location it occurred if relevant): |
| | 13. | What steps have been taken to address this event? |
| | 14. | What steps have been taken to prevent further occurrences? |
| D. | FORI | M COMPLETION |
| | 15. | Date form completed: |
| | 1.0 | Data form reviewed: |
| | 16. | ID of person reviewing this form: |




Enterics for Global Health: Shigella Surveillance Study (EFGH)

#### **Lab Case Report Form Appendix**



#### Table of Contents

| CRF Number | CRF Name |
|------------|----------------------------------------------------------------|
| 15 | Specimen Accession |
| 16 | Stool Culture Results – Rectal Swab |
| 16a | Shigella Serotyping & AST Results – Rectal Swab |
| 17 | Stool Culture Results - Whole Stool (Gambia & Bangladesh only) |
| 17a | Shigella Serotyping & AST - Whole Stool |

**Purpose:** To capture specimen accession and storage information for all biological specimens collected in EFGH. Note: temperature excursions are asked separately for rectal swabs (asked only for rectal swab #1 as it is assumed all swabs are shipped together) and whole stools in case whole stool is shipped separate from swabs.

| all swabs are shipped together) and whole stools in case whole stool is shipped separate from swabs. | | |
|---|---|---|
| Inci | Instructions: Complete this form for all enrolled participants. | |
| 1115 | instructions: complete this form for all enrolled participants. | |
| | PLEASE PLACE PARTICIPANT LABEL HERE (OPTIONAL): | |
| Α. | DAD | TICIPANT INFORMATION |
| ۸. | 1. | Participant ID |
| | 2. | EFGH country site: |
| | ۷. | Bangladesh |
| | | Pakistan Peru The Gambia |
| | 3. | Enrollment facility ID: |
| | 4. | Visit specimens were collected at |
| | | Enrollment (complete all sections) |
| | | Week 4 (complete Sections G & H only) |
| В. | RECT | TAL SWAB 1 (DRY) (enrollment visit only) |
| | 5. | Is there a dry rectal swab (swab 1) available for this participant? |
| | | Yes |
| | | □ No (skip to Section C) |
| | 6. | Date sample received at central lab: _ - - 2 0 (dd-mm-yyyy) |
| | 7. | Time sample received at central lab: _ : (hh : min, 24:00 hr) |
| | 8. | Specimen ID: Not applicable |
| | | What type of temperature monitor was used for the rectal swab shipment? Note it is assumed that all |
| | 9. | rectal swabs utilize the same temperature monito |
| | | ☐ WarmMark |
| | | 3M (skip to Q11) |
| | | No monitor available (skip to Q12) |
| | 10. | Temperature excursion for 3 rectal swab shipment (based on WarmMark monitor read): |
| | | Not reached (no color change on WarmMark monitor) |
| | | ☐ Brief |
| | | ☐ Moderate |
| | | ☐ Prolonged |
| | | Answer Q10, then skip to Q12 |
| | 11. | Temperature excursion for 3 rectal swab shipment (based on 3M monitor read): |
| | | 0 (No excursion) |
| | | 0-1 (30 minutes-9 hours) |
| | | 2 (10-20 hours) |
| | | ☐ 3 (21-30 hours) |
| | | 4 (31-40 hours) |
| | | 5 (41+ hours) |
| | 12. | Is the dry rectal swab (swab 1) acceptable for accessioning? |
| | | Ves (skin to 013) |

| | | No, not acceptable for accessioning (answer Q12a, skip to Section C) |
|---|---|---|
| | | 12a. If not acceptable, why? (select all that apply) |
| | | Improperly labelled |
| | | Sample containers did not arrive tighly shut |
| | | Other (specify): |
| | 13. | Date rectal swab was placed in -80°C freezer: - - 2 0 _ (dd-mm-yyyy) |
| | 14. | Time rectal swab was placed in -80°C freezer: : (hh : min, 24:00 hr) |
| | | Comments (optional): |
| C. | REC | TAL SWAB 2 (MODIFIED BGS) (enrollment visit only) |
| | 15. | Is there a mBGS rectal swab (swab 2) available for this participant? |
| | | Yes |
| | | No (skip to Section D) |
| | 16. | Date samples received at central lab: _ - - 2 0 (dd-mm-yyyy) |
| | 17. | Time samples received at central lab: _ : (hh: min, 24:00 hr) |
| | 18. | Specimen ID: Not applicable |
| | 19. | Is the mBGS rectal swab (swab 2) acceptable for accessioning? |
| | | Yes (skip to Q20) |
| | | No, not acceptable for accessioning |
| | | 19a. If not acceptable, why? (select all that apply) |
| | | Improperly labelled |
| | | Sample containers did not arrive tighly shut |
| | | Other (specify): |
| | | Comments (optional): |
| D. | REC | TAL SWAB 3 (CARY-BLAIR) (enrollment visit only) |
| | 20. | Is there a Cary-Blair rectal swab (swab 3) available for this participant? |
| | | Yes |
| | | No (skip to Section E) |
| | 21. | Date samples received at central lab: - - 2 0 (dd-mm-yyyy) |
| | 22. | Time samples received at central lab: : (hh: min, 24:00 hr) |
| | 23. | Specimen ID: Not applicable |
| | 24. | Is the Cary-Blair rectal swab (swab 3) acceptable for accessioning? |
| | | Yes (skip to Q25) |
| | | No, not acceptable for accessioning |
| | | 24a. If not acceptable, why? (select all that apply) |
| | | Improperly labelled |
| | | Sample containers did not arrive tighly shut |
| | | Other (specify): |
| | | Comments (optional): |
| | \A/L1 | <br>DLE STOOL SAMPLE (enrollment visit or within 24 hours [home collection- applicable to Bangladesh, The |
| E. | | ole Stool Sample (enrollment visit or within 24 nours (nome collection- applicable to Bangiaaesh, The<br>hbia, Peru, Malawi, and Pakistan sites]) |
| | 25. | Is there a whole stool sample available for this participant? |

| | | Yes |
|---|---|---|
| | | □ No (skip to Section G) |
| | | Specimen ID: Not applicable |
| | 26. | Was the whole stool shipped together or separately from the rectal swab? |
| | | Same shipment (skip to Q32) |
| | | Different shipment |
| | 27. | Date samples received at central lab: - - 2 0 (dd-mm-yyyy) |
| | 28. | Time samples received at central lab: : (hh: min, 24:00 hr) |
| | 29. | What type of temperature monitor was used for the whole stool shipment? |
| | | WarmMark |
| | | 3M (skip to Q31) |
| | | No monitor available (skip to Q32) |
| | 30. | Temperature excursion for whole stool shipment (based on WarmMark monitor read): |
| | | Not reached (no color change on WarmMark monitor) |
| | | ☐ Brief |
| | | ☐ Moderate |
| | | ☐ Prolonged |
| | | Answer Q30, then skip to Q32 |
| | 31. | Temperature excursion for whole stool shipment (based on 3M monitor read): |
| | | 0 (No excursion) |
| | | 0-1 (30 minutes-9 hours) |
| | | 2 (10-20 hours) |
| | | 3 (21-30 hours) |
| | | 4 (31-40 hours) |
| | | 5 (41+ hours) |
| | 32. | Is the whole stool sample acceptable for accessioning? |
| | | Yes (skip to Q33) |
| | | No, not acceptable for accessioning (answer Q32a then skip to Section F [Gambia and Bangladesh |
| | | sites only] or Section G [other sites]) |
| | | 32a. If not acceptable, why? (select all that apply) (answer Q32a then skip to Section F) |
| | | Improperly labelled |
| | | Sample containers did not arrive tighly shut |
| | | Other (specify): |
| | 33. | Number of vials of whole stool being stored: (1-5) |
| | 34. | Weight of the 1 <sup>st</sup> stored vial of stool (back up qPCR sample): mg (between 180-220mg) |
| | 35. | Date whole stool was placed in -80°C freezer - - 2 0 _ (dd-mm-yyyy) |
| | 36. | Time whole stool was placed in -80°C : (hh: min, 24:00 hr) |
| | | freezer |
| | | Comments (optional): |
| | | Skip to Section G |
| F. | | DLE STOOL SAMPLE FOR WHOLE STOOL CULTURE (Bangladesh and The Gambia sites only; enrollment stool only) |
| | 37. | Is there a mBGS whole stool sample available for this participant? |

| | | Yes | |
|---|---|---|---|
| | | No (skip to Section G) | |
| | 38. | Date samples received at central lab: | _ - - 2 0 (dd-mm-yyyy) |
| | 39. | Time samples received at central lab: | _ : (hh : min, 24:00 hr) |
| | 40. | Specimen ID: | Not applicable |
| | 41. | Is the whole stool sample acceptable for accessioning? | |
| | | Yes (skip to Q43) | |
| | | No, not acceptable for accessioning | |
| | | 42. If not acceptable, why? (select all that appl | y) |
| | | Improperly labelled | |
| | | Sample containers did not arrive tighly s | hut |
| | | Other (specify): | |
| | | Comments (optional): | |
| G. | DRIE | D BLOOD SPOT (enrollment & Week 4 visit only) | |
| | 43. | Is a dried blood spot (DBS) card available for this p | participant? |
| | | Yes | |
| | | ☐ No (skip to Section H) | |
| | 44. | Date samples received at central lab: | _ - - 2 0 (dd-mm-yyyy) |
| | 45. | Time samples received at central lab: | _ : (hh : min, 24:00 hr) |
| | 46. | Specimen ID: Not applicable | |
| | 47. | Is the DBS acceptable for accessioning? | |
| | | Yes (skip to Q48) | |
| | | No, not acceptable for accessioning (answer 4) | 7a, skip to Section H) |
| | | 47a. If not acceptable, why? (select all that appl | (y) |
| | | Improperly labelled | |
| | | Sample containers did not arrive tighly s | hut |
| | | Other (specify): | |
| | 48. | Date DBS card placed in ~4°C storage: | _ - - 2 0 (dd-mm-yyyy) |
| | 49. | Time DBS card placed in ~4°C storage: | _ : (hh : min, 24:00 hr) |
| | | Comments (optional): | |
| Н. | FOR | RM COMPLETION | |
| | 50. | ID of person completing this form: | Date form completed: |
| | | | _ _ - |
| | 51. | ID of person reviewing this form: | Date form reviewed: |
| | | | _ - - 2 0 (dd-mm-yyyy) |
| | 52. | ID of person entering this form: | Date form entered:<br> _ - - 2 0 (dd-mm-yyyy) |
| | 53. | ID of person conducting data verification: | Date of data verification: |
| | 55. | | |
| | | | _ - - 2 0 (dd-mm-yyyy) |

**Purpose:** To capture information about clinical microbiology results from <u>rectal swab</u> samples

**Instructions:** This form is to be completed as a final reporting of Shigella isolates and is to be completed for each child (even if no Shigella was isolated). The related form (16a) is to be completed if Shigella is isolated.

| PLA | CE PA | RTICIPANT LABEL HERE (OPTIONAL): | | |
|---|---|---|---|---|
| A. | SAM | MPLE INFORMATION | | |
| | 1. | Participant ID | | |
| | 2. | Date form initated: | | - - 2 0 (dd-mm-yyyy) |
| | 3. | Time form initiated: | | : (hh : min, 24:00 hr) |
| | 4. | Time of inoculation onto primary media: | ll | : (hh : min, 24:00 hr) |
| В. | LACT | OSE FERMENTER | | |
| | 5. | Were lactose fermenter (LF) colonies isolat | ed? | |
| | | Yes | | |
| | | □ No (skip to Q9) | | |
| | 6. | Confirm that up to 10 lactose fermenter colonies were stored at minus 80°C: | | |
| | | Yes (skip to Q9) | | |
| | | □ No | | |
| | | 5a. If no, why not? | | |
| | 7. | Date LF colonies were placed in minus 80°C | Cfreezer: | - - 2 0 (dd-mm-yyyy) |
| | 8. | Time LF colonies were placed in minus 80°C | C freezer: | : (hh: min, 24:00 hr) |
| C. | SHIG | EELLA ISOLATES (complete based on final Shi | | |
| | 9. | Number of unique <i>Shigella</i> serotypes: | | |
| D. | FORI | isolate, please fill out the serotype and AST M COMPLETION | results in Jo | orm 16a) |
| <u> </u> | 10. | ID of person completing this form: | 1 1 | Date form completed: |
| | 11. | To or person completing this form. | | _ - - 2 0 (dd-mm-yyyy) Date form reviewed: |
| | 11. | ID of person reviewing this form: | .11 | _ - - 2 0 (dd-mm-yyyy) |
| | 12. | ID of person entering this form: | I | Date form entered: |
| | | | | _ - - 2 0 (dd-mm-yyyy) |
| | 13. | ID of person conducting data verification: | | Date of data verification:<br> _ - - 2 0 _ (dd-mm-yyyy) |

**Purpose:** To capture information about Shigella isolates from <u>rectal swab</u> samples

**Instructions:** This form is to be completed as a final reporting of Shigella isolates and is to be completed for each child from which Shigella was isolated. This form will be missing for children without Shigella isolated.

| PLA | PLACE PARTICIPANT LABEL HERE (OPTIONAL): | | | | | |
|---|---|---|---|---|---|---|
| A. | SAM | PLE INFORMATION | | | | |
| | 1. | Participant ID | _ | _ | | |
| | 2. | Date form initated: | - | - 2 0 _ | (dd-mm-yyyy, | ) |
| | 3. | Time form initiated: | : | (hh : min, 2 | 4:00 hr) | |
| В. | SHIG | ELLA ISOLATES (comple | ete based on final # c | of unique Shigella isola | ites) | |
| | | | | Isolate 1 | | |
| | 4. | Specimen ID of <b>1</b> st uni | ique isolate: | | Not applicab | ole |
| | 5. | From which media wa | as the 1 <sup>st</sup> unique isola | ate grown: | | |
| | | ☐ Modified BGS | | | | |
| | | Cary-Blair | | | | |
| | | Both (only tick "bo | oth" if exact same spe | ecies, serotype, and zo | ne sizes) | |
| | 6. | Shigella serogroup: | | | | |
| | | S. dysenteriae | S. flexneri S. b | oydii 🗌 S. sonnei 🛭 | <u>Undetermined</u> | |
| | | 6a. <i>S. flexneri</i> serotyp | e: | | | |
| | | ☐ 1a | 1b | 1d | 2a | ☐ 2b |
| | | ☐ 3a | 3b | 4a | ☐ 4b | ☐ 5a |
| | | ☐ 5b | <u> </u> | □x | ☐ Y | ☐ Non-typable |
| | | Other (specify): | | | | |
| | 7. | Date of 1 <sup>st</sup> unique isolate recovery: - - 2 0 (dd-mm-yyyy) | | | | |
| | 8. | Time of 1st unique isolate recovery: : (hh : min, 24:00 hr) | | | | |
| | 9. | Date of AST test on 1 <sup>st</sup> unique isolate: - - 2 0 (dd-mm-yyyy) Same as date of recovery (Q7) | | | | |
| | 10. | Time of AST test on 15 | st unique isolate: | _ : <i>(h</i> | h : min, 24:00 hr) | |
| | 11. | Antibiotic susceptibili | ty testing results: | | | |
| | | Antibiotic Zone (mm) Interpretation | | | | |

| | Ampicillin | _ | S I R | | |
|---|---|---|---|---|---|
| <br> | Azithromycin | _ | S I R | Not interpreta | able ( <i>obtain MIC</i> ) |
| | Ceftriaxone | | S I R | | |
| | Ciprofloxacin<br>Nalidixic acid | | | | |
| | Pivemicellinam | <u> </u> | S I I R | | |
| | Trimethoprim/ | <u> </u> | | | |
| | sulfamethoxazole | | S I R | | |
| 12. | Azithromycin MIC (if zone si | ze is not interpr | etable) | . [ | Not applicable |
| 13. | Date 1 <sup>st</sup> isolate was placed in | n minus 80°C fr | eezer: _ - _<br>(dd-mm-yyyy) | - 2 0 _<br>Same as date | <br>of recovery <i>(Q7)</i> |
| <br>14. | Time 1 <sup>st</sup> isolate was placed i | n minus 80°C fı | | (hh : min, . | |
| <u> </u> | | 1. | solate 2 | | |
| 15. | Specimen ID of <b>2</b> <sup>nd</sup> <b>unique</b> is | solate: | | Not applica | able |
| <br>16. | From which media was the 2 | 2 <sup>nd</sup> unique isola | te grown: | | |
| | Modified BGS | | | | |
| | Cary-Blair | | | | |
| | Both | | | | |
| 17. | Shigella serogroup: | | | | |
| | S. dysenteriae S. flexneri S. boydii S. sonnei Undetermined | | | | |
| | S. flexneri serotype: | | | | |
| | ☐ 1a ☐ 1 | b | ☐ 1d | 2a | ☐ 2b |
| | ☐ 3a ☐ 3 | b | ☐ 4a | 4b | ☐ 5a |
| | ☐ 5b ☐ 6 | | □x | Y | ☐ Non-typable |
| | Other (specify): | | | | |
| 18. | Date of 2 <sup>nd</sup> unique isolate re | covery: _ | - - 2 | 0 <i>(dd-m</i> | пт-уууу) |
| 19. | Time of 2 <sup>nd</sup> unique isolate recovery: : (hh : min, 24:00 hr) | | | | |
| 20. | Date of AST test on 2 <sup>nd</sup> unique isolate: - - 2 0 (dd-mm-yyyy) Same as date of recovery (Q18) | | | | |
| 21. | Time of AST test on 2 <sup>nd</sup> unique isolate: : (hh : min, 24:00 hr) | | | | |
| 22. | Antibiotic susceptibility test | ing: | | | |
| | Antibiotic | Zone (mm) | MIC | Interp | oretation |
| | Ampicillin | | S I R | | |
| | Azithromycin | | S I R | Not interpret | table ( <i>obtain MIC</i> ) |
| | Ceftriaxone | | | | |

| | | Ciprofloxacin | III | S I R |
|---|---|---|---|---|
| | | Nalidixic acid | III | S I I R |
| | | Pivemicellinam | III | S I I R |
| | | Trimethoprim/<br>sulfamethoxazole | 111 | S 🔲 I 🔲 R |
| | 23. | Azithromycin MIC (if zone s | ize is not interpretable | ) Not applicable |
| | 24. | Date 2 <sup>nd</sup> isolate was placed | • | - - 2 0 <br>(dd-mm-yyyy) |
| | 25. | Time 2 <sup>nd</sup> was placed in min | us 80 freezer: _ | _ : (hh : min, 24:00 hr) |
| | | | | ased on number of additional isolates and serotyping, repeating forms when entering into REDCap. |
| D. | FOR | M COMPLETION | | |
| | 26. | ID of person completing thi | s form: | Date form completed:<br> |
| | 27. | ID of person reviewing this | form: | Date form reviewed: _ - _ _ 2 0 (dd-mm-yyyy) |
| | 28. | ID of person entering this fo | orm: | Date form entered: _ - _ - 2 0 _ _ (dd-mm-yyyy) |
| | 29. | ID of person conducting da | ta verification: | Date of data verification: |
| İ | | 111 | | |

**Appendix:** print out and complete this form for every nth isolate if >2 isolates recovered

| Isolate number: | | | | |
|---|---|---|---|---|
| Specimen ID of isolate | Specimen ID of isolate: Not applicable | | | |
| From which media wa | s the isolate grown: | | | |
| Modified BGS | | | | |
| Cary-Blair | | | | |
| Both | | | | |
| Shigella serogroup: | | | | |
| S. dysenteriae | S. flexneri S. b | oydii 🗌 S. sonnei 🛭 | Undetermine | <u>ed</u> |
| S. flexneri serotype: | | | | |
| 1a | ☐ 1b | 1d | 2a | 2b |
| 3a | 3b | 4a | 4b | 5a |
| 5b | ☐ 6 | Пх | Y | ☐ Non-typable |
| Other (specify): | | | | |
| Date of isolate recove | ry: - | _ - 2 0 | (dd-mm-yy | yyy) |
| Time of isolate recove | ery: : | _ (hh : min, 24:00 | 0 hr) | |
| Date of AST test on is | olate: - | _ - 2 0 | | -уууу) |
| T' CACT I I | | Same as date of recov | | |
| | | (hh : min, 24 | ::00 nr)<br> | |
| Antibiotic susceptibili | | | | |
| Antibiotic | Zone (mm | | | Interpretation |
| Ampicillin | | S | I ∐ R | Not intermediate |
| Azithromycin | | S L | I LR | Not interpretable (obtain MIC) |
| Ceftriaxone S | | | | |
| Ciprofloxacin | | S | I 🗌 R | |
| Nalidixic acid _ _ _ S | | | | |
| Pivemicellinam S | | | | |
| Trimethoprim/ sulfamethoxazole | | | | |
| Azithromycin MIC (if zone size is not interpretable) . . Not applicable | | | | |
| Date isolate was placed in minus 80 freezer: - - 2 0 | | | | |
| Time isolate was placed in minus 80 freezer: : (hh: min, 24:00 hr) | | | | |

## Enterics for Global Health – Shigella Surveillance Study (EFGH) Implementing Institution Name (Country Site) CRF 17 - Stool Culture Results - Whole Stool

**Purpose:** To capture information about clinical microbiology results from whole stool samples (only applicable in Bangladesh & The Gambia).

**Instructions:** This form is to be completed as a final reporting of Shigella isolates and is to be completed for each child (even if no Shigella was isolated) with a whole stool sample transported in Cary-Blair media in the Gambia and Bangladesh The related form (17a) is to be completed if Shigella is isolated.

| PLACE PARTICIPANT LABEL HERE (OPTIONAL): | | | | |
|---|---|---|---|---|
| A. | SAM | PLE INFORMATION | | |
| | 1. | Participant ID | ll_ | |
| | 2. | Date form initiated: | | - - 2 0 (dd-mm-yyyy) |
| | 3. | Time form initiated: | | : (hh : min, 24:00 hr) |
| | 4. | Time of inoculation onto primary media: | 11_ | : (hh : min, 24:00 hr) |
| В. | SHIGELLA ISOLATES (complete based on final Shigella serotypes) | | | |
| | 5. | Number of unique Shigella serotypes: (0 | | -20). For each unique isolate, please fill out the |
| | J. | serotype and AST results in form 17a | | |
| C. | FORI | DRM COMPLETION | | |
| | _ | ID of person completing this form: | | Date form completed: |
| | 6. | | | - - 2 0 (dd-mm-yyyy) |
| | 7. | ID of person reviewing this form: | | Date form reviewed: |
| | /. | | | _ - - 2 0 (dd-mm-yyyy) |
| | Q | 8. ID of person entering this form: | | Date form entered: |
| | 0. | | | _ - - 2 0 _ (dd-mm-yyyy) |
| | 9. | ID of person conducting data verification: | | Date of data verification: |
| | Э. | | | _ - - 2 0 _ (dd-mm-yyyy) |

**Purpose:** To capture information about Shigella isolates from whole stool samples (only applicable in Bangladesh & The Gambia).

**Instructions:** This form is to be completed as a final reporting of Shigella isolates from whole stool and is to be completed for each child from which Shigella was isolated. This form will be missing for children without Shigella isolated.

| PLACE PARTICIPANT LABEL HERE (OPTIONAL): | | | | | | |
|---|---|---|---|---|---|---|
| A. | SAM | SAMPLE INFORMATION | | | | |
| | 1. | Participant ID | | _ | | |
| | 2. | Date form initiated: | - | - 2 0 _ | (dd-mm-yyyy | ) |
| | 3. | Time form initiated: | : | (hh : min, 2 | 4:00 hr) | |
| В. | SHIG | <b>SELLA ISOLATES</b> (complete l | pased on final # c | of unique Shigella isoa | tes) | |
| | | | I | Isolate 1 | | |
| | 4. | Specimen ID of 1st unique | isolate: | | Not applicat | ole |
| | 5. | Shigella serogroup: | | | | |
| | | S. dysenteriae S. j | lexneri 🗌 S. bo | oydii 🗌 S. sonnei 🛭 | Undetermined | |
| | | S. flexneri serotype: | | | | |
| | | ☐ 1a | 1b | ☐ 1d | 2a | 2b |
| | | ☐ 3a ☐ | 3b | ☐ 4a | ☐ 4b | 5a |
| | | 5b | 6 | □x | ☐ Y | ☐ Non-typable |
| | | Other (specify): | | | | |
| | 6. | Date of 1st unique isolate recovery: - - 2 0 (dd-mm-yyyy) | | | | |
| | 7. | Time of 1 <sup>st</sup> unique isolate recovery: : (hh : min, 24:00 hr) | | | | |
| | 8. | Date of AST test on 1 <sup>st</sup> unique isolate: - - 2 0 (dd-mm-yyyy) Same as date of recovery (Q6) | | | | |
| | 9. | Time of AST test on 1 <sup>st</sup> unique isolate: : (hh: min, 24:00 hr) | | | | |
| | 10. | Antibiotic susceptibility testing results: | | | | |
| | | Antibiotic | Zone (mm) | Interpretation | | |
| | | Ampicillin | 111 | S I R | | |
| | | Azithromycin | 111 | □ S □ I □ R | ☐ Not interpretab | le ( <i>obtain MIC</i> ) |

| | Ceftriaxone | lll | □S □I □R | | |
|---|---|---|---|---|---|
| | Ciprofloxacin | III | □ S □ I □ R | | |
| | Nalidixic acid | | □S □I □R | | |
| | Pivemicellinam | _ | □ S □ I □ R | | |
| | Trimethoprim/<br>sulfamethoxazole | | S I R | | |
| 11. | Azithromycin MIC (if zone | size is not interpr | etable) | . <u></u> | ] Not applicable |
| 12. | Date 1 <sup>st</sup> isolate was placed in minus 80 freezer: - - 2 0 (dd-mm-yyyy) Same as date of recovery (Q6) | | | | |
| 13. | Time 1 <sup>st</sup> isolate was placed | in minus 80 free | zer: : | _ (hh : min, 24: | 00 hr) |
| | | Is | olate 2 | | |
| 14. | Specimen ID of <b>2</b> <sup>nd</sup> <b>unique</b> | isolate: | | Not applica | able |
| 15. | Shigella serogroup: | | | | |
| | S. dysenteriae S. fl | exneri 🗌 S. bo | ydii 🗌 S. sonnei 📗 | <u>Undetermined</u> | |
| | S. flexneri serotype: | | | | |
| | ☐ 1a | 1b | ☐ 1d | 2a | 2b |
| | 3a | 3b | 4a | 4b | 5a |
| | 5b | 6 | □x | Y | ☐ Non-typable |
| | Other (specify): | | | | |
| 16. | Date of 2 <sup>nd</sup> unique isolate i | ecovery: _ | - - 2 | 0 (dd-m | іт-уууу) |
| 17. | Time of 2 <sup>nd</sup> unique isolate | recovery: _ | : (hh: | min, 24:00 hr) | |
| 18. | Date of AST test on 2 <sup>nd</sup> unique isolate: - - 2 0 (dd-mm-yyyy) Same as date of recovery (Q16) | | | | |
| 19. | Time of AST test on 2 <sup>nd</sup> unique isolate: : (hh: min, 24:00 hr) | | | | |
| 20. | Antibiotic susceptibility testing: | | | | |
| | Antibiotic | Zone (mm) | MIC | Interpr | etation |
| | Ampicillin | | S I R | | |
| | Azithromycin | | □ S □ I □ R | ☐ Not interpret | able ( <i>obtain MIC</i> ) |
| | Ceftriaxone | 11 | □ S □ I □ R | | |
| | Ciprofloxacin | | S I R | | |
| | Nalidixic acid | | S I R | | |
| | Pivemicellinam | | S I R | | |

| | | Trimethoprim/ sulfamethoxazole | S |
|---|---|---|---|
| | 21. | Azithromycin MIC (if zone size is not interpretable) | Not applicable |
| | 22. | Date 2 <sup>nd</sup> isolate was placed in minus 80 freezer: _ (c | ld-mm-yyyy) |
| | | | Same as date of recovery (Q16) |
| | 23. | Time 2 <sup>nd</sup> was placed in minus 80 freezer: _ | : (hh: min, 24:00 hr) |
| C. | EODI | M COMPLETION | |
| C. | ION | VI CONFEETION | |
| C. | 24. | ID of person completing this form: | Date form completed: |
| C. | | | Date form completed: _ - - 2 0 (dd-mm-yyyy) |
| C. | | ID of person completing this form: | - |
| С. | 24. | | _ - - 2 0 _ (dd-mm-yyyy) |
| С. | 24. | ID of person completing this form: ID of person reviewing this form: | _ - - 2 0 (dd-mm-yyyy) Date form reviewed: |
| C. | 24. | ID of person completing this form: | _ - - 2 0 (dd-mm-yyyy) Date form reviewed: - - 2 0 (dd-mm-yyyy) |
| C. | 24. | ID of person completing this form: ID of person reviewing this form: | _ - - 2 0 (dd-mm-yyyy) Date form reviewed: _ - _ - 2 0 (dd-mm-yyyy) Date form entered: |

**Appendix:** print out and complete this form for every nth isolate if >2 isolates recovered

| Isolate number: | | | | |
|---|---|---|---|---|
| Specimen ID of isolate: Not applicable | | | | |
| From which media wa | s the isolate grown: | | | |
| ☐ Modified BGS | | | | |
| Cary-Blair | | | | |
| Both | | | | |
| Shigella serogroup: | | | | |
| S. dysenteriae | ] S. flexneri 🔲 S. b | ooydii 🗌 S. sonnei | Undetermine Undetermine | <u>ed</u> |
| S. flexneri serotype: | | | | |
| 1a | ☐ 1b | 1d | 2a | 2b |
| 3a | ☐ 3b | 4a | ☐ 4b | ☐ 5a |
| 5b | <u> </u> | □х | Y | ☐ Non-typable |
| Other (specify): | <u> </u> | | <u> </u> | |
| Date of isolate recove | ery: - | _ - 2 0 | (dd-mm-y | vyy) |
| Time of isolate recove | ery: : | _ (hh : min, 24: | 00 hr) | |
| Date of AST test on is | ·==-·· | - 2 0 _ | (dd-mm | - <i>yyyy)</i> |
| Time of AST test on is | | ate of recovery | 21:00 hr) | |
| | | | 24.00 III ) | |
| Antibiotic susceptibili | | | | |
| Antibiotic | Zone (mm | | IIC | Interpretation |
| Ampicillin | | S | JI ∐ R | <u> </u> |
| Azithromycin | | <u> </u> S <u> </u> | JI ∐ R<br>Ji □ B | |
| Ceftriaxone | ll_ | | JI ∐ R<br>Ji □ B | |
| Ciprofloxacin S S R | | | | |
| Nalidixic acid S ☐ I ☐ R Pivemicellinam | | | | |
| Trimethoprim/ | | | | |
| sulfamethoxazole S I R | | | | |
| Azithromycin MIC (if zone size is not interpretable) . . Not applicable | | | | |
| Date isolate was placed in minus 80 freezer: - - 2 0 (dd-mm-yyyy) | | | | |
| Time isolate was placed in minus 80 freezer: : (hh: min, 24:00 hr) | | | | |



- 11. Lee G, Penataro Yori P, Paredes Olortegui M, et al. An instrument for the assessment of diarrhoeal severity based on a longitudinal community-based study. *BMJ Open* 2014; **4**(6): e004816.
- 12. WHO Department of Nutrition for Health and Development. WHO Anthro Survey Analyser. WHO 2019. Geneva, Switzerland. https://whonutrition.shinyapps.io/anthro
- 13. Dilruba, N, Blackwelder, WC, Sommerfelt, H, et al. Pathogens Associated With Linear Growth Faltering in Children With Diarrhea and Impact of Antibiotic Treatment: The Global Enteric Multicenter Study. *JID* 2021; **224**(Supp 7)" S848-55.
- 14. Stenberg K, Lauer JA, Gkountouras G, Fitzpatrick C, Stanciole A. Econometric estimation of WHO-CHOICE country-specific costs for inpatient and outpatient health service delivery. *Cost Eff Resour Alloc* 2018; **16**: 11.
- 15. Manning WG, Mullahy J. Estimating log models: to transform or not to transform? *J Health Econ* 2001; **20**(4): 461-94.